## STATISTICAL ANALYSIS PLAN FOR CLINICAL STUDY REPORT

A PHASE 2B RANDOMIZED, ACTIVE-CONTROLLED, STAGED, OPEN-LABEL TRIAL TO INVESTIGATE SAFETY AND EFFICACY OF BMS-955176 IN COMBINATION WITH DOLUTEGRAVIR AND ATAZANAVIR (WITH OR WITHOUT RITONAVIR) IN TREATMENT-EXPERIENCED HIV-1 INFECTED ADULTS

PROTOCOL AI468048

**VERSION #2.0** 

# **TABLE OF CONTENTS**

| STATIST | TICAL ANALYSIS PLAN FOR CLINICAL STUDY REPORT | 1 |
|---|---|---|
| TABLE ( | OF CONTENTS | 2 |
| LIST OF | TABLES | 5 |
| 1 | BACKGROUND AND RATIONALE | 6 |
| 2 | OBJECTIVES | 7 |
| 2.1 | Study Design | 7 |
| 2.2 | Treatment Assignment | 9 |
| 2.3 | Blinding and Unblinding | 9 |
| 2.4 | Protocol Amendments | 9 |
| 3 | ENDPOINTS | 10 |
| 3.1 | Primary | 10 |
| 3.2 | Secondary | 11 |
| 3.3 | Exploratory | 11 |
| 4 | ENDPOINTS | 12 |
| 4.1 | Primary Endpoints | 12 |
| 4.2 | Secondary Endpoints | 12 |
| 4.3 | Exploratory Endpoints | 12 |
| 5 | SAMPLE SIZE AND POWER | 13 |
| 6 | STUDY PERIODS, TREATMENT REGIMENS AND POPULATIONS FOR ANALYSES | 13 |
| 6.1 | Study Periods | 13 |
| 6.2 | Treatment Regimens | 13 |
| 6.3 | Populations for Analyses | 14 |
| 7 | STATISTICAL ANALYSIS | 14 |
| 7.1 | General Methods | 14 |
| 7.2 | Study Conduct | 15 |
| 7.3 | Study Population | 15 |
| 7.3.1 | Subject Disposition | 15 |
| 7.3.2 | Demographics and Other Characteristics | 16 |
| 7.3.2.1 | Demographics and Other Baseline Characteristics | 16 |
| 7.3.2.2 | Pre-treatment CDC Class C AIDS Events | 19 |
| 7.3.2.3 | Previous Medication | 19 |

| 7.3.2.4 | Baseline Resistance | 19 |
|---|---|---|
| 7.4 | Extent of Exposure | 20 |
| 7.4.1 | Study Therapy | 20 |
| 7.4.2 | Discontinuation of Study Therapy | 21 |
| 7.4.3 | Interruption or Delay of Study Therapy | 21 |
| 7.4.4 | Concomitant Therapy | 21 |
| 7.5 | Efficacy | 21 |
| 7.5.1 | Primary Efficacy Endpoint: Proportion of Subjects with Plasma HIV-1 RNA < 40c/mL at the Week 24 Snapshot | 21 |
| 7.5.1.1 | Summaries of Primary Efficacy Endpoint Within Subgroups | 22 |
| 7.5.2 | Secondary Efficacy Endpoints | 23 |
| 7.5.2.1 | Proportion of Subjects with Plasma HIV-1 RNA < 40c/mL at Weeks 48 and 96 | 23 |
| 7.5.2.2 | Proportion of Subjects with Plasma HIV-1 RNA < 200c/mL at the Week 24, 48 and 96 Snapshot | 23 |
| 7.5.2.3 | Change from Baseline in Plasma HIV-1 RNA (log <sub>10</sub> ) over Time | 23 |
| 7.5.2.4 | Changes from Baseline in CD4+ and CD8+ T-cell Count over Time | 23 |
| 7.5.2.5 | Newly-emergent Genotypic Substitutions, $IC_{50}$ Fold Changes from Baseline and Newly-emergent Gag Polymorphisms | 24 |
| 7.5.3 | Exploratory Efficacy Endpoints | 25 |
| 7.5.3.1 | Proportion of Subjects with Plasma HIV-1 RNA within Certain Range over Time | 25 |
| 7.5.3.2 | Efficacy Summaries by Baseline Gag Polymorphisms | 25 |
| 7.5.4 | Futility Analysis | 25 |
| 7.6 | Safety | 26 |
| 7.6.1 | Overall Adverse Events | 26 |
| 7.6.2 | Deaths | 27 |
| 7.6.3 | Serious Adverse Events | 27 |
| 7.6.4 | Serious Adverse Events Emerging After Switch to Continuation Therapy | 27 |
| 7.6.5 | Non-Serious Adverse Events | 27 |
| 7.6.6 | Adverse Events Leading to Discontinuation of Therapy | 28 |
| 7.6.7 | Adverse Events Leading to Discontinuation of Therapy After Switch to Continuation Therapy | 28 |
| 7.6.8 | Adverse Events by Relationship | 28 |

| 7.6.9 | Advers | e Events by Intensity | 28 |
|---|---|---|---|
| 7.6.10 | CDC C | Class C AIDS Events | 28 |
| 7.6.11 | Advers | e Events of Special Interest | 28 |
| 7.6.12 | Multip | le Adverse Events | 28 |
| 7.6.13 | Clinica | ıl Laboratory Evaluations | 29 |
| 7.6.13.1 | Labora | itory Abnormalities | 29 |
| 7.6.13.2 | Labora | tory Tests over Time | 29 |
| 7.6.14 | Electro | ocardiograms | 30 |
| 7.6.15 | Vital S | igns | 30 |
| 7.7 | Clinica | l Biomarker Assessments | 31 |
| 7.8 | Integra | ted Summaries | 31 |
| 7.9 | Outcon | nes Research | 32 |
| 7.9.1 | EQ-5D | )-3L | 32 |
| 7.9.2 | FAHI | | 33 |
| 7.10 | Pharma | acokinetics | 34 |
| 8 | CONV | ENTIONS | 35 |
| 8.1 | Deriva | tion of Baseline and On-Treatment Parameters Using Visit Windows | 35 |
| 8.1.1 | Baselir | 1e | 35 |
| 8.1.2 | On-Tre | eatment Parameters | 35 |
| 8.2 | Derive | d Dates | 37 |
| 8.3 | Derive | d Parameters | 37 |
| 8.4 | Study | Гһегару | 37 |
| 8.5 | Conco | mitant Medications | 38 |
| 8.6 | Counti | ng Rules for Adverse Events | 38 |
| 8.7 | Pharma | acokinetic Evaluations | 39 |
| 8.7.1 | Decimo | al Places for Pharmacokinetic Data | 39 |
| 8.7.2 | Pharm | acokinetic Summaries | 39 |
| 9 | REFER | RENCES | 40 |
| APPEND | IX 1 | SNAPSHOT ALGORITHM | 41 |
| APPEND | IX 2 | GENOTYPIC AND PHENOTYPIC RESISTANCE | 43 |
| APPEND | IX 3 | TIME TO LOSS OF VIROLOGIC RESPONSE | 47 |
| APPEND | IX 4 | EQ-5D-3L SCORING PROGRAM - U.S. WEIGHTED | 49 |
| APPENDIX 5 EO-5D-3L SCORING PROGRAM - V | | EO-5D-3L SCORING PROGRAM - U.K. WEIGHTED | 52 |

| 10 R | REFERENCES | 53 |
|---|---|---|
| | OOCUMENT HISTORY | |
| | LIST OF TABLES | |
| Table 7.3.2.1 | -1: Demographic Characteristics | 16 |
| Table 7.3.2.1 | -2: Baseline Disease Characteristics | 17 |
| Table 7.3.2.1 | -3: Other Baseline Characteristics | 18 |
| Table 7.6.1-1 | : Adverse Event Summaries | 26 |
| Table 8.1.2-1 | : Visit Windows | 36 |
| Table 9-1: | Snapshot Algorithm Analysis Visit Windows | 41 |
| Table 9-2: | Genotypic Substitutions | 43 |
| Table 9-3: | Cut-offs used by Monogram Biosciences to Determine Reduced Susceptibility | 45 |
| Table 11-1: | Document History | 53 |

#### 1 BACKGROUND AND RATIONALE

Despite advances in prevention and care, HIV/AIDS remains a significant epidemic in both the US and worldwide. AIDS remains the 6th leading cause of death, internationally. Globally, approximately 35 million people were living with HIV infection in 2013. A number of these patients include those who are treatment-experienced. Note: the use of the term "treatment-experienced" herein refers to subjects who have failed at least one or two antiretroviral (ARV) regimens and who may be harboring drug resistant virus (current or archived) to at least one drug class.

In contrast to current HIV treatment guidelines for treatment-naïve patients, the recommended composition of combination antiretroviral therapy (cART) is far less uniform for treatment-experienced subjects. The level of detail in the DHHS and EACS guidelines leads to a lack of uniformity in treatment for patients in later lines of therapy. Moreover, drug related toxicities (both short and longer term) in treatment-experienced subjects necessitate vigilance and continued monitoring. Thus, there is a need for new and efficacious agents with novel mechanisms of action (MOA) and favorable safety/tolerability profiles. Given the aging HIV-1 infected population and overall fewer number of ARV options for treatment-experienced patients, there is a need for a more simplified regimen that may have a better long-term safety profile such as that of a nucleoside- and booster-sparing cART regimen. This study evaluates the merits of a nucleoside-sparing cART regimen and a nucleoside/booster-sparing cART regimen in Stage 1 and 2, respectively.

Given the afore-mentioned challenges with existing treatment in ARV treatment-experienced adults, the two primary objectives of this two stage, Phase 2b study are to: 1) To study the efficacy of one dose (120mg) of BMS-955176 (a novel HIV-1 maturation inhibitor) when given in combination with atazanavir boosted with ritonavir (ATV/r) 300/100mg and dolutegravir (DTG) 50mg in Stage 1, and 2) to study the efficacy of two doses (120 and 180mg) of BMS-955176 when given in combination with unboosted ATV 400mg and DTG 50mg in Stage 2.

Ultimately this Phase 2b clinical trial will provide supportive data in the context of a therapeutic dose of BMS-955176 and the clinical safety/efficacy/resistance of the proposed component(s) of a single tablet regimen (STR, that is also a nucleoside/ritonavir sparing ARV strategy) for Phase 3 trial development in HIV-1 infected treatment-experienced subjects. Specifically, two arms in Stage 2 will contain the individual ARV components of a potential STR: BMS-955176, ATV, and DTG.

#### **Research Hypothesis:**

This Phase 2b study will evaluate whether the combination of BMS-955176 with ATV (with or without RTV) and DTG is efficacious, safe, and well-tolerated in HIV-1 infected treatment-experience adults.

## **Schedule of Analyses:**

A first interim analysis will be conducted after approximately 50% of the randomized subjects have completed 24 weeks of therapy in Stage 1. This analysis will use the BMS equivalent of SDTM (Study Data Tabulation Model) data to facilitate the development of models for population pharmacokinetics, exposure-response relationships and viral kinetics.

A second interim analysis will be conducted after the last subject has completed 24 weeks of therapy in Stage 1. This will be a complete analysis of the available efficacy, safety and resistance data.

An interim analysis might be conducted after the last randomized subject in Stage 1 is on tratment for 48 weeks in case the continuation dose couldn't be selected based on the Week 24 results

An interim analysis will be conducted after the last randomized subject in Stage 2 is on treatment for 24 weeks. The expectation is that the last subject in Stage 1 will have completed the Week 96 visit by that time.

An interim analysis will be conducted after the last randomized subject in Stage 2 completes the Week 48 visit. The analyses related to the first 48 weeks of treatment for Stage 2 will be performed.

The final analysis will be conducted after the last randomized subject in Stage 2 completes the Week 96 visit.

#### 2 OBJECTIVES

# 2.1 Study Design

This is a randomized, active-controlled, staged, open-label clinical trial.

The screening period begins on the day the subject signs on the informed consent form. If the subject meets all eligibility criteria, the subject is to be randomized within the 42-day screening period.

Approximately 200 treatment-experienced HIV-1 subjects will be randomized to one of five treatment arms (approximately 40 per arm) in a staged fashion.

The data from the Week 24 analysis of Stage 1 and AI468038, including safety, efficacy and pharmacokinetics, will be examined to trigger the start of Stage 2 and confirm the two doses of BMS-955176 for study in Stage 2.

#### Stage 1:

In Stage 1, approximately 80 subjects will be randomly assigned 1:1 to one of two treatment arms and on Day 1, they will begin dosing with:

• Arm 1: BMS-955176 120mg QD + ATV/r 300/100mg QD + DTG 50mg QD, or

• Arm 2: TDF 300mg QD + ATV/r 300/100mg QD + DTG 50mg QD.

### Stage 2:

In Stage 2, approximately 120 subjects will be randomly assigned 1:1:1 to one of three treatment arms and on Day 1, they will begin dosing with:

- Arm 3: BMS-955176 120 mg QD + ATV 400 mg QD + DTG 50 mg QD, or
- Arm 4: BMS-955176 180 mg QD + ATV 400 mg QD + DTG 50 mg QD, or
- Arm 5: TDF 300 mg QD + ATV/r 300/100 mg QD + DTG 50 mg QD.

Subjects in all arms will have the opportunity to participate in an elective Intensive PK substudy visit at Week 2 (window for visit: Day 12-16). Approximately 60 subjects, 12 subjects from each arm, are expected to participate in the substudy; BMS may allow the substudy to over-enroll in an effort to have a sufficient number of complete datasets.

Subjects are expected to be treated for the duration of 96 weeks. After Day 1 and the optional Intensive PK visit at Week 2, subjects are required to attend 12 more in-clinic study visits over the 96-week treatment period, as follows:

- Visits are conducted every 4 weeks from Week 4 through Week 16
- Visits are conducted every 8 weeks from Week 24 through Week 48
- Visits are conducted every 12 weeks from Week 60 through Week 96

# **Selection of Continuation Dose and Switch for Stage 1**

Once all subjects in Stage 1 have reached Week 24, BMS will conduct an interim analysis of efficacy, safety, resistance and pharmacokinetics. An analysis of virologic futility will also occur at Week 24. If Arm 1 meets criteria for virologic futility at Week 24, the clinical trial will be terminated.

Based upon the Week 24 analysis of Arms 1 and 2, combined with the Week 24 analysis of all arms in the parallel AI468038 study, a continuation dose of BMS-955176 for Arm 1 will be selected for subjects in Arm 1. Subjects in the BMS-955176 treatment arm 1 may subsequently be transitioned to a selected continuation dose of BMS-955176. Subjects in the Arm containing TDF (i.e., Arm 2) will continue with the TDF treatment regimen. The assigned backbone will remain unaltered. The Week 24 efficacy, safety and pharmacokinetic analyses from Stage 1 and study AI468038 will also trigger the start of Stage 2. If the continuation dose cannot be clearly identified using the Week 24 data, the study will continue in original fashion until an analysis of the Week 48 data can be performed and the continuation dose is selected. If a continuation dose cannot be selected based upon the Week 24 data, this does not preclude the ability to start recruitment of Stage 2.

After the continuation dose is selected and once all of the logistics have been completed globally, the transition of the subjects in Arm 1 to the continuation dose will occur. It is anticipated that this transition will occur on or after all subjects have reached Week 48.

## Selection of Continuation Dose and Switch for Stage 2

Once all subjects in Stage 2 have reached Week 24, BMS will conduct an interim analysis of efficacy, safety, resistance and pharmacokinetics. An analysis of virologic futility will also occur at Week 24. If a BMS-955176 dose arm meets criteria for virologic futility at Week 24, subjects in said arm will begin dosing with the next highest available remaining dose of BMS-955176.

The totality of data from AI468038 and AI468048 (Stage 1 and 2) will be used to select a continuation dose of BMS-955176 for Arms 3 and 4. Subjects in the BMS-955176 treatment arms 3 and 4 will subsequently be transitioned to the selected continuation dose of BMS-955176. It is anticipated that this transition may occur on or after all subjects in Stage 2 have reached Week 48. The assigned backbone will not change. Subjects in the TDF-containing arm (i.e., Arm 5) will continue with their assigned treatment regimen.

# 2.2 Treatment Assignment

Approximately 200 treatment-experienced HIV-1 subjects will be randomized to one of five treatment arms (approximately 40 per arm) in a staged fashion.

#### Stage 1:

In Stage 1, approximately 80 subjects will be randomly assigned 1:1 to one of two treatment arms:

- Arm 1: BMS-955176 120mg QD + ATV/r 300/100mg QD + DTG 50mg QD, or
- Arm 2: TDF 300mg QD + ATV/r 300/100mg QD + DTG 50mg QD.

#### Stage 2:

In Stage 2, approximately 120 subjects will be randomly assigned 1:1:1 to one of three treatment arms:

- Arm 3: BMS-955176 120mg QD + ATV 400mg QD + DTG 50mg QD, or
- Arm 4: BMS-955176 180mg QD + ATV 400mg QD + DTG 50mg QD, or
- Arm 5: TDF 300mg QD + ATV/r 300/100mg QD + DTG 50mg QD.

## 2.3 Blinding and Unblinding

This is an open-label study.

#### 2.4 Protocol Amendments

The following protocol amendments and administrative letters have been processed and changes that may affect the statistical analysis are listed below:

- Amendment 1 (Jan 28, 2015 site specific):
  - Permit the collection and storage of blood samples for use in future exploratory pharmacogenetic research.

- Amendment 2 (Jan 28, 2015 country specific, Brazil)
  - To comply with the Brazilian law in force regarding post study access to therapy.
- Amendment 3 (Feb 13, 2015 country specific, Argentina)
  - In response to a request from the Argentinean Health Authority: in case of pregnancy the study drug should be permanently discontinued.
- Amendment 4 (March 19, 2015)
  - Incorporated information that more clarifies the Week 24 data (consisting of efficacy, safety and pharmacokinetic data) to be used to confirm the doses for Stage 2 and to trigger the start of Stage 2 of the study relative to other analyses conducted under the protocol for other purposes.
  - Removed the requirement that all sparse PK samples need to be collected as pre-AM dose samples. Only one visit Weeks 4-24 (as opposed to all visits Week 4-24) needs to be performed in the morning and to have the blood collected as a pre-AM dose sampling.
- Amendment 5 (June 3, 2015)
  - To mitigate the risk of randomizing subjects infected with HIV-1 with an unknown efficacy profile, exclusion criteria have been modified to now exclude subjects with Clade AE as well as those subjects who have failed a previous boosted PI- or Integrase strand transfer inhibitor (INSTI)-containing regimen for which resistance analyses were not conducted at the time of failure.
  - Pregnancy was added as a reason to be discontinued from the study and the practice of Rescreening was more clearly defined, an administrative change was made to clearly indicate that AIDS History is taken at Screening.
  - At Week 24, a Time to Loss of Virologic Response analysis will be conducted as a sensitivity analysis that compliments the snapshot analysis, and a definition of virologic rebound was added.
- Amendment 6 (July 15, 2015 country specific: Argentina)
  - Section 3.2: Eliminate bullet d) in order to be consistent with local regulations.

#### 3 ENDPOINTS

#### 3.1 Primary

#### **Primary Objective Stage 1**

• To assess the antiviral efficacy of BMS-955176 120mg, and a TDF 300mg-containing arm, each when given in combination with ATV/r 300/100mg and DTG 50mg by determining the proportion of treatment-experienced subjects with plasma HIV-1 RNA < 40c/mL at Week 24 in Stage 1.

### **Primary Objective Stage 2**

To assess the antiviral efficacy of two doses (120 and 180mg) of BMS-955176, each when given in combination with unboosted ATV 400mg and DTG 50mg, and to assess the antiviral efficacy of TDF 300mg when given in combination with ATV/r 300/100mg and DTG 50mg

by determining the proportion of treatment-experienced subjects with plasma HIV-1 RNA < 40c/mL at Week 24 in Stage 2.

## 3.2 Secondary

- To assess the antiviral efficacy of BMS-955176 Arms, and TDF-containing regimens (TDF + ATV/r + DTG), by determining the proportion of treatment-experienced subjects with plasma HIV-1 RNA < 40c/mL at Weeks 48 and 96
- To assess the antiviral efficacy of BMS-955176 Arms, and TDF-containing regimens, by determining the proportion of treatment-experienced subjects with plasma HIV-1 RNA < 200c/mL at Weeks 24, 48, 96
- To assess the emergence of HIV drug resistance in samples selected for drug resistance testing
- To assess efficacy of BMS-955176 Arms, and TDF-containing regimens, by using the mean changes from baseline in log<sub>10</sub> HIV-1 RNA, CD4+ T-cell counts, and percentage of CD4+ T-cells
- To assess the safety and tolerability of BMS-955176 in treatment-experienced subjects by measuring frequency of SAEs and AEs leading to discontinuation
- To assess disease progression as measured by the occurrence of new AIDS defining events (CDC Class C events)
- To characterize the pharmacokinetics of BMS-955176 when co-administered with ATV (with or without ritonavir) and DTG in treatment-experienced HIV-1 infected subjects.

# 3.3 Exploratory

- To determine the effect of BMS-955176 Arms, and TDF-containing regimens, on renal clinical parameters and biomarkers through Weeks 48 and 96
- To determine the effect of BMS-955176 Arms, and TDF-containing regimens, on bone biomarkers through Weeks 12 and 24
- To assess the impact of baseline (pre-therapy) Gag polymorphisms on the efficacy of BMS-955176 by determining the proportion of treatment-experienced subjects with plasma HIV-1 RNA < 40c/mL, HIV-1 RNA < 200c/mL, and the changes from baseline in log<sub>10</sub> HIV-1 RNA at Weeks 24, 48 and 96, by baseline polymorphisms
- To characterize the steady-state plasma PK of DTG when co-administered with BMS-955176 and ATV (with or without RTV) in treatment-experienced subjects. The effect of BMS-955176 on DTG PK in the presence of ATV (without RTV) may be assessed relative to historical data
- To compare steady-state exposures of DTG when co-administered with BMS-955176 and ATV/RTV to DTG when co-administered with TDF and ATV/RTV
- To characterize the PK of ATV when co-administered with DTG and BMS-955176, with or without RTV
- To explore PK/PD and PK/viral kinetic (VK) relationships between BMS-955176, ATV, and/or DTG exposure and both efficacy and safety endpoints

• To assess the impact of the study therapies on health-related quality of life measures.

#### 4 ENDPOINTS

# 4.1 Primary Endpoints

- Proportion of subjects with plasma HIV-1 RNA < 40c/mL at Week 24 for Stage 1, assessed using the snapshot algorithm
- Proportion of subjects with plasma HIV-1 RNA < 40c/mL at Week 24 for Stage 2, assessed using the snapshot algorithm

## 4.2 Secondary Endpoints

- Proportion of subjects with plasma HIV-1 RNA < 40c/mL at Weeks 48 and 96, assessed using the snapshot algorithm
- Proportion of subjects with plasma HIV-1 RNA < 200c/mL at Weeks 24, 48 and 96, assessed using the snapshot algorithm
- Emergence of HIV drug resistance among samples selected for drug resistance testing will be assessed using the most recent version of the IAS-USA list of HIV-1 drug resistance mutations
- Changes from baseline in log<sub>10</sub> HIV-1 RNA and in CD4+ T-cell counts, and changes in the percentage of CD4+ T-cells over time will be assessed using on-treatment laboratory results, and pre-specified visit windows
- Frequency of SAEs and AEs leading to discontinuation will be tabulated directly from the case report forms (CRFs). The summary will count the number of subjects that have at least one event
- Occurrence of new AIDS defining events will be tabulated from the CRFs. The summary will count the number of subjects that have at least one event
- Steady state PK parameters of BMS-955176: C<sub>max</sub>, T<sub>max</sub>, C<sub>tau</sub>, C<sub>0</sub> and AUC(TAU) will be assessed using the intensive PK data, collected at Week 2 from a subset of subjects

# 4.3 Exploratory Endpoints

- Changes from baseline in renal biomarkers over time will be assessed using on-treatment laboratory results, and pre-specified visit windows
- Changes from baseline in bone biomarkers over time will be assessed using on-treatment laboratory results, and pre-specified visit windows
- Proportion of subjects with plasma HIV-1 RNA < c/mL and HIV-1 RNA < 200c/mL at Weeks 24, 48 and 96, by baseline polymorphism, will be assessed using the snapshot algorithm. The changes from baseline in log<sub>10</sub> HIV-1 RNA at Weeks 24, 48 and 96, by baseline polymorphism will be assessed using on-treatment laboratory results, and prespecified visit windows.
- Steady-state PK parameters of DTG: C<sub>max</sub>, T<sub>max</sub>, C<sub>tau</sub>, C<sub>0</sub> and AUC(TAU) will be assessed using the intensive PK data, collected at Week 2 from a subset of subjects

- Steady-state PK parameters of ATV:  $C_{max}$ ,  $T_{max}$ ,  $C_{tau}$ ,  $C_0$  and AUC(TAU) will be assessed using the intensive PK data, collected at Week 2 from a subset of subjects
- Population PK modeling to obtain population-derived average steady state exposure of BMS-955176 that will be used in exposure-response and PK/VK assessments. The population PK, exposure-response, and viral kinetic analyses will be described in a separate analysis plan.
- Quality of life is assessed using the EQ-5D-3L and the Functional Assessment of HIV Infection (FAHI) instruments.

#### 5 SAMPLE SIZE AND POWER

This is an estimation study, without statistical testing, and hence there are no power considerations.

It is expected that response rate for the primary endpoint for all five arms will be somewhere around 80%. With this response rate, and 40 subjects per arm, an exact Clopper-Pearson 95% confidence interval would run from roughly 64% to 91%.

# 6 STUDY PERIODS, TREATMENT REGIMENS AND POPULATIONS FOR ANALYSES

# 6.1 Study Periods

This study consists of the following periods:

- Screening (or Pre-randomization) Period: begins on the day the subject signs the informed consent and continues through Day 1 prior to dosing. The screening period last about 42 days.
- Open-label Treatment Period (or On-treatment Period): begins on the first day of open-label therapy and ends after 96 weeks of dosing or early termination, whichever comes first.

#### 6.2 Treatment Regimens

The treatment regimens are defined as follows:

- As-randomized refers to the treatment regimen assigned at randomization. Accrual, disposition, demographic and baseline characteristics, protocol deviations and efficacy results will be presented as-randomized.
- As-treated refers to the actual treatment regimen received. Subjects who receive an incorrect study therapy for the entire period of treatment are grouped according to the first incorrect study regimen received. Otherwise, subjects are grouped according to their randomized treatment regimen. Subjects who never receive study therapy, have their as-treated treatment regimen coded as "missing". Results for exposure, concomitant medication, resistance, safety and PK parameters, and outcomes research scales will be presented as-treated.

## 6.3 Populations for Analyses

Populations for analyses consist of enrolled, randomized and treated subjects:

- Enrolled subjects are those who signed an informed consent form and were assigned a Patient Identification number (PID).
- Randomized subjects are enrolled subjects who received a treatment assignment from the IVRS. The randomized subjects will be used to assess subject disposition.
- Treated subjects (also referred to as mITT analysis set) are randomized subjects who received at least 1 dose of study therapy. The treated subjects will be used to assess demography and baseline characteristics, protocol deviations, exposure, concomitant medication, efficacy, resistance, safety and outcomes research scales.
- PK population is defined as all treated subjects who have any available concentration-time data. The evaluable PK population is a sub-population including all treated subjects who have adequate PK profiles.

#### 7 STATISTICAL ANALYSIS

This section describes the analyses for the Week 24 primary analysis and the Week 48 and 96 secondary analyses.

Analyses do not exclude data obtained after the start of prohibited medication, unless otherwise specified.

#### 7.1 General Methods

This is an estimation study. Formal comparisons of treatment arms will not be performed except for the virologic futility analyses performed at Week 24 of Stage 1 and Stage 2 (see Section 7.5.4).

Presentations will present treatment arms as the original treatment arms, before the potential movement to the continuation BMS-955176 dose. Data from Arms 2 and 5 will not be pooled unless otherwise specified. Separate outputs will be created for each stage unless otherwise specified.

Categorical variables will be tabulated with counts and percentages.

Continuous variables will be summarized with univariate statistics.

Subjects must have a baseline measurement and at least one on-treatment measurement to be evaluable for change from baseline analyses. All data will be displayed for statistics that do not depend on a baseline measurement.

Laboratory parameters will be summarized using SI and US values and units.

Statistical analyses are carried out in SAS version 9.1.3 (Statistical Analysis System, SAS Institute, North Caroline, USA) or higher, unless otherwise indicated.

# 7.2 Study Conduct

Protocol deviations that are programmable from the database and that could potentially affect the interpretability of the study results are deemed relevant protocol deviations. Relevant protocol deviations occurring during the study, are determined prior to unblinding. The proportion of subjects with relevant protocol deviations through the analysis time point is summarized by treatment arm and overall for the treated subjects.

The list of relevant deviations is provided below:

- Subjects with Screening plasma HIV-1 RNA < 400c/mL
- Subjects with Screening CD4 T-cell count < 50cells/mm<sup>3</sup>
- Subjects with Screening Estimated eGFR < 60mL/min (CKD-EPI formula)
- Subjects resistant to study drugs (unboosted ATV, FC < 2.2; DTG; and TDF) based on Screening genotype/phenotype report(s)
- Subjects who received the wrong study medication
- Subjects who took prohibited concomitant medications, as specified in the protocol, for more than 3 consecutive days.
- Subjects with gaps in study medication dosing greater than 3 consecutive days.

# 7.3 Study Population

# 7.3.1 Subject Disposition

The disposition of subjects will be summarized separately for the pre-randomization period and the on-treatment period.

The pre-randomization status will be summarized for all enrolled subjects. This summary will include the number of subjects enrolled, randomized, not randomized and the reasons for not being randomized.

The end of Week 96 subject status will be summarized by treatment arm and overall for the randomized subjects. This summary will include the number of subjects randomized, completing Week 96 and not completing Week 96. The reasons for not completing Week 96 will also be included.

A separate output will summarize the number of subjects in each population.

Subjects enrolled and randomized will be summarized by country and study site. Enrollment by age group is summarized analogously. Age groups are: in utero; preterm newborn (gestational age < 37 weeks); newborns (0 to 27 days); infants and toddlers (28 days to 23 months); children (2 to 11 years); adolescents (12 to 17 years); adults (18 to 64 years); adults (65 to 84 years); adults ( $\ge 85$  years).

# 7.3.2 Demographics and Other Characteristics

All baseline presentations will identify subjects with missing measurements. In tabulations of categorical variables, percentages are based on subjects with measurements.

# 7.3.2.1 Demographics and Other Baseline Characteristics

Demographic and other baseline characteristics (including disease characteristics) will be summarized by as-randomized treatment arm and overall for the treated subjects. Available demographic characteristics will also be summarized for subjects enrolled but not randomized.

**Table 7.3.2.1-1:** Demographic Characteristics

| Characteristic | Summarized as | Categories |
|---|---|---|
| Gender | Categorical | Male, Female |
| Age | Continuous and Categorical | < 50 , ≥ 50 years |
| Race | Categorical | White, |
| | | Black/African American, |
| | | American Indian/Alaska Native, |
| | | Asian, |
| | | Native Hawaiian/Other Pacific Islander, |
| | | Other |
| Ethnicity (US only) | Categorical | Hispanic/Latino |
| | | Non Hispanic/Latino |
| Geographic Region | Categorical | Europe |
| | | Asia |
| | | Australia |
| | | South America |
| | | North America |
| | | Africa |

 Table 7.3.2.1-2:
 Baseline Disease Characteristics

| Characteristic | Summarized as | Categories |
|---|---|---|
| Plasma HIV-1 RNA | Continuous (log <sub>10</sub> c/mL) and | <30,000c/mL |
| | Categorical | 30,000 to < 100,000c/mL |
| | | 100,000 to < 500,000c/ mL |
| | | ≥ 500,000c/mL |
| CD4+ T-cell count | Continuous and Categorical | <50cells/mm <sup>3</sup> |
| | | 50 to < 100cells/mm <sup>3</sup> |
| | | 100 to $\leq$ 200 cells/mm <sup>3</sup> |
| | | 200 to $\leq$ 350cells/mm <sup>3</sup> |
| | | $350 \text{ to} < 500 \text{cells/mm}^3$ |
| | | $\geq$ 500cells/mm <sup>3</sup> |
| CD4+ T-cell percentage | Continuous | |
| CD8+ T-cell count | Continuous | |
| HIV-1 Subtype | Categorical | |
| IC <sub>50</sub> for BMS-955176 | Continuous | |
| IC50 Fold Change for | Categorical | < 1.0 |
| BMS-955176 | | 1.0 to < 5 |
| | | 5 to < 10 |
| | | 10 to < 100 |
| | | 100 to < 500 |
| | | >= 500 |

**Table 7.3.2.1-3:** Other Baseline Characteristics

| Characteristic | Summarized as | Categories |
|---|---|---|
| Height | Continuous | |
| Weight | Continuous | |
| BMI | Continuous | |
| Hematology: | Categorical | Normal, Grade 1, Grade 2, Grade 3, Grade 4 |
| Hemoglobin, | | |
| Absolute Neutrophil Count(ANC), | | |
| Platelets, | | |
| White Blood Cell Count (WBC) | | |
| Liver Function Tests: | Categorical | Normal, Grade 1, Grade 2, Grade 3, Grade 4 |
| Alanine Aminotransferase (ALT), | | |
| Aspartate Aminotransferase (AST), | | |
| Albumin, serum, low | | |
| Alkaline Phosphatase, | | |
| Total Bilirubin | | |
| Enzymes: | Categorical | Normal, Grade 1, Grade 2, Grade 3, Grade 4 |
| Creatinine Kinase (CK), | | |
| Lipase | | |
| Renal Function Tests: | Categorical | Normal, Grade 1, Grade 2, Grade 3, Grade 4 |
| Creatinine, | _ | |
| Creatinine Clearance (eGFR), | | |
| Uric Acid | | |
| Electrolytes: | Categorical | Normal, Grade 1, Grade 2, Grade 3, Grade 4, |
| Bicarbonate, serum, low | - | |
| Calcium, serum, high | | |
| Calcium, serum, low | | |
| Potassium, serum, high | | |
| Potassium, serum, low | | |
| Sodium, serum, high | | |
| Sodium, serum, low | | |
| Fasting Lipids: | Categorical | Normal, Grade 1, Grade 2, Grade 3, Grade 4 |
| Total Cholesterol, | - | |
| LDL-Cholesterol, | | |
| Triglycerides | | |
| Fasting Glucose: | Categorical | Normal, Grade 1, Grade 2, Grade 3, Grade 4, |
| Glucose, serum, high | <b>5</b> | , |
| Glucose, serum, low | | |

Baseline laboratory values are graded using the DAIDS Toxicity Grades tables as presented in Appendix 3 of the protocol.

Physical examination findings at baseline will be summarized by randomized treatment group and overall.

#### 7.3.2.2 Pre-treatment CDC Class C AIDS Events

Pre-treatment CDC Class C AIDS events (as collected on the AIDS defining events CRF page) will be summarized by as-treated treatment arm and overall for the treated subjects. Pre-treatment events are those with an onset before the start of any study therapy. Documented clinical diagnoses are used to define AIDS (see Protocol Appendix 2).

#### 7.3.2.3 Previous Medication

Previous medications are defined as those medications that are taken before the start of any study therapy. Previous medications will be summarized by as-treated treatment arm and overall for the treated subjects. Medications are presented alphabetically by anatomic class, therapeutic class and generic name. The WHO dictionary is used to code the non-study medication.

### 7.3.2.4 Baseline Resistance

Phenotypic resistance to a drug is defined as a fold change (i.e., ratio of the 50% inhibitory concentration ( $IC_{50}$ ) of the clinical isolate to the  $IC_{50}$  of the reference strain) which is greater than the cut-off for reduced susceptibility.

The number of subjects with phenotypic resistance at baseline will be summarized for all treated subjects, for subjects who had on-study resistance testing done and for treated subjects that are identified as protocol defined virologic failures (see Protocol Section 5.4.1.3) using the following, mutually exclusive categories:

- No resistance to drugs in any class
- ≥ 1 NRTI
- ≥ 1 NNRTI
- ≥ 1 PI
- ≥1 INI
- $\geq 1$  NRTI and  $\geq 1$  NNRTI
- $\geq 1 \text{ NRTI and } \geq 1 \text{ PI}$
- $\geq 1 \text{ NRTI and } \geq 1 \text{ INI}$
- $\geq 1$  NNRTI and  $\geq 1$  PI
- $\geq 1$  NNRTI and  $\geq 1$  INI
- $\geq 1$  PI and  $\geq 1$  INI
- $\geq 1$  NRTI and  $\geq 1$  NNRTI and  $\geq 1$  PI
- $\geq 1$  NRTI and  $\geq 1$  NNRTI and  $\geq 1$  INI

- $\geq 1 \text{ NRTI and } \geq 1 \text{ PI and } \geq 1 \text{ INI}$
- $\geq 1$  NNRTI and  $\geq 1$  PI and  $\geq 1$  INI
- $\geq 1$  NRTI and  $\geq 1$  NNRTI and  $\geq 1$  PI and  $\geq 1$  INI

The number of subjects with phenotypic resistance will also be summarized by class and drug name.

The genotypic resistance profile at baseline will be summarized by treatment arm for all treated subjects, for subjects who had on-study resistance testing done and for treated subjects that are identified as protocol defined virologic failures. Tabulations will present genotypable isolates, those with PI substitutions from genotypable isolates, those with selected RT substitutions from genotypable isolates, and those with integrase substitutions from genotypable isolates using the most current version of the International AIDS Society-USA (IAS-USA) list (see APPENDIX 2). The genotypic resistance profile at baseline will also be summarized by baseline HIV subtype for all treated subjects.

In addition, baseline gag polymorphisms at positions 362, 364, 369 and 370 (relative to the wild type HxB2) will be summarized by treatment arm. This list of positions might be updated. The summary will report single mutations and combinations of mutations. The baseline gag polymorphisms at selected positions will also be summarized by baseline HIV subtype for all treated subjects.

Any deviation from the wild type virus (HxB2) in baseline gag sequencing will be summarized for treated subjects by treatment arm. This summary will also be provided by baseline HIV subtype.

The summaries for gag will be provided for treated subjects, for treated subjects who had onstudy resistance testing done and for treated subjects that are identified as protocol defined virologic failures.

## 7.4 Extent of Exposure

Extent of exposure is presented for treated subjects by as-treated treatment arm.

## 7.4.1 Study Therapy

Time (in days) on study therapy will be summarized by treatment arm. Time on study therapy is defined as the difference between the earliest last dose date of any component of the treatment arm and the first dose date of study treatment plus 1 day.

Time on study therapy and average daily dose will be summarized for each individual drug component by treatment arm. Time on an individual drug component is defined as the number of days between the first dose date and the last dose date of the drug. The average daily dose is the total amount of drug in grams divided by the number of days between the first dose date and the last dose date of the drug.

The time on BMS-955176 and average daily dose after the switch to the continuation dose will be summarized for subjects who switched to the continuation dose after Week 24, rather than starting on the continuation dose at the time of randomization. Time on BMS-955176 continuation dose is defined as the difference between the last dose date of continuation dosing and the first dose date of continuation dosing plus 1 day.

# 7.4.2 Discontinuation of Study Therapy

Time (in days) on any study therapy will be described by a Kaplan-Meier curve and life table with the Kaplan-Meier estimates.

Discontinuations from study therapy are considered events in this analysis. For subjects who have not discontinued, time on study therapy is censored at the last recorded dose stop date of any study therapy. For the purpose of this analysis, we will consider the start date and event/censor date regardless of any interruptions.

# 7.4.3 Interruption or Delay of Study Therapy

Interruptions of study therapy greater than 3 consecutive days will be summarized by treatment arm and for each drug in the regimen. Interruptions are identified from complete dosing records in which either the number of units per day or the number of doses per day is zero.

# 7.4.4 Concomitant Therapy

Concomitant medications are defined as those taken at any time on or after the start date of study therapy and before or on the last dose date of study therapy. Concomitant medications will be summarized by treatment arm and overall for the treated subjects. Medications are presented alphabetically by anatomic class, therapeutic class and generic name. The WHO dictionary is used to code the non-study medication.

## 7.5 Efficacy

Efficacy endpoints are evaluated for treated subjects by as-randomized treatment arm during the treatment period through a specific analysis week. Measurements obtained on treatment and before or on the analysis week date (see Section 8.2) will be included.

# 7.5.1 Primary Efficacy Endpoint: Proportion of Subjects with Plasma HIV-1 RNA < 40c/mL at the Week 24 Snapshot

The primary efficacy endpoint is the proportion of subjects with plasma HIV-1 RNA < 40c/mL at the Week 24 snapshot. The primary analysis will be based on a modified ITT (mITT) approach. A sensitivity analysis will be conducted using an observed values approach. The two approaches will be implemented as follows:

• Modified ITT: The numerator will be based on subjects with plasma HIV-1 RNA < 40c/mL at Week 24. The denominator will be based on all treated subjects.

• Observed values: Similar to the mITT approach, the numerator will be based on subjects with plasma HIV-1 RNA < 40c/mL at Week 24. However, the denominator will be based on treated subjects with plasma HIV-1 RNA at Week 24.

Response rates will be tabulated by treatment arm with exact (Clopper-Pearson) binomial 95% confidence intervals.

This endpoint is assessed with the snapshot algorithm. The snapshot algorithm is described in detail in Appendix 1 of the CDER (2013) draft guidance<sup>1</sup> on developing antiretroviral drugs (see also APPENDIX 1 of this SAP). If the draft guidance is superseded, and development timelines permit any needed changes, the instructions from the new guidance should be followed.

The main principle of the snapshot analysis is that the primary efficacy endpoint is intended to be primarily a virologic endpoint and not a clinical endpoint. The snapshot algorithm follows a "Virology First" hierarchy. The hierarchy for assessing percentages is "HIV-1 RNA < Limit of Detection" or "HIV-1 RNA ≥ Limit of Detection" first for any given time window followed by reasons for "No Virologic Data in the Window".

The snapshot approach algorithm is based on the event occurring within a visit window which is outlined in Section 8.1.

#### Optimized Background Therapy (OBT) Substitutions

Changes in background therapy are not allowed per protocol. Subjects who do change their dose for TDF in the event of treatment-limiting renal toxicity will be considered virologic failure if they have HIV-1 RNA > 40 at the time of the change.

Movement of a subject to the continuation dose of BMS-955176 will not be a cause for classifying a subject as a virologic failure.

The snapshot analysis must include a table that is of the same format shown in Table B (line 1209) of the draft guidance. A more detailed presentation that breaks down the FDA categories into finer detail, may also be provided. The snapshot analysis will be accompanied by a detailed listing that facilitates finding the patients in each category described in the table.

The snapshot analysis is supplemented by a Time to Loss of Virologic Response (TLOVR) analysis at Weeks 24. Analyses are presented for the randomized treatment groups both separately and combined. TLOVR analyses are described in APPENDIX 3.

# 7.5.1.1 Summaries of Primary Efficacy Endpoint Within Subgroups

The primary efficacy endpoint will be summarized within the following subgroups using the mITT and the observed values approach:

- Baseline viral load:  $< 100,000 \text{c/mL}, \ge 100,000 \text{c/mL}$
- Baseline CD4 category:  $< 100 \text{cells/mm}^3$ ,  $100 \text{ to} < 200 \text{cells/mm}^3$ ,  $200 \text{ to} < 350 \text{cells/mm}^3$ ,  $350 \text{ to} < 500 \text{cells/mm}^3$ ,  $\ge 500 \text{cells/mm}^3$
- Gender

- Race
- HIV-1 clade

## 7.5.2 Secondary Efficacy Endpoints

# 7.5.2.1 Proportion of Subjects with Plasma HIV-1 RNA < 40c/mL at Weeks 48 and 96

The proportion of subjects with HIV1 RNA < 40c/mL at Weeks 48 and 96 will be assessed analogously to the primary efficacy endpoint using the snapshot algorithm. Summaries within subgroups identified for the primary analysis will be provided for Week 48 and 96 using the mITT and the observed values approach. Also a time to loss of virologic response analysis will be done.

# 7.5.2.2 Proportion of Subjects with Plasma HIV-1 RNA < 200c/mL at the Week 24, 48 and 96 Snapshot

The proportion of subjects with plasma HIV-1 RNA < 200c/mL at Week 24, 48 and 96 will be summarized using mITT and the observed values approach, analogously to the primary efficacy endpoint using the snapshot algorithm. No summaries within subgroups will be provided.

## 7.5.2.3 Change from Baseline in Plasma HIV-1 RNA (log<sub>10</sub>) over Time

The change from baseline in plasma HIV-1 RNA (log<sub>10</sub>) will be summarized over time for the treated subjects using observed values. The mean changes from baseline will be plotted at each scheduled visit (except Week 2) through Week 96 by treatment arm, with error bars representing 1 standard error. The change from baseline in plasma HIV-1 RNA (log<sub>10</sub>) at Week 24, 48 and 96 will be presented graphically using box plots. The change from baseline will also be provided for the subgroups identified for the primary analysis.

# 7.5.2.4 Changes from Baseline in CD4+ and CD8+ T-cell Count over Time

CD4+ and CD8+ T-cell counts and changes from baseline will be summarized at each scheduled visit through Week 96 by treatment arm using observed values. The mean changes from baseline will be plotted at each scheduled visit through Week 96 by treatment arm, with error bars representing 1 standard error. The change from baseline in CD4+ and CD8/ T-cell counts at Week 24, 48 and 96 will be presented graphically using box plots. Also the percentage of CD4+ T-cells and changes from baseline will be summarized at each scheduled visit through Week 96. The change from baseline will also be provided for the subgroups identified for the primary analysis.

# 7.5.2.5 Newly-emergent Genotypic Substitutions, IC<sub>50</sub> Fold Changes from Baseline and Newly-emergent Gag Polymorphisms

Viral resistance is measured using the "PhenoSense GT plus Integrase" assay from Monogram (LabCorp). The PhenoSense GT plus Integrase is used to determine both genotypic and phenotypic resistance to Nucleoside Reverse Transcriptase Inhibitors (NRTIs), Non-Nucleoside Reverse Transcriptase Inhibitors (NNRTIs), Integrase Inhibitors (INIs), and Protease Inhibitors (PIs). The "PhenoSense Gag" assay is used for determining phenotypic susceptibility to BMS-955176. HIV-1 Gag sequencing data will be obtained from the NGS-Gag Quantitative Sequencing (QS) assay.

Genotypic substitutions and phenotypic resistance profiles focus on subjects with on-treatment isolates.

Newly emergent phenotypic resistance to a drug is defined as a baseline fold change  $\leq$  the cut-off for reduced susceptibility and an on-treatment fold change > the cut-off for reduced susceptibility. The newly emergent phenotypic resistance profile (using all on-treatment isolates) will be tabulated by treatment arm for treated subjects with on-treatment resistance testing done.

Newly emergent phenotypic resistance to BMS-955176 is defined as a baseline fold change IC50  $\leq$  3 and an on-treatment fold change IC50 > 3. The newly emergent phenotypic resistance to BMS-955176 (using all on-treatment isolates) will be tabulated by treatment arm for treated subjects with on-treatment resistance testing done.

Newly emergent genotypic substitutions (using all on-treatment isolates) are tabulated by treatment arm for treated subjects with on-treatment resistance testing done. The presentation will be similar to the one for baseline genotypic substitutions.

The maximum change from baseline in BMS-955176 IC $_{50}$  and the maximum BMS-955176 fold change IC $_{50}$  (FC-IC50) through Week 96 will be summarized for all treated subjects with ontreatment phenotypic resistance profile. In addition, the proportion of subjects with a > 3 fold increase from baseline in BMS-955176 FC-IC50 (i.e., BMS-955176 FC-IC50 on-treatment divided by BMS-955176 FC-IC50 at baseline > 3) will be summarized. The Gag polymorphisms will be summarized for subjects with a > 3 fold increase from baseline in BMS-955176 FC-IC50. These summaries will use all of the data present in the database at the time of lock.

Newly emergent Gag polymorphisms at the selected positions will be summarized by treatment arm for treated subjects with on-treatment resistance testing done, overall and by baseline HIV subtype. In addition, any newly emergent Gag deviation will be summarized for treated subjects with on-treatment resistance testing done, overall and by baseline HIV subtype.

All summaries described in this section will also be provided for treated subjects that are identified as protocol defined virologic failures.

Protocol Defined Virologic Failure (PDVF) is defined by a subject meeting one of the following criteria (see Protocol, Section 5.4.1.2):

- Confirmed > 1 log10c/mL increase in HIV-1 RNA at any time above nadir level where nadir is ≥ 40c/mL
- Confirmed HIV-1 RNA ≥ 400c/mL after Week 24
- Confirmed HIV-1 RNA  $\geq 40 \text{c/mL}$  if prior suppression to < 40 c/mL
- Failure to have the last on-treatment HIV-1 RNA to < 400c/mL within Week 24, 48, or 96 week snapshot window
- Failure to achieve > 1 log10c/mL decrease in HIV-1 RNA by Week 8

# 7.5.3 Exploratory Efficacy Endpoints

# 7.5.3.1 Proportion of Subjects with Plasma HIV-1 RNA within Certain Range over Time

The proportion of subjects with HIV-1 RNA:

- < 40c/mL
- 40 to < 100 c/mL
- 100 to < 200 c/mL
- 200 to < 400 c/mL
- > 400 c/mL

will be presented by visit using the observed values approach.

### 7.5.3.2 Efficacy Summaries by Baseline Gag Polymorphisms

To assess the impact of baseline gag polymorphisms the following efficacy endpoints will be summarized by all combinations of baseline gag polymorphisms at selected positions:

- Proportion of subjects with plasma HIV-1 RNA < 40c/mL at Weeks 24, 48 and 96
- Proportion of subjects with plasma HIV-1 RNA < 200c/mL at Weeks 24, 48 and 96
- Change from baseline in log<sub>10</sub> HIV-1 RNA at Weeks 4, 8, 12, 24, 48 and 96

## 7.5.4 Futility Analysis

An analysis of virologic futility will be performed at Week 24 when the last randomized subject in Stage 1 completes the Week 24 visit. This analysis will be conducted to evaluate whether the BMS-955176 arm shows significantly worse antiviral efficacy than the TDF arm. The proportion of subjects with HIV-1 RNA < 40c/mL at Week 24 will be evaluated using the FDA snapshot algorithm. The comparison of the BMS-955176 arm to the TDF arm will be made with one-sided Fisher's exacts test, conducted at the 0.01 probability level.

An analysis of virologic futility will also be performed at Week 24 when the last randomized subject in Stage 2 completes the Week 24 visit. This analysis will be conducted to evaluate

whether the BMS-955176 arms show significantly worse antiviral efficacy than the TDF arm in Stage 2. The proportion of subjects with HIV-1 RNA < 40c/mL at Week 24 will be evaluated using the snapshot algorithm. The comparisons of Arms 3 and 4 (BMS-955176) to Arm 5 (TDF) will each be made with a one-sided, Fisher's exact test, conducted at the 0.01 probability level.

# 7.6 Safety

Safety endpoints include the frequency of adverse events (AEs), serious adverse events (SAEs), non-serious adverse events, CDC Class C AIDS events, adverse events leading to discontinuations, deaths and other significant adverse events as reported on case report forms. Other safety endpoints include laboratory abnormalities, changes in laboratory parameters, changes in vital signs and physical measurements, and ECGs. Safety endpoints will not be evaluated through a specific analysis week. All safety data available in the database at the time of the lock will be included.

Safety summaries are provided for treated subjects by as-treated treatment arm, unless otherwise specified.

#### 7.6.1 Overall Adverse Events

Adverse events will be classified by primary System Organ Class (SOC) and Preferred Term (PT) according to the latest version of the Medical Dictionary for Regulatory Activities (MedDRA) in production at BMS at the time of database lock.

AEs and SAEs with an onset on or after the start of study therapy through 30 days after the last dose of study therapy will be considered as occurring during study therapy. These will be summarized and presented by SOC and PT both in descending order of frequency over all treatment arms, unless otherwise specified.

**Table 7.6.1-1:** Adverse Event Summaries

| Endpoint | <b>During Study Therapy</b> | During Study Therapy, after<br>Switch to Continuation Dose |
|---|---|---|
| SAEs | X | X |
| SAEs leading to death <sup>a</sup> | X | |
| SAEs related to study therapy and leading to death <sup>a</sup> | X | |
| Non-SAEs $\geq$ 5% <sup>a</sup> | X | |
| AEs leading to discontinuation of study therapy | X | X |
| AEs - All Grades | X | |
| AEs - Grade 2 to 4 | X | |
| AEs- Grade 3 to 4 | X | |

**Table 7.6.1-1:** Adverse Event Summaries

| Endpoint | During Study Therapy | During Study Therapy, after<br>Switch to Continuation Dose |
|---|---|---|
| Related AEs - All Grades | X | |
| Related AEs - Grade 2 to 4 | X | |
| Related AEs - Grade 3 to 4 | X | |
| CDC Class C AIDS Events | X | |
| Events of Special Interest | X | |
| Exposure-adjusted Events ≥ 5% | X | |
| Exposure-adjusted SAEs <sup>a</sup> | X | |
| Exposure-adjusted SAEs related to study therapy <sup>a</sup> | X | |
| Exposure-adjusted non-SAEs $\geq 5\%$ <sup>a</sup> | X | |

ClinicalTrials.gov or EudraCT reporting requirement

#### 7.6.2 Deaths

All deaths recorded on the status page, the AE page or SAE page of the CRF will be considered in the analyses. A listing of all deaths that occur will be produced for the enrolled subjects.

#### 7.6.3 Serious Adverse Events

SAEs occurring during study therapy will be summarized by SOC and PT. SAEs leading to death and SAEs related to study therapy and leading to death will be summarized in a similar way.

A listing of all SAEs will be produced, displaying all SAEs (including pre-treatment events) for enrolled subjects.

# 7.6.4 Serious Adverse Events Emerging After Switch to Continuation Therapy

For subjects who switched to a continuation dose after Week 24, rather than starting on a continuation dose at the time of randomization, SAEs with an onset after the start date of continuation therapy through 30 days after the last dose of study therapy, will be summarized by SOC and PT.

#### 7.6.5 Non-Serious Adverse Events

Non-serious adverse events occurring in at least 5% of the subjects treated will be summarized by SOC and PT.

# 7.6.6 Adverse Events Leading to Discontinuation of Therapy

Adverse events leading to discontinuation will be summarized by SOC and PT.

# 7.6.7 Adverse Events Leading to Discontinuation of Therapy After Switch to Continuation Therapy

For subjects who switched to a continuation dose after Week 24, rather than starting on a continuation dose at the time of randomization, AEs leading to discontinuation with an onset after the start date of continuation therapy will be summarized by SOC and PT.

## 7.6.8 Adverse Events by Relationship

Drug-related adverse events are those with 'related' or missing relationship to study drug. Drug-related adverse events will be summarized by SOC and PT.

## 7.6.9 Adverse Events by Intensity

Adverse events and drug-related adverse events with the following grades:

- all Grades,
- Grade 2 to Grade 4,
- Grade 3 to Grade 4,

will be summarized by SOC and PT.

Adverse events with missing intensity are included only in the summaries for all grades. If a subject has an adverse event with different intensities over time, then only the greatest intensity will be presented.

#### 7.6.10 CDC Class C AIDS Events

CDC Class C AIDS events will be summarized and presented by SOC and PT.

#### 7.6.11 Adverse Events of Special Interest

Separate summaries will be provided for the following events of special interest: gastrointestinal events. The list of events will be identified before database lock. The definition of gastrointestinal events will be based on existing Standardized MedDRA Queries (SMQs) if existing SMQs support the events of special interest requirements. If needed, a customized SMQ (cSMQ) will be developed. Gastrointestinal events will be summarized by SOC and PT.

## 7.6.12 Multiple Adverse Events

Several descriptive summaries of adverse events that take into account the number of occurrences that an AE was reported by individual subjects will be provided. In order to prepare these summaries, the CRF data will be processed according to standard BMS algorithms to categorize each line of subject data as a new occurrence or a continuation of an existing event.

This determination will be based upon onset and resolution dates. Each line of subject data will represent the maximum severity observed as well as the last known assessed relationship to study medication by the investigator.

This data will be presented as the rate per 100 years of patient exposure. Exposure to study medication will be calculated according to approved standard BMS algorithms as well.

As an example, if 5 subjects report 7 unique episodes of headache and had a combined cumulative exposure of 20 years to study medication, the incidence rate is reported as 7 / 20 \* 100 or 35 cases per 100 patient years of exposure.

For adverse events with multiple occurrences, the following will be provided:

- A table showing the total number and rate (exposure adjusted) of occurrences for general AEs occurring in at least 5% of the subjects treated.
- A listing displaying the unique instances of all AEs (i.e., after duplicates have been eliminated and overlapping and contiguous occurrences of the same event have been collapsed).

Exposure-adjusted summaries will also be provided for SAEs, SAEs related to study therapy and non-SAEs.

## 7.6.13 Clinical Laboratory Evaluations

Laboratory parameters will be presented using SI and US values and units.

## 7.6.13.1 Laboratory Abnormalities

The incidence of laboratory abnormalities presenting the worst toxicity grade during the treatment period will be tabulated by treatment arm for all grades (Grades 1, 2, 3, 4) and Grades 3 and 4.

Subjects with at least 1 measurement after the start of study therapy will be included in the summaries. Abnormalities are determined from laboratory measurements analyzed at the central or local laboratory. Grading categories for laboratory tests are determined using the DAIDS grading system (see Appendix 3 of the protocol).

This incidence will be further summarized by baseline toxicity grade.

Treatment emergent abnormalities by toxicity grade (increased to Grades 1, 2, 3, 4, and any grade) will also be summarized by baseline toxicity grade (normal, Grade 1 to 4, not reported) and total analogously. Treatment emergent abnormalities are those with a higher on-treatment toxicity grade than the baseline toxicity grade (including not reported baseline).

## 7.6.13.2 Laboratory Tests over Time

All summaries of laboratory data over time will use observed values. Visit windows are defined in Section 8.

Observed values and changes from baseline in creatinine and creatinine clearance will be summarized at each scheduled visit by treatment arm.

Observed values, changes from baseline and percent changes from baseline will be summarized over time for the following laboratory tests:

- Fasting Total cholesterol,
- Fasting HDL-cholesterol
- Fasting LDL-cholesterol,
- Fasting Triglycerides.
- Total:HDL cholesterol ratio

Values obtained after the start of serum lipid-reducing agents will be excluded from these lipid summaries. Mean percent changes from baseline using observed values will be plotted at each scheduled visit with error bars representing 1 standard error of the reported statistic.

## 7.6.14 Electrocardiograms

QRS, PR and QTc Fridericia intervals and changes from baseline will be summarized over time by treatment arm using observed values. Standard 95% confidence intervals for mean changes from baseline will also be provided.

The subject's longest interval observed during the treatment period for these ECG parameters will be summarized categorically by treatment arm using the following categories:

- QRS interval:  $< 100, 100 \text{ to} < 110, 110 \text{ to} < 120, 120 \text{ to} < 130, 130 \text{ to} < 140, <math>\ge 140 \text{msec}$ ;
- PR interval: < 200, 200 to < 220, 220 to < 240, 240 to < 260, 260 to < 280, 280 to < 300, ≥ 300msec;
- QTcF interval: < 400, 400 to < 425, 425 to < 450, 450 to < 460, 460 to < 470, 470 to < 480, 480 to < 490,  $\ge 490$ msec.

The largest change from baseline in these intervals observed during the treatment period is also summarized categorically by treatment arm using the following categories:

- $\triangle QRS$ : < 0, 0 to < 10, 10 to < 20, 20 to < 30, 30 to < 40,  $\ge$  40msec;
- $\Delta PR$ : < 0, 0 to < 20, 20 to < 40, 40 to < 60, 60 to < 80,  $\geq$  80msec;
- $\triangle QTcF$ : < 0, 0 to < 10, 10 to < 20, 20 to < 30, 30 to < 40,  $\geq$  40msec.

#### 7.6.15 Vital Signs

All summaries of vital signs over time will use observed values. Visit windows are defined in Section 8. Observed values and changes from baseline will be summarized over time. For blood pressure and heart rate, only sitting assessments will be included in the summaries.

Observed values and changes from baseline for body weight and BMI will be summarized over time.

#### 7.7 Clinical Biomarker Assessments

Renal and bone biomarkers values, changes from baseline and percent changes from baseline will be summarized over time using observed values. Visit windows are defined in Section 8.

The renal biomarkers include urinary beta-2-microglobulin/creatinine and fractional excretion of phosphorous (FeP), defined as

• 100 \* [(urine phos x serum creatinine) / (serum phos x urine creatinine)]

The bone biomarkers include: N-terminal Propertide of Type 1 procollagen (P1NP) and Cross-linked C-telopeptide of Type 1 collagen (CTx).

The median change from baseline in FeP over time will be plotted with error bars representing IQR. The median percent change from baseline in P1NP, CTx and urinary beta-2-microglobulin/creatinine over time will be plotted in a similar way.

# 7.8 Integrated Summaries

For the final analysis (i.e., when the last subject in Stage 2 completed the Week 96 visit), a number of integrated summaries will be provided. These outputs will include 4 columns: one for each of the treatment arms 1, 3 and 4 and one for the TDF containing arms (arms 2 and 5) combined.

The following information will be summarized:

- Week 96 subject status (see Section 7.3.1)
- Demography and baseline disease characteristics (see Section 7.3.2.1)
- Baseline resistance (see Section 7.3.2.4):
  - The number of treated subjects with phenotypic resistance using the earlier mentioned mutually exclusive categories, and by class and drug name.
  - The genotypic resistance profile for all treated subjects.
  - The baseline gag polymorphisms at selected positions.
- Time on study therapy (see Section 7.4.1)
- Newly emergent resistance for treated subjects with on-treatment resistance testing done (see Section 7.5.2.5):
  - Newly emergent phenotypic resistance profile
  - Newly emergent phenotypic resistance to BMS-955176
  - Newly emergent genotypic substitutions
  - Newly emergent Gag polymorphisms at the selected positions
  - Any newly emergent deviation from the wild type virus in Gag sequencing
- Safety (see Section 7.6):
  - Overall AE summary
  - SAEs

- AEs leading to discontinuation
- Grade 2-4 related AEs
- Grade 3-4 AEs
- CDC Class C events
- Gastrointestinal events
- Grade 3-4 laboratory toxicities

#### 7.9 Outcomes Research

#### 7.9.1 EQ-5D-3L

As described in the SAP for BMS study CN162-007, the EuroQol (EQ-5D-3L) provides a simple but effective standardized measure of a subject's quality of life and health state classification<sup>2</sup>. It is intended to provide both a compact descriptive profile and a single index value that will be used in the clinical and economic evaluation of health care. The questionnaire consists of 2 parts, which together are used to build a composite picture of the respondent's health status.

In the first part, the "health state classification", the respondent is asked to indicate his/her current health state, by ticking the most appropriate of three statements about each of the 5 quality of life dimensions: mobility, self-care, usual activity, pain/discomfort, and anxiety/depression. Each of the 3 statements represents an increasing level of severity (1 = no problem, 2 = some or moderate problems, 3 = unable, or extreme problems). The string of five numbers, one for each dimension, indicates the aggregate health state. For example: "11111" indicates perfect health and "33333" indicates the worst health state.

The second part, "Visual Analogue Scale Thermometer", evaluates the respondent's current health-related quality of life by means of a 20cm visual analogue scale (VAS) with endpoints at 100 (best imaginable health state) and 0 (worst imaginable health state).

The scores obtained from the 5 health state dimensions (first part of the questionnaire) will be converted to a US centric utility score based on the algorithm described by Shaw et al<sup>3</sup>. This utility score has range score from -0.019 (worse health state) to a maximum of 1.000 (best health state). APPENDIX 4 contains SAS code for calculating the US centric EQ-5D-3L utility score.

The scores obtained from the 5 health state dimensions will also be converted to a UK centric utility score based on the algorithm described by Dolan<sup>4</sup>. APPENDIX 5 contains SAS code for calculating the UK utility scores.

For both the US centric and UK centric utility scores, values and changes from baseline are summarized as continuous parameters at baseline and all applicable, on-treatment analysis visits. Subjects must have paired measurements at baseline and the analysis visit to be evaluable.

#### 7.9.2 FAHI

The FAHI consists of 5 subscales: Physical Well-Being, Emotional Well-Being, Function and Global Well-Being, Social Well-Being, and Cognitive functioning. Each scale consists of a number of questions, each of which has 5 possible responses: 0, 1, 2, 3 and 4.

A detailed description of the FAHI structure and scoring algorithm is contained in internal BMS document, "FAHI Source Doc (16-DEC-2014).PDF", which is available upon request. A summary of the scoring algorithm is provided below.

Negatively stated items are reversed by subtracting the response from 4. After reversing proper items, all subscale items are summed to a total which is the subscale score. Higher scores indicate better the quality of life. The score for each scale is the prorated sum of the items answered. Thus, if a scale has 10 items, and only 6 are answered, the results of the six questions answered are summed and multiplied by 10. The result is then divided by 6.

- The Physical Well-Being section of the questionnaire contains 13 questions, however only 10 of them are used in scoring the scale. These are questions GP1-GP7, BMT6, HI7 and HI12. Before computing the score for this scale, all of the responses are reversed by subtracting the response from 4.
- The Emotional Well-Being scale consists of 10 items. Before computing the score for this scale, all of the responses are reversed by subtracting the response from 4.
- The Function and Global Well-Being scale consists of 13 items. Only one item, GE3, is reversed before the scale is scored.
- The Social Well-Being scale consists of 8 items. None of these items are reversed before the scale is scored.
- The Cognitive Functioning scale consists of three items. Two of these items, HI8 and HI9, are reversed before the scale is scored.

The scoring of any of the FAHI sub-scales is only considered valid as long as more than 50% of the subscale questions have been answered.

The total score for the FAHI is the sum of prorated scores from each of the five subscales. The overall score for the FAHI is considered valid if all of the subscales are considered to be valid.

The analysis data set includes the overall score and each of the subscale scores by visit for each subject as well as indicator variables that show if the validity condition has been met for each of the subscales, as well as the FAHI overall. Calculations for the FAHI total score and subscale scores use only valid data.

FAHI total scores are summarized as continuous parameters at baseline and all applicable ontreatment analysis visits.

#### 7.10 Pharmacokinetics

The following intensive PK parameters will be summarized (using mean, SD, median, minimum, maximum, geometric mean and %CV) for BMS-955176, DTG and ATV by treatment arm:

- C<sub>max</sub>: maximum observed plasma concentration
- T<sub>max</sub>: time of maximum observed plasma concentration
- C<sub>tau</sub>: observed plasma concentration at the end of a dosing interval
- C<sub>0</sub>: observed pre-dose plasma concentration
- AUC(TAU) area under the concentration-time curve in one dosing interval

The Pharmacokinetic (PK) population will be used for all listings. Evaluable PK population will be used for summary statistics and statistical analyses.

Subject plasma concentration-time profiles will be listed and summarized by treatment arm and nominal collection time for each analyte. Plots of individual plasma concentration profiles over time will be provided. Overlay of individual plasma concentration profiles over time will be provided by treatment arm. Plots of mean (+SD) plasma concentration profiles versus time will be presented for each analyte, and all treatments will be superimposed on the same plot for the analyte.

All individual PK parameters will be listed for each analyte including any exclusions and reasons for exclusion from summaries. Summary statistics will be tabulated for each PK parameter by treatment arm. Geometric means and coefficients of variation will be presented for Cmax, AUC(TAU),  $C_{tau}$ , and  $C_0$ . Medians and ranges will be presented for Tmax.

The effect of BMS-955176 on the exposure of DTG (in the presence of ATV/RTV 300/100mg) will be estimated by the geometric mean ratio, with 90% confidence interval, of the exposure data in Arm 1 over the reference ATV/r arm (Arm 2). These estimates will be generated using general linear models fitted to log-transformed data. The effect of BMS-955176 on the exposure of DTG (in the presence of ATV 400mg) will be estimated by the geometric mean ratio, with 90% confidence intervals, of the exposure data in Arm 3 and Arm 4, separately, over historical data. These estimates will be generated using general linear models fitted to log-transformed data.

The population PK, exposure-response and viral kinetic analyses will be described in a separate analysis plan. Intensive and sparse pharmacokinetic data will be used in population PK, PK/PD and PK/VK.

#### 8 CONVENTIONS

# 8.1 Derivation of Baseline and On-Treatment Parameters Using Visit Windows

## 8.1.1 Baseline

Baseline parameters are derived from pre-treatment measurements. Pre-treatment measurements are included for subjects in the following ways:

- For treated subjects: measurements are included through the start of study therapy.
- For randomized subjects who never received study therapy: measurements are included through randomization.
- For enrolled subjects who were never randomized: all available measurements are included.

The following algorithm details the derivation of baseline parameters:

- CD4+ and CD8+ T-cells: the last value on or before the start of study therapy. If there are multiple measurements on the same day from central and local laboratories, then the value from the central laboratory is selected.
- Genotypic and phenotypic parameters: identified from the last typable resistance test on or before the start of study therapy. HIV subtype is identified from the first resistance test at which subtype was assessed. If there are multiple tests on the same day, the last test run is chosen.
- All other parameters: the last value measured on or before the start of study therapy is selected. If there are multiple measurements on the same day, the value with the latest entry date/time is chosen:
  - HIV-1 RNA: Values are assigned a value of 1 more (or 1 less) if an inequality ">" ("<") is present. Values outside the upper (or lower) limit of quantification are assigned a value or 1 more (or 1 less) than the limit. Only values from the central laboratory will be used.

#### 8.1.2 On-Treatment Parameters

Time is measured from the first dose of study therapy.

On-treatment parameters are derived from measurements after the start of study therapy through the last dose of study therapy plus 4 days for efficacy, biomarkers and outcomes research scales, plus 10 days for resistance parameters and plus 30 days for safety.

For the primary and secondary efficacy endpoints of proportion of subjects with plasma HIV-1 RNA < 40c/mL at Weeks 24, 48 and 96, the snapshot algorithm and related window definition will be applied. The snapshot windows shown in the Table 8.1.2-1 below differ from those proposed by the FDA by 1 day. The FDA windowing appears to have the first study day as Day 0, while the table below has the first study day as Day 1.

The windows for other parameters are based on the midpoint between planned study visits. For analysis through Week 96, the visit windows are presented in the following table:

Table 8.1.2-1: Visit Windows

| Visit | Target Day | HIV-1 RNA (Snapshot<br>Algorithm) | Other Parameters |
|-------|------------|-----------------------------------|------------------|
| B/L | 1 | | ≤1 |
| 2 | 15 | | 2 - 21 |
| 4 | 29 | | 22 - 43 |
| 8 | 57 | | 44 - 71 |
| 12 | 85 | | 72 - 99 |
| 16 | 113 | | 100 - 141 |
| 24 | 169 | 127 - 210<br>(18-30 wks) | 142 - 197 |
| 32 | 225 | | 198 - 253 |
| 40 | 281 | | 254 - 309 |
| 48 | 337 | 295 - 378<br>(42-54 wks) | 310 - 379 |
| 60 | 421 | | 380 - 463 |
| 72 | 505 | | 464 - 547 |
| 84 | 589 | | 548 - 631 |
| 96 | 673 | 631-714<br>(90-102 wks) | 632 - 715 |

#### Study days are calculated as:

- Measurement date first date of study therapy + 1 day, if measurement date if on or after start date of study therapy.
- Measurement date first date of study therapy, if measurement date is before start date of study therapy.

Weeks are study days divided by 7.

The following conventions are used to select the value to be used in the analysis:

• HIV-1 RNA: analysis of the proportion of subjects with plasma HIV-1 RNA < 40c/mL at Week 24, 48 and 96 use the last plasma HIV-1 RNA value in the pre-defined visit window following the snapshot algorithm. For all other analyses or summaries of HIV-1 RNA, the value in the visit window that is closest to the target day of the planned visit (as determined by the absolute differences in days between the planned visit and the assessment date) will be used. In case of ties between observations located on different sides of the target day, the earlier assessment will be used. In case of ties located on the same side of the target day
(i.e., more than one value for the same day but different time), the value with the earlier entry date/time will be used. Only values from the central laboratory will be used.

- Values are assigned a value of 1 more (or 1 less) if an inequality ">" (or "<") is present.</li>
   Values outside the upper (or lower) limit of quantification are assigned a value of 1 more (or 1 less) than the limit.
- For other laboratory and non-laboratory parameters: if a subject has more than one measurement included within a window, the assessment closest to the target day will be used. In case of ties between observations located on different sides of the target day, the earlier assessment will be used. In case of ties located on the same side of the target day (i.e., more than one value for the same day but different time), the value with the earlier entry date/time will be used.

#### 8.2 Derived Dates

- Start date of any study therapy is the earliest start date of BMS-955176, TDF, ATV, RTV or DTG identified from dosing records with non-missing start date. This date is used to identify treated subjects and to distinguish pre-treatment from any on-study measurements.
- Start date of continuation dosing of study therapy for BMS-955176 is the earliest start date of the continuation dose(s) of BMS-955176 with non-missing daily dose and non-missing start date. This date is used to identify treated subjects receiving the continuation dose(s) of BMS-955176 and to distinguish on-study measurements in the original dosing period from on-study measurements in the continuation dosing period.
- Start date of serum lipid-reducing agents is the earliest start date of any concomitant or post-treatment medication from the therapeutic class 'serumlipidreducing agent'. This date is used to exclude data in longitudinal lipid analyses during treatment.
- <u>Analysis week date</u> is the start date of study therapy plus the upperbound of the window defining the analysis week minus 1 day (see <u>Section 8.1</u>). This date is used to include data through the analysis week.

#### 8.3 Derived Parameters

When deriving a parameter that requires more than one test measurement, the parameter must be derived using measurements from the same collection date, accession number and site code for each test.

# 8.4 Study Therapy

Time on therapy for each individual drug component is calculated from the first and last dates of dosing, regardless the interruptions. The first date of dosing is the minimum of the dosing start dates, and the last date of dosing is the maximum of dosing stop dates.

#### 8.5 Concomitant Medications

Start and stop date of all concomitant medications are collected on the CRF. In order to classify medication as prior, current or concomitant, partial, missing or invalid start and stop dates will be imputed where possible as follows:

- If the reported start date is missing or invalid and the informed consent date is not missing or invalid, then the imputed start date is set equal to the informed consent date. If the consent date is missing or invalid and the birth date is not missing or invalid, then the imputed start date is set equal to the birth date. If the start date, the consent date and the birth date are all invalid or missing, then the imputed start date is set equal to missing.
- If the reported start date is partially entered, then the imputed start date is set equal to the earliest possible reported start date based on the partial entered reported start date.
- If the reported end date is missing, continuing, unknown or invalid, then the imputed end date is set equal to the most recent database extraction date.
- If the reported end date of the medication is partial, then the imputed end date is set equal to the last possible reported end date based on the partial entered reported end date.

Imputed dates will not appear on the listings of non-study medication.

# 8.6 Counting Rules for Adverse Events

Where a subject has the same adverse event, based on preferred term, reported multiple times in a single analysis period, the subject will only be counted once at the preferred term level in adverse event frequency tables.

Where a subject has multiple adverse events within the same system organ class in a single analysis period, the subject will only be counted once at the system organ class level in adverse event frequency tables.

When a subject has the same adverse event, based on preferred term, reported multiple times in a single analysis period, the following criteria, in order of precedence, will be used to select the event to be included in the summary tables:

- Relationship to study medication: related events will take precedence over unrelated events.
- Intensity of the event: more intense events will take precedence over less intense events.
- Onset date and time: earlier onset date/time events will take precedence over late onset date/time events.

When reporting adverse events by intensity, summary tables will also be provided based on the most intense event during the analysis period - independent of relationship to study medication. For these tables, the following criteria, in order of precedence, will be used to select the event to be included in the summary tables:

- Intensity of the event
- Onset date and time

#### 8.7 Pharmacokinetic Evaluations

## 8.7.1 Decimal Places for Pharmacokinetic Data

The number of decimal places displayed in all listings will be determined by the number of decimal places in the raw data.

Unless otherwise specified, minimum and maximum will be reported to the precision as the data collected, one more decimal place for the mean and median, and two more decimal places for the standard deviation. The adjusted geometric mean, geometric mean ratio and the lower and upper limits of confidence interval will be displayed to three decimal places.

#### 8.7.2 Pharmacokinetic Summaries

#### **In-text Tables**

For in-text pharmacokinetic tables, coefficient of variation (% CV) will be reported as integers. For other statistics, values of 100 or higher will be presented as integers, values of 10 - < 100 will be displayed to one decimal place, and values of 1 - < 10 will be displayed to two decimal places. Values less than 1 will be displayed to three decimal places. Ratios will also be displayed to three decimal places.

# **Handling of Non-Quantifiable Concentrations**

For the summaries of plasma concentration-time data, concentrations that are less than the lower limit of quantification (LLOQ) should be displayed as "< LLOQ" in the listings and be treated as missing in summary tables and plots. For the purpose of calculating intensive PK parameters, pre-dose concentrations that are less than LLOQ and concentrations prior to the first quantifiable concentration that are less than LLOQ will be set to zero, and all other concentrations less than LLOQ will be set to missing.

Sparse PK concentrations for PK/PD and PK/VK correlations will be calculated by imputing values less than LLOQ as ½ \* LLOQ.

All available plasma concentration-time data and derived pharmacokinetic parameter values will be included in the PK data set and listed accordingly.

#### **Treatment of Outliers**

Individual plasma concentrations, if deemed to be anomalous, may be excluded from the analysis following a review of available documentation (e.g., bioanalytical report, clinical data). Any such exclusion will be clearly listed in the study report along with justification for exclusion.

Entire plasma concentration-time profiles for a subject may be excluded following review of available documentation (e.g., bioanalytical report, clinical data). However, results of analysis with and without the excluded profiles may be presented in the study report. Any such exclusion will be clearly listed in the study report along with justification for exclusion.

#### **PK Exclusions**

Exclusion of one or more parameters or the entire dataset may be considered due to incomplete profile, or there is no sample around the suspected Cmax. In addition, subjects may be excluded from the analysis if they missed doses, had diarrhea, or vomited at or before a time equal to twice the median Tmax for immediate-release products, or vomited at any time during sampling after the administration of modified-release formulations.

#### 9 REFERENCES

An interim analysis will be conducted after the last randomized subject in Stage 1 is on treatment for 24 weeks. The analyses related to the first 24 weeks of treatment for Stage 1 will be performed.

An interim analysis might be conducted after the last randomized subject in Stage 1 is on tratment for 48 weeks in case the continuation dose couldn't be selected based on the Week 24 results

An interim analysis will be conducted after the last randomized subject in Stage 2 is on treatment for 24 weeks. The expectation is that the last subject in Stage 1 will have completed the Week 96 visit by that time. The analyses related to the first 24 weeks of treatment for Stage 2 will be performed as well as all analyses related to Stage 1 (except the futility analysis).

An interim analysis will be conducted after the last randomized subject in Stage 2 completes the Week 48 visit. The analyses related to the first 48 weeks of treatment for Stage 2 will be performed.

The final analysis will be conducted after the last randomized subject in Stage 2 completes the Week 96 visit. All analyses described in this plan will be performed for both Stages (except the futility analysis). This includes the integrated summaries described in Section 7.8.

## APPENDIX 1 SNAPSHOT ALGORITHM

The snapshot algorithm is described in detail in Appendix A of the CDER (2013) draft guidance on developing antiretroviral drugs<sup>1</sup>. If the draft guidance is superseded, and development timelines permit any needed changes, then the instructions from the new guidance should be followed.

In some sections of the draft guidance, the responder cutoff is listed as HIV-1 RNA "< 50copies/mL". This is a carryover from earlier days when the assay limit of detection was 50. Currently approved assays have lower limits. Hence, in implementing the snapshot algorithm, the assay limit of detection will replace the HIV-1 RNA limit of "< 50copies/mL".

The analysis visit windows that appear in Table A of the draft guidance (line 1205) appear to use Day 0 as the start date. Windows that use Day 1 as the start date are in the following table.

| <b>Table 9-1:</b> | <b>Snapshot Algorithm Analysis Visit Windows</b> |
|-------------------|--------------------------------------------------|
|-------------------|--------------------------------------------------|

| VISIT | Window in Weeks | Days |
|---|---|---|
| W. 1.24 | (Weeks indicate end of study week) | (Inclusive of start & end points) |
| Week 24 | 18 through 30 | 127 through 210 |
| Week 48 | 42 through 54 | 295 through 378 |
| Week 96 | 90 through 102 | 631 through 714 |

Each snapshot analysis includes a summary of virologic outcomes at an analysis visit (e.g., Week 24) that has the same format as Table B (line 1209) of the draft guidance.

Each snapshot analysis may also include a summary of expanded virologic outcomes at an analysis visit. This summary has a similar format to Table B, but also displays the 95% CI for the response category "HIV-1 RNA < 40 c/mL", and breaks down the failure category "HIV RNA  $\geq 40 \text{c/mL}$ " into 4 subcategories. Virologic outcomes are summarized according to the following categories:

- HIV-1 RNA < 40c/mL
- HIV-1 RNA  $\geq 40$ c/mL
  - HIV-1 RNA  $\geq$  40c/mL in Week 24 window
  - Discontinued study/study drug due to lack of efficacy. This includes subjects who discontinued study therapy due to lack of efficacy at any time from Day 1 through the Week 24 window if this resulted in no on-treatment HIV-1 RNA in the window.
  - Discontinued study/study drug due for other reasons. This includes subjects with last on-treatment HIV-1 RNA ≥ 40c/mL who discontinued study therapy due to any reason except AE, death and lack of efficacy at any time from Day 1 through the Week 24 window if this resulted in no on-treatment HIV-1 RNA in the window.

- No virologic data in Week 24 window
  - Discontinued study/study drug due to AE or death. This includes subjects who discontinued study therapy due to AE or death at any time from Day 1 through the Week 24 window if this resulted in no on-treatment HIV-1 RNA in the window.
  - Discontinued study/study drug for other reasons. This includes subjects with last on-treatment HIV-1 RNA < 40c/mL who discontinued study therapy for other reasons (withdrew consent, lost to follow-up, moved, etc.) at any time from Day 1 through the Week 24 window if this resulted in no on-treatment HIV-1 RNA in the window.</li>
  - On study but missing data in window

Each snapshot analysis may also include a by-subject listing that facilitates finding the subjects in each outcome category. The listing includes: subject ID; age/gender/race; as-randomized treatment group; assessment day; HIV-1 RNA on day of assessment; virologic outcome (HIV-1 RNA < 40 c/mL, HIV-1 RNA  $\ge 40 \text{c/mL}$ , or no virologic data in window); virologic outcome specification (see subcategories in the expanded virologic outcome summary); day of discontinuation of study therapy; and the reason for discontinuation of study therapy. The listing is sorted and paged by treatment group. Within treatment group, the subjects are sorted by virologic outcome and then by the virologic outcome specification.

An analysis data set contains at least the information specified starting on line 1346 ("Datasets for Snapshot Approach"). This analysis data set may contain additional variables, and have multiple uses besides the snapshot analysis.

#### APPENDIX 2 GENOTYPIC AND PHENOTYPIC RESISTANCE

#### **Genotypic Resistance**

Genotypic resistance will be assessed by searching for all:

- RT substitutions
- PI substitutions
- Integrase (IN) substitutions

that are listed in the most current version of the International AIDS Society-USA (IAS-USA) list.

The following table was prepared relative to the IAS-USA list from June/July of 2014<sup>5</sup>. The table describes the categories and subcategories, by which the substitutions will be categorized. In the table below, slashes ("/") between amino acid codes do indicate mixtures. The slashes indicate that any of the amino acids in the list qualify as substitutions.

**Table 9-2:** Genotypic Substitutions

| Category | Description of Relevant Substitutions |
|---|---|
| Protease Gene | |
| Any PI substitution | At least one of the PI substitutions listed in the IAS-USA. L10C/F/I/R/V, V11I, G16E, |
| | K20I/M/R/T/V, L24I, |
| | D30N, V32I, L33F/I/V, E34Q, M36I/L/V, |
| | K43T, M46I/L, I47A/V, G48V, |
| | I50L/V, F53L/Y, I54A/L/M/S/T/V, Q58E, |
| | D60E, I62V, L63P, I64L/M/V, H69K/R, |
| | A71I/L/T/V, G73A/C/S/T, T74P, L76V, V77I, |
| | V82A/F/I/L/S/T, N83D, I84V, I85V, N88D/S, L89I/M/V, |
| | L90M, 193L/M |
| Major PI Substitutions | Any of the major PI substitutions listed in the IAS-USA |
| | D30N, V32I, |
| | M46I/L, I47A/V, G48V, |
| | I50L/V, I54L/M, Q58E, |
| | T74P, L76V, |
| | V82A/F/L/S/T, N83D, I84V, N88S, |
| | L90M |
| | Major PI substitutions are sub-tabulated by codon. |
| Minor PI Substitutions | Any of the minor PI substitutions listed in the IAS-USA |
| | L10C/F/I/R/V, V11I, G16E, |

 Table 9-2:
 Genotypic Substitutions

| Category | <b>Description of Relevant Substitutions</b> |
|---|---|
| | K20I/M/R/T/V, L24I, |
| | L33F/I/V, E34Q, M36I/L/V, |
| | K43T, |
| | F53L/Y, I54A/S/V/T, |
| | D60E, I62V, L63P, I64L/M/V, H69K/R, |
| | A71I/L/T/V, G73A/C/S/T, V77I, |
| | V82I, I85V, N88D, L89I/M/V, |
| | I93L/M |
| | Minor PI substitutions are sub-tabulated by codon. |
| Reverse Transcriptase Gene | |
| Any RT substitution | At least one of the nRTI or NNRTI substitutions listed in the IAS-USA RT substitutions are sub-tabulated into nRTI and NNRTI substitutions. |
| nRTI | At least one of the nRTI substitutions listed in the IAS-USA |
| | nRTI substitutions are further sub-tabulated into: 69 Insertion Complex 151 Complex, TAMS and Other. |
| 69 insertion complex | Substitution at codon 69 with a double amino acid insertion and at least one of the following: M41L, A62V, K70R, L210W, T215Y/F, K219Q/E |
| 151 complex | Q151M and at least one of the following: A62V, V75I, F77L, F116Y |
| Thymidine Analogue-<br>Associated Mutations (TAMS) | At least one of the following: M41L, D67N, K70R, L210W, T215Y/F, K219Q/E |
| Other | At least one of the other nRTI substitutions not covered above: K65R/E/N, K70E, L74V, Y115F, M184V/I |
| NNRTI | At least one of the substitutions listed in the IAS-USA for any of the NNRTIs: V90I, A98G, |
| | L100I, K101E/H/P, K103N/S,V106A/I/M, V108I, |
| | E138A/G/K/Q/R, |
| | V179D/F/L/T, |
| | Y181C/I/V, Y188C/L/H, |
| | G190S/A, |
| | H221Y, P225H, F227C,<br>M230I/L. |
| | NNRTI substitutions are tabulated by codon. |
| Integrase Gene | At least one of the substitutions listed in the IAS-USA for integrase inhibitors |
| Any Integrase Substitutions | T66I/A/K |
| | L74M |
| | E92Q/G, T97A |

**Table 9-2:** Genotypic Substitutions

| Category | <b>Description of Relevant Substitutions</b> |
|----------|------------------------------------------------|
| | F121Y |
| | E138A/K |
| | G140A/S |
| | Y143R/H/C, S147G, Q148H/K/R |
| | N155H |
| | Integrase substitutions are tabulated by codon |

# **Phenotypic Resistance**

The phenotypic resistance to a drug is defined as a fold change (i.e., ratio of the 50% inhibitory concentration (IC<sub>50</sub>) of the clinical isolate to the IC<sub>50</sub> of the reference strain) greater than the cutoff for reduced susceptibility. The following table displays cut-offs used by Monogram
Biosciences, Inc. to determine reduced susceptibility to each drug.

The phenotypic resistance status, as determined by Monogram (for ARVs other than BMS-955176) should be available in the clinical database. Hence, programming these cutoffs should be unnecessary.

Note: Monogram may use TFV as a code for tenofovir in phenotypic data files.

Table 9-3: Cut-offs used by Monogram Biosciences to Determine Reduced Susceptibility

| Class | Drug | Reduced Susceptibility Cut-off |
|-------|---------------------------------|--------------------------------|
| PI | Atazanovir (ATV) | 2.2 |
| | Atazanavir/Ritonavir (ATV/r) | 5.2 |
| | Darunavir/Ritonavir (DRV/r) | 10 |
| | Fosamprenavir/Ritonavir (AMP/r) | 4 |
| | Indinavir/Ritonavir (IDV/r) | 10 |
| | Lopinavir/Ritonavir (LPV/r) | 9 |
| | Nelfinavir (NFV) | 3.6 |
| | Ritonavir (RTV) | 2.5 |
| | Saquinavir/Ritonavir (SQV/r) | 2.3 |
| | Tipranavir/Ritonavir (TPV/r) | 2 |
| NNRTI | Delavirdine (DLV) | 6.2 |
| | Efavirenz (EFV) | 3 |
| | Etravirine (ETR) | 2.9 |
| | Nevirapine (NVP) | 4.5 |

Table 9-3: Cut-offs used by Monogram Biosciences to Determine Reduced Susceptibility

| Class | Drug | Reduced Susceptibility Cut-off |
|-------|---------------------|--------------------------------|
| | Rilpivirine (RPV) | 2.5 |
| NRTI | Abacavir (ABC) | 4.5 |
| | Didanosine (ddI) | 1.3 |
| | Emtricitabine (FTC) | 3.5 |
| | Lamivudine (3TC) | 3.5 |
| | Stavudine (d4T) | 1.7 |
| | Tenofovir (TDF) | 1.4 |
| | Zidovudine (ZDV) | 1.9 |
| IN | Raltegravir (RAL) | 2.2 |
| | Dolutegravir (DTG) | 4 |
| | Elvitegravir (EVG) | 3.5 |

#### APPENDIX 3 TIME TO LOSS OF VIROLOGIC RESPONSE

This appendix describes the Time to Loss of Virologic Response (TLOVR) algorithm for analyses at Week 24, 48 and 96. The instructions that follow are based on the FDA guidance from 2002<sup>6</sup>. Guidance from the European Union<sup>7</sup> indicates that snapshot analyses should be supplemented by at TLOVR analysis.

For this study, the TLOVR analyses are done on the mITT data sets. The assay limit used in the TLOVR analysis is the limit of detection.

TLOVR has two components, a time-to-failure (life table) analysis, and a tabulation of treatment outcomes at each particular time point (e.g. Week 24).

The time to failure data are analyzed using the Kaplan-Meier method. The presentation will include a K-M curve, estimates of the response rates at the end of weeks 24, 48 and 96 and 95% confidence intervals for the estimate. The time-to-failure analysis is based on the following rules (FDA, 2002):

- "For 2 and 3 below, discard all visits with no data. In what follows, visit means visit with an observed viral load. All available visits, including off-schedule visits and post-week 96 visits, should be used for the calculation. Data should not be interpolated for visits or time points with missing data.
- Subjects who never achieved confirmed HIV RNA levels below the assay limit (on two consecutive visits) before any of the following events will be considered to have failed at time 0.
  - a) Death
  - b) Introduction of a new antiretroviral drug to the regimen. Exceptions may be made for certain pre-specified changes in background therapy where the reason for change is due to toxicity or intolerance of background therapy and not the study drug or control.
  - c) Last available visit
- For all subjects who have confirmed HIV RNA levels below an assay limit (two consecutive visits below an assay limit), the time to failure is the earliest of the choices below, with modification specified in 4:
  - a) Time of the event as described in 2b
  - b) Time of loss to follow-up
  - c) Time of confirmed levels above an assay limit. Confirmed is defined as two consecutive visits greater than an assay limit or one visit greater than an assay limit followed by loss to follow-up.
  - d) Time of death
- If the time to virologic failure defined above is immediately preceded by a single missing scheduled visit or multiple consecutive missing scheduled visits, the time of virologic failure is replaced by the time of the first such missing visit."

The tabulation of treatment outcomes shows the proportions of success and failure for various reasons. For a subject, the reason for failure is based on the primary reason for the earliest treatment failure. For any visit, subjects who achieved confirmed virologic success, defined as two consecutive visits below the assay limit of detection, but have not failed according the above loss of virologic success algorithm are considered successes. All others should be classified into the appropriate categories, which are shown in the FDA draft guidance.

The visit windows used in tabulating treatment outcomes are the same visit windows used for the snapshot algorithm. For subjects who failed for multiple reasons at the earliest time of failure, the precedence of failure classification is: death, virologic rebound and then premature discontinuation. For example, if virologic rebound and premature discontinuation occur on the same day, then the reason for failure is virologic rebound.

#### APPENDIX 4 EQ-5D-3L SCORING PROGRAM - U.S. WEIGHTED

This SAS scoring algorithm was downloaded on January 20, 2015 from:

http://archive.ahrq.gov/professionals/clinicians-providers/resources/rice/EQ5Dscore.html

 $^{\prime \star}$  EQ-5D U.S. PREFERENCE-WEIGHTED INDEX  $^{\star \prime}$ 

```
/* Author: PPD */
/* Date: May 20, 2004 */
```

/\* Program was written with SAS Release 8.02 for Windows. \*/

/\* The scoring algorithm presented below was taken from: Shaw JW, Johnson JA, Coons SJ. U.S. Valuation of the EQ-5D Health States: Development and Testing of the D1 Valuation Model. Medical Care. Submitted 2004. \*/

/\* This program computes the U.S. preference-weighted index score using self-reported EQ-5D data. It is presumed that the data set includes the following five variables:

| Dimension | Variable Name | Range |
|---|---|---|
| Mobility Self-care Usual activities Pain/discomfort Anxiety/depression | MO<br>SC<br>UA<br>PD<br>AD | 1-3<br>1-3<br>1-3<br>1-3<br>1-3 |

where a 1 indicates no problems, a 2 indicates moderate problems, and a 3 indicates severe problems. The variables containing responses for the five dimensions must be named as above (in capital letters). Missing values should be left blank (ie, a '.' should not be substituted for a missing value). The index score will not be generated when responses are missing for 1 or more of the five dimensions.

In the data step, the user should specify the location (LIBNAME) and name of the data set to be analyzed (DATANAME). It is recommended that the index values be saved to a new data set (NEWDATANAME) in the desired library. \*/

```
/* SAS Data Step */
```

data LIBNAME.DATANAME; set LIBNAME.NEWDATANAME;

```
/* Generate Dummy Variables for Levels 2 and 3 of Five Dimensions */
m1 = 0;
m2 = 0;
s1 = 0;
s2 = 0;
u1 = 0;
u2 = 0;
p1 =0;
p2 = 0;
a1 =0;
a2 = 0;
if MO = 2 then m1 = 1;
if MO = 3 then m2 = 1;
if SC = 2 then s1 = 1;
if SC = 3 then s2 = 1;
if UA = 2 then u1 = 1;
if UA = 3 then u2 = 1;
if PD = 2 then p1 = 1;
if PD = 3 then p2 = 1;
if AD = 2 then a1 = 1;
if AD = 3 then a2 = 1;
/* Generate Interaction Terms (I2, I2-squared, I3, I3-squared) */
m0 = 0 ;
s0 = 0;
u0 = 0;
p0 = 0;
a0 = 0;
if m1 = 0 and m2 = 0 then m0 = 1;
if s1 = 0 and s2 = 0 then s0 = 1;
if u1 = 0 and u2 = 0 then u0 = 1;
if p1 = 0 and p2 = 0 then p0 = 1;
if a1 = 0 and a2 = 0 then a0 = 1;
i2 = m1 + s1 + u1 + p1 + a1;
i2 = i2 - 1;
if i2<0 then i2 = 0;
i22 = i2*i2;
i3 = m2 + s2 + u2 + p2 + a2;
i3 = i3 - 1;
if i3<0 then i3 = 0;
i32 = i3*i3;
/* Generate D1 Term */
i1 = m0 + s0 + u0 + p0 + a0;
d1 = 4 - i1;
if d1<0 then d1 = 0;
```

```
/* Generate Raw Index Score */

pred = .146016*ml + .557685*m2 + .1753425*s1 + .4711896*s2 + .1397295*ul + .3742594*u2 + .1728907*pl + .5371011*p2 + .156223*al + .4501876*a2 + -.1395949*dl + .0106868*i22 + -.1215579*i3 + -.0147963*i32;

EQ index = 1 - pred;

if (MO = .) or (SC = .) or (UA = .) or (PD = .) or (AD = .) then EQ_index = . ;/* Drop Variables Generated by Program */

drop ml m2 sl s2 ul u2 pl p2 al a2 m0 s0 u0 p0 a0 i2 i22 i3 i32 dl pred nvector;

run;
```

#### APPENDIX 5 EQ-5D-3L SCORING PROGRAM - U.K. WEIGHTED

The following SAS code is an example of computing UK centric utility scores. The code was taken from the BMS SAP for study  $CN162-007^2$ .

```
utility = 1;
if mobility=1 then mob=0;
else if mobility=2 then mob=-0.069;
else if mobility=3 then mob=-0.314;
if selfcare=1 then self=0;
else if selfcare=2 then self=-0.104;
else if selfcare=3 then self=-0.214;
if usualact=1 then usual=0;
else if usualact=2 then usual=-0.036;
else if usualact=3 then usual=-0.094;
if paindis=1 then pain=0;
else if paindis=2 then pain=-0.123;
else if paindis=3 then pain=-0.386;
if anxdep=1 then anxiety=0;
else if anxdep=2 then anxiety=-0.071;
else if anxdep=3 then anxiety=-0.236;
utility = utility + mob + self + usual + pain + anxiety;
if mobility in (2,3) or selfcare in (2,3) or usualact in (2,3) or paindis in (2,3) or anxdep in (2,3)
then utility = utility -0.081;
if mobility=3 or selfcare=3 or usualact=3 or paindis=3 or anxdep=3 then utility = utility -0.269;
```

#### 10 REFERENCES

- 1. Guidance for industry: Human Immunodeficiency Virus-1 Infection: Developing Antiretroviral Drugs for Treatment. US Department of Health and Human Services, Food and Drug Administration, Center for Drug Evaluation and Research (CDER). Draft Guidance. June, 2013.
- 2. Statistical Analysis Plan for CN162-007, version 2, BMS DCN 930065069
- 3. Shaw, J.W., et al, 2005, "US Valuation of the EQ-5D Heath States Development and Testing of the D1 Valuation Model", Medical Care, vol. 43, no. 3, 203-220.
- 4. Dolan P. (1997). Modeling valuations for EuroQol health states, Medical Care, 35, 1095-1108
- 5. Johnson V, et al., Update of the Drug Resistance Mutations in HIV-1. Topics in HIV Medicine 2013; 21 (1): 4 12.
- 6. Guidance for industry: Antiretroviral Drugs Using Plasma HIV RNA Measurements Clinical Considerations for Accelerated and Traditional Approval. US Department of Health and Human Services, Food and Drug Administration, Center for Drug Evaluation and Research (CDER). October, 2002.
- 7. Guideline on the clinical development medicinal products for the treatment HIV infection. EMEA/CPMP/EWP/633/02; Rev 3. 2013.

#### 11 DOCUMENT HISTORY

Table 11-1: Document History

| Version<br>Number | Author(s) | Description |
|---|---|---|
| 1.0 | PPD | Original version |
| | | Section 1: update schedule of analyses |
| | | Section 2.4: add protocol amendment 6 |
| | | Section 7.2: add relevant protocol deviation related to screening eGFR |
| | | Section 7.3.2.4: add baseline resistance summaries for treated subjects that are identified as protocol defined virologic failures. |
| 2.0 | PPD | Section 7.5.2.5: Include summary for newly emergent phenotypic resistance to BMS-955176. |
| | | For Gag: add summaries by HIV subtype. |
| | | Section 7.8: was added to describe the integrated outputs |
| | | Section 8.1: correct visit window for Weeks 16 and 24, and remove Week 20 |
| | | Section 9: describe content of the reports in more detail |
| | | Update Table 10-1 based on 2014 IAS-USA |

# Appendix to Reporting Analysis Plan for Study AI468048/205892 ---Final Analysis

Compound Number: BMS-955176/GSK3532795

Study Title A Phase 2b Randomized, Active-Controlled, Staged, Open-Label

Trial to Investigate Safety and Efficacy of BMS-955176 in Combination with Dolutegravir and Atazanavir (with or without Ritonavir) in Treatment-Experienced HIV-1 Infected Adults

**Effective Date:** 09 November 2017 (This appendix should be attached to the

amendment of Reporting and Analysis Plan for study

AI468048/205892 Version 2.0 effective on 15 October 2016).

**Description**: This appendix describes the plan for the final statistical analyses of study AI468048/205892.

#### Author's Name, Title and Functional Area:

PPD Data Analyst Statistician, Clinical Statistics

#### Approved through email by:



Copyright 2017 ViiV Healthcare and the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.


## AI468038/205891

# **TABLE OF CONTENTS**

| | | | | PAGE |
|----|------|----------|----------------|------|
| 1. | CHR | ONOLOG | Y | 3 |
| 2. | FINA | L ANALY | SIS | 3 |
| 3. | LIST | OF DISP | LAYS | 6 |
| | 3.1. | | Population | |
| | | | Tables | |
| | | 3.1.2. | ICH Listings | |
| | | 3.1.3. | Other Listings | 8 |
| | 3.2. | Efficacy | / | 9 |
| | | 3.2.1. | | 9 |
| | | 3.2.2. | ICH Listings | |
| | | 3.2.3. | Other Listings | 10 |
| | 3.3. | Safety. | | 12 |
| | | 3.3.1. | Tables | 12 |
| | | 3.3.2. | ICH Listings | |
| | 3.4. | Virology | y | 19 |
| | | 3.4.1. | Tables | 19 |
| | | 3.4.2. | Other Listings | |

## 1. CHRONOLOGY

15-OCT-2016 Reporting and Analysis Plan for Study AI468048, Version 2.0 09-NOV-2017 Appendix of Analysis Plan for Study AI468048 (Final Analysis)

# 2. FINAL ANALYSIS

Per the company decision to end this study prior to all subjects reaching the primary endpoint, a simplified approach for the final report has been proposed by the project team. Hence the final analyses for AI468048 study as described in this appendix will be performed on subjects who were enrolled into this study, regardless of study stage, and will supersede what have been previously stated in the finalized BMS RAP Version 2.0. In addition, due to the GCP non-compliance of Site P (Dr. Juan Ballesteros in Chile) with ICH GCP E6 (R2) Guidelines, data obtained from this GCP non-compliant site will not be included in the final analyses (e.g., summary tables of selected efficacy and safety data); however, subject data listings will include all subjects enrolled in this study. Subject data listings for the GCP non-compliant Site P will also be provided.

The details of the final reporting and analysis plan are described as below:

#### 1) Analysis Populations

Due to the GCP non-compliance of Site PD data obtained from this GCP non-compliant site will be excluded in the final analyses.

Populations for Analyses for this synoptic report are defined as follows:

- Enrolled subjects are those who signed an informed consent form and were assigned a Patient Identification number (PID).
- Randomized subjects are enrolled subjects who received a treatment assignment from the IVRS and will be used in subject data listings as specified.
- Modified Randomized Subjects are enrolled subjects who received a treatment assignment from the IVRS, excluding subjects from Site PP The modified randomized subjects will be used to assess subject disposition.
- Treated Subjects are randomized subjects who received at least 1 dose of study therapy and will be used in subject data listings as specified.
- Modified Treated Subjects are randomized subjects who received at least 1 dose of study therapy, exclude subjects from Site PP Modified treated subjects will be used to assess demography and baseline characteristics,

protocol deviations, exposure, concomitant medication, efficacy, resistance and safety data.

Pharmacokinetic (PK) population is defined as all treated subjects who
have any available concentration-time data. The evaluable PK population
is a sub-population including all treated subjects who have adequate PK
profiles.

# 2) Demographic and baseline characteristic

This report includes the analyses of demographics, baseline characteristics, and baseline resistance data based on Modified Treated Subjects population. Subject data listings will be based on Treated Subjects population.

The detailed outputs for demographic and baseline characteristic data are listed in the Section 3.1 of List of Displays for Study Population.

#### 3) Simplified report on primary efficacy endpoint

Selected summaries and analyses on primary efficacy endpoint will be performed for this final analysis, based on Modified Treated Subjects population. Subject data listings will be based on Treated Subjects population.

The detailed outputs for primary efficacy endpoint data are listed in the Section 3.2 of List of Displays for Efficacy.

#### 4) Secondary and Exploratory Efficacy Endpoints

Analyses for secondary and exploratory efficacy endpoints, including pharmacokinetic and quality of life endpoints, will not be performed except for HIV-1 RNA, CD4+ counts, and drug resistance endpoints (see additional details in Section 3.4, Virology) which are subject to availability of the data and will be analyzed based on Modified Treated Subjects population. There will be no subgroups and no multivariate analysis performed for secondary and exploratory efficacy endpoints for this final analysis. Subject data listings based on Treated Subjects population except PK data which will be based PK population.

The detailed outputs for primary secondary and exploratory efficacy endpoints are listed in the Section 3.2 of List of Displays for Efficacy.

#### 5) Safety displays

Final safety analysis will be summarized based on Modified Treated Subjects population; however, subject data listings will be based on Treated Subjects population. Subject data listings will be based on Treated Subjects population.

The detailed outputs are listed in the Section 3.3 of List of Displays for Safety.

# 6) Virology

HIV drug resistance data will be summarized based on Modified Treated Subjects population. Subject data listings will be based on Treated Subjects population.

The detailed outputs for HIV drug resistance data are listed in the section of List of Display for Virology.

# 7) General

The display for TLFs will be based on BMS shells and will not utilize HARP for SAC.

The list of displays has been updated as shown below.

# 3. LIST OF DISPLAYS

The data displays will be based on the BMS shell as specified in the column of BMS Table number/File Name/BMS Template, where applicable. The details information on BMS shell can be found in the Analysis Data Presentation Plan revision 2.0 for this study.

The following data display numbering will be applied for RAP generated displays:

| Section | Tables |
|------------------|-------------|
| Study Population | 1.1 to 1.5 |
| Efficacy | 2.1 to 2.4 |
| Safety | 3.1 to 3.46 |
| Virology | 4.1 to 4.9 |
| Section | Listings |
| ICH Listings | 1 to 26 |
| Other Listings | 27 to 44 |

# 3.1. Study Population

## 3.1.1. **Tables**

For Table and listing displays, Treated Subjects, Modified Treated Subjects, Randomized Subjects, and Modified Randomized Subjects populations will be used as specified below.

| Number | Title | BMS Table number/File Name/BMS Template |
|---|---|---|
| 1.1 | End of Study Subject Status Summary | Table S.2.1.1B / rt-ds-statuss1.lst / GS_DS_T_X_005 |
| | Modified Randomized Subjects | |

| Number | Title | BMS Table number/File Name/BMS Template |
|---|---|---|
| 1.2 | Populations for Analysis Summary | Table S.2.1.1C / rt-dm-populations1.lst / |
| | | SS_DM_T_002 |
| 1.3 | Demographic Characteristics Summary | Table S.3.1.1 / rt-dm-summarys1.lst / |
| | Modified Treated Subjects | GS_DM_T_X_002 |
| 1.4 | Summary of Baseline Disease Characteristics | Table S.3.2.1 / rt-dm-diseases1.lst / SS_DM_T_004 |
| | Modified Treated Subjects | |
| 1.5 | Summary of Baseline Physical Measurements | Table S.3.3.1 / rt-pm-bsls1.lst / GS_PM_T_X_001 |
| | Modified Treated Subjects | |

# 3.1.2. ICH Listings

| Number | Title | BMS Table number/File Name/BMS Template |
|---|---|---|
| 1 | End of Study Subject Status | Appendix 2.1.1B / rl-ds-statuss1.lst / |
| | Randomized Subjects | GS_DS_L_X_005 |
| 2 | Randomization Scheme and Codes | Appendix 1.9.1 / rl-ds-randcode.lst / SS_DS_L_001 |
| | Randomized Subjects | |
| 3 | Subjects Excluded from Analysis | Appendix 2.2.1 / rl-dm-excls1.lst / SS_DM_L_001 |
| | Treated Subjects | |
| 4 | Listing of Relevant Protocol Deviations | Table S.2.3.1B / rl-pd-rels1.lst / SS_PD_L_001 |
| | Randomized Subjects | |
| 5 | Demographic Characteristics | Appendix 3.1.1A / rl-dm-demchars1.lst / |
| | Treated Subjects | GS_DM_L_X_001 |

| Number | Title | BMS Table number/File Name/BMS Template |
|---|---|---|
| 6 | Non-Study Medication Previous and Concomitant Medications Treated Subjects | Appendix 4.2.1 / rl-cm-meds1.lst / GS_CM_L_X_006 |

# 3.1.3. Other Listings

| Number | Title | BMS Table number/File Name/BMS Template |
|---|---|---|
| 27 | Listing of Batch Numbers | Appendix 1.7.1 / rl-ex-batch.lst / SS_EX_L_001 |
| | Treated Subjects | |
| 28 | Summary of Baseline Disease Characteristics | Appendix 3.2.1A / rt-dm-diseasenrands1.lst / |
| | Subjects Enrolled but Not Randomized | SS_DM_T_004 |
| 29 | Listing of HIV Disease Characteristics | Appendix 3.2.1B / rl-dm-diseases1.lst / |
| | Treated Subjects | SS_DM_L_002 |
| 30 | Physical Examination | Appendix 3.4.1 / rl-pe-lists1.lst / GS_PE_L_X_001 |
| | Treated Subjects | |
| 31 | General Medical History | Appendix 3.7.1 / rl-mh-list1.lst / GS_MH_L_X_001 |
| | Treated Subjects | |

# 3.2. Efficacy

Summary and analyses for primary efficacy data, secondary efficacy data and exploratory efficacy data, unless indicated in Section 3.2.1 below, will not be presented for the final analysis except for HIV Drug Resistance data from Modified Treated Subjects who underwent resistance testing will be summarized and presented, see additional details in Section 3.4.

Subject data listings will be provided for primary efficacy data, secondary efficacy data, exploratory efficacy data, and available plasma concentration data based on Treated Subjects population in Sections 3.2.2 and 3.2.3.

#### 3.2.1. Tables

| Number | Title | BMS Table number/File Name/BMS Template |
|---|---|---|
| 2.1 | Detailed Summary of HIV-1 RNA < 40 c/mL Proportion of | Table S.5.1.1A / rt-vl-resp40w24s1.lst / |
| | Responders at Week 24 Snapshot | SS_VL_T_001 |
| | Modified Treated Subjects | |
| 2.2 | Summary of HIV-1 RNA < 40 c/mL Proportion of Responders by | Table S.5.1.1E / rt-vl-resp40w24obssubgs1.lst / |
| | Scheduled Assessments Over Time | SS_VL_T_003 |
| | Modified Treated Subjects (Observed) <sup>1</sup> | (By Weeks 24, 48, and 96 instead of By Subgroup) |
| 2.3 | Summary Statistics for Values and Change from Baseline Over Time | Table S.5.7.1A / rt-lb-cd4s1.lst / SS_VL_T_006 |
| | CD4 Cell Count (cells/uL) | (Without "By Subgroup") |
| | Modified Treated Subjects (Observed) <sup>1</sup> | |
| 2.4 | Summary Statistics for Values and Change from Baseline Over Time | Table S.5.8.1A / rt-lb-cd4pcts1.lst / SS_VL_T_006 |
| | CD4 Cell Percentage | (Without "By Subgroup") |
| | Modified Treated Subjects (Observed) <sup>1</sup> | |

| Number Title | BMS Table number/File Name/BMS Template |
|--------------|-----------------------------------------|
|--------------|-----------------------------------------|

<sup>1</sup> Add the following footnote to the tables 2.2-2.4:

Note: Modified Treated Subjects (Observed): Consisting of subjects in the Treated Subjects Population excluding subjects who have no HIV-1 RNA result data in the assessment visit windows due to discontinuation and who discontinued on or after the date of site notification of study termination by the sponsor [October 10, 2016], will be used to evaluate efficacy in a sensitivity analysis.

# 3.2.2. ICH Listings

| Number | Title | BMS Table number/File Name/BMS Template |
|---|---|---|
| 7 | Listing of Outcomes from HIV-1 RNA < 40 c/mL Snapshot | Appendix 5.1.1A / rl-vl-outcome24s1.lst / |
| | Analysis Data for Subjects in the Week 24 Snapshot | SS_VL_L_004 |
| | Treated Subjects | |

# 3.2.3. Other Listings

| Number | Title | BMS Table number/File Name/BMS Template |
|---|---|---|
| 32 | Listing of HIV-1 RNA | Appendix 5.1.1D / rl-vl-vllist1.lst / SS_VL_L_005 |
| | Treated Subjects | |
| 33 | Listing of CD4+ and CD8+ T- Cell Count and Percentages | Appendix 5.1.1E / rl-lb-cd4cd81.lst / SS_VL_L_005 |
| | Treated Subjects | |
| 34 | Listing of BMS-955176 Plasma Concentration – Time Data | Appendix 8.2.1A / rl-pk-cpar1bmss1.lst / |
| | PK Population | MS_PK_L_001 |
| 35 | Listing of ATV Plasma Concentration – Time Data | Appendix 8.2.1B / rl-pk-cpar1atvs1.lst / |
| | PK Population | MS_PK_L_001 |


## Al468038/205891

| Number | Title | BMS Table number/File Name/BMS Template |
|---|---|---|
| 36 | Listing of DTG Plasma Concentration – Time Data | Appendix 8.2.1C / rl-pk-cpar1dtgs1.lst / |
| | PK Population | MS_PK_L_001 |

# 3.3. Safety

The Modified Treated Subjects population will be used in the safety summaries and analyses. All treated subjects will be used in the data listings. Subject data listings will be based on Treated Subjects population.

# 3.3.1. Tables

| Number | Title | BMS Table number/File Name/BMS Template |
|---|---|---|
| 3.1 | Extent of Exposure to BMS-955176 Time on Therapy | Table S.4.1.1A / rt-ex-bmss1.lst / SS_EX_T_001 |
| | Modified Treated Subjects | |
| 3.2 | Extent of Exposure to Tenofovir Time on Therapy | Table S.4.1.1B / rt-ex-tdfs1.lst / SS_EX_T_001 |
| | Modified Treated Subjects | |
| 3.3 | Extent of Exposure to Atazanavir Time on Therapy | Table S.4.1.1C / rt-ex-atvs1.lst / SS_EX_T_001 |
| | Modified Treated Subjects | |
| 3.4 | Extent of Exposure to Dolutegravir Time on Therapy | Table S.4.1.1D / rt-ex-dtgs1.lst / SS_EX_T_001 |
| | Modified Treated Subjects | |
| 3.5 | Extent of Exposure to Ritonavir Time on Therapy | Table S.4.1.1E / rt-ex-rtvs1.lst / SS_EX_T_001 |
| | Modified Treated Subjects | |
| 3.6 | Extent of Exposure to Treatment Regimen Time on Therapy | Table S.4.1.1F / rt-ex-regimens1.lst / SS_EX_T_001 |
| | Modified Treated Subjects | |
| 3.7 | Adverse Events Overall Adverse Events Summary | Table S.6.7.1 rt-ae-overallsums1.lst SS_AE_T_001 |
| | Modified Treated Subjects | |
| 3.8 | Summary of Serious Adverse Events | Table S.6.2.1A / rt-ae-saes1.lst / GS_AE_T_X_001 |
| | Modified Treated Subjects | |
| 3.9 | Summary of Serious Adverse Event With Death As An Outcome | Table S.6.2.1C / rt-ae-saeldeaths1eu.lst / |
| | Modified Treated Subjects | GS_AE_T_X_001 |

| Number | Title | BMS Table number/File Name/BMS Template |
|---|---|---|
| 3.10 | Summary of Drug Related Serious Adverse Event With Death As An | Table S.6.2.2D / rt-ae-relsaeldeaths2eu.lst / |
| | Outcome | GS_AE_T_X_001 |
| | Modified Treated Subjects | |
| 3.11 | Listing of Serious Adverse Events | Table S.6.2.1E / rl-ae-saes1.lst / GS_AE_L_S_001 |
| | Modified Treated Subjects | |
| 3.12 | Death Listing | Table S.6.1.1 / rl-ae-deaths1.lst / SS_AE_L_001 |
| | Enrolled Subjects | |
| 3.13 | Summary of Adverse Events Leading to Discontinuation of Study | Table S.6.3.1A / rt-ae-aediscs1.lst / GS_AE_T_X_001 |
| | Medication | |
| | Modified Treated Subjects | |
| 3.14 | Listing of Adverse Event Leading to Discontinuation of Study | Table S.6.3.1C / rl-ae-discs1.lst / GS_AE_L_X_001 |
| | Medication | |
| | Modified Treated Subjects | |
| 3.15 | Summary of Non-Serious Adverse Events Occurring in at Least 5 | Table S.6.5.1A / rt-ae-nsae5pcts1.lst / |
| | Percent of Treated Subjects | GS_AE_T_X_001 |
| | Modified Treated Subjects | |
| 3.16 | Summary of Grade 1 to 4 Adverse Events | Table S.6.5.1B / rt-ae-grade1to4s1.lst / |
| | Modified Treated Subjects | GS_AE_T_X_001 |
| 3.17 | Summary of Grade 2 to 4 Adverse Events | Table S.6.5.1C / rt-ae-grade2to4s1.lst / |
| | Modified Treated Subjects | GS_AE_T_X_001 |
| 3.18 | Summary of Grade 3 to 4 Adverse Events | Table S.6.5.1D / rt-ae-grade3to4s1.lst / |
| | Modified Treated Subjects | GS_AE_T_X_001 |
| 3.19 | Summary of Grade 1 to 4 Related Adverse Events | Table S.6.5.1E / rt-ae-relateds1.lst / GS_AE_T_X_001 |
| | Modified Treated Subjects | |

| Number | Title | BMS Table number/File Name/BMS Template |
|---|---|---|
| 3.20 | Summary of Grade 2 to 4 Related Adverse Events | Table S.6.5.1F / rt-ae-relgrade2to4s1.lst / |
| | Modified Treated Subjects | GS_AE_T_X_001 |
| 3.21 | Summary of Grade 3 to 4 Related Adverse Events | Table S.6.5.1G / rt-ae-relgrade3to4s1.lst / |
| | Modified Treated Subjects | GS_AE_T_X_001 |
| 3.22 | Summary of CDC Class C AIDS Events | Table S.6.4.1A / rt-ae-cdcaes1.lst / GS_AE_T_X_001 |
| | Modified Treated Subjects | |
| 3.23 | Listing of Adverse Event | Table S.6.4.1B / rl-ae-cdcaes1.lst / GS_AE_L_X_001 |
| | CDC Class C AIDS Events | |
| | Modified Treated Subjects | |
| 3.24 | Summary of Gastrointestinal Events of Special Interest | Table S.6.4.1C / rt-ae-giaes1.lst / GS_AE_T_X_001 |
| | Modified Treated Subjects | |
| 3.25 | Listing of Adverse Event | Table S.6.4.1D / rl-ae-giaes1.lst / GS_AE_L_X_001 |
| | Gastrointestinal Events of Special Interest | |
| | Modified Treated Subjects | |
| 3.26 | Summary of Worst Toxicity Grade | Table S.7.1.1A / rt-lb-toxs1.lst / SS_LB_T_001 |
| | Modified Treated Subjects | |
| 3.27 | Summary of Grade 3-4 Toxicity | Table S.7.1.1B / rt-lb-g34toxs1.lst / SS_LB_T_001 |
| | Modified Treated Subjects | |
| 3.28 | Summary of Treatment-Emergent Abnormalities | Table S.7.1.1C / rt-lb-etoxs1.lst / SS_LB_T_001 |
| | Modified Treated Subjects | |
| 3.29 | Summary Statistics for Renal Function Values and Change | Table S.7.2.1A / rt-lb-renals1.lst / SS_VL_T_006 |
| | from Baseline - SI Units | |
| | Modified Treated Subjects | |

| Number | Title | BMS Table number/File Name/BMS Template |
|---|---|---|
| 3.30 | Summary Statistics for Renal Function Values and Change | Table S.7.2.1B / rt-zl-renals1.lst / SS_VL_T_006 |
| | from Baseline - US Units | |
| | Modified Treated Subjects | |
| 3.31 | Summary Statistics for Fasting Lipid Values and Change from | Table S.7.2.1C / rt-lb-lipidss1.lst / SS_VL_T_006 |
| | Baseline - SI Units | |
| | Modified Treated Subjects | |
| 3.32 | Summary Statistics for Fasting Lipid Values and Change from | Table S.7.2.1D / rt-zl-lipidss1.lst / SS_VL_T_006 |
| | Baseline - US Units | |
| | Modified Treated Subjects | |
| 3.33 | Summary Statistics for Fasting Lipid Values and Percent | Table S.7.2.1E / rt-lb-pchglipidss1.lst / SS_VL_T_006 |
| | Change from Baseline - SI Units | |
| | Modified Treated Subjects | |
| 3.34 | Summary Statistics for Fasting Lipid Values and Percent | Table S.7.2.1F / rt-zl-pchglipidss1.lst / SS_VL_T_006 |
| | Change from Baseline - US Units | |
| | Modified Treated Subjects | |
| 3.35 | Summary Statistics for Renal Biomarker Values and Change from | Table S.7.5.1A / rt-zl-bmrenals1.lst / SS_VL_T_006 |
| | Baseline - US Units | |
| | Modified Treated Subjects | |
| 3.36 | Summary Statistics for Renal Biomarker Values and Change from | Table S.7.5.1B / rt-lb-bmrenals1.lst / SS_VL_T_006 |
| | Baseline - SI Units | |
| | Modified Treated Subjects | |
| 3.37 | Summary Statistics for Renal Biomarker Values and Percent Change | Table S.7.5.1C / rt-zl-pchbmrenals1.lst / |
| | from Baseline - US Units | SS_VL_T_006 |
| | Modified Treated Subjects | |

| Number | Title | BMS Table number/File Name/BMS Template |
|---|---|---|
| 3.38 | Summary Statistics for Renal Biomarker Values and Percent Change | Table S.7.5.1D / rt-lb-pchbmrenals1.lst / |
| | from Baseline - SI Units | SS_VL_T_006 |
| | Modified Treated Subjects | |
| 3.39 | Summary Statistics for Bone Biomarker Values and Change from | Table S.7.5.1E / rt-zl-bmbones1.lst / SS_VL_T_006 |
| | Baseline - US Units | |
| | Modified Treated Subjects | |
| 3.40 | Summary Statistics for Bone Biomarker Values and Change from | Table S.7.5.1F / rt-lb-bmbones1.lst / SS_VL_T_006 |
| | Baseline - SI Units | |
| | Modified Treated Subjects | |
| 3.41 | Summary Statistics for Bone Biomarker Values and Percent Change | Table S.7.5.1G / rt-zl-pchbmbones1.lst / |
| | from Baseline - US Units | SS_VL_T_006 |
| | Modified Treated Subjects | |
| 3.42 | Summary Statistics for Bone Biomarker Values and Percent Change | Table S.7.5.1H / rt-lb-pchbmbones1.lst / |
| | from Baseline - SI Units | SS_VL_T_006 |
| | Modified Treated Subjects | |
| 3.43 | Summary of Electrocardiogram Values and Changes from | Appendix 7.3.1A / rt-eg-sumchgs1.lst / SS_EG_T_003 |
| | Baseline over Time | |
| | Modified Treated Subjects | |
| 3.44 | Summary of Electrocardiogram Change from Baseline Category | Appendix 7.3.1B / rt-eg-changecats1.lst / |
| | Modified Treated Subjects | SS_EG_T_001 |
| 3.35 | Summary of Electrocardiogram Category | Appendix 7.3.1C / rt-eg-cats1.lst / SS_EG_T_002 |
| | Modified Treated Subjects | |

# CONFIDENTIAL

| Number | Title | BMS Table number/File Name/BMS Template |
|---|---|---|
| 3.46 | Summary of Vital Sign Values and Changes from Baseline over | Appendix 7.4.1A / rt-vs-sums1.lst / SS_VL_T_006 |
| | Time | |
| | Modified Treated Subjects | |

# 3.3.2. ICH Listings

| Number | Title | BMS Table number/File Name/BMS Template |
|---|---|---|
| 8 | Listing of Study Medication Exposure by Subject Listing | Appendix 4.1.1A / rl-ex-lists1.lst / SS_EX_L_001 |
| | Treated Subjects | |
| 9 | Listing of Adverse Event | Appendix 6.5.1 / rl-ae-lists1.lst / GS_AEL_X_001 |
| | Treated Subjects | |
| 10 | Listing of Adverse Event Unique Events | Appendix 6.6.1 / rl-ae-uniques1.lst / |
| | Treated Subjects | GS_AE_L_U_002 |
| 11 | Listing of Hematology - SI Units | Appendix 7.1.1A / rl-lb-hems1.lst / SS_LB_L_001 |
| | Treated Subjects | |
| 12 | Listing of Liver Function Tests - SI Units | Appendix 7.1.1B / rl-lb-lfts1.lst / SS_LB_L_001 |
| | Treated Subjects | |
| 13 | Listing of Enzymes - SI Units | Appendix 7.1.1C / rl-lb-enzs1.lst / SS_LB_L_001 |
| | Treated Subjects | |
| 14 | Listing of Renal Function Tests - SI Units | Appendix 7.1.1D / rl-lb-rfts1.lst / SS_LB_L_001 |
| | Treated Subjects | |
| 15 | Listing of Electrolytes - SI Units | Appendix 7.1.1E / rl-lb-elcs1.lst / SS_LB_L_001 |
| | Treated Subjects | |

| Number | Title | BMS Table number/File Name/BMS Template |
|---|---|---|
| 16 | Listing of Fasting Lipids and Glucose – SI Units | Appendix 7.1.1F / rl-lb-flgs1.lst / SS_LB_L_001 |
| | Treated Subjects | |
| 17 | Listing of Hematology - US Unit | Appendix 7.1.1G / rl-zl-hems1.lst / SS_LB_L_001 |
| | Treated Subjects | |
| 18 | Listing of Liver Function Tests - US Unit | Appendix 7.1.1H / rl-zl-lfts1.lst / SS_LB_L_001 |
| | Treated Subjects | |
| 19 | Listing of Enzymes - US Unit | Appendix 7.1.1I / rl-zl-enzs1.lst / SS_LB_L_001 |
| | Treated Subjects | |
| 20 | Listing of Renal Function Tests - US Unit | Appendix 7.1.1J / rl-zl-rfts1.lst / SS_LB_L_001 |
| | Treated Subjects | |
| 21 | Listing of Electrolytes - US Unit | Appendix 7.1.1K / rl-zl-elcs1.lst / SS_LB_L_001 |
| | Treated Subjects | |
| 22 | Listing of Fasting Lipids and Glucose – US Unit | Appendix 7.1.1L / rl-zl-flgs1.lst / SS_LB_L_001 |
| | Treated Subjects | |
| 23 | Listing of Differences in Categorization of SI and US Laboratory | Appendix 7.1.1M / rl-lb-diffunits1.lst / |
| | Test Results Treated Subjects | GS_LB_L_S_008 |
| 24 | Listing of Pregnancy Test | Appendix 7.1.1N / rl-lb-pregs1.lst / GS_LB_L_X_006 |
| | Treated Female Subjects | |
| 25 | Listing of Electrocardiogram | Appendix 7.3.1D / rl-eg-ecgs1.lst / GS_EG_L_X_001 |
| | Treated Subjects | |
| 26 | Listing of Vital Signs | Appendix 7.4.1B / rl-vs-lists1.lst / GS_VS_L_X_006 |
| | Treated Subjects | |

# 3.4. Virology

The Modified Treated Subjects population with available virology data will be used in the summaries and analyses. All treated subjects with available virology data will be used in the data listings.

# 3.4.1. Tables

| Number | Title | BMS Table number/File Name/BMS Template |
|---|---|---|
| 4.1 | Baseline Genotypic Resistance Profile | Table S.3.9.1A / rt-gn-bases1.lst / SS_GN_T_001 |
| | Modified Treated Subjects | |
| 4.2 | Baseline Gag Polymorphisms at Selected Positions | Table S.3.9.1C / rt-gn-bslgags1.lst / SS_GN_T_002 |
| | Modified Treated Subjects | |
| 4.3 | Baseline Gag Polymorphisms at Selected Positions | Table S.3.9.1J / rt-gn-bslgagpdvfs1.lst / SS_GN_T_002 |
| | Modified Treated Subjects Identified as Protocol Defined Virologic | |
| | Failures | |
| 4.4 | Newly Emergent Genotypic Resistance Profile | Table S.5.10.1A / rt-gn-news1.lst / SS_GN_T_001 |
| | Modified Treated Subjects with On-Treatment Genotypic Resistance | |
| | Testing | |
| 4.5 | Newly Emergent Genotypic Resistance Profile | Table S.5.10.1B / rt-gn-newpdvfs1.lst / SS_GN_T_001 |
| | Modified Treated Subjects Identified as Protocol Defined Virologic | |
| | Failures | |
| 4.6 | Emergent Gag Polymorphisms at Selected Positions | Table S.5.10.1C / rt-gn-newgags1.lst / SS_GN_T_002 |
| | Modified Treated Subjects with On-Treatment Gag Sequencing | |
| 4.7 | Emergent Gag Polymorphisms at Selected Positions | Table S.5.10.1D / rt-gn-newgagpdvfs1.lst / |
| | Modified Treated Subjects Identified as Protocol Defined Virologic | SS_GN_T_002 |
| | Failures | |
| Number | Title | BMS Table number/File Name/BMS Template |
|---|---|---|
| 4.8 | Newly Emergent Phenotypic Resistance Profile | Table S.5.10.1G / rt-pn-news1.lst / SS_PN_T_001 |
| | Modified Treated Subjects with On-Treatment Phenotypic Resistance | |
| | Profile | |
| 4.9 | Newly Emergent Phenotypic Resistance Profile | Table S.5.10.1H / rt-pn-newpdvfs1.lst / SS_PN_T_001 |
| | Modified Treated Subjects Identified as Protocol Defined Virologic | |
| | Failures | |

# 3.4.2. Other Listings

| Number | Title | BMS Table number/File Name/BMS Template |
|---|---|---|
| 37 | Listing of Baseline Genotypic Substitutions | Appendix 3.9.1B / rl-gn-bsls1.lst / SS_GN_L_001 |
| | Treated Subjects | |
| 38 | Listing of Baseline Gag Polymorphisms at Selected Positions | Appendix 3.9.1C / rl-gn-gagbsls1.lst / SS_GN_L_002 |
| | Treated Subjects | |
| 39 | Listing of Baseline Gag Deviations from Wild Type Virus | Appendix 3.9.1D / rl-gn-gagbslanys1.lst / |
| | Treated Subjects | SS_GN_L_003 |
| 40 | Listing of Protocol Defined Virologic Failures | Not Available / rl-vl-pdvf.lst / SS_VL_L_006 |
| | Treated Subjects | |
| 41 | Listing of Genotypic Substitutions | Appendix 5.10.1A / rl-gn-ontrts1.lst / SS_GN_L_001 |
| | Treated Subjects with Baseline and On-Treatment Data | |
| 42 | Listing of Gag Polymorphisms at Selected Positions | Appendix 5.10.1B / rl-gn-gagontrts1.lst / |
| | Treated Subjects with Baseline and On-Treatment Data | SS_GN_L_002 |


## Al468038/205891

| Number | Title | BMS Table number/File Name/BMS Template |
|---|---|---|
| 43 | Listing of Newly Emergent Gag Deviations | Appendix 5.10.1C / rl-gn-gagontrts1.lst / |
| | Treated Subjects with Baseline and On-Treatment Data | SS_GN_L_003 |
| 44 | Listing of Phenotypic Resistance | Appendix 5.10.1D / rl-pn-ontrt1.lst / SS_PN_L_001 |
| | Treated Subjects with Baseline and On-Treatment Data | |

# GLOBAL BIOMETRIC SCIENCES ANALYSIS DATA PRESENTATION PLAN

## BMS-955176

# HIV MATURATION INHIBITOR CLINICAL STUDY REPORT FOR AI438-048

**DOCUMENT REVISION: 2.0** 

#### DPP for Al468-048 CSR

#### Version 2.0

| □Initia | al Version (1.0) ${\sf X}$ Significant Revision | n (2.0, etc.) □Minor Revision (1. | 1, etc.) |
|---|---|---|---|
| Prepared by: | Statistician PPD | PPD<br> | Oct 6, 2015 |
| Approved by: | Statistical Programmer (Minor changes are approved by Statistician | Signature<br>per signature above) | Date |
| X<br>Study-Specific<br>DPP | GBS Lead or ED Statistical Lead | Signature | Date |
| | Medical Lead* | Signature | Date |
| Periodic<br>Safety Update | GBS Lead or ED Statistical Lead | Signature | Date |
| DPP | Medical Surveillance Team Chair, GPV&E | Signature | Date |
| Event-Based<br>DPP | GBS Lead or ED Statistical Lead | Signature | Date |
| Core or<br>Integrated | GBS Lead | Signature | Date |
| DPP | Medical Lead | Signature | Date |
| | TA Head, GBS | Signature | Date |
| | Development Lead | Signature | Date |
| Summary of Clinical | TA Head, CP&P | Signature | Date |
| Pharmacology<br>DPP | TA Head, ED GBS | Signature | Date |
| ECTR<br>Standard DPP | GBS Head of ED or designee | Signature | Date |
| | VP, ECTR or designee | Signature | Date |

\*(For ECTR Studies, if there is no Medical Lead, secure approval from the TA Head for Discovery Medicine or Clinical Pharmacology & Pharmacometrics according to the functional area of the Study Director or his/her designee)

10 October 2013 CT DIR GBL 048 FRM 01, Version 01


#### **NEW or MODIFIED**

# **DATA PRESENTATION PLAN**

**APPROVAL PAGE** 

#### DPP for Al468-048 CSR

#### Version 2.0

| □Initia | al Version (1.0) ${\sf X}$ Significant Revisio | on (2.0, etc.) □Minor Revision (1. | 1, etc.) |
|---|---|---|---|
| Deanared by | PPD | | |
| Prepared by: | Statisticlan PPD | . Signature<br>PPD | Date 0ct 15,20 |
| | Statistical Programmer | Signature | Date |
| Approved by: ( | Minor changes are approved by Statisticia | ITPPD | |
| Х | PPD | | 00515,2011 |
| Study-Specific<br>DPP | GBS Lead or ED Statistical Lead | | Date |
| | Medical Lead* | Signature | Date |
| Periodic<br>Safety Update | GBS Lead or ED Statistical Lead | Signature | Date |
| DPP | Medical Surveillance Team Chair, GPV&E | Signature | Date |
| ☐<br>Event-Based | | | |
| DPP | GBS Lead or ED Statistical Lead | Signature | Date |
| ☐<br>Core or | GBS Lead | Signalure | Date |
| Integrated<br>DPP | Medical Lead | Signature | Date |
| | TA Head, GBS | Signature | Date |
| | Development Lead | Signature | Date |
| Summary of Clínical | TA Head, CP&P | Signature | Date |
| Pharmacology<br>DPP | TA Head, ED GBS | Signature | Date |
| ECTR<br>Standard DPP | GBS Head of ED or designee | Signature | Date |
| | VP, ECTR or designee | Signature | Date |

\*(For ECTR Studies, if there is no Medical Lead, secure approval from the TA Head for Discovery Medicine or Clinical Pharmacology & Pharmacometrics according to the functional area of the Study Director or his/her designee)

#### DPP for Al468-048 CSR

## Version 2.0

| □lnitia | l Version (1.0) | X Significant Revision (2.0, | etc.) □Minor | Revision (1.1, etc.) |
|---|---|---|---|---|
| | PPD | | | |

| Prepared by: | | | |
|---|---|---|---|
| | Statistician | Signature | Date |
| | Statistical Programmer | Signature | Date |
| Approved by: ( | (Minor changes are approved by Statistician | | <b></b> |
| | PPD PPD | , por organica | |
| X<br>Study-Specific | GBS Lead or ED Statistical Lead | Signature | Date |
| DPP | | PPD | Dale |
| | PPD | | 10-15-15 |
| | Medical Lead* | Signature | Date |
| | · | | |
| Periodic | GBS Lead or ED Statistical Lead | Signature | Date |
| Safety Update<br>DPP | Madical Consillance Team Chair GDV/8E | Cianatura | |
| — | Medical Surveillance Team Chair, GPV&E | Signature | Date |
| Event-Based | | | |
| DPP | GBS Lead or ED Statistical Lead | Signature | Date |
| Core or | GBS Lead | Signature | Date |
| Integrated<br>DPP | | | |
| טרר | Medical Lead | Signature | Date |
| | TAIL4 ODG | Olympia. | |
| | TA Head, GBS | Signature | Date |
| | Development Lead | Signature | Date |
| | · | | |
| Summary of | TA Head, CP&P | Signature | Date |
| Clinical | | <del>-</del> | |
| Pharmacology<br>DPP | TA Head, ED GBS | Signature | Date |
| ECTR | GBS Head of ED or designee | Signature | Date |
| Standard DPP | | | |
| | VP, ECTR or designee | Signature | Date |

# **REVISION HISTORY**

| Revision | Date | Revised By | Changes Made Reasons for the Change |
|---|---|---|---|
| 1.0 | July 16, 2015 | PPD | Original issue |
| 2.0 | Oct 6, 2015 | PPD | Additional outputs for baseline resistance have been added based on the revised SAP v2.0 (see Tables S.3.9.xH-R) |
| | | | Additional outputs for on-treatment resistance have been added based on the revised SAP v2.0 (see Tables S.5.10.xR-W). |
| | | | Integrated outputs have been added as described in the revised SAP v2.0. |
| | | | Update the schedule of analysis: Week 48 Stage 1 interim analysis only if continuation dose cannot be selected based on Week 24, Stage 1 results. The Week 96 Stage 1 will be performed at the time of Week 24 Stage 2. |

# **TABLE OF CONTENTS**

| ANALY | SIS DATA PRESENTATION PLAN | 1 |
|-------|------------------------------------------------------------|-----|
| TABLE | OF CONTENTS | 3 |
| TABLE | OF CONTENTS: TEMPLATES | 5 |
| 1 | LIST OF DATA PRESENTATIONS | 8 |
| 1.1 | Codes Used for Deliverables | 8 |
| 1.2 | List | 8 |
| 2 | INTRODUCTION | 58 |
| 2.1 | Guidance for DPP Users and Reviewers | 58 |
| 2.2 | Referenced Documents | 58 |
| 3 | GENERAL CRITERIA/CONVENTIONS | 59 |
| 3.1 | Exceptions to Global and/or Departmental Standards | 59 |
| 3.2 | Populations | 59 |
| 3.3 | Conventions | 60 |
| 3.4 | Treatment Information | 60 |
| 3.5 | Graph Criteria/Conventions | 60 |
| 4 | PRESENTATION PLAN TEMPLATES AND METADATA | 62 |
| 4.1 | Administrative Appendices | 62 |
| 4.2 | Study Conduct | 66 |
| 4.2.1 | Protocol Deviations | 66 |
| 4.3 | Study Population | 69 |
| 4.3.1 | Disposition of Subjects | 69 |
| 4.3.2 | Demographics and Baseline Characteristics | 85 |
| 4.3.3 | Medical History and Previous Treatments | 147 |
| 4.4 | Extent Of Exposure. | 153 |
| 4.4.1 | Study Therapy and Treatment Compliance | 153 |
| 4.4.2 | Concomitant Therapy | 170 |
| 4.5 | Efficacy Results | 172 |
| 4.6 | Safety Results | 279 |
| 4.6.1 | All Adverse Events | 279 |
| 4.6.2 | Deaths | 281 |
| 4.6.3 | Serious Adverse Events | 282 |
| 4.6.4 | Adverse Events Leading to Discontinuation of Study Therapy | 289 |

| 4.6.5 | Other Significant Adverse Events | 294 |
|--------|--------------------------------------|-----|
| 4.6.6 | Multiple Adverse Events | 307 |
| 4.6.7 | Clinical Laboratory Evaluations | 316 |
| 4.6.8 | Electrocardiograms | 346 |
| 4.6.9 | Vital Signs and Physical Findings | 354 |
| 4.6.10 | Other Observations Related to Safety | 358 |
| 4.7 | Pharmacokinetic Results | 369 |
| 4.8 | Pharmacodynamic Results | 406 |
| 4.9 | Other Study Results | 406 |

# TABLE OF CONTENTS: TEMPLATES

| Template SS_EX_L_001: Batch Number Listing | 63 |
|---|---|
| Template SS_DS_L_001: Randomization Scheme and Codes | 64 |
| Template SS_DM_T_001: Accrual Summary | 65 |
| Template SS_PD_T_001: Relevant Protocol Deviation Summary | 67 |
| Template SS_PD_L_001: Relevant Protocol Deviation Listing | 68 |
| Template GS_DS_T_T_001: Pre-Randomization Subject Status | 70 |
| Template GS_DS_L_S_001: Pre-randomization Subject Status Listing | 72 |
| Template GS_DM_T_T_005 : Enrollment Summary | 74 |
| Template SS_DM_T_002: Counts and Percentages Table | 76 |
| Template GS_DS_T_X_005 : End of Study Subjects Status | 78 |
| Template GS_DS_L_X_005: End of Study Subject Status by Treatment Group | 80 |
| Template SS_DM_T_002 : Population Summary | 82 |
| Template SS_DM_L_001: Listing of Subjects Excluded from the Efficacy Analysis | 84 |
| Template GS_DM_T_X_002: Demographic Characteristics Summary (incl. 'Not reported' category) | 86 |
| Template GS_DM_T_T_002: Demographic Characteristics Summary (incl. 'Not reported' category) | 89 |
| Template GS_DM_L_X_001: Demographics Listing by Treatment Group | 91 |
| Template SS_DM_T_004 : Baseline Disease Characteristics | 93 |
| Template SS_DM_L_002: Listing of HIV Disease Characteristics | 97 |
| Template GS_PM_T_X_001: Physical Measurements Table | 99 |
| Template GS_PE_T_X_001: Physical Examination by Treatment Group | 101 |
| Template GS_PE_L_X_001 : Physical Examination Listing by Treatment Group | 103 |
| Template SS_GN_T_001: Baseline Genotypic Resistance Profile | 105 |
| Template SS_GN_L_001:Genotypic Resistance Listing | 109 |
| Template SS_GN_T_002: Baseline Gag Polymorphisms at Selected Positions | 111 |
| Template SS_GN_T_003: Baseline Gag Deviations from Wild Type | 119 |
| Template SS_GN_L_002: Gag Listing for Selected Positions | 128 |
| Template SS_GN_L_003: Gag Listing of Deviations from the Wild Type Virus | 130 |
| Template SS_PN_T_001: Baseline Phenotypic Resistance Categories | 132 |
| Template SS_PN_T_002: Phenotypic Resistance by Class and Drug Name | 137 |
| Template SS PN L 001: Phenotypic Resistance Listing | 142 |

| Template GS_LB_T_X_004: Laboratory Toxicity Grade Summary | 144 |
|---|---|
| Template GS_AE_T_X_001: Adverse Event Summary by System Organ Class and Preferred Term | 146 |
| Template GS_MH_T_X_001: Medical History Summary | |
| Template GS_MH_L_X_001: Medical History Listing by Treatment Group | |
| Template GS_CM_T_X_001 : Non-Study Medication Summary | |
| Template SS_EX_T_001: Extent of Exposure Summary | |
| Template GS EX G 001: Kaplan-Meier Plot Grouped by Treatment with Censoring | |
| Template SS_EX_T_002: Time on Study Therapy Life Table | |
| Template SS_EX_T_003: Summary of Interruptions Greater than 3 Days | |
| Template SS_EX_L_001: Study Medication Exposure Listing | 167 |
| Template SS_EX_L_002: Study Medication Listing related to Continuation Dose | 169 |
| Template GS_CM_L_X_006: Non-Study Medication Listing by Treatment Group | 171 |
| Template SS_VL_T_001: Detailed Summary of HIV-1 < Y (by Subgroup) | 173 |
| Template SS_VL_T_002: Summary of HIV-1 < Y (by Subgroup) | 175 |
| Template SS_VL_T_003: Proportion of Responders (Observed) | 199 |
| Template SS_VL_T_004: Treatment Outcomes Table Using the TLOVR Algorithm | 207 |
| Template SS_VL_T_005: Proportion of Subjects with HIV-1 RNA within Certain Range | 213 |
| Template SS_VL_T_006 : Summary Statistics Over Time | 215 |
| Template GS_LB_G_001: Box Plot | 222 |
| Template GS_L_G_002: Longitudinal Line Plot Grouped by Treatment with Horizontal Shift and Reference Line | 231 |
| Template SS_VL_L_004: Listing of Outcomes from Snapshot Analysis | 235 |
| Template SS_VL_L_005: Listing of Viral Load | 239 |
| Template SS_LB_L_002: Listing of CD4 and CD8 | 241 |
| Template SS_PN_T_003: Maximum Change in IC50 Summary | 265 |
| Template SS_PN_T_004: Proportion of Subjects with > 3 Fold Increase in IC50 Fold Change | 270 |
| Template SS_VL_T_007: Proportion of Responders (mITT) - Futility Analysis | 278 |
| Template SS_AE_T_001: Overall Adverse Events Summary | 280 |
| Template SS_AE_L_001: Listing of Death | 282 |
| Template GS_AE_L_S_001: Adverse Event Listing (by Subject) | 287 |
| Template GS_AE_L_X_001: Adverse Event Listing (by Treatment Group) | 292 |

| Template GS_AE_T_M_001: Exposure Adjusted Adverse Events Summary by SOC and | |
|---|---|
| Preferred Term | 308 |
| Template GS_AE_L_U_002: Unique Adverse Event Listing | 314 |
| Template SS_LB_T_001: Laboratory Test Worst Abnormalities Table by Baseline | 317 |
| Template SS_LB_T_002: Laboratory Test Treatment Emergent Abnormalities Table | 320 |
| Template SS_LB_L_001: Laboratory Test Results Listing With Toxicity Grades | 331 |
| Template GS_LB_L_S_008: Differences in Categorization of SI and US units | 343 |
| Template GS_LB_L_X_006: Pregnancy Listing by Treatment Group | 345 |
| Template SS_EG_T_003 : ECG Summary Table with 95% CI | 347 |
| Template SS_EG_T_001 : ECG Change from Baseline Category Summary | 349 |
| Template SS_EG_T_002: ECG Category Summary | 351 |
| Template GS_EG_L_X_001: ECG Listing | 353 |
| Template GS_VS_L_X_006: Vital Signs Listing by Treatment Group | 356 |
| Template MS_PK_T_004: Summary Statistics for PK Parameters | 369 |
| Template MS_PK_T_005: In-text Table for Summary Statistics for PK Parameters | 373 |
| Template MS_PK_T_006: Statistical Analysis for PK Parameters | 377 |
| Template MS_PK_T_007: In-text Table for Statistical Analysis for PK Parameters | 379 |
| Template MS_PK_L_005: Listing for PK Parameters | 382 |
| Template MS_PK_L_001: Listing of Plasma Concentration-Time Data | 386 |
| Template MS_PK_G_002: Individual Plot of Plasma Concentrations vs. Time | 390 |
| Template MS_PK_G_001: Overlay of Individual Matrix Concentration vs. Time | 396 |
| Template MS_PK_G_006: Mean Plot of Matrix Concentration vs. Time | 401 |

## 1 LIST OF DATA PRESENTATIONS

## 1.1 Codes Used for Deliverables

| Code | Description |
|---|---|
| WK24S1 | Interim Analysis Week 24, Stage 1 |
| WK48S1 | Interim Analysis Week 48, Stage 1* |
| WK96S1 | Final Analysis Week 96, Stage 1 (most likely at the time of Interim Analysis Week 24, Stage 2) |
| WK24S2 | Interim Analysis Week 24, Stage 2 |
| WK48S2 | Interim Analysis Week 48, Stage 2 |
| WK96S2 | Final Analysis Week 96, Stage 2 |

<sup>\*</sup> The Week 48, Stage 1 interim analysis would only be performed in case a continuation dose cannot be selected based on the Week 24, Stage 1 interim analysis.

**Note:** in order to make the distinction between the different database locks for each stage, the table numbers should have '-Wkxx' attached to the table numbers mentioned in the rest of the DPP. For example, Table S.2.3.1A will become Table S.2.3.1A-Wk24 for the Stage 1 Week 24 interim analysis. Table S.2.3.2A will become Table S.2.3.2A-Wk48 for the Stage 2 Week 48 analysis.

#### 1.2 **List**

| No. | Table No. | Output File<br>Name | Template ID | Title and Population | Purpose |
|---|---|---|---|---|---|
| 1 | Appendix 1.7.1 | rl-ex-batchs1.lst | SS_EX_L_001 | Listing of Batch Numbers<br>Treated Subjects - Stage 1 | WK24S1,<br>WK48S1, |
| | | | | | WK96S1,<br>WK96S2 |
| 2 | Appendix 1.7.2 | rl-ex-batchs2.lst | SS_EX_L_001 | Listing of Batch Numbers<br>Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 3 | Appendix 1.9.1 | rl-ds-<br>randcodes1.lst | SS_DS_L_001 | Randomization Scheme and<br>Codes<br>Randomized Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 4 | Appendix 1.9.2 | rl-ds-<br>randcodes2.lst | SS_DS_L_001 | Randomization Scheme and<br>Codes<br>Randomized Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 5 | Appendix<br>2.1.1E | rt-dm-accruals1.lst | SS_DM_T_001 | Accrual Summary Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 6 | Appendix 2.1.2E | rt-dm-accruals2.lst | SS_DM_T_001 | Accrual Summary Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |

| No. | Table No. | Output File<br>Name | Template ID | Title and Population | Purpose |
|---|---|---|---|---|---|
| 7 | Table S.2.3.1A | rt-pd-rels1.lst | SS_PD_T_001 | Relevant Protocol Deviation<br>Summary | WK24S1,<br>WK48S1, |
| | | | | Randomized Subjects - Stage 1 | WK96S1,<br>WK96S2 |
| 8 | Table S.2.3.2A | rt-pd-rels2.lst | SS_PD_T_001 | Relevant Protocol Deviation | WK24S2, |
| | | | | Summary<br>Randomized Subjects - Stage 2 | WK48S2,<br>WK96S2 |
| 9 | Table S.2.3.1B | rl-pd-rels1.lst | SS PD L 001 | Listing of Relevant Protocol | WK24S1, |
| | | F | | Deviations | WK48S1, |
| | | | | Randomized Subjects - Stage 1 | WK96S1, |
| 10 | T.11 C.2.2.2D | 1 1 101 | GG DD I 001 | Titi CD 1 (D ) | WK96S2 |
| 10 | Table S.2.3.2B | rl-pd-rels2.lst | SS_PD_L_001 | Listing of Relevant Protocol Deviations | WK24S2,<br>WK48S2, |
| | | | | Randomized Subjects - Stage 2 | WK46S2,<br>WK96S2 |
| 11 | Table S.2.1.1A | rt-ds-prerands1.lst | GS DS T T 001 | Pre-Randomization Subject | WK24S1, |
| | | p | 00_00_0 | Status | WK48S1, |
| | | | | Enrolled Subjects - Stage 1 | WK96S1, |
| | | | | | WK96S2 |
| 12 | Table S.2.1.2A | rt-ds-prerands2.lst | GS_DS_T_T_001 | Pre-Randomization Subject | WK24S2, |
| | | | | Status Enrolled Subjects - Stage 2 | WK48S2,<br>WK96S2 |
| 13 | Appendix | rl-ds-prerands1.lst | GS DS L S 001 | Pre-Randomized Subject Status | WK24S1, |
| 13 | 2.1.1A | 11-us-preranus1.ist | US_DS_L_S_001 | Enrolled Subjects - Stage 1 | WK2451,<br>WK48S1, |
| | 2.1.111 | | | Emoneu Suojeets Suige 1 | WK96S1, |
| | | | | | WK96S2 |
| 14 | Appendix | rl-ds-prerands2.lst | GS_DS_L_S_001 | Pre-Randomized Subject Status | WK24S2, |
| | 2.1.2A | | | Enrolled Subjects - Stage 2 | WK48S2, |
| 1.5 | A di | rt-dm- | CC DM T T 005 | Engellmant Common | WK96S2 |
| 15 | Appendix 2.1.1C | rt-am-<br>enrolls1eu.lst | GS_DM_T_T_005 | Enrollment Summary<br>Number of Subjects at Each | WK24S1,<br>WK48S1, |
| | 2.1.10 | Cinons i cu.ist | | Study Site by Country | WK96S1, |
| | | | | Enrolled Subjects - Stage 1 | WK96S2 |
| 16 | Appendix | rt-dm- | GS_DM_T_T_005 | Enrollment Summary | WK24S2, |
| | 2.1.2C | enrolls2eu.lst | | Number of Subjects at Each | WK48S2, |
| | | | | Study Site by Country | WK96S2 |
| 17 | A a di | | CC DM T 002 | Enrolled Subjects - Stage 2 | WIZ 24C 1 |
| 1 / | Appendix 2.1.1D | rt-dm-<br>enrages1eu.lst | SS_DM_T_002 | Enrollment Summary<br>Number of Subjects per Age | WK24S1,<br>WK48S1, |
| | 2.1.1D | emages reu.ist | | Group | WK46S1,<br>WK96S1, |
| | | | | Enrolled Subjects - Stage 1 | WK96S2 |
| 18 | Appendix | rt-dm- | SS_DM_T_002 | Enrollment Summary | WK24S2, |
| | 2.1.2D | enrages2eu.lst | | Number of Subjects per Age | WK48S2, |
| | | | | Group | WK96S2 |
| 10 | T.1.1. C 2 1 1D | | | Enrolled Subjects - Stage 2 | WWAAC1 |
| 19 | Table S.2.1.1B | rt-ds-statuss1.lst | GS_DS_T_X_005 | End of Study Subject Status | WK24S1, |
| | | | | Summary<br>Randomized Subjects - Stage 1 | WK48S1,<br>WK96S1, |
| | | | | Randonnized Subjects - Stage 1 | WK96S1,<br>WK96S2 |
| 20 | Table S.2.1.2B | rt-ds-statuss2.lst | GS DS T X 005 | End of Study Subject Status | WK24S2, |
| | | | | Summary | WK48S2, |
| | | | | Randomized Subjects - Stage 2 | WK96S2 |

| No. | Table No. | Output File<br>Name | Template ID | Title and Population | Purpose |
|---|---|---|---|---|---|
| 21 | Table S.2.1.3B | rt-ds-statuss12.lst | GS_DS_T_X_005 | End of Study Subject Status<br>Summary<br>Randomized Subjects - Stage 1<br>and 2 | WK96S2 |
| 22 | Appendix<br>2.1.1B | rl-ds-statuss1.lst | GS_DS_L_X_005 | End of Study Subject Status<br>Randomized Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 23 | Appendix 2.1.2B | rl-ds-statuss2.lst | GS_DS_L_X_005 | End of Study Subject Status<br>Randomized Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 24 | Table S.2.1.1C | rt-dm-<br>populations l .lst | SS_DM_T_002 | Populations for Analysis<br>Summary - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 25 | Table S.2.1.2C | rt-dm-<br>populations2.lst | SS_DM_T_002 | Populations for Analysis<br>Summary - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 26 | Appendix 2.2.1 | rl-dm-excls1.lst | SS_DM_L_001 | Subjects Excluded from<br>Efficacy Analysis (mITT)<br>Randomized Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 27 | Appendix 2.2.2 | rl-dm-excls2.lst | SS_DM_L_001 | Subjects Excluded from<br>Efficacy Analysis (mITT)<br>Randomized Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 28 | Table S.3.1.1 | rt-dm-<br>summarys1.lst | GS_DM_T_X_002 | Demographic Characteristics Summary Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 29 | Table S.3.1.2 | rt-dm-<br>summarys2.lst | GS_DM_T_X_002 | Demographic Characteristics Summary Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 30 | Table S.3.1.3 | rt-dm-<br>summarys12.lst | GS_DM_T_X_002 | Demographic Characteristics Summary Treated Subjects - Stage 1 and 2 | WK96S2 |
| 31 | Appendix 3.1.1B | rt-dm-<br>sumenrolls1.lst | GS_DM_T_T_002 | Demographic Characteristics Summary Subjects Enrolled but Not Randomized - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 32 | Appendix 3.1.2B | rt-dm-<br>sumenrolls2.lst | GS_DM_T_T_002 | Demographic Characteristics Summary Subjects Enrolled but Not Randomized - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 33 | Appendix<br>3.1.1A | rl-dm-<br>demchars1.lst | GS_DM_L_X_001 | Demographic Characteristics<br>Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 34 | Appendix 3.1.2A | rl-dm-<br>demchars2.lst | GS_DM_L_X_001 | Demographic Characteristics<br>Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |

| No. | Table No. | Output File<br>Name | Template ID | Title and Population | Purpose |
|---|---|---|---|---|---|
| 35 | Table S.3.2.1 | rt-dm-diseases1.lst | SS_DM_T_004 | Summary of Baseline Disease<br>Characteristics<br>Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1, |
| 36 | Table S.3.2.2 | rt-dm-diseases2.lst | SS_DM_T_004 | Summary of Baseline Disease Characteristics Treated Subjects - Stage 2 | WK96S2<br>WK24S2,<br>WK48S2,<br>WK96S2 |
| 37 | Table S.3.2.3 | rt-dm-<br>diseases12.lst | SS_DM_T_004 | Summary of Baseline Disease Characteristics Treated Subjects - Stage 1 and 2 | WK96S2 |
| 38 | Appendix 3.2.1A | rt-dm-<br>diseasenrands1.lst | SS_DM_T_004 | Summary of Baseline Disease Characteristics Subjects Enrolled but Not Randomized - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 39 | Appendix 3.2.2A | rt-dm-<br>diseasenrands2.lst | SS_DM_T_004 | Summary of Baseline Disease Characteristics Subjects Enrolled but Not Randomized - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 40 | Appendix<br>3.2.1B | rl-dm-diseases1.lst | SS_DM_L_002 | Listing of HIV Disease Characteristics Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 41 | Appendix 3.2.2B | rl-dm-diseases2.lst | SS_DM_L_002 | Listing of HIV Disease Characteristics Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 42 | Table S.3.3.1 | rt-pm-bsls1.lst | GS_PM_T_X_001 | Physical Measurements Summary Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 43 | Table S.3.3.2 | rt-pm-bsls2.lst | GS_PM_T_X_001 | Physical Measurements Summary Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 44 | Table S.3.4.1 | rt-pe-bslsums1.lst | GS_PE_T_X_001 | Physical Examination Summary Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 45 | Table S.3.4.2 | rt-pe-bslsums2.lst | GS_PE_T_X_001 | Physical Examination Summary<br>Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 46 | Appendix 3.4.1 | rl-pe-lists1.lst | GS_PE_L_X_001 | Physical Examination<br>Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 47 | Appendix 3.4.2 | rl-pe-lists2.lst | GS_PE_L_X_001 | Physical Examination<br>Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 48 | Table S.3.9.1A | rt-gn-bases1.lst | SS_GN_T_001 | Baseline Genotypic Resistance Profile Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 49 | Table S.3.9.2A | rt-gn-bases2.lst | SS_GN_T_001 | Baseline Genotypic Resistance<br>Profile<br>Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |

| No. | Table No. | Output File<br>Name | Template ID | Title and Population | Purpose |
|---|---|---|---|---|---|
| 50 | Table S.3.9.3A | rt-gn-bases12.lst | SS_GN_T_001 | Baseline Genotypic Resistance Profile | WK96S2 |
| <i>7</i> 1 | A 1' | , | CC CN T 001 | Treated Subjects - Stage 1 and 2 | WW2401 |
| 51 | Appendix | rt-gn- | SS_GN_T_001 | Baseline Genotypic Resistance | WK24S1, |
| | 3.9.1A | basebysubtypes1.ls | | Profile | WK48S1, |
| | | ι | | By HIV Subtype | WK96S1, |
| 52 | Annandin | ut on | CC CN T 001 | Treated Subjects - Stage 1 | WK96S2 |
| 32 | Appendix 3.9.2A | rt-gn- | SS_GN_T_001 | Baseline Genotypic Resistance<br>Profile | WK24S2, |
| | 3.9.2A | basebysubtypes2.ls | | | WK48S2,<br>WK96S2 |
| | | ι | | By HIV Subtype Treated Subjects - Stage 2 | W K9052 |
| 53 | Table S.3.9.1B | rt-gn-baseots1.lst | SS_GN_T_001 | Baseline Genotypic Resistance | WK24S1, |
| 33 | 14010 5.5.7.11 | 1t-gii-0ascots1.ist | 35_011_1_001 | Profile | WK2451,<br>WK48S1, |
| | | | | Treated Subjects with On- | WK96S1, |
| | | | | Treatment Resistance Testing - | WK96S2 |
| | | | | Stage 1 | W112 0B2 |
| 54 | Table S.3.9.2B | rt-gn-baseots2.lst | SS GN T 001 | Baseline Genotypic Resistance | WK24S2, |
| | 14010 5.5.5.2 | 10 gii 0460002.160 | 22_01\_1_001 | Profile | WK48S2, |
| | | | | Treated Subjects with On- | WK96S2 |
| | | | | Treatment Resistance Testing - | |
| | | | | Stage 2 | |
| 55 | Appendix | rl-gn-bsls1.lst | SS GN L 001 | Listing of Baseline Genotypic | WK24S1, |
| | 3.9.1B | 8 11 1 11 | | Substitutions | WK48S1, |
| | | | | Treated Subjects - Stage 1 | WK96S1, |
| | | | | , , , | WK96S2 |
| 56 | Appendix | rl-gn-bsls2.lst | SS_GN_L_001 | Listing of Baseline Genotypic | WK24S2, |
| | 3.9.2B | _ | | Substitutions | WK48S2, |
| | | | | Treated Subjects - Stage 2 | WK96S2 |
| 57 | Table S.3.9.1C | rt-gn-bslgags1.lst | SS_GN_T_002 | Baseline Gag Polymorphisms at | WK24S1, |
| | | | | Selected Positions | WK48S1, |
| | | | | Treated Subjects - Stage 1 | WK96S1, |
| | | | | | WK96S2 |
| 58 | Table S.3.9.2C | rt-gn-bslgags2.lst | SS_GN_T_002 | Baseline Gag Polymorphisms at | WK24S2, |
| | | | | Selected Positions | WK48S2, |
| | | | | Treated Subjects - Stage 2 | WK96S2 |
| 59 | Table S.3.9.3C | rt-gn-bslgags12.lst | SS_GN_T_002 | Baseline Gag Polymorphisms at | WK96S2 |
| | | | | Selected Positions | |
| | | | | Treated Subjects - Stage 1 and 2 | |
| 60 | Table S.3.9.1D | rt-gn- | SS_GN_T_002 | Baseline Gag Polymorphisms at | WK24S1, |
| | | bslgagbysubtypes1 | | Selected Positions | WK48S1, |
| | | .lst | | By HIV Subtype | WK96S1, |
| <i>C</i> 1 | T-1-0202D | 4 | CC CN T 000 | Treated Subjects - Stage 1 | WK96S2 |
| 61 | Table S.3.9.2D | rt-gn- | SS_GN_T_002 | Baseline Gag Polymorphisms at | WK24S2, |
| | | bslgagbysubtypes2 | | Selected Positions | WK48S2, |
| | | .lst | | By HIV Subtype | WK96S2 |
| 62 | Table C 2 0 2D | sub c | CC CN T 002 | Treated Subjects - Stage 2 | WWOGGO |
| 62 | Table S.3.9.3D | rt-gn- | SS_GN_T_002 | Baseline Gag Polymorphisms at | WK96S2 |
| | | bslgagbysubtypes1 | | Selected Positions By HIV Subtype | |
| | | 2.lst | | | |
| | | | | Treated Subjects - Stage 1 and 2 | |

| No. | Table No. | Output File<br>Name | Template ID | Title and Population | Purpose |
|---|---|---|---|---|---|
| 63 | Table S.3.9.1H | rt-gn-<br>bslgagontrts1.lst | SS_GN_T_002 | Baseline Gag Polymorphisms at Selected Positions Treated Subjects with On- Treatment Resistance Testing - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 64 | Table S.3.9.2H | rt-gn-<br>bslgagontrts2.lst | SS_GN_T_002 | Baseline Gag Polymorphisms at Selected Positions Treated Subjects with On- Treatment Resistance Testing - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 65 | Table S.3.9.3H | rt-gn-<br>bslgagontrts12.lst | SS_GN_T_002 | Baseline Gag Polymorphisms at Selected Positions Treated Subjects with On- Treatment Resistance Testing - Stage 1 and 2 | WK96S2 |
| 66 | Table S.3.9.1I | rt-gn-<br>bslgagontrtbysubty<br>pes1.lst | SS_GN_T_002 | Baseline Gag Polymorphisms at Selected Positions By HIV Subtype Treated Subjects with On- Treatment Resistance Testing - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 67 | Table S.3.9.2I | rt-gn-<br>bslgagontrtbysubty<br>pes2.lst | SS_GN_T_002 | Baseline Gag Polymorphisms at Selected Positions By HIV Subtype Treated Subjects with On- Treatment Resistance Testing - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 68 | Table S.3.9.3I | rt-gn-<br>bslgagontrtbysubty<br>pes12.lst | SS_GN_T_002 | Baseline Gag Polymorphisms at Selected Positions By HIV Subtype Treated Subjects with On- Treatment Resistance Testing - Stage 1 and 2 | WK96S2 |
| 69 | Table S.3.9.1J | rt-gn-<br>bslgagpdvfs1.lst | SS_GN_T_002 | Baseline Gag Polymorphisms at Selected Positions Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 70 | Table S.3.9.2J | rt-gn-<br>bslgagpdvfs2.lst | SS_GN_T_002 | Baseline Gag Polymorphisms at<br>Selected Positions<br>Treated Subjects Identified as<br>Protocol Defined Virologic<br>Failures - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 71 | Table S.3.9.3J | rt-gn-<br>bslgagpdvfs12.lst | SS_GN_T_002 | Baseline Gag Polymorphisms at<br>Selected Positions<br>Treated Subjects Identified as<br>Protocol Defined Virologic<br>Failures - Stage 1 and 2 | WK96S2 |

| No. | Table No. | Output File<br>Name | Template ID | Title and Population | Purpose |
|---|---|---|---|---|---|
| 72 | Table S.3.9.1K | rt-gn-<br>bslgagpdvfbysubty<br>pes1.lst | SS_GN_T_002 | Baseline Gag Polymorphisms at Selected Positions By HIV Subtype Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 73 | Table S.3.9.2K | rt-gn-<br>bslgagpdvfbysubty<br>pes2.lst | SS_GN_T_002 | Baseline Gag Polymorphisms at Selected Positions By HIV Subtype Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 74 | Table S.3.9.3K | rt-gn-<br>bslgagpdvfbysubty<br>pes12.lst | SS_GN_T_002 | Baseline Gag Polymorphisms at Selected Positions By HIV Subtype Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 1 and 2 | WK96S2 |
| 75 | Table S.3.9.1E | rt-gn-<br>bslgaganys1.lst | SS_GN_T_003 | Baseline Gag Deviations from<br>Wild Type Virus<br>Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 76 | Table S.3.9.2E | rt-gn-<br>bslgaganys2.lst | SS_GN_T_003 | Baseline Gag Deviations from<br>Wild Type Virus<br>Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 77 | Table S.3.9.3E | rt-gn-<br>bslgaganys12.lst | SS_GN_T_003 | Baseline Gag Deviations from<br>Wild Type Virus<br>Treated Subjects - Stage 1 and 2 | WK96S2 |
| 78 | Table S.3.9.1L | rt-gn-<br>bslgaganybysubtyp<br>es1.lst | SS_GN_T_003 | Baseline Gag Deviations from Wild Type Virus By HIV Subtype Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 79 | Table S.3.9.2L | rt-gn-<br>bslgaganybysubtyp<br>es2.lst | SS_GN_T_003 | Baseline Gag Deviations from Wild Type Virus By HIV Subtype Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 80 | Table S.3.9.3L | rt-gn-<br>bslgaganybysubtyp<br>es12.lst | SS_GN_T_003 | Baseline Gag Deviations from Wild Type Virus By HIV Subtype Treated Subjects - Stage 1 and 2 | WK96S2 |
| 81 | Table S.3.9.1M | rt-gn-<br>bslgaganyontrts1.ls<br>t | SS_GN_T_003 | Baseline Gag Deviations from Wild Type Virus Treated Subjects with On- Treatment Resistance Testing - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 82 | Table S.3.9.2M | rt-gn-<br>bslgaganyontrts2.ls<br>t | SS_GN_T_003 | Baseline Gag Deviations from Wild Type Virus Treated Subjects with On- Treatment Resistance Testing - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |

| No. | Table No. | Output File<br>Name | Template ID | Title and Population | Purpose |
|---|---|---|---|---|---|
| 83 | Table S.3.9.3M | rt-gn-<br>bslgaganyontrts12.<br>lst | SS_GN_T_003 | Baseline Gag Deviations from Wild Type Virus Treated Subjects with On- Treatment Resistance Testing - Stage 1 and 2 | WK96S2 |
| 84 | Table S.3.9.1N | rt-gn-<br>bslgaganyontrtbysu<br>btypes1.lst | SS_GN_T_003 | Baseline Gag Deviations from Wild Type Virus By HIV Subtype Treated Subjects with On- Treatment Resistance Testing - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 85 | Table S.3.9.2N | rt-gn-<br>bslgaganyontrtbysu<br>btypes2.lst | SS_GN_T_003 | Baseline Gag Deviations from Wild Type Virus By HIV Subtype Treated Subjects with On- Treatment Resistance Testing - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 86 | Table S.3.9.3N | rt-gn-<br>bslgaganyontrtbysu<br>btypes12.lst | SS_GN_T_003 | Baseline Gag Deviations from Wild Type Virus By HIV Subtype Treated Subjects with On- Treatment Resistance Testing - Stage 1 and 2 | WK96S2 |
| 87 | Table S.3.9.10 | rt-gn-<br>bslgaganypdvfs1.ls<br>t | SS_GN_T_003 | Baseline Gag Deviations from Wild Type Virus Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 88 | Table S.3.9.2O | rt-gn-<br>bslgaganypdvfs2.ls<br>t | SS_GN_T_003 | Baseline Gag Deviations from Wild Type Virus Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 89 | Table S.3.9.3O | rt-gn-<br>bslgaganypdvfs12.1<br>st | SS_GN_T_003 | Baseline Gag Deviations from Wild Type Virus Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 1 and 2 | WK96S2 |
| 90 | Table S.3.9.1P | rt-gn-<br>bslgaganypdvfbysu<br>btypes1.lst | SS_GN_T_003 | Baseline Gag Deviations from Wild Type Virus By HIV Subtype Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 91 | Table S.3.9.2P | rt-gn-<br>bslgaganypdvfbysu<br>btypes2.lst | SS_GN_T_003 | Baseline Gag Deviations from Wild Type Virus By HIV Subtype Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |

| No. | Table No. | Output File<br>Name | Template ID | Title and Population | Purpose |
|---|---|---|---|---|---|
| 92 | Table S.3.9.3P | rt-gn-<br>bslgaganypdvfbysu<br>btypes12.lst | SS_GN_T_003 | Baseline Gag Deviations from Wild Type Virus By HIV Subtype Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 1 and 2 | WK96S2 |
| 93 | Appendix<br>3.9.1C | rl-gn-gagbsls1.lst | SS_GN_L_002 | Listing of Baseline Gag Polymorphisms at Selected Positions Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 94 | Appendix<br>3.9.2C | rl-gn-gagbsls2.lst | SS_GN_L_002 | Listing of Baseline Gag Polymorphisms at Selected Positions Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 95 | Appendix<br>3.9.1D | rl-gn-<br>gagbslanys1.lst | SS_GN_L_003 | Listing of Baseline Gag Deviations from Wild Type Virus Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 96 | Appendix<br>3.9.2D | rl-gn-<br>gagbslanys2.lst | SS_GN_L_003 | Listing of Baseline Gag Deviations from Wild Type Virus Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 97 | Table S.3.9.1F | rt-pn-bsls1.lst | SS_PN_T_001 | Baseline Phenotypic Resistance Categories Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 98 | Table S.3.9.2F | rt-pn-bsls2.lst | SS_PN_T_001 | Baseline Phenotypic Resistance Categories Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 99 | Table S.3.9.3F | rt-pn-bsls12.lst | SS_PN_T_001 | Baseline Phenotypic Resistance<br>Categories<br>Treated Subjects - Stage 1 and 2 | WK96S2 |
| 100 | Table S.3.9.1G | rt-pn-bslots1.lst | SS_PN_T_001 | Baseline Phenotypic Resistance Categories Treated Subjects with On- Treatment Resistance Testing - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 101 | Table S.3.9.2G | rt-pn-bslots2.lst | SS_PN_T_001 | Baseline Phenotypic Resistance Categories Treated Subjects with On- Treatment Resistance Testing - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 102 | Table S.3.9.3G | rt-pn-bslots12.lst | SS_PN_T_001 | Baseline Phenotypic Resistance Categories Treated Subjects with On- Treatment Resistance Testing - Stage 1 and 2 | WK96S2 |
| 103 | Table S.3.9.1Q | rt-pn-bslpdvfs1.lst | SS_PN_T_001 | Baseline Phenotypic Resistance Categories Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |

| No. | Table No. | Output File<br>Name | Template ID | Title and Population | Purpose |
|---|---|---|---|---|---|
| 104 | Table S.3.9.2Q | rt-pn-bslpdvfs2.lst | SS_PN_T_001 | Baseline Phenotypic Resistance Categories Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 105 | Table S.3.9.3Q | rt-pn-<br>bslpdvfs12.lst | SS_PN_T_001 | Baseline Phenotypic Resistance Categories Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 1 and 2 | WK96S2 |
| 106 | Table S.3.9.1H | rt-pn-bsldrugs1.lst | SS_PN_T_002 | Baseline Phenotypic Resistance<br>by Class and Drug Name<br>Treated Subjects - Stage 1 | WK24S1,<br>WK48S1<br>WK96S1,<br>WK96S2 |
| 107 | Table S.3.9.2H | rt-pn-bsldrugs2.lst | SS_PN_T_002 | Baseline Phenotypic Resistance<br>by Class and Drug Name<br>Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 108 | Table S.3.9.3H | rt-pn-<br>bsldrugs12.lst | SS_PN_T_002 | Baseline Phenotypic Resistance<br>by Class and Drug Name<br>Treated Subjects - Stage 1 and 2 | WK96S2 |
| 109 | Table S.3.9.1I | rt-pn-<br>bslotrtdrugs1.lst | SS_PN_T_002 | Baseline Phenotypic Resistance<br>by Class and Drug Name<br>Treated Subjects with On-<br>Treatment Phenotypic<br>Resistance Testing - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 110 | Table S.3.9.2I | rt-pn-<br>bslotrtdrugs2.lst | SS_PN_T_002 | Baseline Phenotypic Resistance<br>by Class and Drug Name<br>Treated Subjects with On-<br>Treatment Phenotypic<br>Resistance Testing - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 111 | Table S.3.9.3I | rt-pn-<br>bslotrtdrugs12.lst | SS_PN_T_002 | Baseline Phenotypic Resistance<br>by Class and Drug Name<br>Treated Subjects with On-<br>Treatment Phenotypic<br>Resistance Testing - Stage 1 and | WK96S2 |
| 112 | Table S.3.9.1R | rt-pn-<br>bsldrugpdvfs1.lst | SS_PN_T_002 | Baseline Phenotypic Resistance by Class and Drug Name Treated Subjects with On- Treatment Phenotypic Resistance Testing Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 113 | Table S.3.9.2R | rt-pn-<br>bsldrugpdvfs2.lst | SS_PN_T_002 | Baseline Phenotypic Resistance by Class and Drug Name Treated Subjects with On- Treatment Phenotypic Resistance Testing Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |

| No. | Table No. | Output File<br>Name | Template ID | Title and Population | Purpose |
|---|---|---|---|---|---|
| 114 | Table S.3.9.3R | rt-pn-<br>bsldrugpdvfs12.lst | SS_PN_T_002 | Baseline Phenotypic Resistance by Class and Drug Name Treated Subjects with On- Treatment Phenotypic Resistance Testing Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 1 and 2 | WK96S2 |
| 115 | Appendix<br>3.9.1E | rl-pn-bsls1.lst | SS_PN_L_001 | Listing of Baseline Phenotypic<br>Resistance<br>Treated Subjects - Stage 1 | WK24S1,<br>WK48S1<br>WK96S1,<br>WK96S2 |
| 116 | Appendix 3.9.2E | rl-pn-bsls2.lst | SS_PN_L_001 | Listing of Baseline Phenotypic<br>Resistance<br>Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 117 | Table S.3.5.1 | rt-lb-bsltoxs1.lst | GS_LB_T_X_004 | Baseline Laboratory Test Results Summary of Toxicity Grade Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 118 | Table S.3.5.2 | rt-lb-bsltoxs2.lst | GS_LB_T_X_004 | Baseline Laboratory Test Results Summary of Toxicity Grade Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 119 | Table S.3.6.1 | rt-ae-preaidss1.lst | GS_AE_T_X_001 | Adverse Events Summary Pre-treatment AIDS Events Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 120 | Table S.3.6.2 | rt-ae-preaidss2.lst | GS_AE_T_X_001 | Adverse Events Summary Pre-treatment AIDS Events Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 121 | Table S.3.7.1 | rt-mh-sums1.lst | GS_MH_T_X_001 | General Medical History<br>Summary<br>Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 122 | Table S.3.7.2 | rt-mh-sums2.lst | GS_MH_T_X_001 | General Medical History<br>Summary<br>Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 123 | Appendix 3.7.1 | rl-mh-lists1.lst | GS_MH_L_X_001 | General Medical History Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 124 | Appendix 3.7.2 | rl-mh-lists2.lst | GS_MH_L_X_001 | General Medical History<br>Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 125 | Table S.3.8.1 | rt-cm-premeds1.lst | GS_CM_T_X_001 | Non-Study Medication Summary Previous Medication Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 126 | Table S.3.8.2 | rt-cm-premeds2.lst | GS_CM_T_X_001 | Non-Study Medication Summary Previous Medication Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |

| No. | Table No. | Output File<br>Name | Template ID | Title and Population | Purpose |
|---|---|---|---|---|---|
| 127 | Table S.4.1.1A | rt-ex-bmss1.lst | SS_EX_T_001 | Extent of Exposure to BMS- | WK24S1, |
| | | | | 955176 | WK48S1, |
| | | | | Time on Therapy | WK96S1, |
| | | | | Treated Subjects - Stage 1 | WK96S2 |
| 128 | Table S.4.1.2A | rt-ex-bmss2.lst | SS EX T 001 | Extent of Exposure to BMS- | WK24S2, |
| | | | | 955176 | WK48S2, |
| | | | | Time on Therapy | WK96S2 |
| | | | | Treated Subjects - Stage 2 | |
| 129 | Table S.4.1.1B | rt-ex-tdfs1.lst | SS_EX_T_001 | Extent of Exposure to Tenofovir | WK24S1, |
| | | | | Time on Therapy | WK48S1, |
| | | | | Treated Subjects - Stage 1 | WK96S1, |
| | | | | | WK96S2 |
| 130 | Table S.4.1.2B | rt-ex-tdfs2.lst | SS_EX_T_001 | Extent of Exposure to Tenofovir | WK24S2, |
| | | | | Time on Therapy | WK48S2, |
| | | | | Treated Subjects - Stage 2 | WK96S2 |
| 131 | Table S.4.1.1C | rt-ex-atvs1.lst | SS_EX_T_001 | Extent of Exposure to | WK24S1, |
| | | | | Atazanavir | WK48S1, |
| | | | | Time on Therapy | WK96S1, |
| | | | | Treated Subjects - Stage 1 | WK96S2 |
| 132 | Table S.4.1.2C | rt-ex-atvs2.lst | SS_EX_T_001 | Extent of Exposure to | WK24S2, |
| | | | | Atazanavir | WK48S2, |
| | | | | Time on Therapy | WK96S2 |
| | | | | Treated Subjects - Stage 2 | |
| 133 | Table S.4.1.1D | rt-ex-dtgs1.lst | SS_EX_T_001 | Extent of Exposure to | WK24S1, |
| | | | | Dolutegravir | WK48S1, |
| | | | | Time on Therapy | WK96S1, |
| | | | | Treated Subjects - Stage 1 | WK96S2 |
| 134 | Table S.4.1.2D | rt-ex-dtgs2.lst | SS_EX_T_001 | Extent of Exposure to | WK24S2, |
| | | | | Dolutegravir | WK48S2, |
| | | | | Time on Therapy | WK96S2 |
| | | | | Treated Subjects - Stage 2 | |
| 135 | Table S.4.1.1E | rt-ex-rtvs1.lst | SS_EX_T_001 | Extent of Exposure to Ritonavir | WK24S1, |
| | | | | Time on Therapy | WK48S1, |
| | | | | Treated Subjects - Stage 1 | WK96S1, |
| 106 | T 11 C 4 1 2 F | | CC FW T 001 | E + CE + Pi | WK96S2 |
| 136 | Table S.4.1.2E | rt-ex-rtvs2.lst | SS_EX_T_001 | Extent of Exposure to Ritonavir | WK24S2, |
| | | | | Time on Therapy | WK48S2, |
| 127 | Table 0 4 1 12 | | CC PV T AA1 | Treated Subjects - Stage 2 | WK96S2 |
| 137 | Table S.4.1.1F | rt-ex-regimens1.lst | SS_EX_T_001 | Extent of Exposure to Treatment | WK24S1, |
| | | | | Regimen Time on Therapy | WK48S1, |
| | | | | Treated Subjects - Stage 1 | WK96S1,<br>WK96S2 |
| 138 | Table S.4.1.2F | rt-ex-regimens2.lst | SS EX T 001 | Extent of Exposure to Treatment | WK24S2, |
| 130 | 1 αυις 5.4.1.2Γ | 11-01-10gillions2.18t | 35_LA_1_001 | Regimen | WK24S2,<br>WK48S2, |
| | | | | Time on Therapy | WK46S2,<br>WK96S2 |
| | | | | Treated Subjects - Stage 2 | W K9032 |
| 139 | Table S.4.1.3F | rt-ex- | SS_EX_T_001 | Extent of Exposure to Treatment | WK96S2 |
| 139 | 1 4015 3.4.1.35 | regimens12.lst | 33_EA_1_001 | Regimen | W 13032 |
| | | 105111011312.131 | | Time on Therapy | |
| | | | | Treated Subjects - Stage 1 and 2 | |
| <u> </u> | L | | | Treated Subjects - Stage 1 and 2 | |

| No. | Table No. | Output File<br>Name | Template ID | Title and Population | Purpose |
|---|---|---|---|---|---|
| 140 | Table S.4.1.1G | rt-ex-conts1.lst | SS_EX_T_001 | Extent of Exposure to BMS-<br>955176 after Switch to<br>Continuation Dose<br>Time on Therapy<br>Treated Subjects who Switched<br>to Continuation Dose - Stage 1 | WK96S1,<br>WK96S2 |
| 141 | Table S.4.1.2G | rt-ex-conts2.lst | SS_EX_T_001 | Extent of Exposure to BMS-<br>955176 after Switch to<br>Continuation Dose<br>Time on Therapy<br>Treated Subjects who Switched<br>to Continuation Dose - Stage 2 | WK96S2 |
| 142 | Figure S.4.1.1 | rg-ex-kms1 | GS_EX_G_001 | Time on Study Therapy<br>Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 143 | Figure S.4.1.2 | rg-ex-kms2 | GS_EX_G_001 | Time on Study Therapy Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 144 | Table S.4.1.1H | rt-ex-kms1.lst | SS_EX_T_002 | Time of Study Therapy Life Table (Kaplan-Meier Estimates) Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 145 | Table S.4.1.2H | rt-ex-kms2.lst | SS_EX_T_002 | Time of Study Therapy Life Table (Kaplan-Meier Estimates) Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 146 | Table S.4.1.1I | rt-ex-interrupts1.lst | SS_EX_T_003 | Summary of Interruptions in<br>Study Therapy Greater than 3<br>Days<br>Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 147 | Table S.4.1.2I | rt-ex-interrupts2.lst | SS_EX_T_003 | Summary of Interruptions in<br>Study Therapy Greater than 3<br>Days<br>Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 148 | Appendix<br>4.1.1A | rl-ex-lists1.lst | SS_EX_L_001 | Study Medication Exposure by Subject Listing Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 149 | Appendix<br>4.1.2A | rl-ex-lists2.lst | SS_EX_L_001 | Study Medication Exposure by<br>Subject Listing<br>Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 150 | Appendix 4.1.1B | rl-ex-listcdoses1.lst | SS_EX_L_002 | Listing of Time on Original and Continuation Dose Treated Subjects - Stage 1 | WK96S1,<br>WK96S2 |
| 151 | Appendix 4.1.2B | rl-ex-listcdoses2.lst | SS_EX_L_002 | Listing of Time on Original and<br>Continuation Dose<br>Treated Subjects - Stage 2 | WK96S2 |
| 152 | Table S.4.2.1 | rt-cm-conmeds1.lst | GS_CM_T_X_001 | Non-Study Medication Summary Concomitant Medication Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |

| No. | Table No. | Output File<br>Name | Template ID | Title and Population | Purpose |
|---|---|---|---|---|---|
| 153 | Table S.4.2.2 | rt-cm-conmeds2.lst | GS_CM_T_X_001 | Non-Study Medication Summary Concomitant Medication Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 154 | Appendix 4.2.1 | rl-cm-meds1.lst | GS_CM_L_X_006 | Non-Study Medication Previous and Concomitant Medications Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 155 | Appendix 4.2.2 | rl-cm-meds2.lst | GS_CM_L_X_006 | Non-Study Medication Previous and Concomitant Medications Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 156 | Table S.5.1.1A | rt-vl-<br>resp40w24s1.lst | SS_VL_T_001 | Detailed Summary of HIV-1 RNA < 40 c/mL Proportion of Responders at Week 24 Snapshot Treated Subjects (mITT) - Stage | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 157 | Table S.5.1.2A | rt-vl-<br>resp40w24s2.lst | SS_VL_T_001 | Detailed Summary of HIV-1 RNA < 40 c/mL Proportion of Responders at Week 24 Snapshot Treated Subjects (mITT) - Stage | WK24S2,<br>WK48S2,<br>WK96S2 |
| 158 | Table S.5.1.1C | rt-vl-<br>sumresp40w24s1.1<br>st | SS_VL_T_002 | Summary of HIV-1 RNA < 40 c/mL Proportion of Responders at Week 24 Snapshot Treated Subjects (mITT) - Stage | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 159 | Table S.5.1.2C | rt-vl-<br>sumresp40w24s2.1<br>st | SS_VL_T_002 | Summary of HIV-1 RNA < 40 c/mL Proportion of Responders at Week 24 Snapshot Treated Subjects (mITT) - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 160 | Table S.5.1.1B | rt-vl-<br>resp40w24subgs1.1<br>st | SS_VL_T_001 | Detailed Summary of HIV-1 RNA < 40 c/mL Proportion of Responders at Week 24 Snapshot By Subgroup Treated Subjects (mITT) - Stage | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 161 | Table S.5.1.2B | rt-vl-<br>resp40w24subgs2.l<br>st | SS_VL_T_001 | Detailed Summary of HIV-1 RNA < 40 c/mL Proportion of Responders at Week 24 Snapshot By Subgroup Treated Subjects (mITT) - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |

| No. | Table No. | Output File<br>Name | Template ID | Title and Population | Purpose |
|---|---|---|---|---|---|
| 162 | Table S.5.2.1A | rt-vl-<br>resp40w48s1.lst | SS_VL_T_001 | Detailed Summary of HIV-1 RNA < 40 c/mL Proportion of Responders at Week 48 Snapshot Treated Subjects (mITT) - Stage | WK96S1,<br>WK96S2 |
| 163 | Table S.5.2.2A | rt-vl-<br>resp40w48s2.lst | SS_VL_T_001 | Detailed Summary of HIV-1 RNA < 40 c/mL Proportion of Responders at Week 48 Snapshot Treated Subjects (mITT) - Stage 2 | WK48S2,<br>WK96S2 |
| 164 | Table S.5.2.1C | rt-vl-<br>sumresp40w48s1.l<br>st | SS_VL_T_002 | Summary of HIV-1 RNA < 40 c/mL Proportion of Responders at Week 48 Snapshot Treated Subjects (mITT) - Stage | WK96S1,<br>WK96S2 |
| 165 | Table S.5.2.2C | rt-vl-<br>sumresp40w48s2.l<br>st | SS_VL_T_002 | Summary of HIV-1 RNA < 40 c/mL Proportion of Responders at Week 48 Snapshot Treated Subjects (mITT) - Stage 2 | WK48S2,<br>WK96S2 |
| 166 | Table S.5.2.1B | rt-vl-<br>resp40w48subgs1.l<br>st | SS_VL_T_001 | Detailed Summary of HIV-1 RNA < 40 c/mL Proportion of Responders at Week 48 Snapshot By Subgroup Treated Subjects (mITT) - Stage | WK96S1,<br>WK96S2 |
| 167 | Table S.5.2.2B | rt-vl-<br>resp40w48subgs2.l<br>st | SS_VL_T_001 | Detailed Summary of HIV-1 RNA < 40 c/mL Proportion of Responders at Week 48 Snapshot By Subgroup Treated Subjects (mITT) - Stage 2 | WK48S2,<br>WK96S2 |
| 168 | Table S.5.3.1A | rt-vl-<br>resp40w96s1.lst | SS_VL_T_001 | Detailed Summary of HIV-1 RNA < 40 c/mL Proportion of Responders at Week 96 Snapshot Treated Subjects (mITT) - Stage | WK96S1,<br>WK96S2 |
| 169 | Table S.5.3.2A | rt-vl-<br>resp40w96s2.lst | SS_VL_T_001 | Detailed Summary of HIV-1 RNA < 40 c/mL Proportion of Responders at Week 96 Snapshot Treated Subjects (mITT) - Stage 2 | WK96S2 |

| No. | Table No. | Output File<br>Name | Template ID | Title and Population | Purpose |
|---|---|---|---|---|---|
| 170 | Table S.5.3.1C | rt-vl-<br>sumresp40w96s1.l<br>st | SS_VL_T_002 | Summary of HIV-1 RNA < 40 c/mL Proportion of Responders at Week 96 Snapshot Treated Subjects (mITT) - Stage | WK96S1,<br>WK96S2 |
| 171 | Table S.5.3.2C | rt-vl-<br>sumresp40w96s2.l<br>st | SS_VL_T_002 | Summary of HIV-1 RNA < 40 c/mL Proportion of Responders at Week 96 Snapshot Treated Subjects (mITT) - Stage | WK96S2 |
| 172 | Table S.5.3.1B | rt-vl-<br>resp40w96subgs1.1<br>st | SS_VL_T_001 | Detailed Summary of HIV-1 RNA < 40 c/mL Proportion of Responders at Week 96 Snapshot By Subgroup Treated Subjects (mITT) - Stage | WK96S1,<br>WK96S2 |
| 173 | Table S.5.3.2B | rt-vl-<br>resp40w96subgs2.1<br>st | SS_VL_T_001 | Detailed Summary of HIV-1 RNA < 40 c/mL Proportion of Responders at Week 96 Snapshot By Subgroup Treated Subjects (mITT) - Stage | WK96S2 |
| 174 | Table S.5.4.1A | rt-vl-<br>resp200w24s1.lst | SS_VL_T_001 | Detailed Summary of HIV-1 RNA < 200 c/mL Proportion of Responders at Week 24 Snapshot Treated Subjects (mITT) - Stage | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 175 | Table S.5.4.2A | rt-vl-<br>resp200w24s2.lst | SS_VL_T_001 | Detailed Summary of HIV-1 RNA < 200 c/mL Proportion of Responders at Week 24 Snapshot Treated Subjects (mITT) - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 176 | Table S.5.4.1B | rt-vl-<br>resp200w24bpolys<br>1.lst | SS_VL_T_001 | Detailed Summary of HIV-1 RNA < 200 c/mL Proportion of Responders at Week 24 Snapshot By Baseline Gag Polymorphism Treated Subjects (mITT) - Stage | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 177 | Table S.5.4.2B | rt-vl-<br>resp200w24bpolys<br>2.lst | SS_VL_T_001 | Detailed Summary of HIV-1 RNA < 200 c/mL Proportion of Responders at Week 24 Snapshot By Baseline Gag Polymorphism Treated Subjects (mITT) - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |

| No. | Table No. | Output File<br>Name | Template ID | Title and Population | Purpose |
|---|---|---|---|---|---|
| 178 | Table S.5.4.1C | rt-vl-<br>resp200w48s1.lst | SS_VL_T_001 | Detailed Summary of HIV-1 RNA < 200 c/mL Proportion of Responders at Week 48 Snapshot Treated Subjects (mITT) - Stage | WK96S1,<br>WK96S2 |
| 179 | Table S.5.4.2C | rt-vl-<br>resp200w48s2.lst | SS_VL_T_001 | Detailed Summary of HIV-1 RNA < 200 c/mL Proportion of Responders at Week 48 Snapshot Treated Subjects (mITT) - Stage 2 | WK48S2,<br>WK96S2 |
| 180 | Table S.5.4.1D | rt-vl-<br>resp200w48bpolys<br>1.lst | SS_VL_T_001 | Detailed Summary of HIV-1 RNA < 200 c/mL Proportion of Responders at Week 48 Snapshot By Baseline Gag Polymorphism Treated Subjects (mITT) - Stage | WK96S1,<br>WK96S2 |
| 181 | Table S.5.4.2D | rt-vl-<br>resp200w48bpolys<br>2.lst | SS_VL_T_001 | Detailed Summary of HIV-1 RNA < 200 c/mL Proportion of Responders at Week 48 Snapshot By Baseline Gag Polymorphism Treated Subjects (mITT) - Stage | WK48S2,<br>WK96S2 |
| 182 | Table S.5.4.1E | rt-vl-<br>resp200w96s1.lst | SS_VL_T_001 | Detailed Summary of HIV-1 RNA < 200 c/mL Proportion of Responders at Week 96 Snapshot Treated Subjects (mITT) - Stage | WK96S1,<br>WK96S2 |
| 183 | Table S.5.4.2E | rt-vl-<br>resp200w96s2.lst | SS_VL_T_001 | Detailed Summary of HIV-1 RNA < 200 c/mL Proportion of Responders at Week 96 Snapshot Treated Subjects (mITT) - Stage | WK96S2 |
| 184 | Table S.5.4.1F | rt-vl-<br>resp200w96bpolys<br>1.lst | SS_VL_T_001 | Detailed Summary of HIV-1 RNA < 200 c/mL Proportion of Responders at Week 96 Snapshot By Baseline Gag Polymorphism Treated Subjects (mITT) - Stage | WK96S1,<br>WK96S2 |
| 185 | Table S.5.4.2F | rt-vl-<br>resp200w96bpolys<br>2.lst | SS_VL_T_001 | Detailed Summary of HIV-1 RNA < 200 c/mL Proportion of Responders at Week 96 Snapshot By Baseline Gag Polymorphism Treated Subjects (mITT) - Stage 2 | WK96S2 |

| No. | Table No. | Output File<br>Name | Template ID | Title and Population | Purpose |
|---|---|---|---|---|---|
| 186 | Table S.5.1.1D | rt-vl-<br>resp40w24obss1.ls | SS_VL_T_003 | Summary of HIV-1 RNA < 40 c/mL | WK24S1,<br>WK48S1, |
| | | t | | Proportion of Responders at<br>Week 24 | WK96S1,<br>WK96S2 |
| | | | | Treated Subjects (Observed) -<br>Stage 1 | W15 052 |
| 187 | Table S.5.1.2D | rt-vl-<br>resp40w24obss2.ls | SS_VL_T_003 | Summary of HIV-1 RNA < 40 c/mL | WK24S2,<br>WK48S2, |
| | | t | | Proportion of Responders at<br>Week 24 | WK4652,<br>WK96S2 |
| | | | | Treated Subjects (Observed) - Stage 2 | |
| 188 | Table S.5.1.1E | rt-vl- | SS_VL_T_003 | Summary of HIV-1 RNA < 40 | WK24S1, |
| | | resp40w24obssubg<br>s1.lst | | c/mL Proportion of Responders at | WK48S1,<br>WK96S1, |
| | | 51.15t | | Week 24 | WK96S2 |
| | | | | By Subgroup Treated Subjects (Observed) - | |
| | | | | Stage 1 | |
| 189 | Table S.5.1.2E | rt-vl- | SS_VL_T_003 | Summary of HIV-1 RNA < 40 | WK24S2, |
| | | resp40w24obssubg | | c/mL | WK48S2, |
| | | s2.lst | | Proportion of Responders at Week 24 | WK96S2 |
| | | | | By Subgroup | |
| | | | | Treated Subjects (Observed) - | |
| 100 | T-1-1- C 5 2 1D | | GG VII T 002 | Stage 2 | WWO(C1 |
| 190 | Table S.5.2.1D | rt-vl-<br>resp40w48obss1.ls | SS_VL_T_003 | Summary of HIV-1 RNA < 40 c/mL | WK96S1,<br>WK96S2 |
| | | t | | Proportion of Responders at | WIC/052 |
| | | | | Week 48 | |
| | | | | Treated Subjects (Observed) - | |
| | | | | Stage 1 | |
| 191 | Table S.5.2.2D | rt-vl- | SS_VL_T_003 | Summary of HIV-1 RNA < 40 | WK48S2, |
| | | resp40w48obss2.ls | | c/mL<br>Proportion of Responders at | WK96S2 |
| | | ľ | | Week 48 | |
| | | | | Treated Subjects (Observed) - | |
| | | | | Stage 2 | |
| 192 | Table S.5.2.1E | rt-vl- | SS_VL_T_003 | Summary of HIV-1 RNA < 40 | WK96S1, |
| | | resp40w48obssubs | | c/mL | WK96S2 |
| | | 1.lst | | Proportion of Responders at Week 48 | |
| | | | | By Subgroup | |
| | | | | Treated Subjects (Observed) - | |
| | | | | Stage 1 | |
| 193 | Table S.5.2.2E | rt-vl- | SS_VL_T_003 | Summary of HIV-1 RNA < 40 | WK48S2, |
| | | resp40w48obssubg | | c/mL | WK96S2 |
| | | s2.1st | | Proportion of Responders at | |
| | | | | Week 48 By Subgroup | |
| | | | | Treated Subjects (Observed) - | |
| | | | | Stage 2 | |

| No. | Table No. | Output File<br>Name | Template ID | Title and Population | Purpose |
|---|---|---|---|---|---|
| 194 | Table S.5.3.1D | rt-vl-<br>resp40w96obss1.ls<br>t | SS_VL_T_003 | Summary of HIV-1 RNA < 40 c/mL Proportion of Responders at Week 96 Treated Subjects (Observed) - Stage 1 | WK96S1,<br>WK96S2 |
| 195 | Table S.5.3.2D | rt-vl-<br>resp40w96obss2.ls<br>t | SS_VL_T_003 | Summary of HIV-1 RNA < 40 c/mL Proportion of Responders at Week 96 Treated Subjects (Observed) - Stage 2 | WK96S2 |
| 196 | Table S.5.3.1E | rt-vl-<br>resp40w96obssubg<br>s1.lst | SS_VL_T_003 | Summary of HIV-1 RNA < 40 c/mL Proportion of Responders at Week 96 By Subgroup Treated Subjects (Observed) - Stage 1 | WK96S1,<br>WK96S2 |
| 197 | Table S.5.3.2E | rt-vl-<br>resp40w96obssubg<br>s2.lst | SS_VL_T_003 | Summary of HIV-1 RNA < 40 c/mL Proportion of Responders at Week 96 By Subgroup Treated Subjects (Observed) - Stage 2 | WK96S2 |
| 198 | Table S.5.5.1A | rt-vl-tlovr24s1.lst | SS_VL_T_004 | Summary of Treatment Outcomes at Week 24 Using the TLOVR Algorithm Treated Subjects - Stage 1 | WK24S1 |
| 199 | Table S.5.5.2A | rt-vl-tlovr24s2.lst | SS_VL_T_004 | Summary of Treatment Outcomes at Week 24 Using the TLOVR Algorithm Treated Subjects - Stage 2 | WK24S2 |
| 200 | Table S.5.5.1B | rt-vl-tlovr48s1.lst | SS_VL_T_004 | Summary of Treatment Outcomes at Week 48 Using the TLOVR Algorithm Treated Subjects - Stage 1 | WK48S1 |
| 201 | Table S.5.5.2B | rt-vl-tlovr48s2.lst | SS_VL_T_004 | Summary of Treatment Outcomes at Week 48 Using the TLOVR Algorithm Treated Subjects - Stage 2 | WK48S2 |
| 202 | Table S.5.5.1C | rt-vl-tlovr96s1.lst | SS_VL_T_004 | Summary of Treatment Outcomes at Week 96 Using the TLOVR Algorithm Treated Subjects - Stage 1 | WK96S1,<br>WK96S2 |
| 203 | Table S.5.5.2C | rt-vl-tlovr96s2.lst | SS_VL_T_004 | Summary of Treatment Outcomes at Week 96 Using the TLOVR Algorithm Treated Subjects - Stage 2 | WK96S2 |

| No. | Table No. | Output File<br>Name | Template ID | Title and Population | Purpose |
|---|---|---|---|---|---|
| 204 | Table S.5.5.1D | rt-vl-klmtlovrs1.lst | SS_EX_T_002 | Summary of Time to Loss of<br>Virologic Response<br>Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 205 | Table S.5.5.2D | rt-vl-klmtlovrs2.lst | SS_EX_T_002 | Summary of Time to Loss of<br>Virologic Response<br>Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 206 | Figure S.5.5.1E | rg-vl-kmtlovrs1 | GS_EX_G_001 | Time to Loss of Virologic Response Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 207 | Figure S.5.5.2E | rg-vl-kmtlovrs2 | GS_EX_G_001 | Time to Loss of Virologic<br>Response<br>Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 208 | Table S.5.6.1A | rt-vl-props1.lst | SS_VL_T_005 | Proportion of Subjects with<br>HIV-1 RNA within Several<br>Ranges<br>Treated Subjects (Observed) -<br>Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 209 | Table S.5.6.2A | rt-vl-props2.lst | SS_VL_T_005 | Proportion of Subjects with HIV-1 RNA within Several Ranges Treated Subjects (Observed) - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 210 | Table S.5.6.1B | rt-vl-sumchgs1.lst | SS_VL_T_006 | Summary Statistics for Values<br>and Change from Baseline Over<br>Time<br>HIV-1 RNA (log10 c/mL)<br>Overall and by Subgroup<br>Treated Subjects (Observed) -<br>Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 211 | Table S.5.6.2B | rt-vl-sumchgs2.lst | SS_VL_T_006 | Summary Statistics for Values<br>and Change from Baseline Over<br>Time<br>HIV-1 RNA (log10 c/mL)<br>Overall and by Subgroup<br>Treated Subjects (Observed) -<br>Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 212 | Table S.5.7.1A | rt-lb-cd4s1.lst | SS_VL_T_006 | Summary Statistics for Values<br>and Change from Baseline Over<br>Time<br>CD4 Cell Count (cells/uL)<br>Overall and by Subgroup<br>Treated Subjects (Observed) -<br>Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 213 | Table S.5.7.2A | rt-lb-cd4s2.lst | SS_VL_T_006 | Summary Statistics for Values<br>and Change from Baseline Over<br>Time<br>CD4 Cell Count (cells/uL)<br>Overall and by Subgroup<br>Treated Subjects (Observed) -<br>Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |

| No. | Table No. | Output File<br>Name | Template ID | Title and Population | Purpose |
|---|---|---|---|---|---|
| 214 | Table S.5.8.1A | rt-lb-cd4pcts1.lst | SS_VL_T_006 | Summary Statistics for Values<br>and Change from Baseline Over<br>Time<br>CD4 Cell Percentage<br>Overall and by Subgroup<br>Treated Subjects (Observed) -<br>Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 215 | Table S.5.8.2A | rt-lb-cd4pcts2.lst | SS_VL_T_006 | Summary Statistics for Values<br>and Change from Baseline Over<br>Time<br>CD4 Cell Percentage<br>Overall and by Subgroup<br>Treated Subjects (Observed) -<br>Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 216 | Table S.5.9.1A | rt-lb-cd8s1.lst | SS_VL_T_006 | Summary Statistics for Values<br>and Change from Baseline Over<br>Time<br>CD8 Cell Count (cells/ul)<br>Overall and by Subgroup<br>Treated Subjects (Observed) -<br>Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 217 | Table S.5.9.2A | rt-lb-cd8s2.lst | SS_VL_T_006 | Summary Statistics for Values<br>and Change from Baseline Over<br>Time<br>CD8 Cell Count (cells/ul)<br>Overall and by Subgroup<br>Treated Subjects (Observed) -<br>Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 218 | Figure S.5.6.1C | rg-vl-box24s1 | GS_LB_G_001 | HIV-1 RNA (log10 c/mL) Change from Baseline to Week 24 Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 219 | Figure S.5.6.2C | rg-vl-box24s2 | GS_LB_G_001 | HIV-1 RNA (log10 c/mL) Change from Baseline to Week 24 Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 220 | Figure S.5.6.1D | rg-vl-box48s1 | GS_LB_G_001 | HIV-1 RNA (log10 c/mL) Change from Baseline to Week 48 Treated Subjects - Stage 1 | WK96S1,<br>WK96S2 |
| 221 | Figure S.5.6.2D | rg-vl-box48s2 | GS_LB_G_001 | HIV-1 RNA (log10 c/mL) Change from Baseline to Week 48 Treated Subjects - Stage 2 | WK48S2,<br>WK96S2 |
| 222 | Figure S.5.6.1E | rg-vl-box96s1 | GS_LB_G_001 | HIV-1 RNA (log10 c/mL) Change from Baseline to Week 96 Treated Subjects - Stage 1 | WK96S1,<br>WK96S2 |
| 223 | Figure S.5.6.2E | rg-vl-box96s2 | GS_LB_G_001 | HIV-1 RNA (log10 c/mL) Change from Baseline to Week 96 Treated Subjects - Stage 2 | WK96S2 |

| No. | Table No. | Output File<br>Name | Template ID | Title and Population | Purpose |
|---|---|---|---|---|---|
| 224 | Figure S.5.7.1B | rg-lb-cd4box24s1 | GS_LB_G_001 | CD4 Cell Count (cells/uL) Change from Baseline to Week 24 Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 225 | Figure S.5.7.2B | rg-lb-cd4box24s2 | GS_LB_G_001 | CD4 Cell Count (cells/uL) Change from Baseline to Week 24 Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 226 | Figure S.5.7.1C | rg-lb-cd4box48s1 | GS_LB_G_001 | CD4 Cell Count (cells/uL) Change from Baseline to Week 48 Treated Subjects - Stage 1 | WK96S1,<br>WK96S2 |
| 227 | Figure S.5.7.2C | rg-lb-cd4box48s2 | GS_LB_G_001 | CD4 Cell Count (cells/uL) Change from Baseline to Week 48 Treated Subjects - Stage 2 | WK48S2,<br>WK96S2 |
| 228 | Figure S.5.7.1D | rg-lb-cd4box96s1 | GS_LB_G_001 | CD4 Cell Count (cells/uL) Change from Baseline to Week 96 Treated Subjects - Stage 1 | WK96S1,<br>WK96S2 |
| 229 | Figure S.5.7.2D | rg-lb-cd4box96s2 | GS_LB_G_001 | CD4 Cell Count (cells/uL) Change from Baseline to Week 96 Treated Subjects - Stage 2 | WK96S2 |
| 230 | Figure S.5.9.1B | rg-lb-cd8box24s1 | GS_LB_G_001 | CD8 Cell Count (cells/uL) Change from Baseline to Week 24 Treated Subjects -Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 231 | Figure S.5.9.2B | rg-lb-cd8box24s2 | GS_LB_G_001 | CD8 Cell Count (cells/uL) Change from Baseline to Week 24 Treated Subjects -Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 232 | Figure S.5.9.1C | rg-lb-cd8box48s1 | GS_LB_G_001 | CD8 Cell Count (cells/uL) Change from Baseline to Week 48 Treated Subjects - Stage 1 | WK96S1,<br>WK96S2 |
| 233 | Figure S.5.9.2C | rg-lb-cd8box48s2 | GS_LB_G_001 | CD8 Cell Count (cells/uL) Change from Baseline to Week 48 Treated Subjects - Stage 2 | WK48S2,<br>WK96S2 |
| 234 | Figure S.5.9.1D | rg-lb-cd8box96s1 | GS_LB_G_001 | CD8 Cell Count (cells/uL) Change from Baseline to Week 96 Treated Subjects - Stage 1 | WK96S1,<br>WK96S2 |
| 235 | Figure S.5.9.2D | rg-lb-cd8box96s2 | GS_LB_G_001 | CD8 Cell Count (cells/uL) Change from Baseline to Week 96 Treated Subjects - Stage 2 | WK96S2 |
| 236 | Figure S.5.6.1F | rg-vl-times1 | GS_LB_G_002 | HIV-1 RNA (log10 c/mL) Mean<br>Change from Baseline Over<br>Time<br>Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |

| No. | Table No. | Output File<br>Name | Template ID | Title and Population | Purpose |
|---|---|---|---|---|---|
| 237 | Figure S.5.6.2F | rg-vl-times2 | GS_LB_G_002 | HIV-1 RNA (log10 c/mL) Mean<br>Change from Baseline Over<br>Time<br>Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 238 | Figure S.5.7.1E | rg-lb-cd4times1 | GS_LB_G_002 | CD4 (cells/uL) Mean Change<br>from Baseline Over Time<br>Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 239 | Figure S.5.7.2E | rg-lb-cd4times2 | GS_LB_G_002 | CD4 (cells/uL) Mean Change<br>from Baseline Over Time<br>Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 240 | Figure S.5.9.1E | rg-lb-cd8times1 | GS_LB_G_002 | CD8 (cells/uL) Mean Change<br>from Baseline Over Time<br>Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 241 | Figure S.5.9.2E | rg-lb-cd8times2 | GS_LB_G_002 | CD8 (cells/uL) Mean Change<br>from Baseline Over Time<br>Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 242 | Appendix<br>5.1.1A | rl-vl-<br>outcome24s1.lst | SS_VL_L_004 | Listing of Outcomes from HIV-<br>1 RNA < 40 c/mL Snapshot<br>Analysis<br>Data for Subjects in the Week<br>24 Snapshot<br>Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 243 | Appendix<br>5.1.2A | rl-vl-<br>outcome24s2.lst | SS_VL_L_004 | Listing of Outcomes from HIV- 1 RNA < 40 c/mL Snapshot Analysis Data for Subjects in the Week 24 Snapshot Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 244 | Appendix<br>5.1.1B | rl-vl-<br>outcome48s1.lst | SS_VL_L_004 | Listing of Outcomes from HIV-<br>1 RNA < 40 c/mL Snapshot<br>Analysis<br>Data for Subjects in the Week<br>48 Snapshot<br>Treated Subjects - Stage 1 | WK96S1,<br>WK96S2 |
| 245 | Appendix<br>5.1.2B | rl-vl-<br>outcome48s2.lst | SS_VL_L_004 | Listing of Outcomes from HIV-<br>1 RNA < 40 c/mL Snapshot<br>Analysis<br>Data for Subjects in the Week<br>48 Snapshot<br>Treated Subjects - Stage 2 | WK48S2,<br>WK96S2 |
| 246 | Appendix<br>5.1.1C | rl-vl-<br>outcome96s1.lst | SS_VL_L_004 | Listing of Outcomes from HIV-<br>1 RNA < 40 c/mL Snapshot<br>Analysis<br>Data for Subjects in the Week<br>96 Snapshot<br>Treated Subjects - Stage 1 | WK96S1,<br>WK96S2 |

| No. | Table No. | Output File<br>Name | Template ID | Title and Population | Purpose |
|---|---|---|---|---|---|
| 247 | Appendix<br>5.1.2C | rl-vl-<br>outcome96s2.lst | SS_VL_L_004 | Listing of Outcomes from HIV-<br>1 RNA < 40 c/mL Snapshot<br>Analysis<br>Data for Subjects in the Week<br>96 Snapshot<br>Treated Subjects - Stage 2 | WK96S2 |
| 248 | Appendix 5.1.1D | rl-vl-vllists1.lst | SS_VL_L_005 | Listing of HIV-1 RNA Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 249 | Appendix 5.1.2D | rl-vl-vllists2.lst | SS_VL_L_005 | Listing of HIV-1 RNA Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 250 | Appendix<br>5.1.1E | rl-lb-cd4cd8s1.lst | SS_VL_L_005 | Listing of CD4+ and CD8+ T-<br>Cell Count and Percentages<br>Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 251 | Appendix 5.1.2E | rl-lb-cd4cd8s2.lst | SS_VL_L_005 | Listing of CD4+ and CD8+ T-<br>Cell Count and Percentages<br>Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 252 | Table<br>S.5.10.1A | rt-gn-news1.lst | SS_GN_T_001 | Newly Emergent Genotypic Resistance Profile Treated Subjects with On- Treatment Genotypic Resistance Testing - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 253 | Table<br>S.5.10.2A | rt-gn-news2.lst | SS_GN_T_001 | Newly Emergent Genotypic Resistance Profile Treated Subjects with On- Treatment Genotypic Resistance Testing - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 254 | Table<br>S.5.10.3A | rt-gn-news12.lst | SS_GN_T_001 | Newly Emergent Genotypic Resistance Profile Treated Subjects with On- Treatment Genotypic Resistance Testing - Stage 1 and 2 | WK96S2 |
| 255 | Table S.5.10.1B | rt-gn-<br>newpdvfs1.lst | SS_GN_T_001 | Newly Emergent Genotypic Resistance Profile Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 256 | Table S.5.10.2B | rt-gn-<br>newpdvfs2.lst | SS_GN_T_001 | Newly Emergent Genotypic Resistance Profile Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 257 | Table S.5.10.3B | rt-gn-<br>newpdvfs12.lst | SS_GN_T_001 | Newly Emergent Genotypic Resistance Profile Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 1 and 2 | WK96S2 |
| No. | Table No. | Output File<br>Name | Template ID | Title and Population | Purpose |
|---|---|---|---|---|---|
| 258 | Appendix<br>5.10.1A | rl-gn-ontrts1.lst | SS_GN_L_001 | Listing of Genotypic Substitutions Treated Subjects with Baseline and On-Treatment Data - Stage | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 259 | Appendix<br>5.10.2A | rl-gn-ontrts2.lst | SS_GN_L_001 | Listing of Genotypic Substitutions Treated Subjects with Baseline and On-Treatment Data - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 260 | Table S.5.10.1C | rt-gn-newgags1.lst | SS_GN_T_002 | Emergent Gag Polymorphisms<br>at Selected Positions<br>Treated Subjects with On-<br>Treatment Gag Sequencing -<br>Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 261 | Table S.5.10.2C | rt-gn-newgags2.lst | SS_GN_T_002 | Emergent Gag Polymorphisms<br>at Selected Positions<br>Treated Subjects with On-<br>Treatment Gag Sequencing -<br>Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 262 | Table S.5.10.3C | rt-gn-<br>newgags12.lst | SS_GN_T_002 | Emergent Gag Polymorphisms<br>at Selected Positions<br>Treated Subjects with On-<br>Treatment Gag Sequencing -<br>Stage 1 and 2 | WK96S2 |
| 263 | Table S.5.10.1R | rt-gn-<br>newgagbysubtypes<br>1.lst | SS_GN_T_002 | Emergent Gag Polymorphisms at Selected Positions By HIV Subtype Treated Subjects with On- Treatment Gag Sequencing - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 264 | Table S.5.10.2R | rt-gn-<br>newgagbysubtypes<br>2.lst | SS_GN_T_002 | Emergent Gag Polymorphisms<br>at Selected Positions<br>By HIV Subtype<br>Treated Subjects with On-<br>Treatment Gag Sequencing -<br>Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 265 | Table S.5.10.3R | rt-gn-<br>newgagbysubtypes<br>12.lst | SS_GN_T_002 | Emergent Gag Polymorphisms<br>at Selected Positions<br>By HIV Subtype<br>Treated Subjects with On-<br>Treatment Gag Sequencing -<br>Stage 1 and 2 | WK96S2 |
| 266 | Table<br>S.5.10.1D | rt-gn-<br>newgagpdvfs1.lst | SS_GN_T_002 | Emergent Gag Polymorphisms<br>at Selected Positions<br>Treated Subjects Identified as<br>Protocol Defined Virologic<br>Failures - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 267 | Table<br>S.5.10.2D | rt-gn-<br>newgagpdvfs2.lst | SS_GN_T_002 | Emergent Gag Polymorphisms<br>at Selected Positions<br>Treated Subjects Identified as<br>Protocol Defined Virologic<br>Failures - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |

| No. | Table No. | Output File<br>Name | Template ID | Title and Population | Purpose |
|---|---|---|---|---|---|
| 268 | Table<br>S.5.10.3D | rt-gn-<br>newgagpdvfs12.lst | SS_GN_T_002 | Emergent Gag Polymorphisms<br>at Selected Positions<br>Treated Subjects Identified as<br>Protocol Defined Virologic<br>Failures - Stage 1 and 2 | WK96S2 |
| 269 | Table S.5.10.1S | rt-gn-<br>newgagpdvfbysubt<br>ypes1.lst | SS_GN_T_002 | Emergent Gag Polymorphisms at Selected Positions By HIV Subtype Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 270 | Table S.5.10.2S | rt-gn-<br>newgagpdvfbysubt<br>ypes2.lst | SS_GN_T_002 | Emergent Gag Polymorphisms at Selected Positions By HIV Subtype Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 271 | Table S.5.10.3S | rt-gn-<br>newgagpdvfbysubt<br>ypes12.lst | SS_GN_T_002 | Emergent Gag Polymorphisms at Selected Positions By HIV Subtype Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 1 and 2 | WK96S2 |
| 272 | Appendix<br>5.10.1B | rl-gn-gagontrts1.lst | SS_GN_L_002 | Listing of Gag Polymorphisms<br>at Selected Positions<br>Treated Subjects with Baseline<br>and On-Treatment Data - Stage | WK24S1,<br>WK48S1<br>WK96S1,<br>WK96S2 |
| 273 | Appendix<br>5.10.2B | rl-gn-gagontrts2.lst | SS_GN_L_002 | Listing of Gag Polymorphisms<br>at Selected Positions<br>Treated Subjects with Baseline<br>and On-Treatment Data - Stage | WK24S2,<br>WK48S2,<br>WK96S2 |
| 274 | Table S.5.10.1E | rt-gn-anygags1.lst | SS_GN_T_003 | Newly Emergent Gag Deviations Treated Subjects with On- Treatment Gag Sequencing - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 275 | Table S.5.10.2E | | SS_GN_T_003 | Newly Emergent Gag Deviations Treated Subjects with On- Treatment Gag Sequencing - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 276 | Table S.5.10.3E | rt-gn-anygags12.lst | SS_GN_T_003 | Newly Emergent Gag Deviations Treated Subjects with On- Treatment Gag Sequencing - Stage 1 and 2 | WK96S2 |

| No. | Table No. | Output File<br>Name | Template ID | Title and Population | Purpose |
|---|---|---|---|---|---|
| 277 | Table S.5.10.1T | rt-gn-<br>anygagbysubtypes<br>1.lst | SS_GN_T_003 | Newly Emergent Gag Deviations By HIV Subtype Treated Subjects with On- Treatment Gag Sequencing - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 278 | Table S.5.10.2T | rt-gn-<br>anygagbysubtypes<br>2.lst | SS_GN_T_003 | Newly Emergent Gag Deviations By HIV Subtype Treated Subjects with On- Treatment Gag Sequencing - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 279 | Table S.5.10.3T | rt-gn-<br>anygagbysubtypes<br>12.lst | SS_GN_T_003 | Newly Emergent Gag Deviations By HIV Subtype Treated Subjects with On- Treatment Gag Sequencing - Stage 1 and 2 | WK96S2 |
| 280 | Table S.5.10.1F | rt-gn-<br>anygagpdvfs1.lst | SS_GN_T_003 | Newly Emergent Gag Deviations Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 281 | Table S.5.10.2F | rt-gn-<br>anygagpdvfs2.lst | SS_GN_T_003 | Newly Emergent Gag Deviations Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 282 | Table S.5.10.3F | rt-gn-<br>anygagpdvfs12.lst | SS_GN_T_003 | Newly Emergent Gag Deviations Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 1 and 2 | WK96S2 |
| 283 | Table<br>S.5.10.1U | rt-gn-<br>anygagpdvfbysubt<br>ypes1.lst | SS_GN_T_003 | Newly Emergent Gag Deviations By HIV Subtype Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 284 | Table<br>S.5.10.2U | rt-gn-<br>anygagpdvfbysubt<br>ypes2.lst | SS_GN_T_003 | Newly Emergent Gag Deviations By HIV Subtype Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 285 | Table<br>S.5.10.3U | rt-gn-<br>anygagpdvfbysubt<br>ypes12.lst | SS_GN_T_003 | Newly Emergent Gag Deviations By HIV Subtype Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 1 and 2 | WK96S2 |

| No. | Table No. | Output File<br>Name | Template ID | Title and Population | Purpose |
|---|---|---|---|---|---|
| 286 | Appendix 5.10.1C | rl-gn-gagontrts1.lst | SS_GN_L_003 | Listing of Newly Emergent Gag<br>Deviations | WK24S1,<br>WK48S1, |
| | | | | Treated Subjects with Baseline | WK96S1,<br>WK96S2 |
| | | | | and On-Treatment Data - Stage | W K9052 |
| 287 | Appendix | rl-gn-gagontrts2.lst | SS_GN_L_003 | Listing of Newly Emergent Gag | WK24S2, |
| | 5.10.2C | | | Deviations Treated Subjects with Baseline | WK48S2,<br>WK96S2 |
| | | | | and On-Treatment Data - Stage | WR/052 |
| 288 | Table | rt-pn-news1.lst | SS_PN_T_001 | Newly Emergent Phenotypic | WK24S1, |
| | S.5.10.1G | | | Resistance Profile | WK48S1, |
| | | | | Treated Subjects with On-<br>Treatment Phenotypic | WK96S1,<br>WK96S2 |
| | | | | Resistance Profile - Stage 1 | W K 9032 |
| 289 | Table | rt-pn-news2.lst | SS PN T 001 | Newly Emergent Phenotypic | WK24S2, |
| | S.5.10.2G | 1 | | Resistance Profile | WK48S2, |
| | | | | Treated Subjects with On- | WK96S2 |
| | | | | Treatment Phenotypic | |
| 290 | Table | rt-pn-news12.lst | SS PN T 001 | Resistance Profile - Stage 2 Newly Emergent Phenotypic | WK96S2 |
| 290 | S.5.10.3G | rt-pn-news12.ist | 35_PN_1_001 | Resistance Profile | W K9052 |
| | 5.5.10.50 | | | Treated Subjects with On- | |
| | | | | Treatment Phenotypic | |
| | | | | Resistance Profile - Stage 1 and | |
| 291 | Table | rt-pn- | SS PN T 001 | Newly Emergent Phenotypic | WK24S1, |
| | S.5.10.1H | newpdvfs1.lst | | Resistance Profile | WK48S1, |
| | | - | | Treated Subjects Identified as | WK96S1, |
| | | | | Protocol Defined Virologic | WK96S2 |
| 202 | T-1.1. | | CC DN T 001 | Failures - Stage 1 | WW24G2 |
| 292 | Table<br>S.5.10.2H | rt-pn-<br>newpdvfs2.lst | SS_PN_T_001 | Newly Emergent Phenotypic Resistance Profile | WK24S2,<br>WK48S2, |
| | 5.5.10.211 | newpavi32.ist | | Treated Subjects Identified as | WK96S2, |
| | | | | Protocol Defined Virologic | |
| | | | | Failures - Stage 2 | |
| 293 | Table | rt-pn- | SS_PN_T_001 | Newly Emergent Phenotypic | WK96S2 |
| | S.5.10.3H | newpdvfs12.lst | | Resistance Profile | |
| | | | | Treated Subjects Identified as<br>Protocol Defined Virologic | |
| | | | | Failures - Stage 1 and 2 | |
| 294 | Table S.5.10.11 | rt-pn- | SS PN T 002 | Newly Emergent Phenotypic | WK24S1, |
| | | newdrugs1.lst | | Resistance by Class and Drug | WK48S1, |
| | | | | Name | WK96S1, |
| | | | | Treated Subjects with On- | WK96S2 |
| | | | | Treatment Phenotypic | |
| 295 | Table S.5.10.2I | rt-pn- | SS PN T 002 | Resistance Profile - Stage 1 Newly Emergent Phenotypic | WK24S2, |
| 293 | 1 4010 5.3.10.21 | newdrugs2.lst | 55_111_1_002 | Resistance by Class and Drug | WK48S2, |
| | | | | Name | WK96S2, |
| | | | | Treated Subjects with On- | |
| | | | | Treatment Phenotypic | |
| | | | | Resistance Profile - Stage 2 | |

| No. | Table No. | Output File<br>Name | Template ID | Title and Population | Purpose |
|---|---|---|---|---|---|
| 296 | Table S.5.10.3I | rt-pn-<br>newdrugs12.lst | SS_PN_T_002 | Newly Emergent Phenotypic Resistance by Class and Drug Name Treated Subjects with On- Treatment Phenotypic | WK96S2 |
| | | | | Resistance Profile - Stage 1 and 2 | |
| 297 | Table S.5.10.1J | rt-pn-<br>newdrugpdvfs1.lst | SS_PN_T_002 | Newly Emergent Phenotypic Resistance by Class and Drug Name Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 298 | Table S.5.10.2J | rt-pn-<br>newdrugpdvfs2.lst | SS_PN_T_002 | Newly Emergent Phenotypic Resistance by Class and Drug Name Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 299 | Table S.5.10.3J | rt-pn-<br>newdrugpdvfs12.ls<br>t | SS_PN_T_002 | Newly Emergent Phenotypic Resistance by Class and Drug Name Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 1 and 2 | WK96S2 |
| 300 | Appendix 5.10.1D | rl-pn-ontrts1.lst | SS_PN_L_001 | Listing of Phenotypic Resistance<br>Treated Subjects with Baseline<br>and On-Treatment Data - Stage | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 301 | Appendix<br>5.10.2D | rl-pn-ontrts2.lst | SS_PN_L_001 | Listing of Phenotypic Resistance<br>Treated Subjects with Baseline<br>and On-Treatment Data - Stage<br>2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 302 | Table<br>S.5.10.1K | rt-pn-maxic50s1.lst | SS_PN_T_003 | Maximum Change from Baseline Summary for BMS- 955176 IC50 Treated Subjects with On- Treatment Phenotypic Resistance Profile - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 303 | Table<br>S.5.10.2K | rt-pn-maxic50s2.lst | SS_PN_T_003 | Maximum Change from Baseline Summary for BMS- 955176 IC50 Treated Subjects with On- Treatment Phenotypic Resistance Profile - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 304 | Table S.5.10.1L | rt-pn-<br>maxic50pdvfs1.lst | SS_PN_T_003 | Maximum Change from Baseline Summary for BMS- 955176 IC50 Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |

| No. | Table No. | Output File<br>Name | Template ID | Title and Population | Purpose |
|---|---|---|---|---|---|
| 305 | Table S.5.10.2L | rt-pn-<br>maxic50pdvfs2.1st | SS_PN_T_003 | Maximum Change from Baseline Summary for BMS- 955176 IC50 Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 306 | Table<br>S.5.10.1M | rt-pn-<br>maxic50fcs1.lst | SS_PN_T_003 | Summary for Maximum BMS-<br>955176 IC50 Fold Change<br>Treated Subjects with On-<br>Treatment Phenotypic<br>Resistance Profile - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 307 | Table<br>S.5.10.2M | rt-pn-<br>maxic50fcs2.lst | SS_PN_T_003 | Summary for Maximum BMS-<br>955176 IC50 Fold Change<br>Treated Subjects with On-<br>Treatment Phenotypic<br>Resistance Profile - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 308 | Table<br>S.5.10.1N | rt-pn-<br>maxic50fcpdvfs1.l<br>st | SS_PN_T_003 | Summary for Maximum BMS-<br>955176 IC50 Fold Change<br>Treated Subjects Identified as<br>Protocol Defined Virologic<br>Failures - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 309 | Table<br>S.5.10.2N | rt-pn-<br>maxic50fcpdvfs2.l<br>st | SS_PN_T_003 | Summary for Maximum BMS-<br>955176 IC50 Fold Change<br>Treated Subjects Identified as<br>Protocol Defined Virologic<br>Failures - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 310 | Table<br>S.5.10.10 | rt-pn-props1.lst | SS_PN_T_004 | Proportion of Subjects with<br>Greater than 3 Fold Increase in<br>BMS-955176 IC50 Fold Change<br>Treated Subjects with Baseline<br>and On-Treatment Phenotypic<br>Resistance Profile - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 311 | Table<br>S.5.10.2O | rt-pn-props2.lst | SS_PN_T_004 | Proportion of Subjects with<br>Greater than 3 Fold Increase in<br>BMS-955176 IC50 Fold Change<br>Treated Subjects with Baseline<br>and On-Treatment Phenotypic<br>Resistance Profile - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 312 | Table<br>S.5.10.3O | rt-pn-props12.lst | SS_PN_T_004 | Proportion of Subjects with<br>Greater than 3 Fold Increase in<br>BMS-955176 IC50 Fold Change<br>Treated Subjects with Baseline<br>and On-Treatment Phenotypic<br>Resistance Profile - Stage 1 and<br>2 | WK96S2 |

| No. | Table No. | Output File<br>Name | Template ID | Title and Population | Purpose |
|---|---|---|---|---|---|
| 313 | Table S.5.10.1P | rt-pn-<br>proppdvfs1.lst | SS_PN_T_004 | Proportion of Subjects with Greater than 3 Fold Increase in BMS-955176 IC50 Fold Change Treated Subjects Identified as Protocol Defined Virologic Failures with Baseline and On-Treatment Phenotypic Resistance Profile - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 314 | Table S.5.10.2P | rt-pn-<br>proppdvfs2.lst | SS_PN_T_004 | Proportion of Subjects with Greater than 3 Fold Increase in BMS-955176 IC50 Fold Change Treated Subjects Identified as Protocol Defined Virologic Failures with Baseline and On-Treatment Phenotypic Resistance Profile - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 315 | Table S.5.10.3P | rt-pn-<br>proppdvfs12.lst | SS_PN_T_004 | Proportion of Subjects with<br>Greater than 3 Fold Increase in<br>BMS-955176 IC50 Fold Change<br>Treated Subjects Identified as<br>Protocol Defined Virologic<br>Failures<br>with Baseline and On-Treatment<br>Phenotypic Resistance Profile -<br>Stage 1 and 2 | WK96S2 |
| 316 | Table<br>S.5.10.1V | rt-pn-<br>propnews1.lst | SS_PN_T_004 | Proportion of Subjects with<br>Newly Emergent Phenotypic<br>Resistance to BMS-955176<br>Treated Subjects with Baseline<br>and On-Treatment Phenotypic<br>Resistance Profile - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 317 | Table<br>S.5.10.2V | rt-pn-<br>propnews2.lst | SS_PN_T_004 | Proportion of Subjects with<br>Newly Emergent Phenotypic<br>Resistance to BMS-955176<br>Treated Subjects with Baseline<br>and On-Treatment Phenotypic<br>Resistance Profile - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 318 | Table<br>S.5.10.3V | rt-pn-<br>propnews12.lst | SS_PN_T_004 | Proportion of Subjects with<br>Newly Emergent Phenotypic<br>Resistance to BMS-955176<br>Treated Subjects with Baseline<br>and On-Treatment Phenotypic<br>Resistance Profile - Stage 1 and | WK96S2 |

| No. | Table No. | Output File<br>Name | Template ID | Title and Population | Purpose |
|---|---|---|---|---|---|
| 319 | Table<br>S.5.10.1W | rt-pn-<br>propnewpdvfs1.lst | SS_PN_T_004 | Proportion of Subjects with Newly Emergent Phenotypic Resistance to BMS-955176 Treated Subjects Identified as Protocol Defined Virologic Failures with Baseline and On-Treatment Phenotypic Resistance Profile - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 320 | Table<br>S.5.10.2W | rt-pn-<br>propnewpdvfs2.lst | SS_PN_T_004 | Proportion of Subjects with Newly Emergent Phenotypic Resistance to BMS-955176 Treated Subjects Identified as Protocol Defined Virologic Failures with Baseline and On-Treatment Phenotypic Resistance Profile - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 321 | Table<br>S.5.10.3W | rt-pn-<br>propnewpdvfs12.ls<br>t | SS_PN_T_004 | Proportion of Subjects with Newly Emergent Phenotypic Resistance to BMS-955176 Treated Subjects Identified as Protocol Defined Virologic Failures with Baseline and On-Treatment Phenotypic Resistance Profile - Stage 1 and 2 | WK96S2 |
| 322 | Table<br>S.5.10.1Q | rt-gn-<br>newgagincs1.lst | SS_GN_T_002 | Emergent Gag Polymorphisms Treated Subjects with Greater than 3 Fold Increase in BMS- 955176 IC50 Fold Change- Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 323 | Table<br>S.5.10.2Q | rt-gn-<br>newgagincs2.lst | SS_GN_T_002 | Emergent Gag Polymorphisms Treated Subjects with Greater than 3 Fold Increase in BMS- 955176 IC50 Fold Change- Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 324 | Table<br>S.5.10.3Q | rt-gn-<br>newgagincs12.lst | SS_GN_T_002 | Emergent Gag Polymorphisms Treated Subjects with Greater than 3 Fold Increase in BMS- 955176 IC50 Fold Change- Stage 1 and 2 | WK96S2 |
| 325 | Table S.5.11.1 | rt-vl-futw24s1.lst | SS_VL_T_007 | Test for Virologic Futility Based<br>on HIV-1 RNA < 40 c/mL<br>Proportion of Responders at<br>Week 24 (mITT)<br>Treated Subjects - Stage 1 | WK24S1 |
| 326 | Table S.5.11.2 | rt-vl-futw24s2.lst | SS_VL_T_007 | Test for Virologic Futility Based<br>on HIV-1 RNA < 40 c/mL<br>Proportion of Responders at<br>Week 24 (mITT)<br>Treated Subjects - Stage 2 | WK24S2 |

| No. | Table No. | Output File<br>Name | Template ID | Title and Population | Purpose |
|---|---|---|---|---|---|
| 327 | Table S.6.7.1 | rt-ae-<br>overallsums1.lst | SS_AE_T_001 | Adverse Events Overall Adverse Events Summary Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 328 | Table S.6.7.2 | rt-ae-<br>overallsums2.lst | SS_AE_T_001 | Adverse Events Overall Adverse Events Summary Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 329 | Table S.6.7.3 | rt-ae-<br>overallsums12.lst | SS_AE_T_001 | Adverse Events Overall Adverse Events Summary Treated Subjects - Stage 1 and 2 | WK96S2 |
| 330 | Table S.6.1.1 | rl-ae-deaths1.lst | SS_AE_L_001 | Death Listing<br>Enrolled Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 331 | Table S.6.1.2 | rl-ae-deaths2.lst | SS_AE_L_001 | Death Listing Enrolled Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 332 | Table S.6.2.1A | rt-ae-saes1.lst | GS_AE_T_X_001 | Adverse Event Summary Serious Adverse Events Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 333 | Table S.6.2.2A | rt-ae-saes2.lst | GS_AE_T_X_001 | Adverse Event Summary Serious Adverse Events Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 334 | Table S.6.2.3A | rt-ae-saes12.lst | GS_AE_T_X_001 | Adverse Event Summary Serious Adverse Events Treated Subjects - Stage 1 and 2 | WK96S2 |
| 335 | Table S.6.2.1B | rt-ae-saeconts1.lst | GS_AE_T_X_001 | Adverse Event Summary Serious Adverse Events After Switch to Continuation Dose Treated Subjects - Stage 1 | WK96S1,<br>WK96S2 |
| 336 | Table S.6.2.2B | rt-ae-saeconts2.lst | GS_AE_T_X_001 | Adverse Event Summary Serious Adverse Events After Switch to Continuation Dose Treated Subjects - Stage 2 | WK96S2 |
| 337 | Table S.6.2.1C | rt-ae-<br>saeldeaths1eu.lst | GS_AE_T_X_001 | Adverse Event Summary Serious Adverse Event With Death As An Outcome Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 338 | Table S.6.2.2C | rt-ae-<br>saeldeaths2eu.lst | GS_AE_T_X_001 | Adverse Event Summary Serious Adverse Event With Death As An Outcome Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 339 | Table S.6.2.1D | rt-ae-<br>relsaeldeaths1eu.lst | GS_AE_T_X_001 | Adverse Event Summary Drug Related Serious Adverse Event With Death As An Outcome Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |

| No. | Table No. | Output File<br>Name | Template ID | Title and Population | Purpose |
|---|---|---|---|---|---|
| 340 | Table S.6.2.2D | rt-ae-<br>relsaeldeaths2eu.lst | GS_AE_T_X_001 | Adverse Event Summary Drug Related Serious Adverse Event With Death As An Outcome Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 341 | Table S.6.2.1E | rl-ae-saes1.lst | GS_AE_L_S_001 | Adverse Event Serious Adverse Events Enrolled Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 342 | Table S.6.2.2E | rl-ae-saes2.lst | GS_AE_L_S_001 | Adverse Event Serious Adverse Events Enrolled Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 343 | Table S.6.3.1A | rt-ae-aediscs1.lst | GS_AE_T_X_001 | Adverse Event Summary Adverse Events Leading to Discontinuation of Study Medication Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 344 | Table S.6.3.2A | rt-ae-aediscs2.lst | GS_AE_T_X_001 | Adverse Event Summary Adverse Events Leading to Discontinuation of Study Medication Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 345 | Table S.6.3.3A | rt-ae-aediscs12.lst | GS_AE_T_X_001 | Adverse Event Summary Adverse Events Leading to Discontinuation of Study Medication Treated Subjects - Stage 1 and 2 | WK96S2 |
| 346 | Table S.6.3.1B | rt-ae-<br>aediscconts1.lst | GS_AE_T_X_001 | Adverse Event Summary Adverse Events Leading to Discontinuation of Study Medication After Switch to Continuation Dose Treated Subjects - Stage 1 | WK96S1,<br>WK96S2 |
| 347 | Table S.6.3.2B | rt-ae-<br>aediscconts2.lst | GS_AE_T_X_001 | Adverse Event Summary Adverse Events Leading to Discontinuation of Study Medication After Switch to Continuation Dose Treated Subjects - Stage 2 | WK96S2 |
| 348 | Table S.6.3.1C | rl-ae-discs1.lst | GS_AE_L_X_001 | Adverse Event Adverse Events Leading to Discontinuation of Study Medication Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 349 | Table S.6.3.2C | rl-ae-discs2.lst | GS_AE_L_X_001 | Adverse Event Adverse Events Leading to Discontinuation of Study Medication Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |

| No. | Table No. | Output File<br>Name | Template ID | Title and Population | Purpose |
|---|---|---|---|---|---|
| 350 | Table S.6.5.1A | rt-ae-nsae5pcts1.lst | GS_AE_T_X_001 | Adverse Event Summary Non-Serious Adverse Events Occurring in at Least 5 Percent of Treated Subjects Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 351 | Table S.6.5.2A | rt-ae-nsae5pcts2.lst | GS_AE_T_X_001 | Adverse Event Summary Non-Serious Adverse Events Occurring in at Least 5 Percent of Treated Subjects Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 352 | Table S.6.5.1B | rt-ae-<br>grade1to4s1.lst | GS_AE_T_X_001 | Adverse Event Summary Grade 1 to 4 Adverse Events Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 353 | Table S.6.5.2B | rt-ae-<br>grade1to4s2.lst | GS_AE_T_X_001 | Adverse Event Summary Grade 1 to 4 Adverse Events Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 354 | Table S.6.5.1C | rt-ae-<br>grade2to4s1.lst | GS_AE_T_X_001 | Adverse Event Summary Grade 2 to 4 Adverse Events Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 355 | Table S.6.5.2C | rt-ae-<br>grade2to4s2.lst | GS_AE_T_X_001 | Adverse Event Summary Grade 2 to 4 Adverse Events Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 356 | Table S.6.5.1D | rt-ae-<br>grade3to4s1.lst | GS_AE_T_X_001 | Adverse Event Summary Grade 3 to 4 Adverse Events Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 357 | Table S.6.5.2D | rt-ae-<br>grade3to4s2.lst | GS_AE_T_X_001 | Adverse Event Summary Grade 3 to 4 Adverse Events Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 358 | Table S.6.5.3D | rt-ae-<br>grade3to4s12.lst | GS_AE_T_X_001 | Adverse Event Summary Grade 3 to 4 Adverse Events Treated Subjects - Stage 1 and 2 | WK96S2 |
| 359 | Table S.6.5.1E | rt-ae-relateds1.lst | GS_AE_T_X_001 | Adverse Event Summary Grade 1 to 4 Related Adverse Events Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 360 | Table S.6.5.2E | rt-ae-relateds2.lst | GS_AE_T_X_001 | Adverse Event Summary Grade 1 to 4 Related Adverse Events Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 361 | Table S.6.5.1F | rt-ae-<br>relgrade2to4s1.lst | GS_AE_T_X_001 | Adverse Event Summary Grade 2 to 4 Related Adverse Events Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 362 | Table S.6.5.2F | rt-ae-<br>relgrade2to4s2.lst | GS_AE_T_X_001 | Adverse Event Summary Grade 2 to 4 Related Adverse Events Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |

| No. | Table No. | Output File<br>Name | Template ID | Title and Population | Purpose |
|---|---|---|---|---|---|
| 363 | Table S.6.5.3F | rt-ae-<br>relgrade2to4s12.lst | GS_AE_T_X_001 | Adverse Event Summary Grade 2 to 4 Related Adverse Events Treated Subjects - Stage 1 and 2 | WK96S2 |
| 364 | Table S.6.5.1G | rt-ae-<br>relgrade3to4s1.lst | GS_AE_T_X_001 | Adverse Event Summary Grade 3 to 4 Related Adverse Events Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 365 | Table S.6.5.2G | rt-ae-<br>relgrade3to4s2.lst | GS_AE_T_X_001 | Adverse Event Summary Grade 3 to 4 Related Adverse Events Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 366 | Appendix 6.5.1 | rl-ae-lists1.lst | GS_AEL_X_001 | Adverse Event Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 367 | Appendix 6.5.2 | rl-ae-lists2.lst | GS_AEL_X_001 | Adverse Event Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 368 | Table S.6.4.1A | rt-ae-cdcaes1.lst | GS_AE_T_X_001 | Adverse Event Summary CDC Class C AIDS Events Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 369 | Table S.6.4.2A | rt-ae-cdcaes2.lst | GS_AE_T_X_001 | Adverse Event Summary CDC Class C AIDS Events Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 370 | Table S.6.4.3A | rt-ae-cdcaes12.lst | GS_AE_T_X_001 | Adverse Event Summary CDC Class C AIDS Events Treated Subjects - Stage 1 and 2 | WK96S2 |
| 371 | Table S.6.4.1B | rl-ae-cdcaes1.lst | GS_AEL_X_001 | Adverse Event CDC Class C AIDS Events Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 372 | Table S.6.4.2B | rl-ae-cdcaes2.lst | GS_AEL_X_001 | Adverse Event CDC Class C AIDS Events Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 373 | Table S.6.4.1C | rt-ae-giaes1.lst | GS_AE_T_X_001 | Adverse Event Summary Gastrointestinal Events of Special Interest Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 374 | Table S.6.4.2C | rt-ae-giaes2.lst | GS_AE_T_X_001 | Adverse Event Summary Gastrointestinal Events of Special Interest Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 375 | Table S.6.4.3C | rt-ae-giaes12.lst | GS_AE_T_X_001 | Adverse Event Summary Gastrointestinal Events of Special Interest Treated Subjects - Stage 1 and 2 | WK96S2 |
| 376 | Table S.6.4.1D | rl-ae-giaes1.lst | GS_AE_L_X_001 | Adverse Event Gastrointestinal Events of Special Interest Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |

| No. | Table No. | Output File<br>Name | Template ID | Title and Population | Purpose |
|---|---|---|---|---|---|
| 377 | Table S.6.4.2D | rl-ae-giaes2.lst | GS_AE_L_X_001 | Adverse Event Gastrointestinal Events of Special Interest Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 378 | Table S.6.6.1A | rt-ae-<br>expadjusts1.lst | GS_AE_T_M_001 | Exposure Adjusted Adverse Events Summary Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 379 | Table S.6.6.2A | rt-ae-<br>expadjusts2.lst | GS_AE_T_M_001 | Exposure Adjusted Adverse Events Summary Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 380 | Table S.6.6.1B | rt-ae-<br>expadjsaes1eu.lst | GS_AE_T_M_001 | Exposure Adjusted Adverse Events Summary Including Multiple Occurrences of Unique Adverse Events Treated Subjects - Stage 1 Serious Adverse Events | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 381 | Table S.6.6.2B | rt-ae-<br>expadjsaes2eu.lst | GS_AE_T_M_001 | Exposure Adjusted Adverse Events Summary Including Multiple Occurrences of Unique Adverse Events Treated Subjects - Stage 2 Serious Adverse Events | WK24S2,<br>WK48S2,<br>WK96S2 |
| 382 | Table S.6.6.1C | rt-ae-<br>expadjrelsaes1eu.ls<br>t | GS_AE_T_M_001 | Exposure Adjusted Adverse Events Summary Including Multiple Occurrences of Unique Adverse Events Treated Subjects - Stage 1 Drug Related Serious Adverse Events | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 383 | Table S.6.6.2C | rt-ae-<br>expadjrelsaes2eu.ls<br>t | GS_AE_T_M_001 | Exposure Adjusted Adverse Events Summary Including Multiple Occurrences of Unique Adverse Events Treated Subjects - Stage 2 Drug Related Serious Adverse Events | WK24S2,<br>WK48S2,<br>WK96S2 |
| 384 | Table S.6.6.1D | rt-ae-<br>expadjnsae5pcts1e<br>u.lst | GS_AE_T_M_001 | Exposure Adjusted Adverse Event Summary Including Multiple Occurrences of Unique Adverse Events Treated Subjects - Stage 1 Non-Serious Adverse Events Using a Global Cutoff of 5 Percent | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 385 | Table S.6.6.2D | rt-ae-<br>expadjnsae5pcts2e<br>u.lst | GS_AE_T_M_001 | Exposure Adjusted Adverse Event Summary Including Multiple Occurrences of Unique Adverse Events Treated Subjects - Stage 2 Non-Serious Adverse Events Using a Global Cutoff of 5 Percent | WK24S2,<br>WK48S2,<br>WK96S2 |

| No. | Table No. | Output File<br>Name | Template ID | Title and Population | Purpose |
|---|---|---|---|---|---|
| 386 | Appendix 6.6.1 | rl-ae-uniques1.lst | GS_AE_L_U_002 | Adverse Event | WK24S1, |
| | | | | Unique Events | WK48S1, |
| | | | | Treated Subjects - Stage 1 | WK96S1, |
| | | | | | WK96S2 |
| 387 | Appendix 6.6.2 | rl-ae-uniques2.lst | GS_AE_L_U_002 | Adverse Event | WK24S2, |
| | | | | Unique Events | WK48S2, |
| | | | | Treated Subjects - Stage 2 | WK96S2 |
| 388 | Table S.7.1.1A | rt-lb-toxs1.lst | SS_LB_T_001 | Laboratory Test Results | WK24S1, |
| | | | | Summary of Worst Toxicity | WK48S1, |
| | | | | Grade | WK96S1, |
| 200 | T 11 0 7 1 0 1 | . 11 | GG I D T 001 | Treated Subjects - Stage 1 | WK96S2 |
| 389 | Table S.7.1.2A | rt-lb-toxs2.lst | SS_LB_T_001 | Laboratory Test Results | WK24S2, |
| | | | | Summary of Worst Toxicity | WK48S2, |
| | | | | Grade | WK96S2 |
| 390 | Table S.7.1.1B | wt lb a24tava1 lat | CC ID T 001 | Treated Subjects - Stage 2 Laboratory Test Results | WW24C1 |
| 390 | 1 able 5.7.1.1B | rt-lb-g34toxs1.lst | SS_LB_T_001 | _ | WK24S1,<br>WK48S1, |
| | | | | Summary of Grade 3-4 Toxicity Treated Subjects - Stage 1 | WK4881,<br>WK96S1, |
| | | | | Treated Subjects - Stage 1 | WK96S1,<br>WK96S2 |
| 391 | Table S.7.1.2B | rt-lb-g34toxs2.lst | SS LB T 001 | Laboratory Test Results | WK24S2, |
| 371 | 1 autc 5.7.1.2D | 11-10-95410352.151 | 35_LD_1_001 | Summary of Grade 3-4 Toxicity | WK48S2, |
| | | | | Treated Subjects - Stage 2 | WK96S2, |
| 392 | Table S.7.1.3B | rt-lb-g34toxs12.lst | SS LB T 001 | Laboratory Test Results | WK96S2 |
| 372 | 1 4010 5.7.1.51 | 11-10-854103512.151 | 55_LD_1_001 | Summary of Grade 3-4 Toxicity | W K 7052 |
| | | | | Treated Subjects - Stage 1 and 2 | |
| 393 | Table S.7.1.1C | rt-lb-etoxs1.lst | SS LB T 001 | Laboratory Test Results | WK24S1, |
| | | | | Summary of Treatment- | WK48S1, |
| | | | | Emergent Abnormalities | WK96S1, |
| | | | | Treated Subjects - Stage 1 | WK96S2 |
| 394 | Table S.7.1.2C | rt-lb-etoxs2.lst | SS_LB_T_001 | Laboratory Test Results | WK24S2, |
| | | | | Summary of Treatment- | WK48S2, |
| | | | | Emergent Abnormalities | WK96S2 |
| | | | | Treated Subjects - Stage 2 | |
| 395 | Table S.7.2.1A | rt-lb-renals1.lst | SS_VL_T_006 | Laboratory Test Results | WK24S1, |
| | | | | Summary Statistics for Renal | WK48S1, |
| | | | | Function Values and Change | WK96S1, |
| | | | | from Baseline - SI Units | WK96S2 |
| 206 | Table S.7.2.2A | # 1b #0# 1 2 1 1 4 | CC VI T OOC | Treated Subjects - Stage 1 | WEDARD |
| 396 | 1 aute 5.7.2.2A | rt-lb-renals2.lst | SS_VL_T_006 | Laboratory Test Results Summary Statistics for Renal | WK24S2,<br>WK48S2, |
| | | | | Function Values and Change | WK46S2,<br>WK96S2 |
| | | | | from Baseline - SI Units | W K9002 |
| | | | | Treated Subjects - Stage 2 | |
| 397 | Table S.7.2.1B | rt-zl-renals1.lst | SS_VL_T_006 | Laboratory Test Results | WK24S1, |
| | | 10 21 10111101.101 | | Summary Statistics for Renal | WK48S1, |
| | | | | Function Values and Change | WK96S1, |
| | | | | from Baseline - US Units | WK96S2 |
| | | | | Treated Subjects - Stage 1 | |
| 398 | Table S.7.2.2B | rt-zl-renals2.lst | SS_VL_T_006 | Laboratory Test Results | WK24S2, |
| | | | | Summary Statistics for Renal | WK48S2, |
| | | | | Function Values and Change | WK96S2 |
| | | | | from Baseline - US Units | |
| | | | | Treated Subjects - Stage 2 | |

| No. | Table No. | Output File<br>Name | Template ID | Title and Population | Purpose |
|---|---|---|---|---|---|
| 399 | Table S.7.2.1C | rt-lb-lipidss1.lst | SS_VL_T_006 | Laboratory Test Results Summary Statistics for Fasting Lipid Values and Change from Baseline - SI Units | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| | | | | Treated Subjects - Stage 1 | |
| 400 | Table S.7.2.2C | rt-lb-lipidss2.lst | SS_VL_T_006 | Laboratory Test Results Summary Statistics for Fasting Lipid Values and Change from Baseline - SI Units Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 401 | Table S.7.2.1D | rt-zl-lipidss1.lst | SS_VL_T_006 | Laboratory Test Results Summary Statistics for Fasting Lipid Values and Change from Baseline - US Units Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 402 | Table S.7.2.2D | rt-zl-lipidss2.lst | SS_VL_T_006 | Laboratory Test Results Summary Statistics for Fasting Lipid Values and Change from Baseline - US Units Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 403 | Table S.7.2.1E | rt-lb-<br>pchglipidss1.lst | SS_VL_T_006 | Laboratory Test Results Summary Statistics for Fasting Lipid Values and Percent Change from Baseline - SI Units Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 404 | Table S.7.2.2E | rt-lb-<br>pchglipidss2.lst | SS_VL_T_006 | Laboratory Test Results Summary Statistics for Fasting Lipid Values and Percent Change from Baseline - SI Units Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 405 | Table S.7.2.1F | rt-zl-<br>pchglipidss1.lst | SS_VL_T_006 | Laboratory Test Results Summary Statistics for Fasting Lipid Values and Percent Change from Baseline - US Units Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 406 | Table S.7.2.2F | rt-zl-<br>pchglipidss2.lst | SS_VL_T_006 | Laboratory Test Results Summary Statistics for Fasting Lipid Values and Percent Change from Baseline - US Units Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 407 | Figure S.7.2.1A | rg-lb-tchols1 | GS_LB_G_002 | Fasting Total Cholesterol<br>(mg/dL) Mean Percent Change<br>from Baseline Over Time<br>Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 408 | Figure S.7.2.2A | rg-lb-tchols2 | GS_LB_G_002 | Fasting Total Cholesterol<br>(mg/dL) Mean Percent Change<br>from Baseline Over Time<br>Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |

| No. | Table No. | Output File<br>Name | Template ID | Title and Population | Purpose |
|---|---|---|---|---|---|
| 409 | Figure S.7.2.1B | rg-lb-ldlcs1 | GS_LB_G_002 | Fasting LDL-Cholesterol<br>(mg/dL) Mean Percent Change<br>from Baseline Over Time<br>Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 410 | Figure S.7.2.2B | rg-lb-ldlcs2 | GS_LB_G_002 | Fasting LDL-Cholesterol<br>(mg/dL) Mean Percent Change<br>from Baseline Over Time<br>Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 411 | Figure S.7.2.1C | rg-lb-hdlcs1 | GS_LB_G_002 | Fasting HDL-Cholesterol<br>(mg/dL) Mean Percent Change<br>from Baseline Over Time<br>Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 412 | Figure S.7.2.2C | rg-lb-hdlcs2 | GS_LB_G_002 | Fasting HDL-Cholesterol (mg/dL) Mean Percent Change from Baseline Over Time Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 413 | Figure S.7.2.1D | rg-lb-trigs1 | GS_LB_G_002 | Fasting Total Triglycerides<br>(mg/dL) Mean Percent Change<br>from Baseline Over Time<br>Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 414 | Figure S.7.2.2D | rg-lb-trigs2 | GS_LB_G_002 | Fasting Total Triglycerides<br>(mg/dL) Mean Percent Change<br>from Baseline Over Time<br>Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 415 | Appendix<br>7.1.1A | rl-lb-hems1.lst | SS_LB_L_001 | Hematology - SI Units<br>Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 416 | Appendix 7.1.2A | rl-lb-hems2.lst | SS_LB_L_001 | Hematology - SI Units<br>Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 417 | Appendix<br>7.1.1B | rl-lb-lfts1.lst | SS_LB_L_001 | Liver Function Tests - SI Units<br>Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 418 | Appendix 7.1.2B | rl-lb-lfts2.lst | SS_LB_L_001 | Liver Function Tests - SI Units<br>Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 419 | Appendix<br>7.1.1C | rl-lb-enzs1.lst | SS_LB_L_001 | Enzymes - SI Units<br>Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 420 | Appendix 7.1.2C | rl-lb-enzs2.lst | SS_LB_L_001 | Enzymes - SI Units<br>Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 421 | Appendix<br>7.1.1D | rl-lb-rfts1.lst | SS_LB_L_001 | Renal Function Tests - SI Units<br>Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 422 | Appendix 7.1.2D | rl-lb-rfts2.lst | SS_LB_L_001 | Renal Function Tests - SI Units<br>Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |

| No. | Table No. | Output File<br>Name | Template ID | Title and Population | Purpose |
|---|---|---|---|---|---|
| 423 | Appendix 7.1.1E | rl-lb-elcs1.lst | SS_LB_L_001 | Electrolytes - SI Units<br>Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1, |
| | | | | | WK96S2 |
| 424 | Appendix | rl-lb-elcs2.lst | SS_LB_L_001 | Electrolytes - SI Units | WK24S2, |
| | 7.1.2E | | | Treated Subjects - Stage 2 | WK48S2,<br>WK96S2 |
| 425 | Appendix | rl-lb-flgs1.lst | SS_LB_L_001 | Fasting Lipids and Glucose - SI | WK24S1, |
| | 7.1.1F | | | Units | WK48S1, |
| | | | | Treated Subjects - Stage 1 | WK96S1, |
| 426 | Appendix | rl-lb-flgs2.lst | SS LB L 001 | Fasting Lipids and Glucose - SI | WK96S2<br>WK24S2, |
| 420 | 7.1.2F | 11-10-11g52.15t | 35_LD_L_001 | Units | WK48S2, |
| | 7.1.21 | | | Treated Subjects - Stage 2 | WK96S2, |
| 427 | Appendix | rl-zl-hems1.lst | SS LB L 001 | Hematology - US Units | WK24S1, |
| | 7.1.1G | | ~~ | Treated Subjects - Stage 1 | WK48S1, |
| | | | | , , , | WK96S1, |
| | | | | | WK96S2 |
| 428 | Appendix | rl-zl-hems2.lst | SS_LB_L_001 | Hematology - US Units | WK24S2, |
| | 7.1.2G | | | Treated Subjects - Stage 2 | WK48S2, |
| | | | | | WK96S2 |
| 429 | Appendix | rl-zl-lfts1.lst | SS_LB_L_001 | Liver Function Tests - US Units | WK24S1, |
| | 7.1.1H | | | Treated Subjects - Stage 1 | WK48S1, |
| | | | | | WK96S1, |
| 120 | A 1: | .1 -1 10 -2 1-4 | CC ID I 001 | Live Fandian Tark HCHaire | WK96S2 |
| 430 | Appendix | rl-zl-lfts2.lst | SS_LB_L_001 | Liver Function Tests - US Units | WK24S2, |
| | 7.1.2H | | | Treated Subjects - Stage 2 | WK48S2,<br>WK96S2 |
| 431 | Appendix | rl-zl-enzs1.lst | SS LB L 001 | Enzymes - US Units | WK24S1, |
| 431 | 7.1.1I | 11 ZI CHZST.ISt | 55_EB_E_001 | Treated Subjects - Stage 1 | WK48S1, |
| | , | | | Treated Subjects Stage 1 | WK96S1, |
| | | | | | WK96S2 |
| 432 | Appendix | rl-zl-enzs2.lst | SS LB L 001 | Enzymes - US Units | WK24S2, |
| | 7.1.2I | | | Treated Subjects - Stage 2 | WK48S2, |
| | | | | | WK96S2 |
| 433 | Appendix | rl-zl-rfts1.lst | SS_LB_L_001 | Renal Function Tests - US Units | WK24S1, |
| | 7.1.1J | | | Treated Subjects - Stage 1 | WK48S1, |
| | | | | | WK96S1, |
| 12.1 | | 1 1 0 01 | GG ID I 001 | D ID II D II D II D II D II D II D II | WK96S2 |
| 434 | Appendix | rl-zl-rfts2.lst | SS_LB_L_001 | Renal Function Tests - US Units | WK24S2, |
| | 7.1.2J | | | Treated Subjects - Stage 2 | WK48S2,<br>WK96S2 |
| 435 | Appendix | rl-zl-elcs1.lst | SS LB L 001 | Electrolytes - US Units | WK24S1, |
| 733 | 7.1.1K | 11-21-01051.151 | 33_LD_L_001 | Treated Subjects - Stage 1 | WK48S1, |
| | /.1.11X | | | Treated Subjects Stage 1 | WK96S1, |
| | | | | | WK96S2 |
| 436 | Appendix | rl-zl-elcs2.lst | SS LB L 001 | Electrolytes - US Units | WK24S2. |
| | 7.1.2K | | | Treated Subjects - Stage 2 | WK48S2. |
| | | | | | WK96S2 |
| 437 | Appendix | rl-zl-flgs1.lst | SS_LB_L_001 | Fasting Lipids and Glucose - US | WK24S1, |
| | 7.1.1L | | _ | Units | WK48S1, |
| | | | | Treated Subjects - Stage 1 | WK96S1, |
| | | | | | WK96S2 |

| No. | Table No. | Output File<br>Name | Template ID | Title and Population | Purpose |
|---|---|---|---|---|---|
| 438 | Appendix 7.1.2L | rl-zl-flgs2.lst | SS_LB_L_001 | Fasting Lipids and Glucose - US Units Units | WK24S2,<br>WK48S2, |
| 439 | Appendix 7.1.1M | rl-lb-diffunits1.lst | GS_LB_L_S_008 | Treated Subjects - Stage 2 Differences in Categorization of SI and US Laboratory Test Results | WK96S2<br>WK24S1,<br>WK48S1,<br>WK96S1, |
| 440 | Appendix 7.1.2M | rl-lb-diffunits2.lst | GS_LB_L_S_008 | Treated Subjects - Stage 1 Differences in Categorization of SI and US Laboratory Test Results Treated Subjects - Stage 2 | WK96S2<br>WK24S2,<br>WK48S2,<br>WK96S2 |
| 441 | Appendix<br>7.1.1N | rl-lb-pregs1.lst | GS_LB_L_X_006 | Pregnancy Test Treated Female Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 442 | Appendix 7.1.2N | rl-lb-pregs2.lst | GS_LB_L_X_006 | Pregnancy Test Treated Female Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 443 | Appendix 7.3.1A | rt-eg-sumchgs1.lst | SS_EG_T_003 | Electrocardiogram Summary of<br>Values and Changes from<br>Baseline over Time<br>Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 444 | Appendix 7.3.2A | rt-eg-sumchgs2.lst | SS_EG_T_003 | Electrocardiogram Summary of<br>Values and Changes from<br>Baseline over Time<br>Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 445 | Appendix<br>7.3.1B | rt-eg-<br>changecats1.lst | SS_EG_T_001 | Electrocardiogram Change from<br>Baseline Category Summary<br>Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 446 | Appendix 7.3.2B | rt-eg-<br>changecats2.lst | SS_EG_T_001 | Electrocardiogram Change from<br>Baseline Category Summary<br>Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 447 | Appendix 7.3.1C | rt-eg-cats1.lst | SS_EG_T_002 | Electrocardiogram Category Summary Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 448 | Appendix 7.3.2C | rt-eg-cats2.lst | SS_EG_T_002 | Electrocardiogram Category Summary Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 449 | Appendix 7.3.1D | rl-eg-ecgs1.lst | GS_EG_L_X_001 | Electrocardiogram Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 450 | Appendix 7.3.2D | rl-eg-ecgs2.lst | GS_EG_L_X_001 | Electrocardiogram Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 451 | Appendix<br>7.4.1A | rt-vs-sums1.lst | SS_VL_T_006 | Vital Sign Summary of Values<br>and Changes from Baseline over<br>Time<br>Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |

| No. | Table No. | Output File<br>Name | Template ID | Title and Population | Purpose |
|---|---|---|---|---|---|
| 452 | Appendix<br>7.4.2A | rt-vs-sums2.lst | SS_VL_T_006 | Vital Sign Summary of Values<br>and Changes from Baseline over<br>Time<br>Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 453 | Appendix<br>7.4.1B | rl-vs-lists1.lst | GS_VS_L_X_006 | Vital Signs Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 454 | Appendix 7.4.2B | rl-vs-lists2.lst | GS_VS_L_X_006 | Vital Signs Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 455 | Appendix<br>7.4.1C | rt-pm-sums1.lst | SS_VL_T_006 | Physical Measurements Summary of Values and Changes from Baseline over Time Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 456 | Appendix<br>7.4.2C | rt-pm-sums2.lst | SS_VL_T_006 | Physical Measurements Summary of Values and Changes from Baseline over Time Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 457 | Table S.7.5.1A | rt-lb-bmrenals1.lst | SS_VL_T_006 | Laboratory Test Results Summary Statistics for Renal Biomarker Values and Change from Baseline - US Units Treated Subjects - Stage 1 | WK96S1,<br>WK96S2 |
| 458 | Table S.7.5.2A | rt-lb-bmrenals2.lst | SS_VL_T_006 | Laboratory Test Results Summary Statistics for Renal Biomarker Values and Change from Baseline - US Units | WK96S2 |
| 459 | Table S.7.5.1B | rt-zl-bmrenals1.lst | SS_VL_T_006 | Treated Subjects - Stage 2 Laboratory Test Results Summary Statistics for Renal Biomarker Values and Change from Baseline - SI Units Treated Subjects - Stage 1 | WK96S1,<br>WK96S2 |
| 460 | Table S.7.5.2B | rt-zl-bmrenals2.lst | SS_VL_T_006 | Laboratory Test Results Summary Statistics for Renal Biomarker Values and Change from Baseline - SI Units Treated Subjects - Stage 2 | WK96S2 |
| 461 | Table S.7.5.1C | rt-lb-<br>pchbmrenals1.lst | SS_VL_T_006 | Laboratory Test Results Summary Statistics for Renal Biomarker Values and Percent Change from Baseline - US Units Treated Subjects - Stage 1 | WK96S1,<br>WK96S2 |
| 462 | Table S.7.5.2C | rt-lb-<br>pchbmrenals2.lst | SS_VL_T_006 | Laboratory Test Results Summary Statistics for Renal Biomarker Values and Percent Change from Baseline - US Units Treated Subjects - Stage 2 | WK96S2 |

| No. | Table No. | Output File<br>Name | Template ID | Title and Population | Purpose |
|---|---|---|---|---|---|
| 463 | Table S.7.5.1D | rt-zl-<br>pchbmrenals1.lst | SS_VL_T_006 | Laboratory Test Results Summary Statistics for Renal Biomarker Values and Percent Change from Baseline - SI Units Treated Subjects - Stage 1 | WK96S1,<br>WK96S2 |
| 464 | Table S.7.5.2D | rt-zl-<br>pchbmrenals2.lst | SS_VL_T_006 | Laboratory Test Results Summary Statistics for Renal Biomarker Values and Percent Change from Baseline - SI Units Treated Subjects - Stage 2 | WK96S2 |
| 465 | Table S.7.5.1E | rt-lb-bmbones1.lst | SS_VL_T_006 | Laboratory Test Results Summary Statistics for Bone Biomarker Values and Change from Baseline - US Units Treated Subjects - Stage 1 | WK24S1 |
| 466 | Table S.7.5.2E | rt-lb-bmbones2.lst | SS_VL_T_006 | Laboratory Test Results Summary Statistics for Bone Biomarker Values and Change from Baseline - US Units Treated Subjects - Stage 2 | WK24S2 |
| 467 | Table S.7.5.1F | rt-zl-bmbones1.lst | SS_VL_T_006 | Laboratory Test Results Summary Statistics for Bone Biomarker Values and Change from Baseline - SI Units Treated Subjects - Stage 1 | WK24S1 |
| 468 | Table S.7.5.2F | rt-zl-bmbones2.lst | SS_VL_T_006 | Laboratory Test Results Summary Statistics for Bone Biomarker Values and Change from Baseline - SI Units Treated Subjects - Stage 2 | WK24S2 |
| 469 | Table S.7.5.1G | rt-lb-<br>pchbmbones1.lst | SS_VL_T_006 | Laboratory Test Results Summary Statistics for Bone Biomarker Values and Percent Change from Baseline - US Units Treated Subjects - Stage 1 | WK24S1 |
| 470 | Table S.7.5.2G | rt-lb-<br>pchbmbones2.lst | SS_VL_T_006 | Laboratory Test Results Summary Statistics for Bone Biomarker Values and Percent Change from Baseline - US Units Treated Subjects - Stage 2 | WK24S2 |
| 471 | Table S.7.5.1H | rt-zl-<br>pchbmbones1.lst | SS_VL_T_006 | Laboratory Test Results Summary Statistics for Bone Biomarker Values and Percent Change from Baseline - SI Units Treated Subjects - Stage 1 | WK24S1 |
| 472 | Table S.7.5.2H | rt-zl-<br>pchbmbones2.lst | SS_VL_T_006 | Laboratory Test Results Summary Statistics for Bone Biomarker Values and Percent Change from Baseline - SI Units Treated Subjects - Stage 2 | WK24S2 |

| No. | Table No. | Output File<br>Name | Template ID | Title and Population | Purpose |
|---|---|---|---|---|---|
| 473 | Figure S.7.5.1A | rg-lb-ub2s1 | GS_LB_G_002 | Urinary Beta-2- Microglobulin/Creatinine Median Percent Change from Baseline Over Time Treated Subjects - Stage 1 | WK24S1 |
| 474 | Figure S.7.5.2A | rg-lb-ub2s2 | GS_LB_G_002 | Urinary Beta-2- Microglobulin/Creatinine Median Percent Change from Baseline Over Time Treated Subjects - Stage 2 | WK24S2 |
| 475 | Figure S.7.5.1B | rg-lb-feps1 | GS_LB_G_002 | Fractional Excretion of Phosphorous Median Change from Baseline Over Time Treated Subjects - Stage 1 | WK24S1 |
| 476 | Figure S.7.5.2B | rg-lb-feps2 | GS_LB_G_002 | Fractional Excretion of Phosphorous Median Change from Baseline Over Time Treated Subjects - Stage 2 | WK24S2 |
| 477 | Figure S.7.5.1C | rg-lb-pchp1nps1 | GS_LB_G_002 | N-Terminal Propeptide of Type 1 Procollagen Median Percent Change from Baseline Over Time Treated Subjects - Stage 1 | WK96S1,<br>WK96S2 |
| 478 | Figure S.7.5.2C | rg-lb-pchp1nps2 | GS_LB_G_002 | N-Terminal Propeptide of Type 1 Procollagen Median Percent Change from Baseline Over Time Treated Subjects - Stage 2 | WK96S2 |
| 479 | Figure S.7.5.1D | rg-lb-pchctxs1 | GS_LB_G_002 | Cross-Linked C-Telopeptide of<br>Type 1 Collagen Median Percent<br>Change from Baseline Over<br>Time<br>Treated Subjects - Stage 1 | WK96S1,<br>WK96S2 |
| 480 | Figure S.7.5.2D | rg-lb-pchctxs2 | GS_LB_G_002 | Cross-Linked C-Telopeptide of<br>Type 1 Collagen Median Percent<br>Change from Baseline Over<br>Time<br>Treated Subjects - Stage 2 | WK96S2 |
| 481 | Table S.8.1.1A | rt-pk-sumbmss1.lst | MS_PK_T_004 | Summary Statistics of BMS-<br>955176 Pharmacokinetic<br>Parameters<br>Evaluable PK Population - Stage | WK24S1 |
| 482 | Table S.8.1.2A | rt-pk-sumbmss2.lst | MS_PK_T_004 | Summary Statistics of BMS-<br>955176 Pharmacokinetic<br>Parameters<br>Evaluable PK Population - Stage | WK24S2 |
| 483 | Table S.8.1.1B | rt-pk-sumatvs1.lst | MS_PK_T_004 | Summary Statistics of ATV Pharmacokinetic Parameters Evaluable PK Population - Stage | WK24S1 |

| No. | Table No. | Output File<br>Name | Template ID | Title and Population | Purpose |
|---|---|---|---|---|---|
| 484 | Table S.8.1.2B | rt-pk-sumatvs2.lst | MS_PK_T_004 | Summary Statistics of ATV Pharmacokinetic Parameters Evaluable PK Population - Stage 2 | WK24S2 |
| 485 | Table S.8.1.1C | rt-pk-sumdtgs1.lst | MS_PK_T_004 | Summary Statistics of DTG Pharmacokinetic Parameters Evaluable PK Population - Stage | WK24S1 |
| 486 | Table S.8.1.2C | rt-pk-sumdtgs2.lst | MS_PK_T_004 | Summary Statistics of DTG Pharmacokinetic Parameters Evaluable PK Population - Stage 2 | WK24S2 |
| 487 | Table 9.2.1A | rt-pk-<br>itsumbmss1.lst | MS_PK_T_005 | Summary Statistics of BMS-<br>955176 Pharmacokinetic<br>Parameters<br>Evaluable PK Population - Stage | WK24S1 |
| 488 | Table 9.2.2A | rt-pk-<br>itsumbmss2.lst | MS_PK_T_005 | Summary Statistics of BMS-<br>955176 Pharmacokinetic<br>Parameters<br>Evaluable PK Population - Stage<br>2 | WK24S2 |
| 489 | Table 9.3.1A | rt-pk-<br>itsumdtgs1.lst | MS_PK_T_005 | Summary Statistics of DTG Pharmacokinetic Parameters Evaluable PK Population - Stage | WK24S1 |
| 490 | Table 9.3.2A | rt-pk-<br>itsumdtgs2.lst | MS_PK_T_005 | Summary Statistics of DTG Pharmacokinetic Parameters Evaluable PK Population - Stage 2 | WK24S2 |
| 491 | Table 9.4.1A | rt-pk-itsumatvs1.lst | MS_PK_T_005 | Summary Statistics of ATV Pharmacokinetic Parameters Evaluable PK Population - Stage | WK24S1 |
| 492 | Table 9.4.2A | rt-pk-itsumatvs2.lst | MS_PK_T_005 | Summary Statistics of ATV Pharmacokinetic Parameters Evaluable PK Population - Stage 2 | WK24S2 |
| 493 | Table<br>S.8.2.5.1A | rt-pk-<br>mixedbmsdtgs1.lst | MS_PK_T_006 | Effect of BMS-955176 on Exposure of DTG PK Parameters DTG Cmax, Ctau and AUC(TAU) BMS-955176 120 mg QD+ ATV/r + DTG versus TDF + ATV/r + DTG Evaluable PK Population - Stage | WK24S1 |

| No. | Table No. | Output File<br>Name | Template ID | Title and Population | Purpose |
|---|---|---|---|---|---|
| 494 | Table<br>S.8.2.5.2A | rt-pk-<br>mixedbms120dtgs2<br>.lst | MS_PK_T_006 | Effect of BMS-955176 on Exposure of DTG PK Parameters DTG Cmax, Ctau and AUC(TAU) BMS-955176 120 mg QD+ ATV + DTG versus Historical Data Evaluable PK Population - Stage | WK24S2 |
| 495 | Table<br>S.8.2.5.2B | rt-pk-<br>mixedbms180dtgs2<br>.lst | MS_PK_T_006 | Effect of BMS-955176 on Exposure of DTG PK Parameters DTG Cmax, Ctau and AUC(TAU) BMS-955176 180 mg QD+ ATV + DTG versus Historical Data Evaluable PK Population - Stage | WK24S2 |
| 496 | Table 9.3.1.1A | rt-pk-<br>itmixedbmss1.lst | MS_PK_T_007 | In-text Table of Effect of BMS- 955176 on Exposure of DTG PK Parameters DTG Cmax, Ctau and AUC(TAU) BMS-955176 120 mg QD+ ATV/r + DTG versus TDF + ATV/r + DTG Evaluable PK Population - Stage | WK24S1 |
| 497 | Table 9.3.1.2A | rt-pk-<br>itmixedbms120s2.1<br>st | MS_PK_T_007 | In-text Table of Effect of BMS- 955176 on Exposure of DTG PK Parameters DTG Cmax, Ctau and AUC(TAU) BMS-955176 120 mg QD+ ATV + DTG versus TDF + ATV/r + DTG Evaluable PK Population - Stage | WK24S2 |
| 498 | Table 9.3.1.2B | rt-pk-<br>itmixedbms180s2.1<br>st | MS_PK_T_007 | In-text Table of Effect of BMS-<br>955176 on Exposure of DTG<br>PK Parameters DTG Cmax,<br>Ctau and AUC(TAU)<br>BMS-955176 180 mg QD+<br>ATV + DTG versus TDF +<br>ATV/r + DTG<br>Evaluable PK Population - Stage | WK24S2 |
| 499 | Appendix<br>8.2.5A | rl-pk-<br>listbms01s1.lst | MS_PK_L_005 | Listing of BMS-955176 Pharmacokinetic Parameters PK Population - Stage 1 | WK24S1 |
| 500 | Appendix<br>8.2.5A | rl-pk-<br>listbms01s2.lst | MS_PK_L_005 | Listing of BMS-955176 Pharmacokinetic Parameters PK Population - Stage 2 | WK24S2 |

| No. | Table No. | Output File<br>Name | Template ID | Title and Population | Purpose |
|---|---|---|---|---|---|
| 501 | Appendix<br>8.2.5B | rl-pk-listatv01s1.lst | MS_PK_L_005 | Listing of ATV Pharmacokinetic Parameters PK Population - Stage 1 | WK24S1 |
| 502 | Appendix<br>8.2.5B | rl-pk-listatv01s2.lst | MS_PK_L_005 | Listing of ATV Pharmacokinetic Parameters PK Population - Stage 2 | WK24S2 |
| 503 | Appendix 8.2.5C | rl-pk-<br>listdtg01s1.lst | MS_PK_L_005 | Listing of DTG Pharmacokinetic Parameters PK Population - Stage 1 | WK24S1 |
| 504 | Appendix 8.2.5C | rl-pk-<br>listdtg01s2.lst | MS_PK_L_005 | Listing of DTG Pharmacokinetic Parameters PK Population - Stage 2 | WK24S2 |
| 505 | Appendix 8.2.1A | rl-pk-<br>cpar1bmss1.lst | MS_PK_L_001 | Listing of BMS-955176 Plasma<br>Concentration – Time Data<br>PK Population - Stage 1 | WK24S1 |
| 506 | Appendix 8.2.1A | rl-pk-<br>cpar1bmss2.lst | MS_PK_L_001 | Listing of BMS-955176 Plasma<br>Concentration – Time Data<br>PK Population - Stage 2 | WK24S2 |
| 507 | Appendix 8.2.1B | rl-pk-cpar1atvs1.lst | MS_PK_L_001 | Listing of ATV Plasma Concentration – Time Data PK Population - Stage 1 | WK24S1 |
| 508 | Appendix 8.2.1B | rl-pk-cpar1atvs2.lst | MS_PK_L_001 | Listing of ATV Plasma Concentration – Time Data PK Population - Stage 2 | WK24S2 |
| 509 | Appendix 8.2.1C | rl-pk-<br>cpar1dtgs1.lst | MS_PK_L_001 | Listing of DTG Plasma Concentration – Time Data PK Population - Stage 1 | WK24S1 |
| 510 | Appendix 8.2.1C | rl-pk-<br>cpar1dtgs2.lst | MS_PK_L_001 | Listing of DTG Plasma Concentration – Time Data PK Population - Stage 2 | WK24S2 |
| 511 | Figure S.8.2.3A | rg-pk-<br>cpar3bmss1.lst | MS_PK_G_002 | Plots of Individual BMS-955176 Plasma Concentration Profiles vs. Time Evaluable PK Population - Stage | WK24S1 |
| 512 | Figure S.8.2.3A | rg-pk-<br>cpar3bmss2.lst | MS_PK_G_002 | Plots of Individual BMS-955176 Plasma Concentration Profiles vs. Time Evaluable PK Population - Stage 2 | WK24S2 |
| 513 | Figure S.8.2.3B | rg-pk-<br>cpar3atvs1.lst | MS_PK_G_002 | Plots of Individual ATV Plasma<br>Concentration Profiles vs. Time<br>Evaluable PK Population- Stage<br>1 | WK24S1 |
| 514 | Figure S.8.2.3B | rg-pk-<br>cpar3atvs2.lst | MS_PK_G_002 | Plots of Individual ATV Plasma<br>Concentration Profiles vs. Time<br>Evaluable PK Population- Stage<br>2 | WK24S2 |
| 515 | Figure S.8.2.3C | rg-pk-<br>cpar3dtgs1.lst | MS_PK_G_002 | Plots of Individual DTG Plasma<br>Concentration Profiles vs. Time<br>Evaluable PK Population - Stage<br>1 | WK24S1 |

| No. | Table No. | Output File<br>Name | Template ID | Title and Population | Purpose |
|---|---|---|---|---|---|
| 516 | Figure S.8.2.3C | rg-pk-<br>cpar3dtgs2.lst | MS_PK_G_002 | Plots of Individual DTG Plasma<br>Concentration Profiles vs. Time<br>Evaluable PK Population - Stage<br>2 | WK24S2 |
| 517 | Figure S.8.2.1A | rg-pk-<br>cpar1bmss1.lst | MS_PK_G_001 | Overlay of Individual BMS-<br>955176 Plasma Concentration<br>Profile vs. Time by Treatment<br>Evaluable PK Population - Stage | WK24S1 |
| 518 | Figure S.8.2.1A | rg-pk-<br>cpar1bmss2.lst | MS_PK_G_001 | Overlay of Individual BMS-<br>955176 Plasma Concentration<br>Profile vs. Time by Treatment<br>Evaluable PK Population - Stage<br>2 | WK24S2 |
| 519 | Figure S.8.2.1B | rg-pk-<br>cparlatvsl.lst | MS_PK_G_001 | Overlay of Individual ATV Plasma Concentration Profile vs. Time by Treatment Evaluable PK Population - Stage | WK24S1 |
| 520 | Figure S.8.2.1B | rg-pk-<br>cpar1atvs2.lst | MS_PK_G_001 | Overlay of Individual ATV Plasma Concentration Profile vs. Time by Treatment Evaluable PK Population - Stage 2 | WK24S2 |
| 521 | Figure S.8.2.1A | rg-pk-<br>cparldtgsl.lst | MS_PK_G_001 | Overlay of Individual DTG Plasma Concentration Profile vs. Time by Treatment Evaluable PK Population - Stage | WK24S1 |
| 522 | Figure S.8.2.1A | rg-pk-<br>cpar1dtgs2.lst | MS_PK_G_001 | Overlay of Individual DTG Plasma Concentration Profile vs. Time by Treatment Evaluable PK Population - Stage 2 | WK24S2 |
| 523 | Figure S.8.2.6A | rg-pk-<br>cpar6bmss1.lst | MS_PK_G_006 | Mean (+SD) BMS-955176 Plasma Concentration Profile vs. Time Evaluable PK Population - Stage | WK24S1 |
| 524 | Figure S.8.2.6A | rg-pk-<br>cpar6bmss2.lst | MS_PK_G_006 | Mean (+SD) BMS-955176 Plasma Concentration Profile vs. Time Evaluable PK Population - Stage 2 | WK24S2 |
| 525 | Figure S.8.2.6B | rg-pk-<br>cpar6atvs1.lst | MS_PK_G_006 | Mean (+SD) ATV Plasma<br>Concentration Profile vs. Time<br>Evaluable PK Population - Stage | WK24S1 |
| 526 | Figure S.8.2.6B | rg-pk-<br>cpar6atvs2.lst | MS_PK_G_006 | Mean (+SD) ATV Plasma<br>Concentration Profile vs. Time<br>Evaluable PK Population - Stage<br>2 | WK24S2 |

| No. | Table No. | Output File<br>Name | Template ID | Title and Population | Purpose |
|---|---|---|---|---|---|
| 527 | Figure S.8.2.6C | rg-pk-<br>cpar6dtgs1.lst | MS_PK_G_006 | Mean (+SD) DTG Plasma<br>Concentration Profile vs. Time<br>Evaluable PK Population - Stage | WK24S1 |
| 528 | Figure S.8.2.6C | rg-pk-<br>cpar6dtgs2.lst | MS_PK_G_006 | Mean (+SD) DTG Plasma<br>Concentration Profile vs. Time<br>Evaluable PK Population - Stage<br>2 | WK24S2 |
| 529 | Appendix<br>10.1.1 | rt-qs-eq5ds1.lst | SS_VL_T_006 | EQ-5D-3L Summary of US and UK Centric Scores and Changes From Baseline Over Time on Treatment Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 530 | Appendix<br>10.1.2 | rt-qs-eq5ds2.lst | SS_VL_T_006 | EQ-5D-3L Summary of US and UK Centric Scores and Changes From Baseline Over Time on Treatment Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |
| 531 | Appendix<br>10.2.1 | rt-qs-fahis1.lst | SS_VL_T_006 | FAHI Summary of Total Scores<br>Over Time on Treatment<br>Treated Subjects - Stage 1 | WK24S1,<br>WK48S1,<br>WK96S1,<br>WK96S2 |
| 532 | Appendix<br>10.2.2 | rt-qs-fahis2.lst | SS_VL_T_006 | FAHI Summary of Total Scores<br>Over Time on Treatment<br>Treated Subjects - Stage 2 | WK24S2,<br>WK48S2,<br>WK96S2 |

#### 2 INTRODUCTION

#### 2.1 Guidance for DPP Users and Reviewers

The Analysis Data Presentation Plan (DPP) contains comprehensive specifications for the development of data displays for an analysis.

#### **Templates and Metadata Tables:**

Within the Analysis DPP, the following templates will reside:

- Global Standard Templates (GS): The layout of these templates is a Global Standard. Global Standard templates will be placed into the DPP without modifications.
- **Project Specific Templates (PS):** The layout of these templates is constructed and described in the Core DPP. Project Specific templates will be placed into the DPP without modifications.
- For Early Development Only Model Document Specific Template (MS): The layout of these templates is constructed and described in the Early Development Standardized DPP Template.
- **Study Specific Templates (SS):** The layout of these templates is constructed for and described in the Analysis DPP.

A **Metadata Table** will contain information on the exact layout for a table, listing or graph.

#### **DPP Conventions:**

Text presented within a template and highlighted in grey:

- is a generic indicator for the type of endpoint or phrase that should replace it (Measure or Period for example)
- represents an optional item for a particular template presentation (P-value or Tablets/Capsules, for example).

The highlighted text in grey will remain as such in the template and the appropriate endpoint or phrase and the specifications to include within a specific table or listing in lieu of the highlighted text in grey will be described in the metadata tables. This will allow multiple tables to refer to the same table template.

#### 2.2 Referenced Documents

The following documents were referenced in the creation of this document.

| Document | Revision |
|---|---|
| GBS General Requirements for Statistical Outputs | v [Click to enter version: x.x] |
| Statistical Analysis Plan | v 2.0 |

### 3 GENERAL CRITERIA/CONVENTIONS

### 3.1 Exceptions to Global and/or Departmental Standards

| Location of Documentation | Standards Document | Exception |
|---|---|---|
| https://external.bms.com<br>/teams/GBS-<br>bms955176/genprogdoc<br>s/Forms/AllItems.aspx | Demographics Domain Requirements<br>Specification | Standards Request #8246: Add countries within geographic regions to Template GS_DM_T_X_002 and GS_DM_T_T_002. Add 2 columns "Geographic Region" and "Country" to end of Template GS_DM_L_X_001. |
| https://external.bms.com<br>/teams/GBS-<br>bms955176/genprogdoc<br>s/Forms/AllItems.aspx | Laboratory Test Results (SI Units) (US Units) Domain Requirements Specifications, Physical Measurements Domain Requirements Specifications, Vital Signs Domain Requirements Specifications | Standards Request #8247, #8251, #8255:<br>Display N, mean, SD, median, IQR for<br>values and changes from baseline over<br>time, with the option to specify absolute<br>or percent changes (see Template<br>SS_VL_T_006). |
| https://external.bms.com<br>/teams/GBS-<br>bms955176/genprogdoc<br>s/Forms/AllItems.aspx | Laboratory Test Results (SI Units) (US Units) Domain Requirements Specifications | Standards Request #8252: Display select lab tests in side-by-side columns in all lab listings, similar to GS_LB_L_S_007, not just LFTs (see Template SS_LB_L_001). |
| https://external.bms.com<br>/teams/GBS-<br>bms955176/genprogdoc<br>s/Forms/AllItems.aspx | Electrocardiogram Domain Requirements<br>Specification | Standards Request #8248: Modify Template GS_EG_T_X_005 to replace min and max with median, Q1, Q3, and add 95% CI for mean change from baseline (see Template SS_EG_T_003). |
| https://external.bms.com<br>/teams/GBS-<br>bms955176/genprogdoc<br>s/Forms/AllItems.aspx | Laboratory Test Results (SI Units) (US Units) Domain Requirements Specifications | Standards Request #8253: Display select toxicities (eg, Grade 1-4) by baseline tox grade categories (all, normal, Grade 1, 2, 3, 4, not reported) with multiple treatment group columns on the same page (see Template SS_LB_T_001). |
| https://external.bms.com<br>/teams/GBS-<br>bms955176/genprogdoc<br>s/Forms/AllItems.aspx | Laboratory Test Results (SI Units) (US Units) Domain Requirements Specifications | Standards Request #8254: Display treatment emergent lab abnormalities (increased to grade 1, increased to grade 2, increased to grade 3, increased to grade 4, increased to any grade) by baseline tox grade categories (all, normal, Grade 1 to 4, not reported) (see Template SS_LB_T_002). |

## 3.2 Populations

| Name as to Appear on<br>Output | Name used in SAP (if different) | Definition when no SAP available |
|---|---|---|
| Enrolled Subjects | | |
| Randomized Subjects | | |
| Treated Subjects | | |

| Name as to Appear on<br>Output | Name used in SAP (if different) | Definition when no SAP available |
|---|---|---|
| PK Population | | |
| Evaluable PK Population | | |

### 3.3 Conventions

[Click to enter text]

### 3.4 Treatment Information

| Drug Name | Column Headers to use in<br>Tables | Order Of<br>Column | Label to use in Listings (if different) |
|---|---|---|---|
| Stage 1: | | | |
| BMS-955176 | BMS-955176 120 mg +<br>ATV/r + DTG | 1 | |
| Tenofovir | TDF 300 mg + ATV/r + DTG | 2 | |
| Stage 2: | | | |
| BMS-955176 | BMS-955176 120 mg + ATV<br>+ DTG | 1 | |
| BMS-955176 | 76 BMS-955176 180 mg + ATV<br>+ DTG | | |
| Tenofovir | TDF 300 mg + ATV/r + DTG | 3 | |
| Stage 1 and 2 combined: | | | |
| BMS-955176 | ST1 BMS-955176 120 mg +<br>ATV/r + DTG | 1 | |
| BMS-955176 | ST2 BMS-955176 120 mg +<br>ATV + DTG | 2 | |
| BMS-955176 | ST2 BMS-955176 180 mg +<br>ATV + DTG | 3 | |
| Stage 1+Stage 2<br>Tenofovir | ST1+ST2 TDF 300 mg +<br>ATV/r + DTG | 4 | |

# 3.5 Graph Criteria/Conventions

| Attribute | Parameter | Value/Line |
|---|---|---|
| Symbol BMS-955176 120 mg + ATV/r + DTG | | Open triangle |
| | BMS-955176 120 mg +<br>ATV + DTG | Open circle |
| | BMS-955176 180 mg +<br>ATV + DTG | Open square |

| Attribute | Parameter | Value/Line |
|------------|------------------------------------|--------------------|
| | TDF 300 mg + ATV/r + DTG | Full circle |
| Line style | BMS-955176 120 mg +<br>ATV/r + DTG | Dotted line |
| | BMS-955176 120 mg +<br>ATV + DTG | Dashed |
| | BMS-955176 180 mg +<br>ATV + DTG | Dashed/Dotted line |
| | TDF 300 mg + ATV/r + DTG | Solid |

- 4 PRESENTATION PLAN TEMPLATES AND METADATA
- 4.1 Administrative Appendices

Template SS\_EX\_L\_001: Batch Number Listing

| Drug | Commercial<br>Batch<br>Number | Subject ID | Age/Gender/Race | Kit<br>Number | Date Kit<br>Assigned<br>by IVRS |
|---|---|---|---|---|---|
| <drug name=""></drug> | XXXXXXXX | PPD | (43/F/B) | XXXXX<br>XXXXX | 10MAR2003<br>10MAR2003 |
| | | | (43/F/B) | XXXXX<br>XXXXX<br>XXXXX | 10MAR2003<br>10MAR2003<br>30FEB2004 |
| <drug name#2=""></drug> | · | | (43/F/B) | XXXXX<br>XXXXX | 10MAR2003<br>10MAR2003 |

| Parameter | Values |
|------------------|--------------------------------|
| Template ID | SS_EX_L_001 |
| Output File Name | rl-ex-batchs1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Appendix 1.7.1 |
| Title 1 | Listing of Batch Numbers |
| Title 2 | Treated Subjects - Stage 1 |

| Parameter | Values |
|------------------|----------------------------|
| Template ID | SS_EX_L_001 |
| Output File Name | rl-ex-batchs2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Appendix 1.7.2 |
| Title 1 | Listing of Batch Numbers |
| Title 2 | Treated Subjects - Stage 2 |

## Template SS\_DS\_L\_001: Randomization Scheme and Codes

| Subject ID<br>(Age/Gender/Race) | Randomized<br>Treatment Group | Randomization<br>Date | As Treated<br>Treatment Group |
|---|---|---|---|
| PPD (59/F/O) | TRT A | 270CT2003 | TRT A |
| PPD (59/F/O) | TRT A | 270CT2003 | TRT B |

| Parameter | Values |
|---|---|
| Template ID | SS_DS_L_001 |
| Output File Name | rl-ds-randcodes1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Appendix 1.9.1 |
| Title 1 | Randomization Scheme and Codes |
| Title 2 | Randomized Subjects - Stage 1 |
| Programming notes | Sorted by site and subject identifier. The listing should also be "paged" by site. |

| Parameter | Values |
|---|---|
| Template ID | SS_DS_L_001 |
| Output File Name | rl-ds-randcodes2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Appendix 1.9.2 |
| Title 1 | Randomization Scheme and Codes |
| Title 2 | Randomized Subjects - Stage 2 |
| Programming notes | Sorted by site and subject identifier. The listing should also be "paged" by site. |

## Template SS\_DM\_T\_001: Accrual Summary

| Site | TRT A | TRT B | TRT C | Total |
|---|---|---|---|---|
| Treatment Initiation Month | N=XXX | N=XXX | N=XXX | N=XXX |
| Site PP | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Calendar Month/Year 1 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Calendar Month/Year 2 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| Site PP Calendar Month/Year 1 Calendar Month/Year 2 | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |
| | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) | XXX (XX.X) |

| Parameter | Values |
|------------------|--------------------------------|
| Template ID | SS_DM_T_001 |
| Output File Name | rt-dm-accruals1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Appendix 2.1.1E |
| Title 1 | Accrual Summary |
| Title 2 | Treated Subjects - Stage 1 |

| Parameter | Values |
|------------------|----------------------------|
| Template ID | SS_DM_T_001 |
| Output File Name | rt-dm-accruals2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Appendix 2.1.2E |
| Title 1 | Accrual Summary |
| Title 2 | Treated Subjects - Stage 2 |

## 4.2 Study Conduct

## 4.2.1 Protocol Deviations

## Template SS\_PD\_T\_001: Relevant Protocol Deviation Summary

| Deviation | Group A | Group B | Group C | Group D | Total |
|---|---|---|---|---|---|
| | N = XX | N = XX | N = XX | N = XX | N = XX |
| ANY DEVIATION | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| INFORMED CONSENT NOT OBTAINED, OR OBTAINED AFTER ENROLLMENT QUALIFYING HIV 1 RNA < 5,000 C/ML OR MISSING PRIOR TO RANDOMIZATION CD4 < 200 CELLS/UL MISSING PRIOR TO RANDOMIZATION PRIOR ANTIRETROVIRAL THERAPY 2 1 WEEK OF EXPOSURE | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |
| | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) | XX (XX.X) |

| Parameter | Values |
|---|---|
| Template ID | SS_PD_T_001 |
| Output File Name | rt-pd-rels1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.2.3.1A |
| Title 1 | Relevant Protocol Deviation Summary |
| Title 2 | Randomized Subjects - Stage 1 |
| Layout notes | Include the relevant protocol deviations listed in the SAP. |

| Parameter | Values |
|---|---|
| Template ID | SS_PD_T_001 |
| Output File Name | rt-pd-rels2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.2.3.2A |
| Title 1 | Relevant Protocol Deviation Summary |
| Title 2 | Randomized Subjects - Stage 2 |
| Layout notes | Include the relevant protocol deviations listed in the SAP. |
### Template SS\_PD\_L\_001: Relevant Protocol Deviation Listing

Subject ID (Age/Gender/Race) Treatment Group

Deviation

(54/M/C) TRT B 

| Parameter | Values |
|---|---|
| Template ID | SS_PD_L_001 |
| Output File Name | rl-pd-rels1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.2.3.1B |
| Title 1 | Listing of Relevant Protocol Deviations |
| Title 2 | Randomized Subjects - Stage 1 |
| Layout notes | Include the relevant protocol deviations listed in the SAP. |
| Programming notes | Sorted by treatment group, site and subject identifier |

| Parameter | Values |
|---|---|
| Template ID | SS_PD_L_001 |
| Output File Name | rl-pd-rels2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.2.3.2B |
| Title 1 | Listing of Relevant Protocol Deviations |
| Title 2 | Randomized Subjects - Stage 2 |
| Layout notes | Include the relevant protocol deviations listed in the SAP. |
| Programming notes | Sorted by treatment group, site and subject identifier |

- 4.3 Study Population
- 4.3.1 Disposition of Subjects

#### Template GS\_DS\_T\_T\_001: Pre-Randomization Subject Status

Protocol: TA123456 Draft Pre-Randomized Subject Status Summary All Enrolled Subjects 

| | Total |
|---|---|
| SUBJECTS ENROLLED | 468 |
| SUBJECTS RANDOMIZED (%) | 445 ( 95.1) |
| SUBJECTS NOT RANDOMIZED (%) | 23 ( 4.9) |
| REASON FOR NOT BEING RANDOMIZED (%) SUBJECT WITHDREW CONSENT POOR/NON-COMPLIANCE SUBJECT NO LONGER MEETS STUDY CRITERIA ADMINISTRATIVE REASON BY SPONSOR OTHER | 4 ( 0.9)<br>3 ( 0.6)<br>12 ( 2.6)<br>1 ( 0.2)<br>3 ( 0.6) |

Percentages based on subjects enrolled Program Source: /wwbdm/ndp/prime/gssr/devtest/sta/test/domain\_example/status1.sas

16NOV2004:10:37:00

| Parameter | Values |
|------------------|-----------------------------------------|
| Template ID | GS_DS_T_T_001 |
| Output File Name | rt-ds-prerands1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.2.1.1A |
| Title 1 | Pre-Randomization Subject Status |
| Title 2 | Enrolled Subjects - Stage 1 |
| Footnote 1 | Percentages based on subjects enrolled. |

| Parameter | Values |
|------------------|---------------------|
| Template ID | GS_DS_T_T_001 |
| Output File Name | rt-ds-prerands2.lst |

| Purpose | VK24S2, WK48S2, WK96S2 |
|------------|-----------------------------------------|
| Table No. | Table S.2.1.2A |
| Title 1 | Pre-Randomization Subject Status |
| Title 2 | Enrolled Subjects - Stage 2 |
| Footnote 1 | Percentages based on subjects enrolled. |

### Template GS\_DS\_L\_S\_001: Pre-randomization Subject Status Listing

Protocol: TA123456 Draft 

Draft Pre-Randomized Subject Status All Enrolled Subjects

| Subject ID | | | |
|---|---|---|---|
| (Áge/Gender/Race) | Date | Randomized | Reason Subject Will Not be Randomized |
| PPD (47/M/C) | 270CT2003 | YES | |
| PPD (31/M/C) | 05NOV2003 | NO | SUBJECT NO LONGER MEETS STUDY CRITERIA: VIRAL LOAD < 50 COPIES AT SCREENING VISIT |
| PPD (24/F/B) | 13FEB2004 | YES | |
| PPD (41/F/C) | 09FEB2004 | NO | SUBJECT WITHDREW CONSENT: SHE IS AFRAID OF BEGINNING A NEW TREATMENT |
| PPD<br>(21/F/B) | 27NOV2003 | YES | |
| PPD<br>(39/M/C) | 090CT2003 | NO | OTHER: SOCIAL SITUATION/PATIENTS WISH |
| PPD (46/M/C) | 05APR2004 | YES | |
| PPD (32/M/C) | 05APR2004 | YES | |
| PPD<br>(38/M/C) | 05APR2004 | NO | LOST TO FOLLOW-UP: 05APR2004 |
| PPD (44/M/C) | 25SEP2003 | YES | |

Program Source: /wwbdm/ndp/prime/gssr/devtest/sta/test/sta lst.sas 07SEP2004:14:35:00

| Parameter | Values |
|------------------|--------------------------------|
| Template ID | GS_DS_L_S_001 |
| Output File Name | rl-ds-prerands1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |

| Table No. | Appendix 2.1.1A |
|-------------------|---------------------------------------|
| Title 1 | Pre-Randomized Subject Status |
| Title 2 | Enrolled Subjects - Stage 1 |
| Programming notes | Sorted by site and subject identifier |

| Parameter | Values |
|-------------------|---------------------------------------|
| Template ID | GS_DS_L_S_001 |
| Output File Name | rl-ds-prerands2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Appendix 2.1.2A |
| Title 1 | Pre-Randomized Subject Status |
| Title 2 | Enrolled Subjects - Stage 2 |
| Programming notes | Sorted by site and subject identifier |

### Template GS\_DM\_T\_T\_005: Enrollment Summary

Protocol: CV123456 

Confidential
Enrollment Summary
Number Of Subjects At Each Study Site By Country

| Country (%) Site Number (%) | ENROLLED<br>N = 200 | RANDOMIZED<br>N = 150 |
|---|---|---|
| AU ALIA PPD | 136 ( 78.0)<br>10 ( 5.0)<br>12 ( 6.0)<br>8 ( 4.0)<br>9 ( 4.5)<br>15 ( 7.5)<br>4 ( 2.0)<br>7 ( 3.5)<br>5 ( 2.5)<br>9 ( 4.5)<br>8 ( 4.0)<br>6 ( 3.0)<br>13 ( 6.5)<br>5 ( 2.5)<br>9 ( 4.5)<br>8 ( 4.0)<br>7 ( 3.5) | 109 ( 72.7) 8 ( 5.3) 9 ( 6.0) 6 ( 4.0) 7 ( 4.7) 12 ( 8.0) 3 ( 2.0) 7 ( 4.7) 5 ( 3.3) 8 ( 5.3) 5 ( 3.3) 5 ( 3.3) 10 ( 6.7) 4 ( 2.7) 8 ( 5.3) 7 ( 4.7) 5 ( 3.3) |
| CANADA<br>PPD | 49 ( 24.5)<br>7 ( 3.5)<br>5 ( 2.5)<br>5 ( 2.5)<br>11 ( 5.5)<br>9 ( 4.5)<br>6 ( 3.0)<br>6 ( 3.0) | 40 ( 26.7)<br>5 ( 3.3)<br>3 ( 2.0)<br>4 ( 2.7)<br>9 ( 6.0)<br>8 ( 5.3)<br>6 ( 4.0)<br>5 ( 3.3) |
| CHILE PPD | 14( 7.0)<br>7 ( 3.5) | 12 ( 8.0)<br>6 ( 4.0) |

-----

Program Source: /gbs/prod/clin/programs/cv/123/456/country.sas

| Parameter | Values |
|-------------|---------------|
| Template ID | GS_DM_T_T_005 |

18FEB2005:10:59:00

| Output File Name | rt-dm-enrolls1eu.lst |
|------------------|--------------------------------------------------|
| Purpose | X24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | pendix 2.1.1C |
| Title 1 | nrollment Summary |
| Title 2 | Number of Subjects at Each Study Site by Country |
| Title 3 | Enrolled Subjects - Stage 1 |

| Parameter | Values |
|---|---|
| Template ID | GS_DM_T_T_005 |
| Output File Name | -dm-enrolls2eu.lst |
| Purpose | 7K24S2, WK48S2, WK96S2 |
| Table No. | Appendix 2.1.2C |
| Title 1 | Enrollment Summary |
| Title 2 | Number of Subjects at Each Study Site by Country |
| Title 3 | Enrolled Subjects - Stage 2 |

### Template SS\_DM\_T\_002: Counts and Percentages Table


<Title 1> <Title 2>

Subgroup: XXXXXXXXX Level: XXXXXXXXXXX

| <pre><col 1="" header=""/> (%) <col 2="" header=""/> (%)</pre> | Group 1<br>N = XXX | Group 2<br>N = XXX |
|---|---|---|
| <pre><event 1=""> <subevent 1=""></subevent></event></pre> | XXX (XXX.X)<br>XXX (XXX.X) | XXX (XXX.X)<br>XXX (XXX.X) |
| <subevent x=""></subevent> | XXX (XXX.X) | XXX (XXX.X) |
| <additional events=""></additional> | | |
| <event x=""> <subevent 1=""></subevent></event> | XXX (XXX.X)<br>XXX (XXX.X) | XXX (XXX.X)<br>XXX (XXX.X) |
| <pre> <subevent x=""></subevent></pre> | XXX (XXX,X) | XXX (XXX.X) |

-----

<Footnote 1>
<Footnote 2>
<Footnote 3>
Program Source: <TBD>

Program Source: <TBD>
DDMMYYYY:HR:MM:SS

| Parameter | Values |
|------------------|--------------------------------|
| Template ID | S_DM_T_002 |
| Output File Name | dm-enrages1eu.lst |
| Purpose | VK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Appendix 2.1.1D |
| Title 1 | Enrollment Summary |

| Title 2 | Jumber of Subjects per Age Group |
|---|---|
| Title 3 | nrolled Subjects - Stage 1 |
| Layout notes | Col 1 Header: Age Group (%). Events 1 through 9 are the following (display even if 0 total counts): IN UTERO; PRETERM NEWBORN (GESTATIONAL AGE < 37 WEEKS); NEWBORNS (0 TO 27 DAYS); INFANTS AND TODDLERS (28 DAYS TO 23 MONTHS); CHILDREN (2 TO 11 YEARS); ADOLESCENTS (12 TO 17 YEARS); ADULTS (18 TO 64 YEARS); FROM 65 TO 84 YEARS; 85 YEARS AND OVER. |

| Parameter | Values |
|---|---|
| Template ID | SS_DM_T_002 |
| Output File Name | rt-dm-enrages2eu.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | ppendix 2.1.2D |
| Title 1 | Enrollment Summary |
| Title 2 | Number of Subjects per Age Group |
| Title 3 | Enrolled Subjects - Stage 2 |
| Layout notes | Col 1 Header: Age Group (%). Events 1 through 9 are the following (display even if 0 total counts): IN UTERO; PRETERM NEWBORN (GESTATIONAL AGE < 37 WEEKS); NEWBORNS (0 TO 27 DAYS); INFANTS AND TODDLERS (28 DAYS TO 23 MONTHS); CHILDREN (2 TO 11 YEARS); ADOLESCENTS (12 TO 17 YEARS); ADULTS (18 TO 64 YEARS); FROM 65 TO 84 YEARS; 85 YEARS AND OVER. |

#### Template GS\_DS\_T\_X\_005: End of Study Subjects Status

Protocol: TA123456 

Draft
End of Study Subject Status Summary
Descriptive text of population basis

| | TRT A | TRT B | TRT C | Total |
|---|---|---|---|---|
| SUBJECTS | 150 | 145 | 150 | 445 |
| SUBJECTS COMPLETING THE STUDY (%) | 146 ( 97.3) | 142 ( 97.9) | 147 ( 98.0) | 435 ( 97.8) |
| SUBJECTS NOT COMPLETING THE STUDY (%) | 4 ( 2.7) | 3 ( 2.1) | 3 ( 2.0) | 10 ( 2.2) |
| REASON FOR NOT COMPLETING THE STUDY (%) LACK OF EFFICACY ADVERSE EVENT SUBJECT WITHDREW CONSENT LOST TO FOLLOW-UP | 1 ( 0.7)<br>2 ( 1.3)<br>1 ( 0.7) | 1 ( 0.7)<br>0<br>1 ( 0.7)<br>1 ( 0.7) | 0<br>1 ( 0.7)<br>2 ( 1.3) | 2 ( 0.4)<br>3 ( 0.7)<br>4 ( 0.9)<br>1 ( 0.2) |

Percentages based on subjects population basis Program Source: /wwbdm/ndp/prime/gssr/devtest/sta/test/domain\_example/status4r.sas

16NOV2004:10:37:00

| Parameter | Values |
|------------------|-------------------------------------|
| Template ID | SS_DS_T_X_005 |
| Output File Name | ds-statuss1.lst |
| Purpose | K24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.2.1.1B |
| Title 1 | End of Study Subject Status Summary |
| Title 2 | Randomized Subjects - Stage 1 |

| Parameter | Values |
|------------------|--------------------|
| Template ID | GS_DS_T_X_005 |
| Output File Name | rt-ds-statuss2.lst |

| Purpose | VK24S2, WK48S2, WK96S2 |
|-----------|-------------------------------------|
| Table No. | e S.2.1.2B |
| Title 1 | End of Study Subject Status Summary |
| Title 2 | Randomized Subjects - Stage 2 |

| Parameter | Values |
|------------------|-------------------------------------|
| Template ID | S_DS_T_X_005 |
| Output File Name | ds-statuss12.lst |
| Purpose | VK96S2 |
| Table No. | Table S.2.1.3B |
| Title 1 | End of Study Subject Status Summary |
| Title 2 | Randomized Subjects - Stage 1 and 2 |

### Template GS\_DS\_L\_X\_005: End of Study Subject Status by Treatment Group

Program Source: /wwbdm/ndp/prime/gssr/devtest/sta/test/sta lst2.sas

Protocol: TA123456 Protocol Pr

End of Study Subject Status
Descriptive text of population basis

Treatment Group: TRT A

| Subject ID<br>(Age/Gender/Race) | Period | Date | Completed<br>Study | Reason Subject Did Not Complete Study |
|---|---|---|---|---|
| PPD<br>(48/M/C) | ON STUDY | 09JUL2004 | YES | |
| PPD (62/F/C) | ON STUDY | 17FEB2004 | NO | ADVERSE EVENT: DUE TO AE OF HYPOTHYROIDISM BY MEDICAL MONITOR |
| PPD (63/F/C) | ON STUDY | 29JUN2004 | NO | SUBJECT WITHDREW CONSENT: TOO LONG OF COMMUTE, LEAVING AREA FOR SUMMER |
| PPD (62/F/C) | ON STUDY | 14MAY2004 | NO | LACK OF EFFICACY: FPG WITH A RESULT OF 15.1 MMOL/L AFTER RETEST |
| PPD (59/F/C) | ON STUDY | | NO | LOST TO FOLLOW-UP |
| PPD (61/F/C) | ON STUDY | 23AUG2004 | YES | |
| PPD (67/M/C) | ON STUDY | 10JUN2004 | NO | DEATH |
| PPD (64/M/C) | ON STUDY | 23AUG2004 | YES | |
| PPD<br>(67/F/C) | ON STUDY | 16APR2004 | NO | POOR/NON-COMPLIANCE: MEDICATION NOT TAKEN ACC. TO INVESTIGATOR'S INSTRUCTION |
| PPD (62/M/C) | ON STUDY | 26AUG2004 | YES | |

| Parameter | Values |
|---------------|--------|
| 1 al allictel | values |

07SEP2004:14:35:00

| Template ID | GS_DS_L_X_005 |
|------------------|--------------------------------|
| Output File Name | rl-ds-statuss1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Appendix 2.1.1B |
| Title 1 | End of Study Subject Status |
| Title 2 | Randomized Subjects - Stage 1 |

| Parameter | Values |
|------------------|-------------------------------|
| Template ID | GS_DS_L_X_005 |
| Output File Name | rl-ds-statuss2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Appendix 2.1.2B |
| Title 1 | End of Study Subject Status |
| Title 2 | Randomized Subjects - Stage 2 |

#### Template SS\_DM\_T\_002: Population Summary

| | Trt A | Trt B | Trt C | Trt D | Total |
|-------------------------|-------|-------|-------|-------|-------|
| RANDOMIZED SUBJECTS (A) | XX | XX | XX | XX | XX |
| TREATED SUBJECTS (B) | XX | XX | XX | XX | XX |

Parameter Values Template ID SS DM T 002 Output File Name rt-dm-populations1.lst WK24S1, WK48S1, WK96S1, WK96S2 Purpose Table No. Table S.2.1.1C Populations for Analysis Summary - Stage 1 Title 1 (A) Randomized subjects in the treatment group to which they were randomized. Footnote 1 (B) Subjects who took at least one dose of study medication in the treatment group to which they were randomized Footnote 2 unless subjects have never received the study medication they were randomized, in which case subjects will be included Footnote 3 in the treatment group based on the first treatment received. Footnote 4

| Parameter | Values |
|---|---|
| Template ID | SS_DM_T_002 |
| Output File Name | rt-dm-populations2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.2.1.2C |
| Title 1 | Populations for Analysis Summary - Stage 2 |
| Footnote 1 | (A) Randomized subjects in the treatment group to which they were randomized. |

| Footnote 2 | (B) Subjects who took at least one dose of study medication in the treatment group to which they were randomized |
|---|---|
| Footnote 3 | unless subjects have never received the study medication they were randomized, in which case subjects will be included |
| Footnote 4 | in the treatment group based on the first treatment received. |

### Template SS\_DM\_L\_001: Listing of Subjects Excluded from the Efficacy Analysis

Treatment Group: TRT A

Subject ID

(Age/Gender/Race) Reason Subject Excluded from Efficacy Analysis Discontinuation Reason

RANDOMIZED, BUT NOT TREATED LOST TO FOLLOW-UP

(48/M/C)

PPD (62/F/C)

RANDOMIZED, BUT NOT TREATED

SUBJECT WITHDREW CONSENT: TOO LONG OF COMMUTE, LEAVING AREA FOR SUMMER

| Parameter | Values |
|---|---|
| Template ID | SS_DM_L_001 |
| Output File Name | rl-dm-excls1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Appendix 2.2.1 |
| Title 1 | Subjects Excluded from Efficacy Analysis (mITT) |
| Title 2 | Randomized Subjects - Stage 1 |
| Programming notes | Reason for being excluded should always be: RANDOMIZED, BUT NOT TREATED. Sorted by treatment group, site and subject identifier. |

| Parameter | Values |
|------------------|-------------------------------------------------|
| Template ID | SS_DM_L_001 |
| Output File Name | rl-dm-excls2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Appendix 2.2.2 |
| Title 1 | Subjects Excluded from Efficacy Analysis (mITT) |
| Title 2 | Randomized Subjects - Stage 2 |

| Programming notes | Reason for being excluded should always be: RANDOMIZED, BUT NOT TREATED. |
|---|---|
| | Sorted by treatment group, site and subject identifier. |

# 4.3.2 Demographics and Baseline Characteristics

Template GS\_DM\_T\_X\_002: Demographic Characteristics Summary (incl. 'Not reported' category)

Protocol: CA259001 Draft
Demographic Characteristics Summary
All Treated Subjects 

| | TRT A | TRT B | TRT C | Total |
|---|---|---|---|---|
| | N = 1113 | N = 1111 | N = 1107 | N = 3331 |
| AGE (Units) N MEAN MEDIAN MIN , MAX Q1 , Q3 STANDARD DEVIATION | 1112<br>72<br>72<br>72<br>0 , 94<br>66 , 77 | 1109<br>71<br>71<br>0 , 95<br>66 , 76<br>7.7 | 1107<br>72<br>71<br>59,94<br>66,77 | 3328<br>72<br>71<br>0,95<br>66,77 |
| AGE CATEGORIZATION (%) < 50 >= 50 NOT REPORTED | 232 ( 17.3) | 248 ( 18.3) | 246 ( 18.0) | 726 ( 17.9) |
| | 880 ( 78.9) | 861 ( 77.1) | 861 ( 78.8) | 2602 ( 78.3) |
| | 1 ( <0.1) | 2 ( 0.2) | 0 | 3 ( <0.1) |
| GENDER (%) MALE FEMALE NOT REPORTED | 445 ( 40.1) | 437 ( 39.1) | 441 ( 39.6) | 1323 ( 39.6) |
| | 666 ( 59.7) | 669 ( 60.4) | 659 ( 59.8) | 1994 ( 60.0) |
| | 2 ( 0.2) | 5 ( 0.4) | 7 ( 0.6) | 14 ( 0.4) |
| RACE (%) WHITE BLACK OR AFRICAN AMERICAN ASIAN OTHER NOT REPORTED | 1041 ( 93.3)<br>26 ( 2.3)<br>4 ( 0.4)<br>42 ( 4.0)<br>0 | 1042 ( 93.3)<br>24 ( 2.1)<br>5 ( 0.4)<br>40 ( 4.1) | 1041 ( 93.4)<br>20 ( 2.5)<br>3 ( 0.3)<br>42 ( 3.8)<br>1 ( <0.1) | 3124 ( 93.3)<br>70 ( 2.3)<br>12 ( 0.4)<br>124 ( 4.0)<br>1 ( <0.1) |
| ETHNICITY (%) HISPANIC/LATINO NOT HISPANIC/LATINO NOT REPORTED | 24 ( 2.4) | 35 ( 3.1) | 33 ( 2.8) | 92 ( 2.8) |
| | 1089 ( 97.6) | 1076 ( 96.9) | 1073 ( 97.1) | 3238 ( 97.2) |
| | 0 | 0 | 1 ( <0.1) | 1 ( <0.1) |

Program Source: /wwbdm/ndp/prime/gssr/devtest/dem/test/dem tbl mod.sas

30DEC2004:14:45:05

| Parameter | Values |
|---|---|
| Template ID | GS_DM_T_X_002 |
| Output File Name | rt-dm-summarys1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.3.1.1 |
| Title 1 | Demographic Characteristics Summary |
| Title 2 | Treated Subjects - Stage 1 |
| Layout notes | See SAP Table 7.3.2.1-1. Add "COUNTRY BY GEOGRAPHIC REGION (%)" after "ETHNICITY (%)". Indent countries 2 spaces underneath regions. |

| Parameter | Values |
|---|---|
| Template ID | GS_DM_T_X_002 |
| Output File Name | rt-dm-summarys2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.3.1.2 |
| Title 1 | Demographic Characteristics Summary |
| Title 2 | Treated Subjects - Stage 2 |
| Layout notes | See SAP Table 7.3.2.1-1. Add "COUNTRY BY GEOGRAPHIC REGION (%)" after "ETHNICITY (%)". Indent countries 2 spaces underneath regions. |

| Parameter | Values |
|------------------|-------------------------------------|
| Template ID | GS_DM_T_X_002 |
| Output File Name | rt-dm-summarys12.lst |
| Purpose | WK96S2 |
| Table No. | Table S.3.1.3 |
| Title 1 | Demographic Characteristics Summary |

| Title 2 | Treated Subjects - Stage 1 and 2 |
|---|---|
| Layout notes | See SAP Table 7.3.2.1-1. Add "COUNTRY BY GEOGRAPHIC REGION (%)" after "ETHNICITY (%)". Indent countries 2 spaces underneath regions. |

#### Template GS\_DM\_T\_T\_002: Demographic Characteristics Summary (incl. 'Not reported' category)

Protocol: CA259001 Praft 

Draft
Demographic Characteristics Summary
All Treated Subjects

| | Total<br>N = 3348 |
|---|---|
| AGE (Units) N MEAN MEDIAN MIN , MAX Q1 , Q3 STANDARD DEVIATION | 3345<br>72<br>71<br>0,95<br>66,77<br>7.2 |
| AGE CATEGORIZATION (%)<br>< 65<br>65 - 85<br>NOT REPORTED | 598 ( 17.9)<br>2620 ( 78.3)<br>3 ( <0.1) |
| GENDER (%)<br>MALE<br>FEMALE<br>NOT REPORTED | 1323 ( 39.6)<br>1994 ( 60.0)<br>14 ( 0.4) |
| RACE (%) WHITE BLACK OR AFRICAN AMERICAN ASIAN OTHER NOT REPORTED | 3124 ( 93.3)<br>78 ( 2.3)<br>12 ( 0.4)<br>133 ( 4.0)<br>1 ( <0.1) |
| THNICITY (%) HISPANIC/LATINO NOT HISPANIC/LATINO NOT REPORTED | 93 ( 2.8)<br>3254 ( 97.2)<br>1 ( <0.1) |

Program Source: /wwbdm/ndp/prime/gssr/devtest/dem/test/dem tbl mod.sas

30DEC2004:14:46:08

| Parameter | Values |
|------------------|--------------------------------|
| Template ID | GS_DM_T_T_002 |
| Output File Name | rt-dm-sumenrolls1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |

| Table No. | Appendix 3.1.1B |
|---|---|
| Title 1 | Demographic Characteristics Summary |
| Title 2 | Subjects Enrolled but Not Randomized - Stage 1 |
| Layout notes | See SAP Table 7.3.2.1-1. Add "COUNTRY BY GEOGRAPHIC REGION (%)" after "ETHNICITY (%)". Indent countries 2 spaces underneath regions. |

| Parameter | Values |
|---|---|
| Template ID | GS_DM_T_T_002 |
| Output File Name | rt-dm-sumenrolls2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Appendix 3.1.2B |
| Title 1 | Demographic Characteristics Summary |
| Title 2 | Subjects Enrolled but Not Randomized - Stage 2 |
| Layout notes | See SAP Table 7.3.2.1-1. Add "COUNTRY BY GEOGRAPHIC REGION (%)" after "ETHNICITY (%)". Indent countries 2 spaces underneath regions. |

## Template GS\_DM\_L\_X\_001: Demographics Listing by Treatment Group

Protocol: CV131148 

Draft
Demographic Characteristics
All Treated Subjects

Treatment Group: TRT A

| Subject ID | Informed<br>Consent<br>Date | Birth<br>Date | Age | Gender | Ethnicity | Race |
|---|---|---|---|---|---|---|
| PPD | 22NOV2002 | PPD 2001 | 1 | MALE | HISPANIC/LATINO | WHITE |
| | 07DEC2003 | <b>PPD</b> 2003 | 10M | MALE | | OTHER: WHITE SOUTH AFRICAN |
| | 12JUN2003 | PPD 2002 | 6M | MALE | HISPANIC/LATINO | WHITE |
| | 17FEB2003 | <b>PPD</b> 2002 | 1 | MALE | NOT HISPANIC/LATINO | WHITE |
| | 24APR2003 | <b>PPD</b> 2001 | 2 | MALE | NOT HISPANIC/LATINO | WHITE |
| | 14MAY2003 | <b>PPD</b> 2000 | 3 | FEMALE | NOT HISPANIC/LATINO | WHITE |
| | 25DEC2001 | <b>PPD</b> 2001 | 2D | FEMALE | NOT HISPANIC/LATINO | WHITE |

Program Source: /wwbdm/ndp/prime/gssr/devtest/dem/test/dem lst.sas

30DEC2004:15:50:44

| Parameter | Values |
|---|---|
| Template ID | GS_DM_L_X_001 |
| Output File Name | rl-dm-demchars1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Appendix 3.1.1A |
| Title 1 | Demographic Characteristics |
| Title 2 | Treated Subjects - Stage 1 |
| Layout notes | Add 2 columns "Country" and "Geographic Region" after "Race". |

| Parameter | Values |
|-------------|---------------|
| Template ID | GS_DM_L_X_001 |

| Output File Name | rl-dm-demchars2.lst |
|---|---|
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Appendix 3.1.2A |
| Title 1 | Demographic Characteristics |
| Title 2 | Treated Subjects - Stage 2 |
| Layout notes | Add 2 columns "Country" and "Geographic Region" after "Race". |

 $Template \ SS\_DM\_T\_004: Baseline \ Disease \ Characteristics$ 

| | Group A<br>N = XX | Group B<br>N = XX | Group C<br>N = XX | Group D<br>N = XX | Total<br>N = XX |
|---|---|---|---|---|---|
| HIV SUBTYPE<br>A<br>B<br><additional subtypes=""></additional> | XX ( XX.X)<br>XX ( XX.X)<br>XX ( XX.X) | XX ( XX.X)<br>XX ( XX.X)<br>XX ( XX.X) | XX ( XX.X)<br>XX ( XX.X)<br>XX ( XX.X) | XX ( XX.X)<br>XX ( XX.X)<br>XX ( XX.X) | XX ( XX.X)<br>XX ( XX.X)<br>XX ( XX.X) |
| Plasma HIV-1 RNA (log10 c,<br>N<br>MEAN<br>MEDIAN<br>MIN , MAX<br>Q1 , Q3<br>STANDARD DEVIATION | XX | XX<br>XX.X<br>XX.X, XX.X<br>XX.X, XX.X<br>XX.X, XX.X | XX<br>XX.X<br>XX.X, XX.X<br>XX.X, XX.X<br>XX.X, XX.X | XX<br>XX.X<br>XX.X<br>XX.X , XX.X<br>XX.X , XX.X<br>XX.X , XX.X | XX<br>XX.X<br>XX.X, XX.X<br>XX.X, XX.X<br>XX.X, XX.X |
| HIV-1 RNA CATEGORIZATION<br>< 30,000 c/mL<br>30,000 to < 100,000 c/m<br>100,000 to < 500,000 c/m<br>≥ 500,000 c/mL<br>NOT REPORTED | XX ( XX.X) L XX ( XX.X) mL XX ( XX.X) XX ( XX.X) XX ( XX.X) | XX ( XX.X)<br>XX ( XX.X)<br>XX ( XX.X)<br>XX ( XX.X)<br>XX ( XX.X) | XX ( XX.X)<br>XX ( XX.X)<br>XX ( XX.X)<br>XX ( XX.X)<br>XX ( XX.X) | XX ( XX.X)<br>XX ( XX.X)<br>XX ( XX.X)<br>XX ( XX.X)<br>XX ( XX.X) | XX ( XX.X)<br>XX ( XX.X)<br>XX ( XX.X)<br>XX ( XX.X)<br>XX ( XX.X) |
| CD4+ T-cell counts (cells,<br>N<br>MEAN<br>MEDIAN<br>MIN , MAX<br>Q1 , Q3<br>STANDARD DEVIATION | /uL) XX XX.X XX.X XX.X, XX.X XX.X, XX.X XX.X, XX.X | XX<br>XX.X<br>XX.X, XX.X<br>XX.X, XX.X<br>XX.X, XX.X | XX<br>XX.X<br>XX.X<br>XX.X , XX.X<br>XX.X , XX.X<br>XX.X , XX.X | XX<br>XX.X<br>XX.X<br>XX.X , XX.X<br>XX.X , XX.X<br>XX.XX | XX<br>XX.X<br>XX.X<br>XX.X, XX.X<br>XX.X, XX.X<br>XX.XX |
| CD4+ T-cell CATEGORIZATION < 50 cells/uL 50 to < 100 cells/uL 100 to < 200 cells/uL 200 to < 350 cells/uL 350 to < 500 cells/uL > 500 cells/uL NOT REPORTED | XX ( XX.X) | XX ( XX.X)<br>XX ( XX.X) | XX ( XX.X)<br>XX ( XX.X) | XX ( XX.X)<br>XX ( XX.X) | XX ( XX.X)<br>XX ( XX.X) |
| CD4+ T-cell percentage<br>N<br>MEAN<br>MEDIAN<br>MIN , MAX<br>Q1 , Q3<br>STANDARD DEVIATION | XX<br>XX.X<br>XX.X<br>XX.X , XX.X<br>XX.X , XX.X<br>XX.X , XX.X | XX<br>XX.X<br>XX.X<br>XX.X , XX.X<br>XX.X , XX.X<br>XX.XX | XX<br>XX.X<br>XX.X<br>XX.X , XX.X<br>XX.X , XX.X | XX<br>XX.X<br>XX.X<br>XX.X , XX.X<br>XX.X , XX.X | XX<br>XX.X<br>XX.X<br>XX.X , XX.X<br>XX.X , XX.X |

| CD8+ T-cell counts (cell: N MEAN MEDIAN MIN , MAX Q1 , Q3 STANDARD DEVIATION | XX<br>XX.X<br>XX.X<br>XX.X, XX.X<br>XX.X, XX.X<br>XX.X, XX.X | XX<br>XX.X<br>XX.X<br>XX.X , XX.X<br>XX.X , XX.X<br>XX.XX | XX<br>XX.X<br>XX.X, XX.X<br>XX.X, XX.X<br>XX.X, XX.X | XX<br>XX.X<br>XX.X<br>XX.X , XX.X<br>XX.X , XX.X<br>XX.XX | XX<br>XX.X<br>XX.X<br>XX.X, XX.X<br>XX.X, XX.X<br>XX.XX |
|---|---|---|---|---|---|
| BMS-955176 IC50 (µM) N MEAN Geometric Mean (Coefficient of Variation MEDIAN | XX<br>XX.X<br>n)<br>XX.X | XX<br>XX.X | XX<br>XX.X | XX<br>XX.X | XX<br>XX.X |
| MIN , MAX<br>Q1 , Q3<br>STANDARD DEVIATION | XX.X , XX.X<br>XX.X , XX.X<br>XX.XX | XX.X , XX.X<br>XX.X , XX.X<br>XX.XX | XX.X , XX.X<br>XX.X , XX.X<br>XX.XX | XX.X , XX.X<br>XX.X , XX.X<br>XX.XX | XX.X , XX.X<br>XX.X , XX.X<br>XX.XX |
| EMS-955176 IC50 FOLD CHAN<br>< 1.0<br>1.0 to < 5.0<br>5.0 to < 10<br>10 to < 100<br>100 to < 500<br>>= 500 | XX ( XX.X)<br>XX ( XX.X) | XX ( XX.X)<br>XX ( XX.X)<br>XX ( XX.X)<br>XX ( XX.X)<br>XX ( XX.X)<br>XX ( XX.X) | XX ( XX.X)<br>XX ( XX.X)<br>XX ( XX.X)<br>XX ( XX.X)<br>XX ( XX.X)<br>XX ( XX.X) | XX ( XX.X)<br>XX ( XX.X)<br>XX ( XX.X)<br>XX ( XX.X)<br>XX ( XX.X)<br>XX ( XX.X) | XX ( XX.X)<br>XX ( XX.X)<br>XX ( XX.X)<br>XX ( XX.X)<br>XX ( XX.X)<br>XX ( XX.X) |
| AIDS STATUS<br>YES<br>NO | xx ( XX.X)<br>xx ( XX.X) | XX ( XX.X)<br>XX ( XX.X) | XX ( XX.X)<br>XX ( XX.X) | XX ( XX.X)<br>XX ( XX.X) | XX ( XX.X)<br>XX ( XX.X) |

\_\_\_\_\_

| Parameter | Values |
|------------------|-----------------------------------------------------|
| Template ID | SS_DM_T_004 |
| Output File Name | rt-dm-diseases1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.3.2.1 |
| Title 1 | Summary of Baseline Disease Characteristics |
| Title 2 | Treated Subjects - Stage 1 |
| Layout notes | Include all HIV subtypes available in the database. |

| Parameter | Values |
|------------------|-----------------------------------------------------|
| Template ID | SS_DM_T_004 |
| Output File Name | rt-dm-diseases2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.3.2.2 |
| Title 1 | Summary of Baseline Disease Characteristics |
| Title 2 | Treated Subjects - Stage 2 |
| Layout notes | Include all HIV subtypes available in the database. |

| Parameter | Values |
|------------------|-----------------------------------------------------|
| Template ID | SS_DM_T_004 |
| Output File Name | rt-dm-diseases12.lst |
| Purpose | WK96S2 |
| Table No. | Table S.3.2.3 |
| Title 1 | Summary of Baseline Disease Characteristics |
| Title 2 | Treated Subjects - Stage 1 and 2 |
| Layout notes | Include all HIV subtypes available in the database. |

| Parameter | Values |
|------------------|------------------------------------------------|
| Template ID | SS_DM_T_004 |
| Output File Name | rt-dm-diseasenrands1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Appendix 3.2.1A |
| Title 1 | Summary of Baseline Disease Characteristics |
| Title 2 | Subjects Enrolled but Not Randomized - Stage 1 |

| Layout notes | Include only the 'Total' column. |
|--------------|-----------------------------------------------------|
| | Include all HIV subtypes available in the database. |

| Parameter | Values |
|------------------|-----------------------------------------------------|
| Template ID | SS_DM_T_004 |
| Output File Name | rt-dm-diseasenrands2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Appendix 3.2.2A |
| Title 1 | Summary of Baseline Disease Characteristics |
| Title 2 | Subjects Enrolled but Not Randomized - Stage 2 |
| Layout notes | Include only the 'Total' column. |
| | Include all HIV subtypes available in the database. |

# Template SS\_DM\_L\_002: Listing of HIV Disease Characteristics

Treatment Group: TRT A

| | Plasma | HIV-1 Level | CD4+ | T-cell count | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Subject ID | Result<br>(log10 c | Category<br>/mL) (c/mL) | Result<br>(cells | | CD4 T-cell<br>(percent) | CD8+<br>cells/uL) | HIV<br>Subtype | IC50<br>(µM) | IC Fold<br>Change |
| PPD | X.X | <30,000 | <br>XX | < 200 | XX | <br>xx | xxxx | <br>XX | ×x |
| | X.X | 30,000 to $< 100,000$ | XX | 350 to < 500 | XX | XX | XXXX | XX | XX |
| | X.X | 100,000 to < 500,000 | XX | 200 to < 350 | XX | XX | XXXX | XX | XX |
| | X.X | ≥ 500 <b>,</b> 000 | XX | 200 to < 350 | XX | XX | XXXX | XX | XX |
| | X.X | ≥ 500,000 | XX | 350 to < 500 | XX | XX | XXXX | XX | XX |
| | X.X | ≥ 500 <b>,</b> 000 | XX | ≥ 500 | XX | XX | XXXX | XX | XX |
| | X.X | ≥ 500,000 | XX | 350 to < 500 | XX | XX | XXXX | XX | XX |
| | ×.× | ≥ 500,000 | XX | 350 to < 500 | XX | XX | XXXX | XX | XX |

\_\_\_\_\_\_

| Parameter | Values |
|-------------------|--------------------------------------------------------|
| Template ID | SS_DM_L_002 |
| Output File Name | rl-dm-diseases1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Appendix 3.2.1B |
| Title 1 | Listing of HIV Disease Characteristics |
| Title 2 | Treated Subjects - Stage 1 |
| Programming notes | Sorted by treatment group, site and subject identifier |

| Parameter | Values |
|------------------|------------------------|
| Template ID | SS_DM_L_002 |
| Output File Name | rl-dm-diseases2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Appendix 3.2.2B |

| Title 1 | Listing of HIV Disease Characteristics |
|---|---|
| Title 2 | eated Subjects - Stage 2 |
| Programming notes | Sorted by treatment group, site and subject identifier |

### Template GS\_PM\_T\_X\_001: Physical Measurements Table

Draft
Physical Measurements Summary
All Treated Subjects Protocol: CA259001 

| Period/Visit | TRT A<br>N = 1366 | TRT B<br>N = 1382 | TRT C<br>N = 1338 | Total<br>N = 4086 |
|---|---|---|---|---|
| SCREENING/DAY -1 | | | | |
| HEIGHT (CM)<br>N<br>MEAN<br>MEDIAN<br>MIN , MAX<br>STANDARD DEVIATION | 1366<br>170.6<br>171.0<br>147.3 , 198.1<br>3.62 | 1382<br>170.6<br>171.0<br>149.0 , 198.1<br>3.73 | 1338<br>170.6<br>171.0<br>143.5 , 198.1<br>3.69 | 4086<br>170.6<br>171.0<br>143.5 , 198.1<br>3.68 |
| WEIGHT (KG)<br>N<br>MEAN<br>MEDIAN<br>MIN , MAX<br>STANDARD DEVIATION | 1366<br>87.7<br>85.3<br>51.0 , 158.1<br>18.63 | 1382<br>88.1<br>86.5<br>41.5 , 149.2<br>21.01 | 1338<br>88.7<br>85.7<br>38.4 , 144.5<br>19.39 | 4086<br>88.2<br>85.7<br>38.4,158.1<br>19.71 |
| BODY MASS INDEX (KG/M2)<br>N<br>MEAN<br>MEDIAN<br>MIN , MAX<br>STANDARD DEVIATION | 1366<br>30.11<br>29.31<br>17.44, 54.07<br>6.252 | 1382<br>30.25<br>29.74<br>14.19 , 51.02<br>7.017 | 1338<br>30.46<br>29.49<br>13.13 , 47.95<br>6.523 | 4086<br>30.27<br>29.48<br>13.13 , 54.07<br>6.607 |

Program Source: /wwbdm/ndp/prime/gssr/devtest/phm/test/domain\_example/phm\_tbl1.sas 15DEC2004:16:21:00

| Parameter | Values |
|------------------|--------------------------------|
| Template ID | GS_PM_T_X_001 |
| Output File Name | rt-pm-bsls1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.3.3.1 |
| Title 1 | Physical Measurements Summary |
| Title 2 | Treated Subjects - Stage 1 |

| Parameter | Values |
|------------------|-------------------------------|
| Template ID | GS_PM_T_X_001 |
| Output File Name | rt-pm-bsls2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.3.3.2 |
| Title 1 | Physical Measurements Summary |
| Title 2 | Treated Subjects - Stage 2 |

# Template GS\_PE\_T\_X\_001: Physical Examination by Treatment Group

Protocol: TA123456 Draft
Physical Examination Summary
All Treated Subjects 

| Period/Visit | TRT A<br>N = 16 | TRT B<br>N = 17 | TRT C<br>N = 17 | Total<br>N = 50 |
|---|---|---|---|---|
| SCREENING/DAY 1 | | | | |
| SUBJECTS WITH ABNORMAL PHYSICAL EXAMINATION (%) | 10 (62.5) | 14 ( 82.4) | 14 ( 82.4) | 38 (76.0) |
| GENERAL APPEARANCE HEAD, EARS, EYES, NOSE, THROAT NECK CARDIOVASCULAR LUNGS ABDOMEN LYMPH NODES GENITOURINARY EXTREMITIES NEUROLOGICAL SKIN MUSCULOSKELETAL OTHER | 0<br>5 ( 31.3)<br>0<br>0<br>1 ( 6.3)<br>0<br>3 ( 18.8)<br>0<br>8 ( 50.0)<br>8 ( 50.0) | 1 ( 5.9) 12 ( 70.6) 0 0 0 2 ( 11.8) 0 2 ( 11.8) 0 10 ( 58.8) 1 ( 5.9) 7 ( 41.2) | 0<br>5 ( 29.4)<br>0<br>0<br>1 ( 5.9)<br>1 ( 5.9)<br>0<br>4 ( 23.5)<br>1 ( 5.9)<br>8 ( 47.1)<br>1 ( 5.9)<br>8 ( 47.1) | 1 ( 2.0) 22 ( 44.0) 0 0 1 ( 2.0) 4 ( 8.0) 0 9 ( 18.0) 1 ( 2.0) 26 ( 52.0) 2 ( 4.0) 23 ( 46.0) |
| SCREENING/DAY 5 | | | | |
| SUBJECTS WITH ABNORMAL PHYSICAL EXAMINATION (%) | 10 (62.5) | 14 ( 82.4) | 14 ( 82.4) | 38 ( 76.0) |
| GENERAL APPEARANCE HEAD, EARS, EYES, NOSE, THROAT NECK CARDIOVASCULAR LUNGS ABDOMEN LYMPH NODES GENITOURINARY EXTREMITIES NEUROLOGICAL SKIN MUSCULOSKELETAL OTHER | 0<br>5 (31.3)<br>0<br>0<br>1 (6.3)<br>0<br>3 (18.8)<br>0<br>8 (50.0)<br>8 (50.0) | 1 ( 5.9) 12 ( 70.6) 0 0 0 2 ( 11.8) 0 2 ( 11.8) 0 10 ( 58.8) 1 ( 5.9) 7 ( 41.2) | 0<br>5 (29.4)<br>0<br>0<br>1 (5.9)<br>1 (5.9)<br>0<br>4 (23.5)<br>1 (5.9)<br>8 (47.1)<br>1 (5.9)<br>8 (47.1) | 1 ( 2.0) 22 ( 44.0) 0 0 1 ( 2.0) 4 ( 8.0) 0 9 ( 18.0) 1 ( 2.0) 26 ( 52.0) 2 ( 4.0) 23 ( 46.0) |

Program Source: /wwbdm/ndp/prime/gssr/devtest/mhx/test/domain\_example/phx\_tbl.sas

21SEP2004:10:31:00

| Parameter | Values |
|------------------|---------------------------------------------------|
| Template ID | GS_PE_T_X_001 |
| Output File Name | rt-pe-bslsums1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.3.4.1 |
| Title 1 | Physical Examination Summary |
| Title 2 | Treated Subjects - Stage 1 |
| Layout notes | Include all examinations present in the database. |

| Parameter | Values |
|------------------|---------------------------------------------------|
| Template ID | GS_PE_T_X_001 |
| Output File Name | rt-pe-bslsums2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.3.4.2 |
| Title 1 | Physical Examination Summary |
| Title 2 | Treated Subjects - Stage 2 |
| Layout notes | Include all examinations present in the database. |

### Template GS\_PE\_L\_X\_001: Physical Examination Listing by Treatment Group

Protocol: TA123456 Draft Page 1 of 958

Draft Physical Examination All Treated Subjects

Treatment Group: DRUG C

| Subject ID<br>(Age/Gender/Race) | Period<br>Visit<br>Exam Date<br>Study Day | Exanimation<br>Criteria | Exam<br>Result | Abnormality |
|---|---|---|---|---|
| PPD<br>(46/M/C) | SCREENING A1 PPD -14 | GENERAL APPEARANCE HEENT NECK CARDIOVASCULAR LUNGS ABDOMEN LYMPH NODES GENITOURINARY EXTREMITIES NEUROLOGICAL SKIN MUSCULOSKELETAL | NORMAL ABNORMAL ABNORMAL NORMAL NORMAL NORMAL NORMAL NOT DONE ABNORMAL NORMAL ABNORMAL ABNORMAL | R EYE MILD NYSTIGMUS NCS CAROTID PULSES DIMINISHED SYMETRICALLY WITHOUT BRUITS NCS MSM GRADE I-II / III NCS BILATERAL TRACE NO PITTING ANKLE EDEMA ABRASION R BENIGN MOLES NEVI & ACROCHORITONS BILAT HAND W/MCP&PIP RA CHNGS, TR SYNOVITIS L MCP 3&4,R MCP 3,4,5,TR SYNOVITIS WRIST BILAT,MILD BILAT TRAPESIUS TIGHTNES SYMETRICALLY, SHOULDERS DECR FROM ABDUCT 90 DEGREES SYMETRICALLY W/ANTERIOR TPS |
| PPD<br>(55/F/C) | PRE-TREAT<br>A3<br>PPD<br>-1 | GENERAL APPEARANCE<br>HEENT<br>NECK<br>CARDIOVASCULAR<br>LUNGS<br>ABDOMEN | NORMAL<br>NORMAL<br>NORMAL<br>NORMAL<br>NORMAL<br>NORMAL | |

Program Source: /wwbdm/ndp/prime/gssr/devtest/phy/test/phy lst.sas 28FEB2005:15:09:00

| Parameter | Values |
|------------------|--------------------------------|
| Template ID | GS_PE_L_X_001 |
| Output File Name | rl-pe-lists1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Appendix 3.4.1 |
|-----------|----------------------------|
| Title 1 | Physical Examination |
| Title 2 | Treated Subjects - Stage 1 |

| Parameter | Values |
|------------------|----------------------------|
| Template ID | GS_PE_L_X_001 |
| Output File Name | rl-pe-lists2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Appendix 3.4.2 |
| Title 1 | Physical Examination |
| Title 2 | Treated Subjects - Stage 2 |

Template SS\_GN\_T\_001: Baseline Genotypic Resistance Profile

Subgroup: XXXXXXXXX Level: XXXXXXXXXXX

| | Group A<br>N = XX | Group B<br>N = XX | Group C<br>N = XX | Group D<br>N=XX |
|---|---|---|---|---|
| TESTED | XX/XX (XX.X) | XX/XX (XX.X) | XX/XX (XX.X) | XX/XX (XX.X) |
| SEQUENCED | XX/XX (XX.X) | XX/XX (XX.X) | XX/XX (XX.X) | XX/XX (XX.X) |
| ANY PI SUBSTITUTIONS PI substitutions#1 PI substitutions#2 PI substitutions#3 PI substitutions#4 <additional substitutions=""></additional> | XX/XX (XX.X)<br>XX/XX (XX.X)<br>XX/XX (XX.X)<br>XX/XX (XX.X)<br>XX/XX (XX.X) | XX/XX (XX.X)<br>XX/XX (XX.X)<br>XX/XX (XX.X)<br>XX/XX (XX.X)<br>XX/XX (XX.X) | XX/XX (XX.X)<br>XX/XX (XX.X)<br>XX/XX (XX.X)<br>XX/XX (XX.X)<br>XX/XX (XX.X) | XX/XX (XX.X)<br>XX/XX (XX.X)<br>XX/XX (XX.X)<br>XX/XX (XX.X)<br>XX/XX (XX.X) |
| SELECTED RT SUBSTITUTIONS nRTI SUBSTITUTIONS nRTI substitutions#1 nRTI substitutions#2 <additional substitutions=""></additional> | XX/XX (XX.X)<br>XX/XX (XX.X)<br>XX/XX (XX.X) | XX/XX (XX.X) XX/XX (XX.X) XX/XX (XX.X) | XX/XX (XX.X) XX/XX (XX.X) XX/XX (XX.X) | XX/XX (XX.X) XX/XX (XX.X) XX/XX (XX.X) |
| NNRTI SUBSTITUTIONS NNRTI substitutions#1 NNRTI substitutions#2 INTEGRASE (RAL) SUBSTITUTIONS RAL substitutions#1 | XX/XX (XX.X)<br>XX/XX (XX.X)<br>XX/XX (XX.X)<br>XX/XX (XX.X) | XX/XX (XX.X)<br>XX/XX (XX.X)<br>XX/XX (XX.X)<br>XX/XX (XX.X) | XX/XX (XX.X)<br>XX/XX (XX.X)<br>XX/XX (XX.X)<br>XX/XX (XX.X) | XX/XX (XX.X)<br>XX/XX (XX.X)<br>XX/XX (XX.X)<br>XX/XX (XX.X) |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_001 |
| Output File Name | rt-gn-bases1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.3.9.1A |
| Title 1 | Baseline Genotypic Resistance Profile |
| Title 2 | Treated Subjects - Stage 1 |
| Footnote 1 | Mutations extracted from data are based on IAS-USA list updated June 2014. |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_001 |
| Output File Name | rt-gn-bases2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.3.9.2A |
| Title 1 | Baseline Genotypic Resistance Profile |
| Title 2 | Treated Subjects - Stage 2 |
| Footnote 1 | Mutations extracted from data are based on IAS-USA list updated June 2014. |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_001 |
| Output File Name | rt-gn-bases12.lst |
| Purpose | WK96S2 |
| Table No. | Table S.3.9.3A |
| Title 1 | Baseline Genotypic Resistance Profile |
| Title 2 | Treated Subjects - Stage 1 and 2 |
| Footnote 1 | Mutations extracted from data are based on IAS-USA list updated June 2014. |

| Parameter | Values |
|------------------|---------------------------------------|
| Template ID | SS_GN_T_001 |
| Output File Name | rt-gn-basebysubtypes1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Appendix 3.9.1A |
| Title 1 | Baseline Genotypic Resistance Profile |

| Title 2 | By HIV Subtype |
|---|---|
| Title 3 | Treated Subjects - Stage 1 |
| Footnote 1 | Mutations extracted from data are based on IAS-USA list updated June 2014. |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_001 |
| Output File Name | rt-gn-basebysubtypes2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Appendix 3.9.2A |
| Title 1 | Baseline Genotypic Resistance Profile |
| Title 2 | By HIV Subtype |
| Title 3 | Treated Subjects - Stage 2 |
| Footnote 1 | Mutations extracted from data are based on IAS-USA list updated June 2014. |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_001 |
| Output File Name | rt-gn-baseots1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.3.9.1B |
| Title 1 | Baseline Genotypic Resistance Profile |
| Title 2 | Treated Subjects with On-Treatment Resistance Testing - Stage 1 |
| Footnote 1 | Mutations extracted from data are based on IAS-USA list updated June 2014. |

| Parameter | Values |
|-------------|-------------|
| Template ID | SS_GN_T_001 |

| Output File Name | rt-gn-baseots2.lst |
|---|---|
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.3.9.2B |
| Title 1 | Baseline Genotypic Resistance Profile |
| Title 2 | Treated Subjects with On-Treatment Resistance Testing - Stage 2 |
| Footnote 1 | Mutations extracted from data are based on IAS-USA list updated June 2014. |

## Template SS\_GN\_L\_001:Genotypic Resistance Listing

| Subject ID<br>(Age/Gender/Race)<br>Treatment Group | Current Treatment | Period<br>Visit<br>Date<br>Study Day | RT Substitutions | PI Substitutions | RAL Substitutions |
|---|---|---|---|---|---|
| PPD<br>(54/F/C)<br>ATV/r/RAL/TDF | PRE-TREATMENT | PRE-TREATMENT SCREENING PPD -42 | Q102K, K103K,<br>K103N, I142I,<br>I142V, C162S,<br>I178L, R211K,<br>A272P, K275R,<br>R277K, Q278H | R41K, Q61H | V72I, S81R,<br>S81S, V113I,<br>T124A, V201I,<br>Y227F, S230N,<br>R231K, V234L,<br>A265V |
| | ATV300mg QD+RTV100mg QD+RAL400mg BID+TDF300mg QD | STAGE 1<br>WE<br>PPD<br>119 | Q102K, K103K,<br>K103N, I142I,<br>I142V, C162S,<br>I178L, R211K,<br>A272P, K275R,<br>R277K, Q278H,<br>P294P, P294S | R41K, Q61H | V72I, V113I,<br>T124A, V201I,<br>Y227F, S230N,<br>R231K, V234L,<br>A265V |
| PPD<br>(62/M/C)<br>ATV/r/RAL/TDF | PRE-TREATMENT | PRE-TREATMENT SCREENING PPD -38 | Q102K, K103N,<br>K122E, K122K,<br>D123D, D123E,<br>D123K, D123N,<br>V179I, V179V,<br>Q207N, H208H,<br>H208Y, R211K,<br>A272P, T286A,<br>V293I, E297K | E35D, M36I,<br>M36M, N37D,<br>R57K, R57R,<br>I62V, L63H,<br>I93L | E10D, M50I,<br>M50M, V72I,<br>L101I, V113I,<br>S119P, T125A,<br>K156N, G193E,<br>G193G, G193K,<br>G193R, V201I,<br>S230N, D232E,<br>V234L, D256E,<br>D278A, Q285P,<br>Q285Q |

ParameterValuesTemplate IDSS\_GN\_L\_001Output File Namerl-gn-bsls1.lstPurposeWK24S1, WK48S1, WK96S1, WK96S2Table No.Appendix 3.9.1BTitle 1Listing of Baseline Genotypic Substitutions

| Title 2 | Treated Subjects - Stage 1 |
|-------------------|----------------------------------------------------|
| Programming notes | Please include only the pre-treatment assessments. |

| Parameter | Values |
|-------------------|----------------------------------------------------|
| Template ID | SS_GN_L_001 |
| Output File Name | rl-gn-bsls2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Appendix 3.9.2B |
| Title 1 | Listing of Baseline Genotypic Substitutions |
| Title 2 | Treated Subjects - Stage 2 |
| Programming notes | Please include only the pre-treatment assessments. |

Template SS\_GN\_T\_002: Baseline Gag Polymorphisms at Selected Positions

Subgroup: XXXXXXXXX Level: XXXXXXXXXXX

| | | Group B<br>N = XX | Group C<br>N = XX | Group D<br>N=XX |
|---|---|---|---|---|
| TESTED | XX/XX (XX.X) | XX/XX (XX.X) | XX/XX (XX.X) | XX/XX (XX.X) |
| SEQUENCED | XX/XX (XX.X) | XX/XX (XX.X) | XX/XX (XX.X) | XX/XX (XX.X) |
| SELECTED SUBSTITUTIONS POSITION 362 POSITION 364 POSITION 369 POSITION 370 | XX/XX (XX.X)<br>XX/XX (XX.X)<br>XX/XX (XX.X)<br>XX/XX (XX.X)<br>XX/XX (XX.X) | | XX/XX (XX.X)<br>XX/XX (XX.X)<br>XX/XX (XX.X)<br>XX/XX (XX.X)<br>XX/XX (XX.X) | XX/XX (XX.X)<br>XX/XX (XX.X)<br>XX/XX (XX.X)<br>XX/XX (XX.X)<br>XX/XX (XX.X) |
| POSITIONS 362 AND 364 POSITIONS 362 AND 369 POSITIONS 362 AND 370 POSITIONS 364 AND 369 POSITIONS 364 AND 370 POSITIONS 369 AND 370 | XX/XX (XX.X) XX/XX (XX.X) XX/XX (XX.X) XX/XX (XX.X) XX/XX (XX.X) XX/XX (XX.X) XX/XX (XX.X) | XX/XX (XX.X) | XX/XX (XX.X)<br>XX/XX (XX.X)<br>XX/XX (XX.X)<br>XX/XX (XX.X)<br>XX/XX (XX.X)<br>XX/XX (XX.X) | XX/XX (XX.X) XX/XX (XX.X) XX/XX (XX.X) XX/XX (XX.X) XX/XX (XX.X) XX/XX (XX.X) XX/XX (XX.X) |
| POSITIONS 362, 364 AND 369<br>POSITIONS 362, 364 AND 370<br>POSITIONS 364, 369 AND 370 | XX/XX (XX.X)<br>XX/XX (XX.X)<br>XX/XX (XX.X) | XX/XX (XX.X)<br>XX/XX (XX.X)<br>XX/XX (XX.X) | XX/XX (XX.X)<br>XX/XX (XX.X)<br>XX/XX (XX.X) | XX/XX (XX.X)<br>XX/XX (XX.X)<br>XX/XX (XX.X) |
| POSITIONS 362, 364, 369 AND 370 | XX/XX (XX.X) | XX/XX (XX.X) | XX/XX (XX.X) | XX/XX (XX.X) |

ParameterValuesTemplate IDSS\_GN\_T\_002Output File Namert-gn-bslgags1.lstPurposeWK24S1, WK48S1, WK96S1, WK96S2Table No.Table S.3.9.1CTitle 1Baseline Gag Polymorphisms at Selected PositionsTitle 2Treated Subjects - Stage 1

| Parameter | Values |
|------------------|--------------------------------------------------|
| Template ID | SS_GN_T_002 |
| Output File Name | rt-gn-bslgags2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.3.9.2C |
| Title 1 | Baseline Gag Polymorphisms at Selected Positions |
| Title 2 | Treated Subjects - Stage 2 |

| Parameter | Values |
|------------------|--------------------------------------------------|
| Template ID | SS_GN_T_002 |
| Output File Name | rt-gn-bslgags12.lst |
| Purpose | WK96S2 |
| Table No. | Table S.3.9.3C |
| Title 1 | Baseline Gag Polymorphisms at Selected Positions |
| Title 2 | Treated Subjects - Stage 1 and 2 |

| Parameter | Values |
|------------------|--------------------------------------------------|
| Template ID | SS_GN_T_002 |
| Output File Name | rt-gn-bslgagbysubtypes1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.3.9.1D |
| Title 1 | Baseline Gag Polymorphisms at Selected Positions |
| Title 2 | By HIV Subtype |
| Title 3 | Treated Subjects - Stage 1 |

| Parameter | Values |
|------------------|--------------------------------------------------|
| Template ID | SS_GN_T_002 |
| Output File Name | rt-gn-bslgagbysubtypes2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.3.9.2D |
| Title 1 | Baseline Gag Polymorphisms at Selected Positions |
| Title 2 | By HIV Subtype |
| Title 3 | Treated Subjects - Stage 2 |

| Parameter | Values |
|------------------|--------------------------------------------------|
| Template ID | SS_GN_T_002 |
| Output File Name | rt-gn-bslgagbysubtypes12.lst |
| Purpose | WK96S2 |
| Table No. | Table S.3.9.3D |
| Title 1 | Baseline Gag Polymorphisms at Selected Positions |
| Title 2 | By HIV Subtype |
| Title 3 | Treated Subjects - Stage 1 and 2 |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_002 |
| Output File Name | rt-gn-bslgagontrts1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.3.9.1H |
| Title 1 | Baseline Gag Polymorphisms at Selected Positions |
| Title 2 | Treated Subjects with On-Treatment Resistance Testing - Stage 1 |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_002 |
| Output File Name | rt-gn-bslgagontrts2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.3.9.2H |
| Title 1 | Baseline Gag Polymorphisms at Selected Positions |
| Title 2 | Treated Subjects with On-Treatment Resistance Testing - Stage 2 |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_002 |
| Output File Name | rt-gn-bslgagontrts12.lst |
| Purpose | WK96S2 |
| Table No. | Table S.3.9.3H |
| Title 1 | Baseline Gag Polymorphisms at Selected Positions |
| Title 2 | Treated Subjects with On-Treatment Resistance Testing - Stage 1 and 2 |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_002 |
| Output File Name | rt-gn-bslgagontrtbysubtypes1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.3.9.1I |
| Title 1 | Baseline Gag Polymorphisms at Selected Positions |
| Title 2 | By HIV Subtype |
| Title 3 | Treated Subjects with On-Treatment Resistance Testing - Stage 1 |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_002 |
| Output File Name | rt-gn-bslgagontrtbysubtypes2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.3.9.2I |
| Title 1 | Baseline Gag Polymorphisms at Selected Positions |
| Title 2 | By HIV Subtype |
| Title 3 | Treated Subjects with On-Treatment Resistance Testing - Stage 2 |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_002 |
| Output File Name | rt-gn-bslgagontrtbysubtypes12.lst |
| Purpose | WK96S2 |
| Table No. | Table S.3.9.3I |
| Title 1 | Baseline Gag Polymorphisms at Selected Positions |
| Title 2 | By HIV Subtype |
| Title 3 | Treated Subjects with On-Treatment Resistance Testing - Stage 1 and 2 |

| Parameter | Values |
|------------------|--------------------------------------------------|
| Template ID | SS_GN_T_002 |
| Output File Name | rt-gn-bslgagpdvfs1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.3.9.1J |
| Title 1 | Baseline Gag Polymorphisms at Selected Positions |

| Title 2 | Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 1 |
|---|---|
| Footnote 1 | Protocol Defined Virologic Failure is defined by a subject meeting one of the following criteria: |
| Footnote 2 | 1) Confirmed > 1 log <sub>10</sub> c/mL increase in HIV-1 RNA at anytime above nadir level where nadir is ≥ 40 c/mL |
| Footnote 3 | 2) Confirmed HIV-1 RNA ≥ 40 c/mL if prior suppression to < 40 c/mL |
| Footnote 4 | 3) Failure to have the last on-treatment HIV-1 RNA to < 400 c/mL within Week 24, 48, or 96 week snapshot window |
| Footnote 5 | 4) Failure to achieve > 1 log <sub>10</sub> c/mL decrease in HIV-1 RNA by Week 8 |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_002 |
| Output File Name | rt-gn-bslgagpdvfs2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.3.9.2J |
| Title 1 | Baseline Gag Polymorphisms at Selected Positions |
| Title 2 | Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 2 |
| Footnote 1 | Protocol Defined Virologic Failure is defined by a subject meeting one of the following criteria: |
| Footnote 2 | 1) Confirmed > 1 log <sub>10</sub> c/mL increase in HIV-1 RNA at anytime above nadir level where nadir is ≥ 40 c/mL |
| Footnote 3 | 2) Confirmed HIV-1 RNA ≥ 40 c/mL if prior suppression to < 40 c/mL |
| Footnote 4 | 3) Failure to have the last on-treatment HIV-1 RNA to < 400 c/mL within Week 24, 48, or 96 week snapshot window |
| Footnote 5 | 4) Failure to achieve > 1 log <sub>10</sub> c/mL decrease in HIV-1 RNA by Week 8 |

| Parameter | Values |
|------------------|-------------------------|
| Template ID | SS_GN_T_002 |
| Output File Name | rt-gn-bslgagpdvfs12.lst |
| Purpose | WK96S2 |
| Table No. | Table S.3.9.3J |

| Title 1 | Baseline Gag Polymorphisms at Selected Positions |
|---|---|
| Title 2 | Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 1 and 2 |
| Footnote 1 | Protocol Defined Virologic Failure is defined by a subject meeting one of the following criteria: |
| Footnote 2 | 1) Confirmed > 1 log <sub>10</sub> c/mL increase in HIV-1 RNA at anytime above nadir level where nadir is ≥ 40 c/mL |
| Footnote 3 | 2) Confirmed HIV-1 RNA ≥ 40 c/mL if prior suppression to < 40 c/mL |
| Footnote 4 | 3) Failure to have the last on-treatment HIV-1 RNA to < 400 c/mL within Week 24, 48, or 96 week snapshot window |
| Footnote 5 | 4) Failure to achieve > 1 log <sub>10</sub> c/mL decrease in HIV-1 RNA by Week 8 |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_002 |
| Output File Name | rt-gn-bslgagpdvfbysubtypes1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.3.9.1K |
| Title 1 | Baseline Gag Polymorphisms at Selected Positions |
| Title 2 | By HIV Subtype |
| Title 3 | Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 1 |
| Footnote 1 | Protocol Defined Virologic Failure is defined by a subject meeting one of the following criteria: |
| Footnote 2 | 1) Confirmed > 1 log <sub>10</sub> c/mL increase in HIV-1 RNA at anytime above nadir level where nadir is ≥ 40 c/mL |
| Footnote 3 | 2) Confirmed HIV-1 RNA ≥ 40 c/mL if prior suppression to < 40 c/mL |
| Footnote 4 | 3) Failure to have the last on-treatment HIV-1 RNA to < 400 c/mL within Week 24, 48, or 96 week snapshot window |
| Footnote 5 | 4) Failure to achieve > 1 log <sub>10</sub> c/mL decrease in HIV-1 RNA by Week 8 |

| Parameter | Values |
|------------------|---------------------------------|
| Template ID | SS_GN_T_002 |
| Output File Name | rt-gn-bslgagpdvfbysubtypes2.lst |

| Purpose | WK24S2, WK48S2, WK96S2 |
|---|---|
| Table No. | Table S.3.9.2K |
| Title 1 | Baseline Gag Polymorphisms at Selected Positions |
| Title 2 | By HIV Subtype |
| Title 3 | Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 2 |
| Footnote 1 | Protocol Defined Virologic Failure is defined by a subject meeting one of the following criteria: |
| Footnote 2 | 1) Confirmed > 1 log <sub>10</sub> c/mL increase in HIV-1 RNA at anytime above nadir level where nadir is ≥ 40 c/mL |
| Footnote 3 | 2) Confirmed HIV-1 RNA ≥ 40 c/mL if prior suppression to < 40 c/mL |
| Footnote 4 | 3) Failure to have the last on-treatment HIV-1 RNA to < 400 c/mL within Week 24, 48, or 96 week snapshot window |
| Footnote 5 | 4) Failure to achieve > 1 log <sub>10</sub> c/mL decrease in HIV-1 RNA by Week 8 |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_002 |
| Output File Name | rt-gn-bslgagpdvfbysubtypes12.lst |
| Purpose | WK96S2 |
| Table No. | Table S.3.9.3K |
| Title 1 | Baseline Gag Polymorphisms at Selected Positions |
| Title 2 | By HIV Subtype |
| Title 3 | Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 1 and 2 |
| Footnote 1 | Protocol Defined Virologic Failure is defined by a subject meeting one of the following criteria: |
| Footnote 2 | 1) Confirmed > 1 log <sub>10</sub> c/mL increase in HIV-1 RNA at anytime above nadir level where nadir is ≥ 40 c/mL |
| Footnote 3 | 2) Confirmed HIV-1 RNA ≥ 40 c/mL if prior suppression to < 40 c/mL |
| Footnote 4 | 3) Failure to have the last on-treatment HIV-1 RNA to < 400 c/mL within Week 24, 48, or 96 week snapshot window |
| Footnote 5 | 4) Failure to achieve > 1 log <sub>10</sub> c/mL decrease in HIV-1 RNA by Week 8 |

## Template SS\_GN\_T\_003: Baseline Gag Deviations from Wild Type

Subgroup: XXXXXXXXX Level: XXXXXXXXXXX

| | Group A | Group B | Group C | Group D |
|---|---|---|---|---|
| | N = XX | N = XX | N = XX | N=XX |
| TESTED | XX/XX (XX.X) | XX/XX (XX.X) | XX/XX (XX.X) | XX/XX (XX.X) |
| SEQUENCED | XX/XX (XX.X) | XX/XX (XX.X) | XX/XX (XX.X) | XX/XX (XX.X) |
| ANY DEVIATION DEV 1 DEV 2 DEV 3 DEV 4 | XX/XX (XX.X) | XX/XX (XX.X) | XX/XX (XX.X) | XX/XX (XX.X) |
| | XX/XX (XX.X) | XX/XX (XX.X) | XX/XX (XX.X) | XX/XX (XX.X) |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_003 |
| Output File Name | rt-gn-bslgaganys1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.3.9.1E |
| Title 1 | Baseline Gag Deviations from Wild Type Virus |
| Title 2 | Treated Subjects - Stage 1 |
| Layout notes | Include any deviation from the wild type virus detected in the database. |

| Parameter | Values |
|------------------|------------------------|
| Template ID | SS_GN_T_003 |
| Output File Name | rt-gn-bslgaganys2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |

| Table No. | Table S.3.9.2E |
|---|---|
| Title 1 | Baseline Gag Deviations from Wild Type Virus |
| Title 2 | Treated Subjects - Stage 2 |
| Layout notes | Include any deviation from the wild type virus detected in the database. |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_003 |
| Output File Name | rt-gn-bslgaganys12.lst |
| Purpose | WK96S2 |
| Table No. | Table S.3.9.3E |
| Title 1 | Baseline Gag Deviations from Wild Type Virus |
| Title 2 | Treated Subjects - Stage 1 and 2 |
| Layout notes | Include any deviation from the wild type virus detected in the database. |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_003 |
| Output File Name | rt-gn-bslgaganybysubtypes1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.3.9.1L |
| Title 1 | Baseline Gag Deviations from Wild Type Virus |
| Title 2 | By HIV Subtype |
| Title 3 | Treated Subjects - Stage 1 |
| Layout notes | Include any deviation from the wild type virus detected in the database. |

| Template ID | SS_GN_T_003 |
|---|---|
| Output File Name | rt-gn-bslgaganybysubtypes2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.3.9.2L |
| Title 1 | Baseline Gag Deviations from Wild Type Virus |
| Title 2 | By HIV Subtype |
| Title 3 | Treated Subjects - Stage 2 |
| Layout notes | Include any deviation from the wild type virus detected in the database. |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_003 |
| Output File Name | rt-gn-bslgaganybysubtypes12.lst |
| Purpose | WK96S2 |
| Table No. | Table S.3.9.3L |
| Title 1 | Baseline Gag Deviations from Wild Type Virus |
| Title 2 | By HIV Subtype |
| Title 3 | Treated Subjects - Stage 1 and 2 |
| Layout notes | Include any deviation from the wild type virus detected in the database. |

| Parameter | Values |
|------------------|----------------------------------------------|
| Template ID | SS_GN_T_003 |
| Output File Name | rt-gn-bslgaganyontrts1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.3.9.1M |
| Title 1 | Baseline Gag Deviations from Wild Type Virus |

| Title 2 | Treated Subjects with On-Treatment Resistance Testing - Stage 1 |
|---|---|
| Layout notes | Include any deviation from the wild type virus detected in the database. |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_003 |
| Output File Name | rt-gn-bslgaganyontrts2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.3.9.2M |
| Title 1 | Baseline Gag Deviations from Wild Type Virus |
| Title 2 | Treated Subjects with On-Treatment Resistance Testing - Stage 2 |
| Layout notes | Include any deviation from the wild type virus detected in the database. |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_003 |
| Output File Name | rt-gn-bslgaganyontrts12.lst |
| Purpose | WK96S2 |
| Table No. | Table S.3.9.3M |
| Title 1 | Baseline Gag Deviations from Wild Type Virus |
| Title 2 | Treated Subjects with On-Treatment Resistance Testing - Stage 1 and 2 |
| Layout notes | Include any deviation from the wild type virus detected in the database. |

| Parameter | Values |
|------------------|-------------------------------------|
| Template ID | SS_GN_T_003 |
| Output File Name | rt-gn-bslgaganyontrtbysubtypes1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |

| Table No. | Table S.3.9.1N |
|---|---|
| Title 1 | Baseline Gag Deviations from Wild Type Virus |
| Title 2 | By HIV Subtype |
| Title 3 | Treated Subjects with On-Treatment Resistance Testing - Stage 1 |
| Layout notes | Include any deviation from the wild type virus detected in the database. |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_003 |
| Output File Name | rt-gn-bslgaganyontrtbysubtypes2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.3.9.2N |
| Title 1 | Baseline Gag Deviations from Wild Type Virus |
| Title 2 | By HIV Subtype |
| Title 3 | Treated Subjects with On-Treatment Resistance Testing - Stage 2 |
| Layout notes | Include any deviation from the wild type virus detected in the database. |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_003 |
| Output File Name | rt-gn-bslgaganyontrtbysubtypes12.lst |
| Purpose | WK96S2 |
| Table No. | Table S.3.9.3N |
| Title 1 | Baseline Gag Deviations from Wild Type Virus |
| Title 2 | By HIV Subtype |
| Title 3 | Treated Subjects with On-Treatment Resistance Testing - Stage 1 and 2 |
| Layout notes | Include any deviation from the wild type virus detected in the database. |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_003 |
| Output File Name | rt-gn-bslgaganypdvfs1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.3.9.1O |
| Title 1 | Baseline Gag Deviations from Wild Type Virus |
| Title 2 | Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 1 |
| Footnote 1 | Protocol Defined Virologic Failure is defined by a subject meeting one of the following criteria: |
| Footnote 2 | 1) Confirmed > 1 log <sub>10</sub> c/mL increase in HIV-1 RNA at anytime above nadir level where nadir is ≥ 40 c/mL |
| Footnote 3 | 2) Confirmed HIV-1 RNA ≥ 40 c/mL if prior suppression to < 40 c/mL |
| Footnote 4 | 3) Failure to have the last on-treatment HIV-1 RNA to < 400 c/mL within Week 24, 48, or 96 week snapshot window |
| Footnote 5 | 4) Failure to achieve > 1 log <sub>10</sub> c/mL decrease in HIV-1 RNA by Week 8 |
| Layout notes | Include any deviation from the wild type virus detected in the database. |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_003 |
| Output File Name | rt-gn-bslgaganypdvfs2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.3.9.2O |
| Title 1 | Baseline Gag Deviations from Wild Type Virus |
| Title 2 | Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 2 |
| Footnote 1 | Protocol Defined Virologic Failure is defined by a subject meeting one of the following criteria: |
| Footnote 2 | 1) Confirmed > 1 log <sub>10</sub> c/mL increase in HIV-1 RNA at anytime above nadir level where nadir is ≥ 40 c/mL |

| Footnote 3 | 2) Confirmed HIV-1 RNA ≥ 40 c/mL if prior suppression to < 40 c/mL |
|---|---|
| Footnote 4 | 3) Failure to have the last on-treatment HIV-1 RNA to < 400 c/mL within Week 24, 48, or 96 week snapshot window |
| Footnote 5 | 4) Failure to achieve > 1 log <sub>10</sub> c/mL decrease in HIV-1 RNA by Week 8 |
| Layout notes | Include any deviation from the wild type virus detected in the database. |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_003 |
| Output File Name | rt-gn-bslgaganypdvfs12.lst |
| Purpose | WK96S2 |
| Table No. | Table S.3.9.3O |
| Title 1 | Baseline Gag Deviations from Wild Type Virus |
| Title 2 | Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 1 and 2 |
| Footnote 1 | Protocol Defined Virologic Failure is defined by a subject meeting one of the following criteria: |
| Footnote 2 | 1) Confirmed > 1 log <sub>10</sub> c/mL increase in HIV-1 RNA at anytime above nadir level where nadir is ≥ 40 c/mL |
| Footnote 3 | 2) Confirmed HIV-1 RNA ≥ 40 c/mL if prior suppression to < 40 c/mL |
| Footnote 4 | 3) Failure to have the last on-treatment HIV-1 RNA to < 400 c/mL within Week 24, 48, or 96 week snapshot window |
| Footnote 5 | 4) Failure to achieve > 1 log <sub>10</sub> c/mL decrease in HIV-1 RNA by Week 8 |
| Layout notes | Include any deviation from the wild type virus detected in the database. |

| Parameter | Values |
|------------------|----------------------------------------------|
| Template ID | SS_GN_T_003 |
| Output File Name | rt-gn-bslgaganypdvfbysubtypes1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.3.9.1P |
| Title 1 | Baseline Gag Deviations from Wild Type Virus |

| Title 2 | By HIV Subtype |
|---|---|
| Title 3 | Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 1 |
| Footnote 1 | Protocol Defined Virologic Failure is defined by a subject meeting one of the following criteria: |
| Footnote 2 | 1) Confirmed > 1 log <sub>10</sub> c/mL increase in HIV-1 RNA at anytime above nadir level where nadir is ≥ 40 c/mL |
| Footnote 3 | 2) Confirmed HIV-1 RNA ≥ 40 c/mL if prior suppression to < 40 c/mL |
| Footnote 4 | 3) Failure to have the last on-treatment HIV-1 RNA to < 400 c/mL within Week 24, 48, or 96 week snapshot window |
| Footnote 5 | 4) Failure to achieve > 1 log <sub>10</sub> c/mL decrease in HIV-1 RNA by Week 8 |
| Layout notes | Include any deviation from the wild type virus detected in the database. |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_003 |
| Output File Name | rt-gn-bslgaganypdvfbysubtypes2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.3.9.2P |
| Title 1 | Baseline Gag Deviations from Wild Type Virus |
| Title 2 | By HIV Subtype |
| Title 3 | Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 2 |
| Footnote 1 | Protocol Defined Virologic Failure is defined by a subject meeting one of the following criteria: |
| Footnote 2 | 1) Confirmed > 1 log <sub>10</sub> c/mL increase in HIV-1 RNA at anytime above nadir level where nadir is ≥ 40 c/mL |
| Footnote 3 | 2) Confirmed HIV-1 RNA ≥ 40 c/mL if prior suppression to < 40 c/mL |
| Footnote 4 | 3) Failure to have the last on-treatment HIV-1 RNA to < 400 c/mL within Week 24, 48, or 96 week snapshot window |
| Footnote 5 | 4) Failure to achieve > 1 log <sub>10</sub> c/mL decrease in HIV-1 RNA by Week 8 |
| Layout notes | Include any deviation from the wild type virus detected in the database. |

| Parameter | Values |
|-----------|--------|
|-----------|--------|

| Template ID | SS_GN_T_003 |
|---|---|
| Output File Name | rt-gn-bslgaganypdvfbysubtypes12.lst |
| Purpose | WK96S2 |
| Table No. | Table S.3.9.3P |
| Title 1 | Baseline Gag Deviations from Wild Type Virus |
| Title 2 | By HIV Subtype |
| Title 3 | Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 1 and 2 |
| Footnote 1 | Protocol Defined Virologic Failure is defined by a subject meeting one of the following criteria: |
| Footnote 2 | 1) Confirmed > 1 log <sub>10</sub> c/mL increase in HIV-1 RNA at anytime above nadir level where nadir is ≥ 40 c/mL |
| Footnote 3 | 2) Confirmed HIV-1 RNA ≥ 40 c/mL if prior suppression to < 40 c/mL |
| Footnote 4 | 3) Failure to have the last on-treatment HIV-1 RNA to < 400 c/mL within Week 24, 48, or 96 week snapshot window |
| Footnote 5 | 4) Failure to achieve > 1 log <sub>10</sub> c/mL decrease in HIV-1 RNA by Week 8 |
| Layout notes | Include any deviation from the wild type virus detected in the database. |

## Template SS\_GN\_L\_002: Gag Listing for Selected Positions

| Subject ID<br>(Age/Gender/Race)<br>Treatment Group | HIV<br>Subtype | Current Treatment | Period<br>Visit<br>Date<br>Study Day | Position 362 | Position 364 | Position 369 | Position 370 |
|---|---|---|---|---|---|---|---|
| PPD<br>(54/F/C)<br>ATV/r/RAL/TDF | В | PRE-TREATMENT | PRE-TREATMEN<br>SC<br>PPD | T xxx<br>-42 | xxx | xxx | xxx |
| | | ATV300mg QD+RTV100mg QD+<br>RAL400mg BID+TDF300mg QD | STAGE 1<br>WE<br>PPD | xxx<br>119 | xxx | xxx | xxx |
| PPD<br>(62/M/C)<br>ATV/r/RAL/TDF | С | PRE-TREATMENT | PRE-TREATMEN<br>SCREENING<br>PPD | T xxx<br>-38 | xxx | xxx | xxx |

\_\_\_\_\_

| Parameter | Values |
|---|---|
| Template ID | SS_GN_L_002 |
| Output File Name | rl-gn-gagbsls1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Appendix 3.9.1C |
| Title 1 | Listing of Baseline Gag Polymorphisms at Selected Positions |
| Title 2 | Treated Subjects - Stage 1 |
| Programming notes | Please include only the pre-treatment assessments. |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_L_002 |
| Output File Name | rl-gn-gagbsls2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Appendix 3.9.2C |
| Title 1 | Listing of Baseline Gag Polymorphisms at Selected Positions |
| Title 2 | Treated Subjects - Stage 2 |
| Programming notes | Please include only the pre-treatment assessments. |

Template SS\_GN\_L\_003: Gag Listing of Deviations from the Wild Type Virus

| Subject ID<br>(Age/Gender/Race)<br>Treatment Group | HIV<br>Subtype | Current Treatment | Period<br>Visit<br>Date<br>Study Day | Deviations |
|---|---|---|---|---|
| PPD<br>(54/F/C)<br>ATV/r/RAL/TDF | С | PRE-TREATMENT | PRE-TREATMENT<br>SC<br>PPD<br>-42 | xxx, xxx, xxx, xxx |
| | | ATV300mg QD+RTV100mg QD+<br>RAL400mg BID+TDF300mg QD | STAGE 1<br>WEEK 16<br>PPD 119 | xxx, xxx, xxx, xxx |
| PPD<br>(62/M/C)<br>ATV/r/RAL/TDF | В | PRE-TREATMENT | PRE-TREATMENT SC PPD -38 | XXX |

| Parameter | Values |
|-------------------|---------------------------------------------------------|
| Template ID | SS_GN_L_003 |
| Output File Name | rl-gn-gagbslanys1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Appendix 3.9.1D |
| Title 1 | Listing of Baseline Gag Deviations from Wild Type Virus |
| Title 2 | Treated Subjects - Stage 1 |
| Programming notes | Please include only the pre-treatment assessments. |

| Parameter | Values |
|-------------------|---------------------------------------------------------|
| Template ID | SS_GN_L_003 |
| Output File Name | rl-gn-gagbslanys2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Appendix 3.9.2D |
| Title 1 | Listing of Baseline Gag Deviations from Wild Type Virus |
| Title 2 | Treated Subjects - Stage 2 |
| Programming notes | Please include only the pre-treatment assessments. |

Template SS\_PN\_T\_001: Baseline Phenotypic Resistance Categories

| | Group A<br>N = XX | Group B<br>N = XX | Group C<br>N = XX | Group D<br>N=XX |
|---|---|---|---|---|
| PHENOTYPIC TESTING AT BASELINE | XX/XX (XX.X) | XX/XX (XX.X) | XX/XX (XX.X) | XX/XX (XX.X) |
| PHENOTYPABLE | XX/XX (XX.X) | XX/XX (XX.X) | XX/XX (XX.X) | XX/XX (XX.X) |
| RESISTANCE CATEGORY NO RESISTANCE TO DRUGS IN ANY CLASS 21 NRTI 21 NRTI 21 PI 21 INI (21 NRTI) AND (21 NNRTI) (21 NRTI) AND (21 PI) (21 NRTI) AND (21 INI) (21 NNRTI) AND (21 INI) (21 NNRTI) AND (21 INI) (21 NNRTI) AND (21 INI) (21 NNRTI) AND (21 INI) (21 NNRTI) AND (21 INI) (21 NRTI) AND (21 INI) (21 NRTI) AND (21 NNRTI) AND (21 PI) (21 NRTI) AND (21 NNRTI) AND (21 INI) (21 NRTI) AND (21 PI) AND (21 INI) (21 NNRTI) AND (21 PI) AND (21 INI) (21 NNRTI) AND (21 PI) AND (21 INI) | XX/XX (XX.X) | XX/XX (XX.X) | XX/XX (XX.X) | XX/XX (XX.X) |

-----

| Parameter | Values |
|------------------|-------------------------------------------|
| Template ID | SS_PN_T_001 |
| Output File Name | rt-pn-bsls1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.3.9.1F |
| Title 1 | Baseline Phenotypic Resistance Categories |
| Title 2 | Treated Subjects - Stage 1 |

| Parameter | Values |
|-----------|--------|
|-----------|--------|

| Template ID | SS_PN_T_001 |
|------------------|-------------------------------------------|
| Output File Name | rt-pn-bsls2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.3.9.2F |
| Title 1 | Baseline Phenotypic Resistance Categories |
| Title 2 | Treated Subjects - Stage 2 |

| Parameter | Values |
|------------------|-------------------------------------------|
| Template ID | SS_PN_T_001 |
| Output File Name | rt-pn-bsls12.lst |
| Purpose | WK96S2 |
| Table No. | Table S.3.9.3F |
| Title 1 | Baseline Phenotypic Resistance Categories |
| Title 2 | Treated Subjects - Stage 1 and 2 |

| Parameter | Values |
|---|---|
| Template ID | SS_PN_T_001 |
| Output File Name | rt-pn-bslots1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.3.9.1G |
| Title 1 | Baseline Phenotypic Resistance Categories |
| Title 2 | Treated Subjects with On-Treatment Resistance Testing - Stage 1 |

| Parameter | Values |
|-------------|-------------|
| Template ID | SS_PN_T_001 |

| Output File Name | rt-pn-bslots2.lst |
|---|---|
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.3.9.2G |
| Title 1 | Baseline Phenotypic Resistance Categories |
| Title 2 | Treated Subjects with On-Treatment Resistance Testing - Stage 2 |

| Parameter | Values |
|---|---|
| Template ID | SS_PN_T_001 |
| Output File Name | rt-pn-bslots12.lst |
| Purpose | WK96S2 |
| Table No. | Table S.3.9.3G |
| Title 1 | Baseline Phenotypic Resistance Categories |
| Title 2 | Treated Subjects with On-Treatment Resistance Testing - Stage 1 and 2 |

| Parameter | Values |
|---|---|
| Template ID | SS_PN_T_001 |
| Output File Name | rt-pn-bslpdvfs1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.3.9.1Q |
| Title 1 | Baseline Phenotypic Resistance Categories |
| Title 2 | Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 1 |
| Footnote 1 | Protocol Defined Virologic Failure is defined by a subject meeting one of the following criteria: |
| Footnote 2 | 1) Confirmed > 1 log <sub>10</sub> c/mL increase in HIV-1 RNA at anytime above nadir level where nadir is ≥ 40 c/mL |
| Footnote 3 | 2) Confirmed HIV-1 RNA ≥ 40 c/mL if prior suppression to < 40 c/mL |
| Footnote 4 | 3) Failure to have the last on-treatment HIV-1 RNA to < 400 c/mL within Week 24, 48, or 96 week snapshot window |

| Footnote 5 4) Failure to achieve > 1 log <sub>10</sub> c/mL decrease in HIV-1 RNA by Week 8 |
|---|
|---|

| Parameter | Values |
|---|---|
| Template ID | N_T_001 |
| Output File Name | n-bslpdvfs2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.3.9.2Q |
| Title 1 | eline Phenotypic Resistance Categories |
| Title 2 | Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 2 |
| Footnote 1 | Protocol Defined Virologic Failure is defined by a subject meeting one of the following criteria: |
| Footnote 2 | 1) Confirmed > 1 log <sub>10</sub> c/mL increase in HIV-1 RNA at anytime above nadir level where nadir is ≥ 40 c/mL |
| Footnote 3 | 2) Confirmed HIV-1 RNA ≥ 40 c/mL if prior suppression to < 40 c/mL |
| Footnote 4 | 3) Failure to have the last on-treatment HIV-1 RNA to < 400 c/mL within Week 24, 48, or 96 week snapshot window |
| Footnote 5 | 4) Failure to achieve > 1 log <sub>10</sub> c/mL decrease in HIV-1 RNA by Week 8 |

| Parameter | Values |
|---|---|
| Template ID | SS_PN_T_001 |
| Output File Name | rt-pn-bslpdvfs12.lst |
| Purpose | WK96S2 |
| Table No. | Table S.3.9.3Q |
| Title 1 | Baseline Phenotypic Resistance Categories |
| Title 2 | Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 1 and 2 |
| Footnote 1 | Protocol Defined Virologic Failure is defined by a subject meeting one of the following criteria: |
| Footnote 2 | 1) Confirmed > 1 log <sub>10</sub> c/mL increase in HIV-1 RNA at anytime above nadir level where nadir is ≥ 40 c/mL |
| Footnote 3 | 2) Confirmed HIV-1 RNA ≥ 40 c/mL if prior suppression to < 40 c/mL |

| Footnote 4 | 3) Failure to have the last on-treatment HIV-1 RNA to < 400 c/mL within Week 24, 48, or 96 week snapshot window |
|---|---|
| Footnote 5 | 4) Failure to achieve > 1 log <sub>10</sub> c/mL decrease in HIV-1 RNA by Week 8 |

Template SS\_PN\_T\_002: Phenotypic Resistance by Class and Drug Name

| | TRT A N = 10 | TRT B<br>N = 15 | TRT C<br>N = 14 | TRT D<br>N = 15 | TRT E<br>N = 11 |
|---|---|---|---|---|---|
| PHENOTYPIC TESTING PHENOTYPABLE | | | 14/14 (100.0)<br>14/14 (100.0) | | |
| PHENOTYPE | | 0/14 | 1/14 ( 7.1) | 2/15 ( 13.3)<br>0/15<br>0/15<br>1/15 ( 6.7)<br>0/15<br>0/15<br>0/15<br>0/15<br>0/15<br>1/15 ( 6.7)<br>0/15<br>1/15 ( 6.7) | 0/11 |
| NNRTI<br>DLV<br>EFV<br>ETR<br>NVP | 1/9 ( 11.1)<br>1/9 ( 11.1)<br>1/9 ( 11.1)<br>0/9<br>1/9 ( 11.1) | 1/14 ( 7.1) | 0/14 | 0/15<br>0/15<br>0/15 | 1/11 ( 9.1)<br>1/11 ( 9.1)<br>0/11 |
| NRTI 3TC ABC D4T DDI FTC TFV ZDV | 1/9 ( 11.1)<br>0/9<br>0/9<br>0/9<br>0/9<br>0/9<br>1/9 ( 11.1)<br>1/9 ( 11.1) | 0/14<br>0/14<br>0/14<br>1/14 ( 7.1)<br>0/14 | 0/14<br>0/14<br>0/14<br>1/14 ( 7.1) | 0/15<br>0/15<br>0/15<br>0/15<br>0/15<br>0/15 | 0/11<br>0/11<br>0/11<br>0/11<br>0/11 |

Program Source: /projects/bms208451/stats/primary/prog/tables/rt-pn-new.sas

13MAR2015:05:25:28

| Parameter | Values |
|------------------|-------------------------------------------------------|
| Template ID | SS_PN_T_002 |
| Output File Name | rt-pn-bsldrugs1.lst |
| Purpose | VK24S1, WK48S1 WK96S1, WK96S2 |
| Table No. | Table S.3.9.1H |
| Title 1 | Baseline Phenotypic Resistance by Class and Drug Name |
| Title 2 | Treated Subjects - Stage 1 |

| Parameter | Values |
|------------------|-------------------------------------------------------|
| Template ID | SS_PN_T_002 |
| Output File Name | rt-pn-bsldrugs2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.3.9.2H |
| Title 1 | Baseline Phenotypic Resistance by Class and Drug Name |
| Title 2 | Treated Subjects - Stage 2 |

| Parameter | Values |
|------------------|-------------------------------------------------------|
| Template ID | SS_PN_T_002 |
| Output File Name | rt-pn-bsldrugs12.lst |
| Purpose | WK96S2 |
| Table No. | Table S.3.9.3H |
| Title 1 | Baseline Phenotypic Resistance by Class and Drug Name |
| Title 2 | Treated Subjects - Stage 1 and 2 |

| Template ID | SS_PN_T_002 |
|---|---|
| Output File Name | rt-pn-bslotrtdrugs1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.3.9.1I |
| Title 1 | Baseline Phenotypic Resistance by Class and Drug Name |
| Title 2 | Treated Subjects with On-Treatment Phenotypic Resistance Testing - Stage 1 |

| Parameter | Values |
|---|---|
| Template ID | SS_PN_T_002 |
| Output File Name | rt-pn-bslotrtdrugs2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.3.9.2I |
| Title 1 | Baseline Phenotypic Resistance by Class and Drug Name |
| Title 2 | Treated Subjects with On-Treatment Phenotypic Resistance Testing - Stage 2 |

| Parameter | Values |
|---|---|
| Template ID | SS_PN_T_002 |
| Output File Name | rt-pn-bslotrtdrugs12.lst |
| Purpose | WK96S2 |
| Table No. | Table S.3.9.3I |
| Title 1 | Baseline Phenotypic Resistance by Class and Drug Name |
| Title 2 | Treated Subjects with On-Treatment Phenotypic Resistance Testing - Stage 1 and 2 |

| Parameter | Values |
|-------------|-------------|
| Template ID | SS_PN_T_002 |
| Output File Name | rt-pn-bsldrugpdvfs1.lst |
|---|---|
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.3.9.1R |
| Title 1 | Baseline Phenotypic Resistance by Class and Drug Name |
| Title 2 | Treated Subjects with On-Treatment Phenotypic Resistance Testing |
| Title 3 | Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 1 |
| Footnote 1 | Protocol Defined Virologic Failure is defined by a subject meeting one of the following criteria: |
| Footnote 2 | 1) Confirmed > 1 log <sub>10</sub> c/mL increase in HIV-1 RNA at anytime above nadir level where nadir is ≥ 40 c/mL |
| Footnote 3 | 2) Confirmed HIV-1 RNA ≥ 40 c/mL if prior suppression to < 40 c/mL |
| Footnote 4 | 3) Failure to have the last on-treatment HIV-1 RNA to < 400 c/mL within Week 24, 48, or 96 week snapshot window |
| Footnote 5 | 4) Failure to achieve > 1 log <sub>10</sub> c/mL decrease in HIV-1 RNA by Week 8 |

| Parameter | Values |
|---|---|
| Template ID | SS_PN_T_002 |
| Output File Name | rt-pn-bsldrugpdvfs2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.3.9.2R |
| Title 1 | Baseline Phenotypic Resistance by Class and Drug Name |
| Title 2 | Treated Subjects with On-Treatment Phenotypic Resistance Testing |
| Title 3 | Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 2 |
| Footnote 1 | Protocol Defined Virologic Failure is defined by a subject meeting one of the following criteria: |
| Footnote 2 | 1) Confirmed > 1 log <sub>10</sub> c/mL increase in HIV-1 RNA at anytime above nadir level where nadir is ≥ 40 c/mL |
| Footnote 3 | 2) Confirmed HIV-1 RNA ≥ 40 c/mL if prior suppression to < 40 c/mL |
| Footnote 4 | 3) Failure to have the last on-treatment HIV-1 RNA to < 400 c/mL within Week 24, 48, or 96 week snapshot window |
| Footnote 5 | 4) Failure to achieve > 1 log <sub>10</sub> c/mL decrease in HIV-1 RNA by Week 8 |

| Parameter | Values |
|---|---|
| Template ID | SS_PN_T_002 |
| Output File Name | rt-pn-bsldrugpdvfs12.lst |
| Purpose | WK96S2 |
| Table No. | Table S.3.9.3R |
| Title 1 | Baseline Phenotypic Resistance by Class and Drug Name |
| Title 2 | Treated Subjects with On-Treatment Phenotypic Resistance Testing |
| Title 3 | Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 1 and 2 |
| Footnote 1 | Protocol Defined Virologic Failure is defined by a subject meeting one of the following criteria: |
| Footnote 2 | 1) Confirmed > 1 log <sub>10</sub> c/mL increase in HIV-1 RNA at anytime above nadir level where nadir is ≥ 40 c/mL |
| Footnote 3 | 2) Confirmed HIV-1 RNA ≥ 40 c/mL if prior suppression to < 40 c/mL |
| Footnote 4 | 3) Failure to have the last on-treatment HIV-1 RNA to < 400 c/mL within Week 24, 48, or 96 week snapshot window |
| Footnote 5 | 4) Failure to achieve > 1 log <sub>10</sub> c/mL decrease in HIV-1 RNA by Week 8 |

# Template SS\_PN\_L\_001: Phenotypic Resistance Listing

| Subject ID | Current<br>Treatment/ | | BMS-955176 | RT | | PI | RAL |
|---|---|---|---|---|---|---|---|
| (Age/Gender/Race) Treatment Group | Period/<br>Visit | Date/<br>Study Day | IC50/ IC50<br>Susc Fold Change | | )/ IC50<br>l Change Susc | IC50/ IC50<br>Fold Change Susc | IC50/ IC50<br>Fold Change |
| PPD (43/M/B) BMS-663068 1200 mg QD/ RAL/TDF | PRE-TREATMENT/<br>PRE-TREATMENT/<br>SCREENING | PPD -42 | 0.00017/0.13 | 3TC (S) 3.79 ABC (S) 0.7/ D4T (S) 0.66 DDI (S) 7.52 FTC (S) 1.13 TFV (S) 0.99 ZDW (S) 0.02 DLV (S) 0.04 EFV (S) 0.00 ETR (S) 0.00 NVP (S) 0.13 | '0.95 ATV (S) 5/1.06 ATV/R (S) 2/1.04 DRV/R (S) 3/1.32 IDV/R (S) 6/0.92 LPV/R (S) 29/1.21 NFV (S) 151/1.63 RTV (S) 054/1.24 SQV/R (S) 028/1.39 TPV/R (S) | | 0.00762/0.88 |
| | BMS1200mg QD+<br>RAL400mg BID+<br>TDF300mg QD/<br>STAGE 1/<br>WEEK 4 | <b>PPD</b> 35 | NR/ | EFV (S) 0.00 | 8/1.04 ATV (S)<br>7/1.06 ATV/R (S)<br>8/1.12 DRV/R (S)<br>7/1.26 IDV/R (S)<br>17/1.60 NFV (S)<br>196/1.94 RTV (S)<br>1963/1.50 SQV/R (S)<br>19326/1.55 TPV/R (P) | 0.00414/1.66<br>0.00414/1.66<br>0.00142/1.55<br>0.0119/1.63<br>0.0068/1.25<br>0.0281/2.83<br>0.046/1.97<br>0.0068/1.60 | 0.02064/1.33 |

| Parameter | Values |
|------------------|-------------------------------------------|
| Template ID | SS_PN_L_001 |
| Output File Name | rl-pn-bsls1.lst |
| Purpose | WK24S1, WK48S1 WK96S1, WK96S2 |
| Table No. | Appendix 3.9.1E |
| Title 1 | Listing of Baseline Phenotypic Resistance |
| Title 2 | Treated Subjects - Stage 1 |
| Footnote 1 | Susc = Susceptibility |

| Footnote 2 | P = Partial, R = Resistance, S = Susceptible |
|-------------------|----------------------------------------------------|
| Programming notes | Please include only the pre-treatment assessments. |

| Parameter | Values |
|-------------------|----------------------------------------------------|
| Template ID | SS_PN_L_001 |
| Output File Name | rl-pn-bsls2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Appendix 3.9.2E |
| Title 1 | Listing of Baseline Phenotypic Resistance |
| Title 2 | Treated Subjects - Stage 2 |
| Footnote 1 | Susc = Susceptibility |
| Footnote 2 | P = Partial, R = Resistance, S = Susceptible |
| Programming notes | Please include only the pre-treatment assessments. |

#### Template GS\_LB\_T\_X\_004: Laboratory Toxicity Grade Summary

 Draft

Protocol: BMS234303 Laboratory Test Results Summary of Worst Toxicity Grade All Treated Subjects

| Lab Test Description | Group 1 | Group 2 | Group 3 | Group 4 | Total |
|---|---|---|---|---|---|
| Toxicity Grade | N = 83 | N = 50 | N = 50 | N = 25 | N = 208 |
| BLOOD UREA NITROGEN CRITERION 1 CRITERION 2 NOT REPORTED | 71 ( 85.5) | 10 ( 20.0) | 0 | 0 | 81 (38.9) |
| | 7 ( 8.4) | 5 ( 10.0) | 0 | 0 | 12 (5.8) |
| | 5 ( 0.6) | 35 ( 70.0) | 50 (100.0) | 25 (100.0) | 115 (55.3) |
| LDL-C/HDL-C RATIO (DIRECT) CRITERION 1 CRITERION 2 NOT REPORTED | 33 ( 39.8) | 20 ( 40.0) | 0 | 0 | 53 ( 25.5) |
| | 39 ( 47.0) | 20 ( 40.0) | 0 | 0 | 59 ( 28.4) |
| | 11 ( 13.3) | 10 ( 20.0) | 50 (100.0) | 25 (100.0) | 96 ( 46.1) |
| TOTAL PROTEIN CRITERION 1 CRITERION 2 NOT REPORTED | 75 ( 90.4) | 0 | 10 ( 20.0) | 0 | 85 ( 40.9) |
| | 3 ( 3.6) | 0 | 2 ( 4.0) | 0 | 5 ( 2.4) |
| | 5 ( 0.6) | 50 (100.0) | 38 ( 76.0) | 25 (100.0) | 118 ( 56.7) |
| CHLORIDE CRITERION 1 CRITERION 2 NOT REPORTED | 74 ( 89.2) | 0 | 0 | 20 ( 80.0) | 94 ( 45.2) |
| | 4 ( 4.8) | 0 | 0 | 2 ( 8.0) | 6 ( 2.9) |
| | 5 ( 0.6) | 50 (100.0) | 50 (100.0) | 3 ( 12.0) | 108 ( 51.9) |

Toxicity Scale: Descriptive text of toxicity scale Program Source: /wwbdm/ndp/prime/gssr/devtest/lab/test/labsum.b.sas

07SEP2004:14:35:00

| Parameter | Values |
|---|---|
| Template ID | GS_LB_T_X_004 |
| Output File Name | rt-lb-bsltoxs1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.3.5.1 |
| Title 1 | Baseline Laboratory Test Results Summary of Toxicity Grade |
| Title 2 | Treated Subjects - Stage 1 |

| Footnote 1 | Toxicity Scale: DAIDS |
|---|---|
| Programming notes | The laboratory tests to be included in this output are specified in the SAP. |

| Parameter | Values |
|---|---|
| Template ID | GS_LB_T_X_004 |
| Output File Name | rt-lb-bsltoxs2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.3.5.2 |
| Title 1 | Baseline Laboratory Test Results Summary of Toxicity Grade |
| Title 2 | Treated Subjects - Stage 2 |
| Footnote 1 | Toxicity Scale: DAIDS |
| Programming notes | The laboratory tests to be included in this output are specified in the SAP. |

#### Template GS\_AE\_T\_X\_001: Adverse Event Summary by System Organ Class and Preferred Term

Protocol: CV131154 Confidential Page 1 of 21
Adverse Event Summary
All Treated Subjects

| System Organ Class (%) Preferred Term (%) | TRT A<br>N = 200 | TRT B<br>N = 959 | TRT C<br>N = 482 | Total<br>N = 1641 |
|---|---|---|---|---|
| TOTAL SUBJECTS WITH AN EVENT | 100 ( 50.0) | 866 ( 90.3) | 417 ( 86.5) | 1383 ( 89.0) |
| BLOOD AND LYMPHATIC SYSTEM DISORDERS ANAEMIA LEUKOPENIA EOSINOPHILIA LYMPHADENOPATHY LEUKOCYTOSIS THROMBOCYTOPENIA IRON DEFICIENCY ANAEMIA BONE MARROW TOXICITY ANAEMIA FOLATE DEFICIENCY ANAEMIA OF CHRONIC DISEASE BASOPHILIA BONE MARROW DEPRESSION LYMPH NODE PAIN MONOCYTOSIS NEUTROPENIA THROMBOCYTHAEMIA | 6 ( 3.0)<br>0<br>0<br>0<br>0<br>4 ( 2.0)<br>0<br>0<br>0<br>0<br>0<br>0<br>0 | 51 ( 5.3)<br>17 ( 1.8)<br>17 ( 1.8)<br>5 ( 0.5)<br>0<br>1 ( 0.1)<br>4 ( 0.4)<br>2 ( 0.2)<br>1 ( 0.1) | 39 ( 8.1) 16 ( 3.3) 5 ( 1.0) 3 ( 0.6) 7 ( 1.5) 5 ( 1.0) 1 ( 0.2) 1 ( 0.2) 0 0 0 0 1 ( 0.2) 0 0 | 96 ( 5.9) 33 ( 2.3) 22 ( 1.5) 8 ( 0.6) 7 ( 0.5) 6 ( 0.4) 9 ( 0.5) 3 ( 0.2) 2 ( 0.1) 1 ( <0.1) |
| CARDIAC DISORDERS PALPITATIONS TACHYCARDIA CARDIAC FAILURE CONGESTIVE BRADYCARDIA SINUS BRADYCARDIA ARRHYTHMIA ATRIAL FIBRILLATION | 10 ( 5.0)<br>0<br>5 ( 2.5)<br>5 ( 2.5)<br>0<br>0<br>0 | 54 ( 5.6)<br>21 ( 2.2)<br>13 ( 1.4)<br>3 ( 0.3)<br>4 ( 0.4)<br>1 ( 0.1)<br>1 ( 0.1)<br>2 ( 0.2) | 36 ( 7.5)<br>8 ( 1.7)<br>4 ( 0.8)<br>3 ( 0.6)<br>1 ( 0.2)<br>4 ( 0.8)<br>3 ( 0.6)<br>2 ( 0.4) | 100 ( 6.1)<br>29 ( 2.0)<br>22 ( 1.3)<br>11 ( 0.7)<br>5 ( 0.3)<br>5 ( 0.3)<br>4 ( 0.3)<br>4 ( 0.3) |
| UNASSIGNED<br>UNASSIGNED | 1 ( 0.5)<br>1 ( 0.5) | 0 | 0 | 1 ( <0.1)<br>1 ( <0.1) |

MedDRA Version: 7.1

Program Source: /wwbdm/ndp/prime/msr/devtest/test/sample1.sas

18FEB2005:10:59:00

| Parameter | Values |
|------------------|--------------------------------|
| Template ID | GS_AE_T_X_001 |
| Output File Name | rt-ae-preaidss1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.3.6.1 |
| Title 1 | Adverse Events Summary |
| Title 2 | Pre-treatment AIDS Events |
| Title 3 | Treated Subjects - Stage 1 |
| Footnote 1 | MedDRA Version x.x |

| Parameter | Values |
|------------------|----------------------------|
| Template ID | GS_AE_T_X_001 |
| Output File Name | rt-ae-preaidss2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.3.6.2 |
| Title 1 | Adverse Events Summary |
| Title 2 | Pre-treatment AIDS Events |
| Title 3 | Treated Subjects - Stage 2 |

# 4.3.3 Medical History and Previous Treatments

#### Template GS\_MH\_T\_X\_001: Medical History Summary

Protocol: TA001001 Draft General Medical History Summary All Treated Subjects 

| | TRT A<br>N = 16 | TRT B<br>N = 17 | TRT C<br>N = 17 | Total<br>N = 50 |
|---|---|---|---|---|
| SUBJECTS WITH ABNORMAL MEDICAL HISTORY (%) | 16 (100.0) | 16 ( 94.1) | 16 ( 94.1) | 48 ( 96.0) |
| BODY SYSTEM (%) HEAD, EYES, EARS, NOSE, THROAT CARDIOVASCULAR PERIPHERAL VASCULAR RESPIRATORY GASTROINTESTINAL HEPATOBILIARY RENAL GENITOURINARY ENDOCRINE-METABOLIC HEMATOLOGIC-LYMPHATIC MUSCULOSKELETAL DERMATOLOGIC NEUROLOGIC PSYCHIATRIC ALLERGIES NEOPLASIA ALCOHOL USE TOBACCO USE DRUG ABUSE OTHER | 12 ( 75.0) 3 ( 18.8) 0 2 ( 12.5) 6 ( 37.5) 2 ( 12.5) 2 ( 12.5) 6 ( 37.5) 16 (100.0) 0 11 ( 68.8) 4 ( 25.0) 8 ( 50.0) 3 ( 18.8) 3 ( 18.8) 1 ( 6.3) 9 ( 56.3) 4 ( 25.0) 0 2 ( 12.5) | 11 (64.7) 5 (29.4) 3 (17.6) 1 (5.9) 5 (29.4) 0 7 (41.2) 16 (94.1) 1 (5.9) 10 (58.8) 6 (35.3) 5 (29.4) 2 (11.8) 3 (17.6) 0 4 (23.5) 6 (35.3) 0 3 (17.6) | 10 ( 58.8) 4 ( 23.5) 0 1 ( 5.9) 5 ( 29.4) 1 ( 5.9) 1 ( 5.9) 6 ( 35.3) 16 ( 94.1) 0 9 ( 52.9) 4 ( 23.5) 6 ( 35.3) 3 ( 17.6) 3 ( 17.6) 0 8 ( 47.1) 5 ( 29.4) 0 2 ( 11.8) | 33 ( 66.0)<br>12 ( 24.0)<br>3 ( 6.0)<br>4 ( 8.0)<br>16 ( 32.0)<br>3 ( 6.0)<br>19 ( 38.0)<br>48 ( 96.0)<br>1 ( 2.0)<br>30 ( 60.0)<br>14 ( 28.0)<br>19 ( 38.0)<br>8 ( 16.0)<br>9 ( 18.0)<br>1 ( 2.0)<br>21 ( 42.0)<br>15 ( 30.0)<br>0 |

| Parameter | Values |
|------------------|---------------------------------|
| Template ID | GS_MH_T_X_001 |
| Output File Name | rt-mh-sums1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.3.7.1 |
| Title 1 | General Medical History Summary |
| Title 2 | Treated Subjects - Stage 1 |

| Parameter | Values |
|------------------|---------------------------------|
| Template ID | GS_MH_T_X_001 |
| Output File Name | rt-mh-sums2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.3.7.2 |
| Title 1 | General Medical History Summary |
| Title 2 | Treated Subjects - Stage 2 |

#### Template GS\_MH\_L\_X\_001: Medical History Listing by Treatment Group

Protocol: CV131148 Protocol Draft Page 1 of 100

General Medical History All Treated Subjects

Treatment Group: TRT A

(83/F/C)

Subject ID
(Age/Gender/Race) System Condition(s)

PPD HEAD, EARS, EYES, NOSE, THROAT CEREBRO VASCULAR

(79/M/C) CARDÍOVASCÚLAR SEE PREVIOUS PAGE
PERIPHERAL VASCULAR PERIPHERAL PULSATIONS NOT PALPABLE

RESPIRATORY NULOL COPD

GASTROINTESTINAL GASTRIC , ULCER - ANAL BLEEDING - RECTUM POLYP & RESECTION

ALLERGIES PENICILLINE

PPD CARDIOVASCULAR CHF

RESPIRATORY BRONCHITIS

GASTROINTESTINAL CHOLELITHIASIS WITH CHOLECYSECTOMY

MUSCULOSKELETAL ARTHROSIS - SPINAL STENOSIS

PSYCHIATRIC DEPRESSION

Program Source: /wwbdm/ndp/prime/gssr/devtest/mhx/test/mhx lst.sas 06APR2004:17:58:02

| Parameter | Values |
|------------------|--------------------------------|
| Template ID | GS_MH_L_X_001 |
| Output File Name | rl-mh-lists1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Appendix 3.7.1 |
| Title 1 | General Medical History |
| Title 2 | Treated Subjects - Stage 1 |

| Parameter | Values |
|------------------|------------------------|
| Template ID | GS_MH_L_X_001 |
| Output File Name | rl-mh-lists2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |

| Table No. | Appendix 3.7.2 |
|-----------|----------------------------|
| Title 1 | General Medical History |
| Title 2 | Treated Subjects - Stage 2 |

#### Template GS\_CM\_T\_X\_001 : Non-Study Medication Summary

Protocol: CV168006 Draft Page 1 of 58

Draft Non-Study Medication Summary Medication Category All Treated Subjects

| Anatomic Class (%) Therapeutic Class (%) Generic Name (%) | TRT A<br>N = 5443 | TRT B<br>N = 6443 | | Total<br>N = 19009 |
|---|---|---|---|---|
| TOTAL SUBJECTS USING MEDICATION | 6134 ( 95.2) | 6134 ( 95.2) | 5884 ( 96.1) | 19009 ( 95.6) |
| ALIMENTARY TRACT & METABOLISM | 431 ( 6.7) | 431 ( 6.7) | 425 ( 6.9) | 1287 ( 6.8) |
| ANABOLIC STEROID PRASTERONE | 0 | 0 | 1 ( <0.1)<br>1 ( <0.1) | 1 ( <0.1)<br>1 ( <0.1) |
| ANTACID ALOH/CACO/MGOH ALOH/MAGTRI ALOH/MGOH ALOH/MGOH ALOH/MGOH/OXETAC ANTACID CACO/FAMO/MGOH CALCIUM CARBONATE DIHYDROXYALUMINIUM SODIUM CARBINATE | 31 ( 0.5)<br>1 ( <0.1)<br>0<br>2 ( <0.1)<br>2 ( <0.1)<br>7 ( <0.1)<br>7 ( <0.1)<br>13 ( 0.2) | 31 ( 0.5)<br>1 ( <0.1)<br>0<br>2 ( <0.1)<br>1 ( <0.1)<br>7 ( 0.1)<br>1 ( <0.1)<br>13 ( 0.2)<br>0 | 46 ( 0.8)<br>0<br>1 ( <0.1)<br>3 ( <0.1)<br>0<br>11 ( 0.2)<br>1 ( <0.1)<br>22 ( 0.4)<br>6 ( 0.1) | 108 ( 0.6)<br>2 ( <0.1)<br>1 ( <0.1)<br>7 ( <0.1)<br>3 ( <0.1)<br>25 ( 0.1)<br>9 ( <0.1)<br>48 ( 0.3)<br>6 ( <0.1) |
| ANTIDIARRHEA/INTEST ANTIINFLAM<br>ANTIDIARRHEAL | 2 ( <0.1)<br>2 ( <0.1) | 2 (< 0.1)<br>2 (< 0.1) | 1 ( <0.1)<br>1 ( <0.1) | 5 ( <0.1)<br>5 ( <0.1) |
| ANTIDIARRHEAL MICROORGANISM<br>LACTOBACILLUS ACIDOPHILUS<br>SACCHAROMYCES BOULARDII | 5 ( <0.1)<br>4 ( <0.1)<br>1 ( <0.1) | 5 ( 0.1)<br>4 ( 0.1)<br>1 (< 0.1) | 3 ( <0.1)<br>3 ( <0.1)<br>0 | 13 ( 0.1)<br>11 ( 0.1)<br>2 ( <0.1) |
| UNASSIGNED<br>UNASSIGNED<br>UNASSIGNED | 2 ( <0.1)<br>1 ( <0.1)<br>1 ( <0.1) | 2 ( <0.1)<br>1 ( <0.1)<br>1 ( <0.1) | 2 ( <0.1)<br>0<br>2 ( <0.1) | 6 ( <0.1)<br>2 ( <0.1)<br>4 ( <0.1) |

Program Source: /wwbdm/ndp/prime/gssr/devtest/checkraw/cmtbl.sas 290CT2004:18:53:00

| Parameter | Values |
|------------------|--------------------------------|
| Template ID | GS_CM_T_X_001 |
| Output File Name | rt-cm-premeds1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |

| Table No. | Table S.3.8.1 |
|---|---|
| Title 1 | Non-Study Medication Summary |
| Title 2 | Previous Medication |
| Title 3 | Treated Subjects - Stage 1 |
| Footnote 1 | Previous medication is defined as any medication that was taken before the start of study medication. |

| Parameter | Values |
|---|---|
| Template ID | GS_CM_T_X_001 |
| Output File Name | rt-cm-premeds2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.3.8.2 |
| Title 1 | Non-Study Medication Summary |
| Title 2 | Previous Medication |
| Title 3 | Treated Subjects - Stage 2 |
| Footnote 1 | Previous medication is defined as any medication that was taken before the start of study medication. |

# 4.4 Extent Of Exposure

# 4.4.1 Study Therapy and Treatment Compliance

# Template SS\_EX\_T\_001: Extent of Exposure Summary

| | Group A<br>N = XX | Group B<br>N = XX | Group C<br>N = XX | Group D<br>N = XX |
|---|---|---|---|---|
| N | XX | XX | XX | XX |
| MEAN | XX.X | XX.X | XX.X | XX.X |
| MEDIAN<br>MINI MAY | XX.X | XX.X | XX.X | XX.X |
| MIN , MAX<br>Q1 , Q3 | XX.X , XX.X<br>XX.X , XX.X | XX.X , XX.X<br>XX.X , XX.X | XX.X , XX.X<br>XX.X , XX.X | XX.X , XX.X<br>XX.X , XX.X |
| STANDARD DEVIATION | XX.XX | XX.XX | XX.XX | XX.XX |
| MEAN DAILY DOSE (mg) | XXX.X | XXX.X | XXX.X | XXX.X |

| Parameter | Values |
|------------------|----------------------------------|
| Template ID | SS_EX_T_001 |
| Output File Name | rt-ex-bmss1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.4.1.1A |
| Title 1 | Extent of Exposure to BMS-955176 |
| Title 2 | Time on Therapy |
| Title 3 | Treated Subjects - Stage 1 |
| Layout notes | Include Mean Daily Dose |

| Parameter | Values |
|------------------|------------------------|
| Template ID | SS_EX_T_001 |
| Output File Name | rt-ex-bmss2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.4.1.2A |

| Title 1 | Extent of Exposure to BMS-955176 |
|--------------|----------------------------------|
| Title 2 | Time on Therapy |
| Title 3 | Treated Subjects - Stage 2 |
| Layout notes | Include Mean Daily Dose |

| Parameter | Values |
|------------------|---------------------------------|
| Template ID | SS_EX_T_001 |
| Output File Name | rt-ex-tdfs1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.4.1.1B |
| Title 1 | Extent of Exposure to Tenofovir |
| Title 2 | Time on Therapy |
| Title 3 | Treated Subjects - Stage 1 |
| Layout notes | Include Mean Daily Dose |

| Parameter | Values |
|------------------|---------------------------------|
| Template ID | SS_EX_T_001 |
| Output File Name | rt-ex-tdfs2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.4.1.2B |
| Title 1 | Extent of Exposure to Tenofovir |
| Title 2 | Time on Therapy |
| Title 3 | Treated Subjects - Stage 2 |
| Layout notes | Include Mean Daily Dose |

| Parameter | Values |
|------------------|----------------------------------|
| Template ID | SS_EX_T_001 |
| Output File Name | rt-ex-atvs1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.4.1.1C |
| Title 1 | Extent of Exposure to Atazanavir |
| Title 2 | Time on Therapy |
| Title 3 | Treated Subjects - Stage 1 |
| Layout notes | Include Mean Daily Dose |

| Parameter | Values |
|------------------|----------------------------------|
| Template ID | SS_EX_T_001 |
| Output File Name | rt-ex-atvs2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.4.1.2C |
| Title 1 | Extent of Exposure to Atazanavir |
| Title 2 | Time on Therapy |
| Title 3 | Treated Subjects - Stage 2 |
| Layout notes | Include Mean Daily Dose |

| Parameter | Values |
|------------------|--------------------------------|
| Template ID | SS_EX_T_001 |
| Output File Name | rt-ex-dtgs1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.4.1.1D |

| Title 1 | Extent of Exposure to Dolutegravir |
|--------------|------------------------------------|
| Title 2 | Time on Therapy |
| Title 3 | Treated Subjects - Stage 1 |
| Layout notes | Include Mean Daily Dose |

| Parameter | Values |
|------------------|------------------------------------|
| Template ID | SS_EX_T_001 |
| Output File Name | rt-ex-dtgs2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.4.1.2D |
| Title 1 | Extent of Exposure to Dolutegravir |
| Title 2 | Time on Therapy |
| Title 3 | Treated Subjects - Stage 2 |
| Layout notes | Include Mean Daily Dose |

| Parameter | Values |
|------------------|---------------------------------|
| Template ID | SS_EX_T_001 |
| Output File Name | rt-ex-rtvs1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.4.1.1E |
| Title 1 | Extent of Exposure to Ritonavir |
| Title 2 | Time on Therapy |
| Title 3 | Treated Subjects - Stage 1 |
| Layout notes | Include Mean Daily Dose |

| Parameter | Values |
|------------------|---------------------------------|
| Template ID | SS_EX_T_001 |
| Output File Name | rt-ex-rtvs2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.4.1.2E |
| Title 1 | Extent of Exposure to Ritonavir |
| Title 2 | Time on Therapy |
| Title 3 | Treated Subjects - Stage 2 |
| Layout notes | Include Mean Daily Dose |

| Parameter | Values |
|------------------|-----------------------------------------|
| Template ID | SS_EX_T_001 |
| Output File Name | rt-ex-regimens1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.4.1.1F |
| Title 1 | Extent of Exposure to Treatment Regimen |
| Title 2 | Time on Therapy |
| Title 3 | Treated Subjects - Stage 1 |
| Layout notes | Do not include Mean Daily Dose |

| Parameter | Values |
|------------------|------------------------|
| Template ID | SS_EX_T_001 |
| Output File Name | rt-ex-regimens2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.4.1.2F |

| Title 1 | xtent of Exposure to Treatment Regimen |
|--------------|----------------------------------------|
| Title 2 | Time on Therapy |
| Title 3 | Treated Subjects - Stage 2 |
| Layout notes | Do not include Mean Daily Dose |

| Parameter | Values |
|------------------|-----------------------------------------|
| Template ID | SS_EX_T_001 |
| Output File Name | rt-ex-regimens12.lst |
| Purpose | WK96S2 |
| Table No. | Table S.4.1.3F |
| Title 1 | Extent of Exposure to Treatment Regimen |
| Title 2 | Time on Therapy |
| Title 3 | Treated Subjects - Stage 1 and 2 |
| Layout notes | Do not include Mean Daily Dose |

| Parameter | Values |
|---|---|
| Template ID | SS_EX_T_001 |
| Output File Name | rt-ex-conts1.lst |
| Purpose | WK96S1, WK96S2 |
| Table No. | Table S.4.1.1G |
| Title 1 | Extent of Exposure to BMS-955176 after Switch to Continuation Dose |
| Title 2 | Time on Therapy |
| Title 3 | Treated Subjects who Switched to Continuation Dose - Stage 1 |
| Layout notes | Include Mean Daily Dose |

| Parameter | Values |
|---|---|
| Template ID | SS_EX_T_001 |
| Output File Name | rt-ex-conts2.lst |
| Purpose | WK96S2 |
| Table No. | Table S.4.1.2G |
| Title 1 | Extent of Exposure to BMS-955176 after Switch to Continuation Dose |
| Title 2 | Time on Therapy |
| Title 3 | Treated Subjects who Switched to Continuation Dose - Stage 2 |
| Layout notes | Include Mean Daily Dose |

Template GS\_EX\_G\_001: Kaplan-Meier Plot Grouped by Treatment with Censoring



Serious Events (incl. Deaths) up to 30 days post-trt included
Non-Serious events up to last day of treatement included. Symbols represent censored observatior
<Special Events> are based upon a predefined list of MEDDRA Preferred Terms.
Program Path: /home/banckenf/sgtest
Program Name: sgissue0005.sas 200CT2008:06:57:24

| Parameter | Values |
|------------------|-------------|
| Template ID | GS_EX_G_001 |
| Output File Name | rg-ex-kms1 |

| Purpose | K24S1, WK48S1, WK96S1, WK96S2 |
|---|---|
| Table No. | re S.4.1.1 |
| Title 1 | Time on Study Therapy |
| Title 2 | Treated Subjects - Stage 1 |
| Layout notes | Y-axis label: Proportion of Subjects on Study Therapy |
| | X-axis label: Time (Weeks) |

| Parameter | Values |
|---|---|
| Template ID | GS_EX_G_001 |
| Output File Name | rg-ex-kms2 |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Figure S.4.1.2 |
| Title 1 | Time on Study Therapy |
| Title 2 | Treated Subjects - Stage 2 |
| Layout notes | Y-axis label: Proportion of Subjects on Study Therapy X-axis label: Time (Weeks) |

Template SS\_EX\_T\_002: Time on Study Therapy Life Table

| Group A (N=194) | | | GROUP B (N=203) | | | GROUP C (N=201) | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Week (a) | n N | Proportion (%)<br># (95% CI) | n | N# | | ortion (%)<br>(95% CI) | n | N# | | ortion (%)<br>95% CI) |
| < 4<br>4 - < 8<br>8 - < 12<br>12 - < 16<br>16 - < 20<br>20 - < 24<br>24 - < 28<br>28 - < 32<br>32 - < 36<br>36 - < 40<br>40 - < 44<br>44 - < 48<br>48 - < 52<br>52 - < 56 | 0 19<br>0 18<br>0 18<br>0 18<br>1 18<br>1 18<br>1 18<br>1 18<br>1 18 | $ \begin{array}{cccccccccccccccccccccccccccccccccccc$ | 0<br>0<br>0<br>5<br>7<br>11<br>13<br>13<br>14<br>15 | 193<br>188<br>179<br>179<br>174<br>169<br>164<br>163<br>161 | 0.0<br>0.0<br>0.0<br>0.0<br>2.7<br>2.7<br>3.8<br>6.0<br>7.1<br>7.7<br>8.3<br>8.3 | (0.0-0.0)<br>(0.0-0.0)<br>(0.0-0.0)<br>(0.0-0.0)<br>(0.4-5.0)<br>(1.0-6.6)<br>(2.6-9.5)<br>(3.4-10.9)<br>(3.4-10.9)<br>(3.8-11.6)<br>(4.3-12.3) | 0<br>0<br>1<br>3<br>5<br>8<br>11<br>18<br>21<br>22<br>25<br>25<br>26<br>26 | 201<br>197<br>194<br>192<br>184<br>181<br>178<br>171<br>163<br>156<br>154<br>150 | 0.0<br>0.0<br>0.5<br>1.6<br>2.6<br>4.2<br>5.9<br>9.8<br>11.5<br>12.0<br>13.8<br>13.8 | ( 0.0- 0.0)<br>( 0.0- 0.0)<br>( 0.0- 1.5)<br>( 0.0- 3.3)<br>( 0.4- 4.9)<br>( 1.4- 7.1)<br>( 2.5- 9.3)<br>( 5.5-14.0)<br>( 6.8-16.1)<br>( 7.3-16.8)<br>( 8.7-18.8)<br>( 8.7-18.8)<br>( 9.5-22.5) |

| Parameter | Values |
|---|---|
| Template ID | SS_EX_T_002 |
| Output File Name | rt-ex-kms1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.4.1.1H |
| Title 1 | Time of Study Therapy Life Table (Kaplan-Meier Estimates) |
| Title 2 | Treated Subjects - Stage 1 |
| Footnote 1 | (a) Cumulative proportion without events at end of interval. |

| Parameter | Values |
|------------------|----------------|
| Template ID | SS_EX_T_002 |
| Output File Name | rt-ex-kms2.lst |

| Purpose | WK24S2, WK48S2, WK96S2 |
|------------|--------------------------------------------------------------|
| Table No. | Table S.4.1.2H |
| Title 1 | Time of Study Therapy Life Table (Kaplan-Meier Estimates) |
| Title 2 | Treated Subjects - Stage 2 |
| Footnote 1 | (a) Cumulative proportion without events at end of interval. |

Template SS\_EX\_T\_003: Summary of Interruptions Greater than 3 Days

| Treatment Regimen | | | | | |
|---|---|---|---|---|---|
| Drug | Group A<br>N = XX | Group B<br>N = XX | | Group D<br>N = XX | Group E<br>N = XX |
| DRUG 1 N MEAN MEDIAN MIN , MAX Q1 , Q3 STANDARD DEVIATION | XX<br>XX.X<br>XX.X<br>XX.X , XX.X<br>XX.X , XX.X<br>XX.XX | XX<br>XX.X<br>XX.X<br>XX.X, XX.X<br>XX.X, XX.X<br>XX.X, XX.X | XX<br>XX.X<br>XX.X<br>XX.X , XX.X<br>XX.X , XX.X<br>XX.X , XX.X | XX<br>XX.X<br>XX.X<br>XX.X, XX.X<br>XX.X, XX.X<br>XX.XX | |
| DRUG 2 N MEAN MEDIAN MIN , MAX Q1 , Q3 STANDARD DEVIATION | XX<br>XX.X<br>XX.X<br>XX.X, XX.X<br>XX.X, XX.X | XX<br>XX.X<br>XX.X, XX.X<br>XX.X, XX.X<br>XX.X, XX.X | XX<br>XX.X<br>XX.X , XX.X<br>XX.X , XX.X<br>XX.X , XX.X | XX<br>XX.X<br>XX.X<br>XX.X, XX.X<br>XX.X, XX.X | XX<br>XX.X<br>XX.X<br>XX.X , XX.X<br>XX.X , XX.X |
| DRUG 3 N MEAN MEDIAN MIN , MAX Q1 , Q3 STANDARD DEVIATION | XX<br>XX.X<br>XX.X<br>XX.X , XX.X<br>XX.X , XX.X | XX<br>XX.X<br>XX.X<br>XX.X, XX.X<br>XX.X, XX.X | XX<br>XX.X<br>XX.X<br>XX.X, XX.X<br>XX.X, XX.X<br>XX.XX | XX<br>XX.X<br>XX.X<br>XX.X , XX.X<br>XX.X , XX.X<br>XX.XX | XX<br>XX.X<br>XX.X<br>XX.X , XX.X<br>XX.X , XX.X<br>XX.XX |

| Parameter | Values |
|---|---|
| Template ID | SS_EX_T_003 |
| Output File Name | rt-ex-interrupts1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.4.1.1I |
| Title 1 | Summary of Interruptions in Study Therapy Greater than 3 Days |
| Title 2 | Treated Subjects - Stage 1 |

| Parameter | Values |
|---|---|
| Template ID | SS_EX_T_003 |
| Output File Name | rt-ex-interrupts2.1st |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.4.1.2I |
| Title 1 | Summary of Interruptions in Study Therapy Greater than 3 Days |
| Title 2 | Treated Subjects - Stage 2 |

# Template SS\_EX\_L\_001: Study Medication Exposure Listing

| Subject Number<br>(Age/Gender/Race)<br>Treatment Group | Drug | Start Date | Stop Date | Daily Dose | Reason for Modification |
|---|---|---|---|---|---|
| PPD<br>(50/M/B)<br>BMS-663068 1200 mg QD/RAL/TDF | BMS-663068 | 04NOV2013 | 04NOV2013 | 0 | DOSING ERROR |
| IND COSCOL IZOU ING QU/IVAII/ IDE | RALTEGRAVIR | 05NOV2013<br>16NOV2013<br>17NOV2013<br>20NOV2013<br>01FEB2014<br>14FEB2014<br>27OCT2011<br>11NOV2012<br>20DEC2012<br>08FEB2013<br>09FEB2013<br>20MAR2013<br>22MAR2013<br>22MAR2013<br>24MAR2013<br>24MAR2013<br>24FEB2014<br>14FEB2014<br>07MAY2014<br>27OCT2011<br>11NOV2012<br>20DEC2012<br>08FEB2013<br>09FEB2013<br>09FEB2013<br>20MAR2013<br>24MAR2013<br>24MAR2013<br>24MAR2013<br>24MAR2013 | 15NOV2013<br>16NOV2013<br>19NOV2013<br>31JAN2014<br>13FEB2014<br>06MAY20114<br>29JUL2014<br>10NOV2012<br>19DEC2012<br>07FEB2013<br>08FEB2013<br>18MAR2013<br>21MAR2013<br>21MAR2013<br>23SEP2013<br>31JAN2014<br>13FEB2014<br>06MAY2014<br>29JUL2014<br>10NOV2012<br>19DEC2012<br>07FEB2013<br>08FEB2013<br>18MAR2013<br>19MAR2013<br>19MAR2013<br>21MAR2013<br>21MAR2013<br>21MAR2013<br>21MAR2013<br>21MAR2013<br>21MAR2013<br>21MAR2013<br>23SEP2013 | 1200<br>0<br>1200<br>1200<br>1200<br>1200<br>1200<br>800<br>0<br>800 | NO CHANGE DOSING ERROR NO CHANGE NO CHANGE NO CHANGE OTHER NO CHANGE NO CHANGE NO CHANGE OTHER NO CHANGE OSING ERROR NO CHANGE DOSING ERROR NO CHANGE DOSING ERROR NO CHANGE DOSING ERROR NO CHANGE DOSING ERROR NO CHANGE OSING ERROR NO CHANGE OTHER NO CHANGE OTHER NO CHANGE OTHER NO CHANGE NO CHANGE NO CHANGE NO CHANGE NO CHANGE NO CHANGE NO CHANGE OSING ERROR NO CHANGE DOSING ERROR NO CHANGE DOSING ERROR NO CHANGE DOSING ERROR NO CHANGE DOSING ERROR NO CHANGE |

| Parameter | Values |
|------------------|------------------|
| Template ID | SS_EX_L_001 |
| Output File Name | rl-ex-lists1.lst |

| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
|-----------|----------------------------------------------|
| Table No. | Appendix 4.1.1A |
| Title 1 | Study Medication Exposure by Subject Listing |
| Title 2 | Treated Subjects - Stage 1 |

| Parameter | Values |
|------------------|----------------------------------------------|
| Template ID | SS_EX_L_001 |
| Output File Name | rl-ex-lists2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Appendix 4.1.2A |
| Title 1 | Study Medication Exposure by Subject Listing |
| Title 2 | Treated Subjects - Stage 2 |

#### Template SS EX L 002: Study Medication Listing related to Continuation Dose

Treatment Group: DRUG C

| Subject Number<br>(Age/Gender/Race) | Tim on<br>Randomized<br>Dose | Date/Study<br>of Switch<br>Continuati | to | Time on<br>Continuation<br>Dose |
|---|---|---|---|---|
| PPD | 280 | PPD | / 281 | 364 |
| PPD | 285 | | / 286 | 370 |
| PPD (50/M/B) | 298 | | / 299 | 351 |

ParameterValuesTemplate IDSS\_EX\_L\_002Output File Namerl-ex-listcdoses1.lstPurposeWK96S1, WK96S2Table No.Appendix 4.1.1BTitle 1Listing of Time on Original and Continuation DoseTitle 2Treated Subjects - Stage 1

| Parameter | Values |
|------------------|---------------------------------------------------|
| Template ID | SS_EX_L_002 |
| Output File Name | rl-ex-listcdoses2.lst |
| Purpose | WK96S2 |
| Table No. | Appendix 4.1.2B |
| Title 1 | Listing of Time on Original and Continuation Dose |
| Title 2 | Treated Subjects - Stage 2 |

# 4.4.2 Concomitant Therapy

| Parameter | Values |
|------------------|--------------------------------|
| Template ID | GS_CM_T_X_001 |
| Output File Name | rt-cm-conmeds1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.4.2.1 |
| Title 1 | Non-Study Medication Summary |
| Title 2 | Concomitant Medication |
| Title 3 | Treated Subjects - Stage 1 |

| Parameter | Values |
|------------------|------------------------------|
| Template ID | GS_CM_T_X_001 |
| Output File Name | rt-cm-conmeds2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.4.2.2 |
| Title 1 | Non-Study Medication Summary |
| Title 2 | Concomitant Medication |
| Title 3 | Treated Subjects - Stage 2 |

#### Template GS\_CM\_L\_X\_006: Non-Study Medication Listing by Treatment Group

Protocol: CV181008 Draft Page 1 of 89

Non-Study Medication Medication Category All Treated Subjects

Treatment Group: TRT A

| Subject ID<br>(Age/Gender/Race) | Period<br>Visit<br>Current Trt | Start<br>Stop<br>Study Day<br>TRD# | | ay | Anatomic Class<br>Therapeutic Class<br>Generic Name<br>Reported Medication | Use |
|---|---|---|---|---|---|---|
| PPD<br>(43/F/B) | SHORT TERM<br>WEEK 1<br>ABC 10 | PPD | 1D | 1 | ALIMENTARY TRACT & METABOLISM<br>ORAL BLOOD GIUCOSE LOWERING DRUG<br>METFORMIN<br>GLUCOPHAGE | OTHER |
| | SHORT TERM<br>WEEK 1<br>ABC 10 | PPD | 1D | 1 | ALIMENTARY TRACT & METABOLISM ORAL BLOOD GLUCOSE LOWERING DRUG GLIPIZIDE GLUCOTROL XL | OTHER |
| | SHORT TERM<br>WEEK 1<br>ABC 10 | PPD | 2D | 2 | NERVOUS SYSTEM OTHER ANALGESIC & ANTIPYRETIC ACETAMINOPHEN TYLENOL | ADVERSE EVENT |
| | SHORT TERM<br>WEEK 1<br>ABC 10 | PPD | 2D | 2 | ALIMENTARY TRACT & METABOLISM ORAL BLOOD GLUCOSE LOWERING DRUG GLIPIZIDE GLUCOTROL XL | OTHER |
| | SHORT TERM<br>WEEK 1<br>ABC 10 | PPD | 2D | 2 | ALIMENTARY TRACT & METABOLISM ORAL BLOOD GLUCOSE LOWERING DRUG METFORMIN GLUCOPHAGE | OTHER |

# Time relative to most recent dose Program Source: /wwbdm/ndp/prime/gssr/devtest/checkraw/cmlist.sas

290CT2004:18:53:00

| Parameter | Values |
|------------------|--------------------------------|
| Template ID | GS_CM_L_X_006 |
| Output File Name | rl-cm-meds1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |

| Table No. | Appendix 4.2.1 |
|-----------|--------------------------------------|
| Title 1 | Non-Study Medication |
| Title 2 | Previous and Concomitant Medications |
| Title 3 | Treated Subjects - Stage 1 |

| Parameter | Values |
|------------------|--------------------------------------|
| Template ID | GS_CM_L_X_006 |
| Output File Name | rl-cm-meds2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Appendix 4.2.2 |
| Title 1 | Non-Study Medication |
| Title 2 | Previous and Concomitant Medications |
| Title 3 | Treated Subjects - Stage 2 |

# 4.5 Efficacy Results

# Template SS\_VL\_T\_001: Detailed Summary of HIV-1 < Y (by Subgroup)

Subgroup: XXXXXXXXX Level: XXXXXXXXXXX

| | BMS-986001<br>100 mg QD/<br>EFV/3TC<br>N = XX | BMS-986001<br>200 mg QD/<br>EFV/3TC<br>N = XX | BMS-986001<br>400 mg QD/<br>EFV/3TC<br>N = XX | TDF/EFV/3TC<br>N = XX |
|---|---|---|---|---|
| NUMBER OF RESPONDERS (A) | 57 (87.7) | 54 (80.6) | 62 ( 93.9) | 88 ( 88.9) |
| 95% CI | (77.2 - 94.5) | (69.1 - 89.2) | (85.2 - 98.3) | (81.0 - 94.3) |
| NUMBER OF VIROLOGIC FAILURES | X (XXX.X) | X (XXX.X) | X (XXX.X) | X (XXX.X) |
| HIV-1 RNA $>= 40$ c/mL (B) | X (XXX.X) | X (XXX.X) | X (XXX.X) | X (XXX.X) |
| DISC. STUDY/STUDY DRUG DUE TO LACK OF EFFICACY (C) | X (XXX.X) | X (XXX.X) | X (XXX.X) | X (XXX.X) |
| DISC. STUDY/STUDY DRUG FOR OTHER REASONS (D) | X (XXX.X) | X (XXX.X) | X (XXX.X) | X (XXX.X) |
| NO VIROLOGIC DATA | | | | |
| DISC. STUDY/STUDY DRUG DUE TO AE OR DEATH (E) | 0 | 4 ( 6.0) | 0 | 2 ( 2.0) |
| DISC. STUDY/STUDY DRUG FOR OTHER REASONS (F) | 0 | 0 | 0 | 2 ( 2.0) |
| MISSING DATA DURING WINDOW BUT ON STUDY | 0 | 0 | 0 | 0 |

\_\_\_\_\_\_

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_001 |
| Output File Name | rt-vl-resp40w24s1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.5.1.1A |
| Title 1 | Detailed Summary of HIV-1 RNA < 40 c/mL |
| Title 2 | Proportion of Responders at Week 24 Snapshot |
| Title 3 | Treated Subjects (mITT) - Stage 1 |
| Footnote 1 | (A) Response is assessed with the snapshot algorithm, which uses the last plasma HIV-1 RNA value in the predefined visit window to classify a subject's response status. |
| Footnote 2 | (B) Includes subjects having HIV-1 RNA >= 40 c/mL within the Week 24 visit window. |
| Footnote 3 | (C) Includes subjects who discontinued due to lack of efficacy at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window. |

| Footnote 4 | (D) Includes subjects who discontinued due to any reasons except AE, death and lack of efficacy at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window and last HIV-1 RNA >= 40 c/mL. |
|---|---|
| Footnote 5 | (E) Includes patients who discontinued due to AE or death at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window |
| Footnote 6 | (F) Other includes: withdrew consent, loss to follow-up, moved etc. with last HIV-1 RNA < 40 c/mL |
| Layout notes | No subgroup presentation |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_001 |
| Output File Name | rt-vl-resp40w24s2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.5.1.2A |
| Title 1 | Detailed Summary of HIV-1 RNA < 40 c/mL |
| Title 2 | Proportion of Responders at Week 24 Snapshot |
| Title 3 | Treated Subjects (mITT) - Stage 2 |
| Footnote 1 | (A) Response is assessed with the snapshot algorithm, which uses the last plasma HIV-1 RNA value in the predefined visit window to classify a subject's response status. |
| Footnote 2 | (B) Includes subjects having HIV-1 RNA >= 40 c/mL within the Week 24 visit window. |
| Footnote 3 | (C) Includes subjects who discontinued due to lack of efficacy at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window. |
| Footnote 4 | (D) Includes subjects who discontinued due to any reasons except AE, death and lack of efficacy at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window and last HIV-1 RNA >= 40 c/mL. |
| Footnote 5 | (E) Includes patients who discontinued due to AE or death at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window |
| Footnote 6 | (F) Other includes: withdrew consent, loss to follow-up, moved etc. with last HIV-1 RNA < 40 c/mL |
| Layout notes | No subgroup presentation |

#### Template SS\_VL\_T\_002: Summary of HIV-1 < Y (by Subgroup)

Subgroup: XXXXXXXXX Level: XXXXXXXXXXX

| | BMS-986001<br>100 mg QD/<br>EFV/3TC<br>N = XX | BMS-986001<br>200 mg QD/<br>EFV/3TC<br>N = XX | BMS-986001<br>400 mg QD/<br>EFV/3TC<br>N = XX | TDF/EFV/3TC<br>N = XX |
|---|---|---|---|---|
| NUMBER OF RESPONDERS (A) 95% CI NUMBER OF VIROLOGIC FAILURES (B) | 57 ( 87.7) | 54 ( 80.6) | 62 ( 93.9) | 88 ( 88.9) |
| | (77.2 - 94.5) | (69.1 - 89.2) | (85.2 - 98.3) | (81.0 - 94.3) |
| | X (XXX.X) | X (XXX.X) | X (XXX.X) | X (XXX.X) |
| NO VIROLOGIC DATA DISC. STUDY/STUDY DRUG DUE TO AE OR DEATH (C) DISC. STUDY/STUDY DRUG FOR OTHER REASONS (D) MISSING DATA DURING WINDOW BUT ON STUDY | 0 | 4 ( 6.0) | 0 | 2 ( 2.0) |
| | 0 | 0 | 0 | 2 ( 2.0) |
| | 0 | 0 | 0 | 0 |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_002 |
| Output File Name | rt-vl-sumresp40w24s1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.5.1.1C |
| Title 1 | Summary of HIV-1 RNA < 40 c/mL |
| Title 2 | Proportion of Responders at Week 24 Snapshot |
| Title 3 | Treated Subjects (mITT) - Stage 1 |
| Footnote 1 | (A) Response is assessed with the snapshot algorithm, which uses the last plasma HIV-1 RNA value in the predefined visit window to classify a subject's response status. |
| Footnote 2 | (B) Includes subjects who are >= 50 copies in the visit window. It also includes subjects who discontinued prior to the visit window for lack or loss of efficacy or any reasons except AE and death at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window and last HIV-1 RNA >= 50 c/mL. |
| Footnote 3 | (C) Includes patients who discontinued due to AE or death at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window |
| Footnote 4 | (D) Other includes: withdrew consent, loss to follow-up, moved etc. with last HIV-1 RNA < 40 c/mL |
|---|---|
| Layout notes | No subgroup presentation |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_002 |
| Output File Name | rt-vl-sumresp40w24s2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.5.1.2C |
| Title 1 | Summary of HIV-1 RNA < 40 c/mL |
| Title 2 | Proportion of Responders at Week 24 Snapshot |
| Title 3 | Treated Subjects (mITT) - Stage 2 |
| Footnote 1 | (A) Response is assessed with the snapshot algorithm, which uses the last plasma HIV-1 RNA value in the predefined visit window to classify a subject's response status. |
| Footnote 2 | (B) Includes subjects who are >= 50 copies in the visit window. It also includes subjects who discontinued prior to the visit window for lack or loss of efficacy or any reasons except AE and death at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window and last HIV-1 RNA >= 50 c/mL. |
| Footnote 3 | (C) Includes patients who discontinued due to AE or death at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window |
| Footnote 4 | (D) Other includes: withdrew consent, loss to follow-up, moved etc. with last HIV-1 RNA < 40 c/mL |
| Layout notes | No subgroup presentation |

| Parameter | Values |
|------------------|-----------------------------------------|
| Template ID | SS_VL_T_001 |
| Output File Name | rt-vl-resp40w24subgs1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.5.1.1B |
| Title 1 | Detailed Summary of HIV-1 RNA < 40 c/mL |

| Title 2 | Proportion of Responders at Week 24 Snapshot |
|---|---|
| Title 3 | By Subgroup |
| Title 4 | Treated Subjects (mITT) - Stage 1 |
| Footnote 1 | (A) Response is assessed with the snapshot algorithm, which uses the last plasma HIV-1 RNA value in the predefined visit window to classify a subject's response status. |
| Footnote 2 | (B) Includes subjects having HIV-1 RNA >= 40 c/mL within the Week 24 visit window. |
| Footnote 3 | (C) Includes subjects who discontinued due to lack of efficacy at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window. |
| Footnote 4 | (D) Includes subjects who discontinued due to any reasons except AE, death and lack of efficacy at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window and last HIV-1 RNA >= 40 c/mL. |
| Footnote 5 | (E) Includes patients who discontinued due to AE or death at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window |
| Footnote 6 | (F) Other includes: withdrew consent, loss to follow-up, moved etc. with last HIV-1 RNA < 40 c/mL |
| Layout notes | Subgroups are: • Baseline HIV-1 RNA < 100,000 c/mL , >=100,000 c/mL • Baseline CD4 < 100, 100 to < 200, 200 to < 350, 350 to < 500, >= 500 cells/uL • Baseline Gag Polymorphism: all combinations of baseline gag polymorphisms at selected positions • Gender: Male, Female • Race: White, Black/African American, American Indian/Alaska Native, Asian, Native Hawaiian/Other Pacific Islander, Other • HIV-1 Clade: Include all clades available in the database |

| Parameter | Values |
|------------------|---------------------------|
| Template ID | SS_VL_T_001 |
| Output File Name | rt-vl-resp40w24subgs2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.5.1.2B |

| Title 1 | Detailed Summary of HIV-1 RNA < 40 c/mL |
|---|---|
| Title 2 | Proportion of Responders at Week 24 Snapshot |
| Title 3 | By Subgroup |
| Title 4 | Treated Subjects (mITT) - Stage 2 |
| Footnote 1 | (A) Response is assessed with the snapshot algorithm, which uses the last plasma HIV-1 RNA value in the predefined visit window to classify a subject's response status. |
| Footnote 2 | (B) Includes subjects having HIV-1 RNA >= 40 c/mL within the Week 24 visit window. |
| Footnote 3 | (C) Includes subjects who discontinued due to lack of efficacy at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window. |
| Footnote 4 | (D) Includes subjects who discontinued due to any reasons except AE, death and lack of efficacy at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window and last HIV-1 RNA >= 40 c/mL. |
| Footnote 5 | (E) Includes patients who discontinued due to AE or death at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window |
| Footnote 6 | (F) Other includes: withdrew consent, loss to follow-up, moved etc. with last HIV-1 RNA < 40 c/mL |
| Layout notes | <ul> <li>Subgroups are:</li> <li>Baseline HIV-1 RNA &lt; 100,000 c/mL , &gt;=100,000 c/mL</li> <li>Baseline CD4 &lt; 100, 100 to &lt; 200, 200 to &lt; 350, 350 to &lt; 500, &gt;= 500 cells/uL</li> <li>Baseline Gag Polymorphism: all combinations of baseline gag polymorphisms at selected positions</li> <li>Gender: Male, Female</li> <li>Race: White, Black/African American, American Indian/Alaska Native, Asian, Native Hawaiian/Other Pacific Islander, Other</li> <li>HIV-1 Clade: Include all clades available in the database</li> </ul> |

| Parameter | Values |
|------------------|-----------------------|
| Template ID | SS_VL_T_001 |
| Output File Name | rt-vl-resp40w48s1.lst |

| Purpose | WK96S1, WK96S2 |
|---|---|
| Table No. | Table S.5.2.1A |
| Title 1 | Detailed Summary of HIV-1 RNA < 40 c/mL |
| Title 2 | Proportion of Responders at Week 48 Snapshot |
| Title 3 | Treated Subjects (mITT) - Stage 1 |
| Footnote 1 | (A) Response is assessed with the snapshot algorithm, which uses the last plasma HIV-1 RNA value in the predefined visit window to classify a subject's response status. |
| Footnote 2 | (B) Includes subjects having HIV-1 RNA >= 40 c/mL within the Week 48 visit window. |
| Footnote 3 | (C) Includes subjects who discontinued due to lack of efficacy at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window. |
| Footnote 4 | (D) Includes subjects who discontinued due to any reasons except AE, death and lack of efficacy at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window and last HIV-1 RNA >= 40 c/mL. |
| Footnote 5 | (E) Includes patients who discontinued due to AE or death at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window |
| Footnote 6 | (F) Other includes: withdrew consent, loss to follow-up, moved etc. with last HIV-1 RNA < 40 c/mL |
| Layout notes | No subgroup presentation |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_001 |
| Output File Name | rt-vl-resp40w48s2.lst |
| Purpose | WK48S2, WK96S2 |
| Table No. | Table S.5.2.2A |
| Title 1 | Detailed Summary of HIV-1 RNA < 40 c/mL |
| Title 2 | Proportion of Responders at Week 48 Snapshot |
| Title 3 | Treated Subjects (mITT) - Stage 2 |
| Footnote 1 | (A) Response is assessed with the snapshot algorithm, which uses the last plasma HIV-1 RNA value in the predefined visit |

| | window to classify a subject's response status. |
|---|---|
| Footnote 2 | (B) Includes subjects having HIV-1 RNA >= 40 c/mL within the Week 48 visit window. |
| Footnote 3 | (C) Includes subjects who discontinued due to lack of efficacy at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window. |
| Footnote 4 | (D) Includes subjects who discontinued due to any reasons except AE, death and lack of efficacy at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window and last HIV-1 RNA >= 40 c/mL. |
| Footnote 5 | (E) Includes patients who discontinued due to AE or death at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window |
| Footnote 6 | (F) Other includes: withdrew consent, loss to follow-up, moved etc. with last HIV-1 RNA < 40 c/mL |
| Layout notes | No subgroup presentation |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_002 |
| Output File Name | rt-vl-sumresp40w48s1.lst |
| Purpose | WK96S1, WK96S2 |
| Table No. | Table S.5.2.1C |
| Title 1 | Summary of HIV-1 RNA < 40 c/mL |
| Title 2 | Proportion of Responders at Week 48 Snapshot |
| Title 3 | Treated Subjects (mITT) - Stage 1 |
| Footnote 1 | (A) Response is assessed with the snapshot algorithm, which uses the last plasma HIV-1 RNA value in the predefined visit window to classify a subject's response status. |
| Footnote 2 | (B) Includes subjects who are >= 50 copies in the visit window. It also includes subjects who discontinued prior to the visit window for lack or loss of efficacy or any reasons except AE and death at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window and last HIV-1 RNA >= 50 c/mL. |
| Footnote 3 | (C) Includes patients who discontinued due to AE or death at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window |
| Footnote 4 | (D) Other includes: withdrew consent, loss to follow-up, moved etc. with last HIV-1 RNA < 40 c/mL |

| Layout notes | No subgroup presentation |
|--------------|--------------------------|
|--------------|--------------------------|

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_002 |
| Output File Name | rt-vl-sumresp40w48s2.lst |
| Purpose | WK48S2, WK96S2 |
| Table No. | Table S.5.2.2C |
| Title 1 | Summary of HIV-1 RNA < 40 c/mL |
| Title 2 | Proportion of Responders at Week 48 Snapshot |
| Title 3 | Treated Subjects (mITT) - Stage 2 |
| Footnote 1 | (A) Response is assessed with the snapshot algorithm, which uses the last plasma HIV-1 RNA value in the predefined visit window to classify a subject's response status. |
| Footnote 2 | (B) Includes subjects who are >= 50 copies in the visit window. It also includes subjects who discontinued prior to the visit window for lack or loss of efficacy or any reasons except AE and death at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window and last HIV-1 RNA >= 50 c/mL. |
| Footnote 3 | (C) Includes patients who discontinued due to AE or death at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window |
| Footnote 4 | (D) Other includes: withdrew consent, loss to follow-up, moved etc. with last HIV-1 RNA < 40 c/mL |
| Layout notes | No subgroup presentation |

| Parameter | Values |
|------------------|----------------------------------------------|
| Template ID | SS_VL_T_001 |
| Output File Name | rt-vl-resp40w48subgs1.lst |
| Purpose | WK96S1, WK96S2 |
| Table No. | Table S.5.2.1B |
| Title 1 | Detailed Summary of HIV-1 RNA < 40 c/mL |
| Title 2 | Proportion of Responders at Week 48 Snapshot |

| Title 3 | By Subgroup |
|---|---|
| Title 4 | Treated Subjects (mITT) - Stage 1 |
| Footnote 1 | (A) Response is assessed with the snapshot algorithm, which uses the last plasma HIV-1 RNA value in the predefined visit window to classify a subject's response status. |
| Footnote 2 | (B) Includes subjects having HIV-1 RNA >= 40 c/mL within the Week 48 visit window. |
| Footnote 3 | (C) Includes subjects who discontinued due to lack of efficacy at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window. |
| Footnote 4 | (D) Includes subjects who discontinued due to any reasons except AE, death and lack of efficacy at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window and last HIV-1 RNA >= 40 c/mL. |
| Footnote 5 | (E) Includes patients who discontinued due to AE or death at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window |
| Footnote 6 | (F) Other includes: withdrew consent, loss to follow-up, moved etc. with last HIV-1 RNA < 40 c/mL |
| Layout notes | <ul> <li>Subgroups are:</li> <li>Baseline HIV-1 RNA &lt; 100,000 c/mL , &gt;=100,000 c/mL</li> <li>Baseline CD4 &lt; 100, 100 to &lt; 200, 200 to &lt; 350, 350 to &lt; 500, &gt;= 500 cells/uL</li> <li>Baseline Gag Polymorphism: all combinations of baseline gag polymorphisms at selected positions</li> <li>Gender: Male, Female</li> <li>Race: White, Black/African American, American Indian/Alaska Native, Asian, Native Hawaiian/Other Pacific Islander, Other</li> <li>HIV-1 Clade: Include all clades available in the database</li> </ul> |

| Parameter | Values |
|------------------|-----------------------------------------|
| Template ID | SS_VL_T_001 |
| Output File Name | rt-vl-resp40w48subgs2.lst |
| Purpose | WK48S2, WK96S2 |
| Table No. | Table S.5.2.2B |
| Title 1 | Detailed Summary of HIV-1 RNA < 40 c/mL |

| Title 2 | Proportion of Responders at Week 48 Snapshot |
|---|---|
| Title 3 | By Subgroup |
| Title 4 | Treated Subjects (mITT) - Stage 2 |
| Footnote 1 | (A) Response is assessed with the snapshot algorithm, which uses the last plasma HIV-1 RNA value in the predefined visit window to classify a subject's response status. |
| Footnote 2 | (B) Includes subjects having HIV-1 RNA >= 40 c/mL within the Week 48 visit window. |
| Footnote 3 | (C) Includes subjects who discontinued due to lack of efficacy at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window. |
| Footnote 4 | (D) Includes subjects who discontinued due to any reasons except AE, death and lack of efficacy at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window and last HIV-1 RNA >= 40 c/mL. |
| Footnote 5 | (E) Includes patients who discontinued due to AE or death at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window |
| Footnote 6 | (F) Other includes: withdrew consent, loss to follow-up, moved etc. with last HIV-1 RNA < 40 c/mL |
| Layout notes | <ul> <li>Subgroups are:</li> <li>Baseline HIV-1 RNA &lt; 100,000 c/mL , &gt;=100,000 c/mL</li> <li>Baseline CD4 &lt; 100, 100 to &lt; 200, 200 to &lt; 350, 350 to &lt; 500, &gt;= 500 cells/uL</li> <li>Baseline Gag Polymorphism: all combinations of baseline gag polymorphisms at selected positions</li> <li>Gender: Male, Female</li> <li>Race: White, Black/African American, American Indian/Alaska Native, Asian, Native Hawaiian/Other Pacific Islander, Other</li> <li>HIV-1 Clade: Include all clades available in the database</li> </ul> |

| Parameter | Values |
|------------------|-----------------------|
| Template ID | SS_VL_T_001 |
| Output File Name | rt-vl-resp40w96s1.lst |
| Purpose | WK96S1, WK96S2 |
| Table No. | Table S.5.3.1A |

| Title 1 | Detailed Summary of HIV-1 RNA < 40 c/mL |
|---|---|
| Title 2 | Proportion of Responders at Week 96 Snapshot |
| Title 3 | Treated Subjects (mITT) - Stage 1 |
| Footnote 1 | (A) Response is assessed with the snapshot algorithm, which uses the last plasma HIV-1 RNA value in the predefined visit window to classify a subject's response status. |
| Footnote 2 | (B) Includes subjects having HIV-1 RNA >= 40 c/mL within the Week 96 visit window. |
| Footnote 3 | (C) Includes subjects who discontinued due to lack of efficacy at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window. |
| Footnote 4 | (D) Includes subjects who discontinued due to any reasons except AE, death and lack of efficacy at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window and last HIV-1 RNA >= 40 c/mL. |
| Footnote 5 | (E) Includes patients who discontinued due to AE or death at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window |
| Footnote 6 | (F) Other includes: withdrew consent, loss to follow-up, moved etc. with last HIV-1 RNA < 40 c/mL |
| Layout notes | No subgroup presentation |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_001 |
| Output File Name | rt-vl-resp40w96s2.lst |
| Purpose | WK96S2 |
| Table No. | Table S.5.3.2A |
| Title 1 | Detailed Summary of HIV-1 RNA < 40 c/mL |
| Title 2 | Proportion of Responders at Week 96 Snapshot |
| Title 3 | Treated Subjects (mITT) - Stage 2 |
| Footnote 1 | (A) Response is assessed with the snapshot algorithm, which uses the last plasma HIV-1 RNA value in the predefined visit window to classify a subject's response status. |
| Footnote 2 | (B) Includes subjects having HIV-1 RNA >= 40 c/mL within the Week 96 visit window. |

| Footnote 3 | (C) Includes subjects who discontinued due to lack of efficacy at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window. |
|---|---|
| Footnote 4 | (D) Includes subjects who discontinued due to any reasons except AE, death and lack of efficacy at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window and last HIV-1 RNA >= 40 c/mL. |
| Footnote 5 | (E) Includes patients who discontinued due to AE or death at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window |
| Footnote 6 | (F) Other includes: withdrew consent, loss to follow-up, moved etc. with last HIV-1 RNA < 40 c/mL |
| Layout notes | No subgroup presentation |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_002 |
| Output File Name | rt-vl-sumresp40w96s1.lst |
| Purpose | WK96S1, WK96S2 |
| Table No. | Table S.5.3.1C |
| Title 1 | Summary of HIV-1 RNA < 40 c/mL |
| Title 2 | Proportion of Responders at Week 96 Snapshot |
| Title 3 | Treated Subjects (mITT) - Stage 1 |
| Footnote 1 | (A) Response is assessed with the snapshot algorithm, which uses the last plasma HIV-1 RNA value in the predefined visit window to classify a subject's response status. |
| Footnote 2 | (B) Includes subjects who are >= 50 copies in the visit window. It also includes subjects who discontinued prior to the visit window for lack or loss of efficacy or any reasons except AE and death at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window and last HIV-1 RNA >= 50 c/mL. |
| Footnote 3 | (C) Includes patients who discontinued due to AE or death at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window |
| Footnote 4 | (D) Other includes: withdrew consent, loss to follow-up, moved etc. with last HIV-1 RNA < 40 c/mL |
| Layout notes | No subgroup presentation |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_002 |
| Output File Name | rt-vl-sumresp40w96s2.lst |
| Purpose | WK96S2 |
| Table No. | Table S.5.3.2C |
| Title 1 | Summary of HIV-1 RNA < 40 c/mL |
| Title 2 | Proportion of Responders at Week 96 Snapshot |
| Title 3 | Treated Subjects (mITT) - Stage 2 |
| Footnote 1 | (A) Response is assessed with the snapshot algorithm, which uses the last plasma HIV-1 RNA value in the predefined visit window to classify a subject's response status. |
| Footnote 2 | (B) Includes subjects who are >= 50 copies in the visit window. It also includes subjects who discontinued prior to the visit window for lack or loss of efficacy or any reasons except AE and death at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window and last HIV-1 RNA >= 50 c/mL. |
| Footnote 3 | (C) Includes patients who discontinued due to AE or death at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window |
| Footnote 4 | (D) Other includes: withdrew consent, loss to follow-up, moved etc. with last HIV-1 RNA < 40 c/mL |
| Layout notes | No subgroup presentation |

| Parameter | Values |
|------------------|----------------------------------------------|
| Template ID | SS_VL_T_001 |
| Output File Name | rt-vl-resp40w96subgs1.lst |
| Purpose | WK96S1, WK96S2 |
| Table No. | Table S.5.3.1B |
| Title 1 | Detailed Summary of HIV-1 RNA < 40 c/mL |
| Title 2 | Proportion of Responders at Week 96 Snapshot |
| Title 3 | By Subgroup |
| Title 4 | Treated Subjects (mITT) - Stage 1 |

| Footnote 1 | (A) Response is assessed with the snapshot algorithm, which uses the last plasma HIV-1 RNA value in the predefined visit window to classify a subject's response status. |
|---|---|
| Footnote 2 | (B) Includes subjects having HIV-1 RNA >= 40 c/mL within the Week 96 visit window. |
| Footnote 3 | (C) Includes subjects who discontinued due to lack of efficacy at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window. |
| Footnote 4 | (D) Includes subjects who discontinued due to any reasons except AE, death and lack of efficacy at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window and last HIV-1 RNA >= 40 c/mL. |
| Footnote 5 | (E) Includes patients who discontinued due to AE or death at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window |
| Footnote 6 | (F) Other includes: withdrew consent, loss to follow-up, moved etc. with last HIV-1 RNA < 40 c/mL |
| Layout notes | <ul> <li>Subgroups are:</li> <li>Baseline HIV-1 RNA &lt; 100,000 c/mL , &gt;=100,000 c/mL</li> <li>Baseline CD4 &lt; 100, 100 to &lt; 200, 200 to &lt; 350, 350 to &lt; 500, &gt;= 500 cells/uL</li> <li>Baseline Gag Polymorphism: all combinations of baseline gag polymorphisms at selected positions</li> <li>Gender: Male, Female</li> <li>Race: White, Black/African American, American Indian/Alaska Native, Asian, Native Hawaiian/Other Pacific Islander, Other</li> <li>HIV-1 Clade: Include all clades available in the database</li> </ul> |

| Parameter | Values |
|------------------|----------------------------------------------|
| Template ID | SS_VL_T_001 |
| Output File Name | rt-vl-resp40w96subgs2.lst |
| Purpose | WK96S2 |
| Table No. | Table S.5.3.2B |
| Title 1 | Detailed Summary of HIV-1 RNA < 40 c/mL |
| Title 2 | Proportion of Responders at Week 96 Snapshot |
| Title 3 | By Subgroup |

| Title 4 | Treated Subjects (mITT) - Stage 2 |
|---|---|
| Footnote 1 | (A) Response is assessed with the snapshot algorithm, which uses the last plasma HIV-1 RNA value in the predefined visit window to classify a subject's response status. |
| Footnote 2 | (B) Includes subjects having HIV-1 RNA >= 40 c/mL within the Week 96 visit window. |
| Footnote 3 | (C) Includes subjects who discontinued due to lack of efficacy at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window. |
| Footnote 4 | (D) Includes subjects who discontinued due to any reasons except AE, death and lack of efficacy at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window and last HIV-1 RNA >= 40 c/mL. |
| Footnote 5 | (E) Includes patients who discontinued due to AE or death at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window |
| Footnote 6 | (F) Other includes: withdrew consent, loss to follow-up, moved etc. with last HIV-1 RNA < 40 c/mL |
| Layout notes | <ul> <li>Subgroups are:</li> <li>Baseline HIV-1 RNA &lt; 100,000 c/mL , &gt;=100,000 c/mL</li> <li>Baseline CD4 &lt; 100, 100 to &lt; 200, 200 to &lt; 350, 350 to &lt; 500, &gt;= 500 cells/uL</li> <li>Baseline Gag Polymorphism: all combinations of baseline gag polymorphisms at selected positions</li> <li>Gender: Male, Female</li> <li>Race: White, Black/African American, American Indian/Alaska Native, Asian, Native Hawaiian/Other Pacific Islander, Other</li> <li>HIV-1 Clade: Include all clades available in the database</li> </ul> |

| Parameter | Values |
|------------------|----------------------------------------------|
| Template ID | SS_VL_T_001 |
| Output File Name | rt-vl-resp200w24s1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.5.4.1A |
| Title 1 | Detailed Summary of HIV-1 RNA < 200 c/mL |
| Title 2 | Proportion of Responders at Week 24 Snapshot |

| Title 3 | Treated Subjects (mITT) - Stage 1 |
|---|---|
| Footnote 1 | (A) Response is assessed with the snapshot algorithm, which uses the last plasma HIV-1 RNA value in the predefined visit window to classify a subject's response status. |
| Footnote 2 | (B) Includes subjects having HIV-1 RNA >= 200 c/mL within the Week 24 visit window. |
| Footnote 3 | (C) Includes subjects who discontinued due to lack of efficacy at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window. |
| Footnote 4 | (D) Includes subjects who discontinued due to any reasons except AE, death and lack of efficacy at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window and last HIV-1 RNA >= 200 c/mL. |
| Footnote 5 | (E) Includes patients who discontinued due to AE or death at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window |
| Footnote 6 | (F) Other includes: withdrew consent, loss to follow-up, moved etc. with last HIV-1 RNA < 200 c/mL |
| Layout notes | No subgroup presentation |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_001 |
| Output File Name | rt-vl-resp200w24s2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.5.4.2A |
| Title 1 | Detailed Summary of HIV-1 RNA < 200 c/mL |
| Title 2 | Proportion of Responders at Week 24 Snapshot |
| Title 3 | Treated Subjects (mITT) - Stage 2 |
| Footnote 1 | (A) Response is assessed with the snapshot algorithm, which uses the last plasma HIV-1 RNA value in the predefined visit window to classify a subject's response status. |
| Footnote 2 | (B) Includes subjects having HIV-1 RNA >= 200 c/mL within the Week 24 visit window. |
| Footnote 3 | (C) Includes subjects who discontinued due to lack of efficacy at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window. |
| Footnote 4 | (D) Includes subjects who discontinued due to any reasons except AE, death and lack of efficacy at any time point from Day 1 |

| | through the time window if this resulted in no virologic data on treatment during the specified window and last HIV-1 RNA >= 200 c/mL. |
|---|---|
| Footnote 5 | (E) Includes patients who discontinued due to AE or death at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window |
| Footnote 6 | (F) Other includes: withdrew consent, loss to follow-up, moved etc. with last HIV-1 RNA < 200 c/mL |
| Layout notes | No subgroup presentation |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_001 |
| Output File Name | rt-vl-resp200w24bpolys1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.5.4.1B |
| Title 1 | Detailed Summary of HIV-1 RNA < 200 c/mL |
| Title 2 | Proportion of Responders at Week 24 Snapshot |
| Title 3 | By Baseline Gag Polymorphism |
| Title 4 | Treated Subjects (mITT) - Stage 1 |
| Footnote 1 | (A) Response is assessed with the snapshot algorithm, which uses the last plasma HIV-1 RNA value in the predefined visit window to classify a subject's response status. |
| Footnote 2 | (B) Includes subjects having HIV-1 RNA >= 200 c/mL within the Week 24 visit window. |
| Footnote 3 | (C) Includes subjects who discontinued due to lack of efficacy at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window. |
| Footnote 4 | (D) Includes subjects who discontinued due to any reasons except AE, death and lack of efficacy at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window and last HIV-1 RNA >= 200 c/mL. |
| Footnote 5 | (E) Includes patients who discontinued due to AE or death at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window |
| Footnote 6 | (F) Other includes: withdrew consent, loss to follow-up, moved etc. with last HIV-1 RNA < 200 c/mL |
| Layout notes | Subgroups are all combinations of baseline gag polymorphisms at selected positions |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_001 |
| Output File Name | rt-vl-resp200w24bpolys2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.5.4.2B |
| Title 1 | Detailed Summary of HIV-1 RNA < 200 c/mL |
| Title 2 | Proportion of Responders at Week 24 Snapshot |
| Title 3 | By Baseline Gag Polymorphism |
| Title 4 | Treated Subjects (mITT) - Stage 2 |
| Footnote 1 | (A) Response is assessed with the snapshot algorithm, which uses the last plasma HIV-1 RNA value in the predefined visit window to classify a subject's response status. |
| Footnote 2 | (B) Includes subjects having HIV-1 RNA >= 200 c/mL within the Week 24 visit window. |
| Footnote 3 | (C) Includes subjects who discontinued due to lack of efficacy at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window. |
| Footnote 4 | (D) Includes subjects who discontinued due to any reasons except AE, death and lack of efficacy at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window and last HIV-1 RNA >= 200 c/mL. |
| Footnote 5 | (E) Includes patients who discontinued due to AE or death at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window |
| Footnote 6 | (F) Other includes: withdrew consent, loss to follow-up, moved etc. with last HIV-1 RNA < 200 c/mL |
| Layout notes | Subgroups are all combinations of baseline gag polymorphisms at selected positions |

| Parameter | Values |
|------------------|------------------------|
| Template ID | SS_VL_T_001 |
| Output File Name | rt-vl-resp200w48s1.lst |
| Purpose | WK96S1, WK96S2 |

| Table No. | Table S.5.4.1C |
|---|---|
| Title 1 | Detailed Summary of HIV-1 RNA < 200 c/mL |
| Title 2 | Proportion of Responders at Week 48 Snapshot |
| Title 3 | Treated Subjects (mITT) - Stage 1 |
| Footnote 1 | (A) Response is assessed with the snapshot algorithm, which uses the last plasma HIV-1 RNA value in the predefined visit window to classify a subject's response status. |
| Footnote 2 | (B) Includes subjects having HIV-1 RNA >= 200 c/mL within the Week 48 visit window. |
| Footnote 3 | (C) Includes subjects who discontinued due to lack of efficacy at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window. |
| Footnote 4 | (D) Includes subjects who discontinued due to any reasons except AE, death and lack of efficacy at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window and last HIV-1 RNA >= 200 c/mL. |
| Footnote 5 | (E) Includes patients who discontinued due to AE or death at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window |
| Footnote 6 | (F) Other includes: withdrew consent, loss to follow-up, moved etc. with last HIV-1 RNA < 200 c/mL |
| Layout notes | No subgroup presentation |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_001 |
| Output File Name | rt-vl-resp200w48s2.lst |
| Purpose | WK48S2, WK96S2 |
| Table No. | Table S.5.4.2C |
| Title 1 | Detailed Summary of HIV-1 RNA < 200 c/mL |
| Title 2 | Proportion of Responders at Week 48 Snapshot |
| Title 3 | Treated Subjects (mITT) - Stage 2 |
| Footnote 1 | (A) Response is assessed with the snapshot algorithm, which uses the last plasma HIV-1 RNA value in the predefined visit window to classify a subject's response status. |

| Footnote 2 | (B) Includes subjects having HIV-1 RNA >= 200 c/mL within the Week 48 visit window. |
|---|---|
| Footnote 3 | (C) Includes subjects who discontinued due to lack of efficacy at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window. |
| Footnote 4 | (D) Includes subjects who discontinued due to any reasons except AE, death and lack of efficacy at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window and last HIV-1 RNA >= 200 c/mL. |
| Footnote 5 | (E) Includes patients who discontinued due to AE or death at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window |
| Footnote 6 | (F) Other includes: withdrew consent, loss to follow-up, moved etc. with last HIV-1 RNA < 200 c/mL |
| Layout notes | No subgroup presentation |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_001 |
| Output File Name | rt-vl-resp200w48bpolys1.lst |
| Purpose | WK96S1, WK96S2 |
| Table No. | Table S.5.4.1D |
| Title 1 | Detailed Summary of HIV-1 RNA < 200 c/mL |
| Title 2 | Proportion of Responders at Week 48 Snapshot |
| Title 3 | By Baseline Gag Polymorphism |
| Title 4 | Treated Subjects (mITT) - Stage 1 |
| Footnote 1 | (A) Response is assessed with the snapshot algorithm, which uses the last plasma HIV-1 RNA value in the predefined visit window to classify a subject's response status. |
| Footnote 2 | (B) Includes subjects having HIV-1 RNA >= 200 c/mL within the Week 48 visit window. |
| Footnote 3 | (C) Includes subjects who discontinued due to lack of efficacy at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window. |
| Footnote 4 | (D) Includes subjects who discontinued due to any reasons except AE, death and lack of efficacy at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window and last HIV-1 RNA >= 200 c/mL. |

| Footnote 5 | (E) Includes patients who discontinued due to AE or death at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window |
|---|---|
| Footnote 6 | (F) Other includes: withdrew consent, loss to follow-up, moved etc. with last HIV-1 RNA < 200 c/mL |
| Layout notes | Subgroups are all combinations of baseline gag polymorphisms at selected positions |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_001 |
| Output File Name | rt-vl-resp200w48bpolys2.lst |
| Purpose | WK48S2, WK96S2 |
| Table No. | Table S.5.4.2D |
| Title 1 | Detailed Summary of HIV-1 RNA < 200 c/mL |
| Title 2 | Proportion of Responders at Week 48 Snapshot |
| Title 3 | By Baseline Gag Polymorphism |
| Title 4 | Treated Subjects (mITT) - Stage 2 |
| Footnote 1 | (A) Response is assessed with the snapshot algorithm, which uses the last plasma HIV-1 RNA value in the predefined visit window to classify a subject's response status. |
| Footnote 2 | (B) Includes subjects having HIV-1 RNA >= 200 c/mL within the Week 48 visit window. |
| Footnote 3 | (C) Includes subjects who discontinued due to lack of efficacy at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window. |
| Footnote 4 | (D) Includes subjects who discontinued due to any reasons except AE, death and lack of efficacy at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window and last HIV-1 RNA >= 200 c/mL. |
| Footnote 5 | (E) Includes patients who discontinued due to AE or death at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window |
| Footnote 6 | (F) Other includes: withdrew consent, loss to follow-up, moved etc. with last HIV-1 RNA < 200 c/mL |
| Layout notes | Subgroups are all combinations of baseline gag polymorphisms at selected positions |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_001 |
| Output File Name | rt-vl-resp200w96s1.lst |
| Purpose | WK96S1, WK96S2 |
| Table No. | Table S.5.4.1E |
| Title 1 | Detailed Summary of HIV-1 RNA < 200 c/mL |
| Title 2 | Proportion of Responders at Week 96 Snapshot |
| Title 3 | Treated Subjects (mITT) - Stage 1 |
| Footnote 1 | (A) Response is assessed with the snapshot algorithm, which uses the last plasma HIV-1 RNA value in the predefined visit window to classify a subject's response status. |
| Footnote 2 | (B) Includes subjects having HIV-1 RNA >= 200 c/mL within the Week 96 visit window. |
| Footnote 3 | (C) Includes subjects who discontinued due to lack of efficacy at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window. |
| Footnote 4 | (D) Includes subjects who discontinued due to any reasons except AE, death and lack of efficacy at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window and last HIV-1 RNA >= 200 c/mL. |
| Footnote 5 | (E) Includes patients who discontinued due to AE or death at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window |
| Footnote 6 | (F) Other includes: withdrew consent, loss to follow-up, moved etc. with last HIV-1 RNA < 200 c/mL |
| Layout notes | No subgroup presentation |

| Parameter | Values |
|------------------|------------------------|
| Template ID | SS_VL_T_001 |
| Output File Name | rt-vl-resp200w96s2.lst |
| Purpose | WK96S2 |
| Table No. | Table S.5.4.2E |

| Title 1 | Detailed Summary of HIV-1 RNA < 200 c/mL |
|---|---|
| Title 2 | Proportion of Responders at Week 96 Snapshot |
| Title 3 | Treated Subjects (mITT) - Stage 2 |
| Footnote 1 | (A) Response is assessed with the snapshot algorithm, which uses the last plasma HIV-1 RNA value in the predefined visit window to classify a subject's response status. |
| Footnote 2 | (B) Includes subjects having HIV-1 RNA >= 200 c/mL within the Week 96 visit window. |
| Footnote 3 | (C) Includes subjects who discontinued due to lack of efficacy at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window. |
| Footnote 4 | (D) Includes subjects who discontinued due to any reasons except AE, death and lack of efficacy at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window and last HIV-1 RNA >= 200 c/mL. |
| Footnote 5 | (E) Includes patients who discontinued due to AE or death at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window |
| Footnote 6 | (F) Other includes: withdrew consent, loss to follow-up, moved etc. with last HIV-1 RNA < 200 c/mL |
| Layout notes | No subgroup presentation |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_001 |
| Output File Name | rt-vl-resp200w96bpolys1.lst |
| Purpose | WK96S1, WK96S2 |
| Table No. | Table S.5.4.1F |
| Title 1 | Detailed Summary of HIV-1 RNA < 200 c/mL |
| Title 2 | Proportion of Responders at Week 96 Snapshot |
| Title 3 | By Baseline Gag Polymorphism |
| Title 4 | Treated Subjects (mITT) - Stage 1 |
| Footnote 1 | (A) Response is assessed with the snapshot algorithm, which uses the last plasma HIV-1 RNA value in the predefined visit window to classify a subject's response status. |

| Footnote 2 | (B) Includes subjects having HIV-1 RNA >= 200 c/mL within the Week 96 visit window. |
|---|---|
| Footnote 3 | (C) Includes subjects who discontinued due to lack of efficacy at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window. |
| Footnote 4 | (D) Includes subjects who discontinued due to any reasons except AE, death and lack of efficacy at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window and last HIV-1 RNA >= 200 c/mL. |
| Footnote 5 | (E) Includes patients who discontinued due to AE or death at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window |
| Footnote 6 | (F) Other includes: withdrew consent, loss to follow-up, moved etc. with last HIV-1 RNA < 200 c/mL |
| Layout notes | Subgroups are all combinations of baseline gag polymorphisms at selected positions |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_001 |
| Output File Name | rt-vl-resp200w96bpolys2.lst |
| Purpose | WK96S2 |
| Table No. | Table S.5.4.2F |
| Title 1 | Detailed Summary of HIV-1 RNA < 200 c/mL |
| Title 2 | Proportion of Responders at Week 96 Snapshot |
| Title 3 | By Baseline Gag Polymorphism |
| Title 4 | Treated Subjects (mITT) - Stage 2 |
| Footnote 1 | (A) Response is assessed with the snapshot algorithm, which uses the last plasma HIV-1 RNA value in the predefined visit window to classify a subject's response status. |
| Footnote 2 | (B) Includes subjects having HIV-1 RNA >= 200 c/mL within the Week 96 visit window. |
| Footnote 3 | (C) Includes subjects who discontinued due to lack of efficacy at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window. |
| Footnote 4 | (D) Includes subjects who discontinued due to any reasons except AE, death and lack of efficacy at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window and last HIV-1 RNA >= |

| | 200 c/mL. |
|---|---|
| Footnote 5 | (E) Includes patients who discontinued due to AE or death at any time point from Day 1 through the time window if this resulted in no virologic data on treatment during the specified window |
| Footnote 6 | (F) Other includes: withdrew consent, loss to follow-up, moved etc. with last HIV-1 RNA < 200 c/mL |
| Layout notes | Subgroups are all combinations of baseline gag polymorphisms at selected positions |

## Template SS\_VL\_T\_003: Proportion of Responders (Observed)

\_\_\_\_\_

| | Group A | Group B | Group C | Group D |
|---|---|---|---|---|
| | N = XX | N = XX | N = XX | N = XX |
| SUBGROUP 1 | | | | |
| NUMBER OF RESPONDERS (a) | XX ( XX.X) | XX ( XX.X) | XX ( XX.X) | XX ( XX.X) |
| 95% CI | (XX.X - XX.X) | (XX.X - XX.X) | (XX.X - XX.X) | (XX.X - XX.X) |
| SUBGROUP 2 | | | | |
| NUMBER OF RESPONDERS (a) | XX ( XX.X) | XX ( XX.X) | XX ( XX.X) | XX ( XX.X) |
| 95% CI | (XX.X - XX.X) | (XX.X - XX.X) | (XX.X - XX.X) | (XX.X - XX.X) |

Parameter Values Template ID  $SS_VL_T_003$ Output File Name rt-vl-resp40w24obss1.lst WK24S1, WK48S1, WK96S1, WK96S2 Purpose Table No. Table S.5.1.1D Summary of HIV-1 RNA < 40 c/mL Title 1 Title 2 Proportion of Responders at Week 24 Title 3 Treated Subjects (Observed) - Stage 1 (a) Response is assessed using the last plasma HIV-1 RNA value in the predefined visit window to classify a subject's response Footnote 1 status. No subgroup presentation Layout notes

| Parameter | Values |
|------------------|--------------------------|
| Template ID | SS_VL_T_003 |
| Output File Name | rt-vl-resp40w24obss2.lst |

| Purpose | WK24S2, WK48S2, WK96S2 |
|---|---|
| Table No. | Table S.5.1.2D |
| Title 1 | Summary of HIV-1 RNA < 40 c/mL |
| Title 2 | Proportion of Responders at Week 24 |
| Title 3 | Treated Subjects (Observed) - Stage 2 |
| Footnote 1 | (a) Response is assessed using the last plasma HIV-1 RNA value in the predefined visit window to classify a subject's response status. |
| Layout notes | No subgroup presentation |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_003 |
| Output File Name | rt-vl-resp40w24obssubgs1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.5.1.1E |
| Title 1 | Summary of HIV-1 RNA < 40 c/mL |
| Title 2 | Proportion of Responders at Week 24 |
| Title 3 | By Subgroup |
| Title 4 | Treated Subjects (Observed) - Stage 1 |
| Footnote 1 | (a) Response is assessed using the last plasma HIV-1 RNA value in the predefined visit window to classify a subject's response status. |
| Layout notes | Subgroups are: • Baseline HIV-1 RNA < 100,000 c/mL , >=100,000 c/mL • Baseline CD4 < 100, 100 to < 200, 200 to < 350, 350 to < 500, >= 500 cells/uL • Gender: Male, Female • Race: White, Black/African American, American Indian/Alaska Native, Asian, Native Hawaiian/Other Pacific Islander, Other |
| | HIV-1 Clade: Include all clades available in the database |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_003 |
| Output File Name | rt-vl-resp40w24obssubgs2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.5.1.2E |
| Title 1 | Summary of HIV-1 RNA < 40 c/mL |
| Title 2 | Proportion of Responders at Week 24 |
| Title 3 | By Subgroup |
| Title 4 | Treated Subjects (Observed) - Stage 2 |
| Footnote 1 | (a) Response is assessed using the last plasma HIV-1 RNA value in the predefined visit window to classify a subject's response status. |
| Layout notes | Subgroups are: • Baseline HIV-1 RNA < 100,000 c/mL , >=100,000 c/mL • Baseline CD4 < 100, 100 to < 200, 200 to < 350, 350 to < 500, >= 500 cells/uL • Gender: Male, Female • Race: White, Black/African American, American Indian/Alaska Native, Asian, Native Hawaiian/Other Pacific Islander, Other • HIV-1 Clade: Include all clades available in the database |

| Parameter | Values |
|------------------|--------------------------|
| Template ID | SS_VL_T_003 |
| Output File Name | rt-vl-resp40w48obss1.lst |
| Purpose | WK96S1, WK96S2 |
| Table No. | Table S.5.2.1D |

| Title 1 | Summary of HIV-1 RNA < 40 c/mL |
|---|---|
| Title 2 | Proportion of Responders at Week 48 |
| Title 3 | Treated Subjects (Observed) - Stage 1 |
| Footnote 1 | (a) Response is assessed using the last plasma HIV-1 RNA value in the predefined visit window to classify a subject's response status. |
| Layout notes | No subgroup presentation |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_003 |
| Output File Name | rt-vl-resp40w48obss2.lst |
| Purpose | WK48S2, WK96S2 |
| Table No. | Table S.5.2.2D |
| Title 1 | Summary of HIV-1 RNA < 40 c/mL |
| Title 2 | Proportion of Responders at Week 48 |
| Title 3 | Treated Subjects (Observed) - Stage 2 |
| Footnote 1 | (a) Response is assessed using the last plasma HIV-1 RNA value in the predefined visit window to classify a subject's response status. |
| Layout notes | No subgroup presentation |

| Parameter | Values |
|------------------|-------------------------------------|
| Template ID | SS_VL_T_003 |
| Output File Name | rt-vl-resp40w48obssubs1.lst |
| Purpose | WK96S1, WK96S2 |
| Table No. | Table S.5.2.1E |
| Title 1 | Summary of HIV-1 RNA < 40 c/mL |
| Title 2 | Proportion of Responders at Week 48 |

| Title 3 | By Subgroup |
|---|---|
| Title 4 | Treated Subjects (Observed) - Stage 1 |
| Footnote 1 | (a) Response is assessed using the last plasma HIV-1 RNA value in the predefined visit window to classify a subject's response status. |
| Layout notes | Subgroups are: • Baseline HIV-1 RNA < 100,000 c/mL , >=100,000 c/mL • Baseline CD4 < 100, 100 to < 200, 200 to < 350, 350 to < 500, >= 500 cells/uL • Gender: Male, Female • Race: White, Black/African American, American Indian/Alaska Native, Asian, Native Hawaiian/Other Pacific Islander, Other • HIV-1 Clade: Include all clades available in the database |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_003 |
| Output File Name | rt-vl-resp40w48obssubgs2.lst |
| Purpose | WK48S2, WK96S2 |
| Table No. | Table S.5.2.2E |
| Title 1 | Summary of HIV-1 RNA < 40 c/mL |
| Title 2 | Proportion of Responders at Week 48 |
| Title 3 | By Subgroup |
| Title 4 | Treated Subjects (Observed) - Stage 2 |
| Footnote 1 | (a) Response is assessed using the last plasma HIV-1 RNA value in the predefined visit window to classify a subject's response status. |
| Layout notes | Subgroups are: |
| | • Baseline HIV-1 RNA < 100,000 c/mL , >=100,000 c/mL |
| | • Baseline CD4 < 100, 100 to < 200, 200 to < 350, 350 to < 500, >= 500 cells/uL |
| | Gender: Male, Female |
| | Race: White, Black/African American, American Indian/Alaska Native, Asian, Native Hawaiian/Other Pacific Islander, |

| Other |
|-----------------------------------------------------------|
| HIV-1 Clade: Include all clades available in the database |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_003 |
| Output File Name | rt-vl-resp40w96obss1.lst |
| Purpose | WK96S1, WK96S2 |
| Table No. | Table S.5.3.1D |
| Title 1 | Summary of HIV-1 RNA < 40 c/mL |
| Title 2 | Proportion of Responders at Week 96 |
| Title 3 | Treated Subjects (Observed) - Stage 1 |
| Footnote 1 | (a) Response is assessed using the last plasma HIV-1 RNA value in the predefined visit window to classify a subject's response status. |
| Layout notes | No subgroup presentation |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_003 |
| Output File Name | rt-vl-resp40w96obss2.lst |
| Purpose | WK96S2 |
| Table No. | Table S.5.3.2D |
| Title 1 | Summary of HIV-1 RNA < 40 c/mL |
| Title 2 | Proportion of Responders at Week 96 |
| Title 3 | Treated Subjects (Observed) - Stage 2 |
| Footnote 1 | (a) Response is assessed using the last plasma HIV-1 RNA value in the predefined visit window to classify a subject's response status. |
| Layout notes | No subgroup presentation |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_003 |
| Output File Name | rt-vl-resp40w96obssubgs1.lst |
| Purpose | WK96S1, WK96S2 |
| Table No. | Table S.5.3.1E |
| Title 1 | Summary of HIV-1 RNA < 40 c/mL |
| Title 2 | Proportion of Responders at Week 96 |
| Title 3 | By Subgroup |
| Title 4 | Treated Subjects (Observed) - Stage 1 |
| Footnote 1 | (a) Response is assessed using the last plasma HIV-1 RNA value in the predefined visit window to classify a subject's response status. |
| Layout notes | Subgroups are: • Baseline HIV-1 RNA < 100,000 c/mL , >=100,000 c/mL |
| | • Baseline CD4 < 100, 100 to < 200, 200 to < 350, 350 to < 500, >= 500 cells/uL |
| | <ul> <li>Gender: Male, Female</li> <li>Race: White, Black/African American, American Indian/Alaska Native, Asian, Native Hawaiian/Other Pacific Islander, Other</li> </ul> |
| | HIV-1 Clade: Include all clades available in the database |

| Parameter | Values |
|------------------|-------------------------------------|
| Template ID | SS_VL_T_003 |
| Output File Name | rt-vl-resp40w96obssubgs2.lst |
| Purpose | WK96S2 |
| Table No. | Table S.5.3.2E |
| Title 1 | Summary of HIV-1 RNA < 40 c/mL |
| Title 2 | Proportion of Responders at Week 96 |

| Title 3 | By Subgroup |
|---|---|
| Title 4 | Treated Subjects (Observed) - Stage 2 |
| Footnote 1 | (a) Response is assessed using the last plasma HIV-1 RNA value in the predefined visit window to classify a subject's response status. |
| Layout notes | <ul> <li>Subgroups are:</li> <li>Baseline HIV-1 RNA &lt; 100,000 c/mL , &gt;=100,000 c/mL</li> <li>Baseline CD4 &lt; 100, 100 to &lt; 200, 200 to &lt; 350, 350 to &lt; 500, &gt;= 500 cells/uL</li> <li>Gender: Male, Female</li> <li>Race: White, Black/African American, American Indian/Alaska Native, Asian, Native Hawaiian/Other Pacific Islander, Other</li> <li>HIV-1 Clade: Include all clades available in the database</li> </ul> |

## $Template \ SS\_VL\_T\_004: Treatment \ Outcomes \ Table \ Using \ the \ TLOVR \ Algorithm$

| Outcome (%) | Trt A<br>N = XXX | Trt B<br>N = XXX |
|---|---|---|
| HIV-1 RNA < 40 C/ML (A)<br>95% CI | XXX (XXX.X)<br>(XXX.X, XXX.X) | XXX (XXX.X)<br>(XXX.X, XXX.X) |
| HIV-1 RNA >= 40 C/ML<br>VIROLOGIC REBOUND (B)<br>NEVER SUPPRESSED THROUGH WEEK 24 (C)<br>DRUG CHANGE DUE TO LACK OF EFFICACY | XXX (XXX.X)<br>XXX (XXX.X)<br>XXX (XXX.X)<br>XXX (XXX.X) | XXX (XXX.X)<br>XXX (XXX.X)<br>XXX (XXX.X)<br>XXX (XXX.X) |
| DEATH | XXX (XXX.X) | XXX (XXX.X) |
| DRUG CHANGE OR DISCONTINUATION DUE TO AE | XXX (XXX.X) | XXX (XXX.X) |
| DRUG CHANGE OR DISCONTINUATION DUE TO OTHER REASONS | XXX (XXX.X) | XXX (XXX.X) |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_004 |
| Output File Name | rt-vl-tlovr24s1.lst |
| Purpose | WK24S1 |
| Table No. | Table S.5.5.1A |
| Title 1 | Summary of Treatment Outcomes at Week 24 Using the TLOVR Algorithm |
| Title 2 | Treated Subjects - Stage 1 |
| Footnote 1 | (A) Virologic response (HIV-1 RNA < 40 c/mL at >= 2 consecutive visits) through Week 24 without intervening failure. |
| Footnote 2 | (B) Virologic response and subsequent HIV-1 RNA >= 40 c/mL at >= 2 consecutive visits or last visit followed by discontinuation of |
| Footnote 3 | study therapy through Week 24. |
| Footnote 4 | (C) Never achieved virologic response through Week 24. |

| Parameter | Values |
|-------------|-------------|
| Template ID | SS_VL_T_004 |

| Output File Name | rt-vl-tlovr24s2.lst |
|---|---|
| Purpose | WK24S2 |
| Table No. | Table S.5.5.2A |
| Title 1 | Summary of Treatment Outcomes at Week 24 Using the TLOVR Algorithm |
| Title 2 | Treated Subjects - Stage 2 |
| Footnote 1 | (A) Virologic response (HIV-1 RNA < 40 c/mL at >= 2 consecutive visits) through Week 24 without intervening failure. |
| Footnote 2 | (B) Virologic response and subsequent HIV-1 RNA >= 40 c/mL at >= 2 consecutive visits or last visit followed by discontinuation of |
| Footnote 3 | study therapy through Week 24. |
| Footnote 4 | (C) Never achieved virologic response through Week 24. |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_004 |
| Output File Name | rt-vl-tlovr48s1.lst |
| Purpose | WK48S1 |
| Table No. | Table S.5.5.1B |
| Title 1 | Summary of Treatment Outcomes at Week 48 Using the TLOVR Algorithm |
| Title 2 | Treated Subjects - Stage 1 |
| Footnote 1 | (A) Virologic response (HIV-1 RNA < 40 c/mL at >= 2 consecutive visits) through Week 48 without intervening failure. |
| Footnote 2 | (B) Virologic response and subsequent HIV-1 RNA >= 40 c/mL at >= 2 consecutive visits or last visit followed by discontinuation of |
| Footnote 3 | study therapy through Week 48. |
| Footnote 4 | (C) Never achieved virologic response through Week 48. |

| Parameter | Values |
|-------------|-------------|
| Template ID | SS_VL_T_004 |

| Output File Name | rt-vl-tlovr48s2.lst |
|---|---|
| Purpose | WK48S2 |
| Table No. | Table S.5.5.2B |
| Title 1 | Summary of Treatment Outcomes at Week 48 Using the TLOVR Algorithm |
| Title 2 | Treated Subjects - Stage 2 |
| Footnote 1 | (A) Virologic response (HIV-1 RNA < 40 c/mL at >= 2 consecutive visits) through Week 48 without intervening failure. |
| Footnote 2 | (B) Virologic response and subsequent HIV-1 RNA >= 40 c/mL at >= 2 consecutive visits or last visit followed by discontinuation of |
| Footnote 3 | study therapy through Week 48. |
| Footnote 4 | (C) Never achieved virologic response through Week 48. |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_004 |
| Output File Name | rt-vl-tlovr96s1.lst |
| Purpose | WK96S1, WK96S2 |
| Table No. | Table S.5.5.1C |
| Title 1 | Summary of Treatment Outcomes at Week 96 Using the TLOVR Algorithm |
| Title 2 | Treated Subjects - Stage 1 |
| Footnote 1 | (A) Virologic response (HIV-1 RNA < 40 c/mL at >= 2 consecutive visits) through Week 96 without intervening failure. |
| Footnote 2 | (B) Virologic response and subsequent HIV-1 RNA >= 40 c/mL at >= 2 consecutive visits or last visit followed by discontinuation of |
| Footnote 3 | study therapy through Week 96. |
| Footnote 4 | (C) Never achieved virologic response through Week 96. |

| Parameter | Values |
|-------------|-------------|
| Template ID | SS_VL_T_004 |

| Output File Name | rt-vl-tlovr96s2.lst |
|---|---|
| Purpose | WK96S2 |
| Table No. | Table S.5.5.2C |
| Title 1 | Summary of Treatment Outcomes at Week 96 Using the TLOVR Algorithm |
| Title 2 | Treated Subjects - Stage 2 |
| Footnote 1 | (A) Virologic response (HIV-1 RNA < 40 c/mL at >= 2 consecutive visits) through Week 96 without intervening failure. |
| Footnote 2 | (B) Virologic response and subsequent HIV-1 RNA >= 40 c/mL at >= 2 consecutive visits or last visit followed by discontinuation of |
| Footnote 3 | study therapy through Week 96. |
| Footnote 4 | (C) Never achieved virologic response through Week 96. |

| Parameter | Values |
|---|---|
| Template ID | SS_EX_T_002 |
| Output File Name | rt-vl-klmtlovrs1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.5.5.1D |
| Title 1 | Summary of Time to Loss of Virologic Response |
| Title 2 | Treated Subjects - Stage 1 |
| Footnote 1 | (a) Cumulative proportion without events at end of interval. |
| Layout notes | Use 4-week intervals |

| Parameter | Values |
|------------------|------------------------|
| Template ID | SS_EX_T_002 |
| Output File Name | rt-vl-klmtlovrs2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |

| Table No. | Table S.5.5.2D |
|--------------|--------------------------------------------------------------|
| Title 1 | Summary of Time to Loss of Virologic Response |
| Title 2 | Treated Subjects - Stage 2 |
| Footnote 1 | (a) Cumulative proportion without events at end of interval. |
| Layout notes | Use 4-week intervals |

| Parameter | Values |
|---|---|
| Template ID | GS_EX_G_001 |
| Output File Name | rg-vl-kmtlovrs1 |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Figure S.5.5.1E |
| Title 1 | Time to Loss of Virologic Response |
| Title 2 | Treated Subjects - Stage 1 |
| Layout notes | <ul> <li>X-axis label: Weeks</li> <li>X-axis tick labels: B/L, 4, 8, and every 4 weeks up to timepoint with data in any group</li> <li>Y-axis label: Percent Without Failure</li> <li>Y-axis ticks: 0 to 100 by 10</li> <li>Censoring symbols: none</li> </ul> |

| Parameter | Values |
|------------------|------------------------------------|
| Template ID | GS_EX_G_001 |
| Output File Name | rg-vl-kmtlovrs2 |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Figure S.5.5.2E |
| Title 1 | Time to Loss of Virologic Response |
| Title 2 | Treated Subjects - Stage 2 |
| Layout notes | X-axis label: Weeks |
|---|---|
| | • X-axis tick labels: B/L, 4, 8, and every 4 weeks up to timepoint with data in any group |
| | Y-axis label: Percent Without Failure |
| | • Y-axis ticks: 0 to 100 by 10 |
| | Censoring symbols: none |

Template SS\_VL\_T\_005: Proportion of Subjects with HIV-1 RNA within Certain Range

Group A Group B Group C Group D N = XXN = XXN = XXN = XXWeeks WEEK 1 < 40 c/mLXX (XX.X) XX (XX.X) XX (XX.X) XX ( XX.X) 40 to < 100 c/mL XX ( XX.X) XX (XX.X) XX (XX.X) XX (XX.X) 100 to < 200 c/mL XX ( XX.X) XX ( XX.X) XX ( XX.X) XX ( XX.X) 200 to < 400 c/mL XX ( XX.X) XX ( XX.X) XX ( XX.X) XX ( XX.X) > 400 c/mLXX ( XX.X) XX ( XX.X) XX ( XX.X) XX (XX.X) WEEK 2 < 40 c/mL XX (XX.X) XX ( XX.X) XX ( XX.X) XX ( XX.X) 40 to < 100 c/mL XX (XX.X) XX (XX.X) XX (XX.X) XX (XX.X) 100 to < 200 c/mL XX ( XX.X) XX ( XX.X) XX ( XX.X) XX ( XX.X) 200 to < 400 c/mL XX ( XX.X) XX ( XX.X) XX ( XX.X) XX ( XX.X) > 400 c/mLXX ( XX.X) XX ( XX.X) XX ( XX.X) XX ( XX.X) WEEK 4 < 40 c/mL XX ( XX.X)XX (XX.X) XX ( XX.X) XX ( XX.X) XX ( XX.X) XX ( XX.X) 40 to < 100 c/mL XX (XX.X) XX (XX.X) 100 to < 200 c/mL XX (XX.X) XX (XX.X) XX (XX.X) XX ( XX.X) 200 to < 400 c/mLXX ( XX.X) XX ( XX.X) XX ( XX.X) XX ( XX.X) > 400 c/mLXX ( XX.X) XX ( XX.X) XX ( XX.X) XX ( XX.X) <additional weeks> < 40 c/mL XX ( XX.X) 40 to < 100 c/mL XX (XX.X) XX (XX.X) XX ( XX.X) XX (XX.X) 100 to < 200 c/mL XX ( XX.X) XX ( XX.X) XX ( XX.X) XX ( XX.X) 200 to < 400 c/mL XX ( XX.X) XX ( XX.X) XX ( XX.X) XX ( XX.X) > 400 c/mL XX ( XX.X) XX ( XX.X) XX ( XX.X) XX ( XX.X)

| Parameter | Values |
|------------------|--------------------------------|
| Template ID | SS_VL_T_005 |
| Output File Name | rt-vl-props1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |

| Table No. | Table S.5.6.1A |
|---|---|
| Title 1 | Proportion of Subjects with HIV-1 RNA within Several Ranges |
| Title 2 | Treated Subjects (Observed) - Stage 1 |
| Programming notes | The following weeks need to be included: baseline, Week 2, 4, 8, 12, 16, 24, 32, 40, 48, 60, 72, 84 and 96. |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_005 |
| Output File Name | rt-vl-props2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.5.6.2A |
| Title 1 | Proportion of Subjects with HIV-1 RNA within Several Ranges |
| Title 2 | Treated Subjects (Observed) - Stage 2 |
| Programming notes | The following weeks need to be included: baseline, Week 2, 4, 8, 12, 16, 24, 32, 40, 48, 60, 72, 84 and 96. |

#### Template SS\_VL\_T\_006: Summary Statistics Over Time

Protocol: AIxxxXXX Page 1 of X

| Period<br>Visit | | | | Percentiles | | | Change From Baseline | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Group | N | Mean | SD | Q1 | Median | Q3 | N | Mean | SD | Q1 | Median | Q3 |
| PRE-TRT B/L Group 1 | XXX | XXX.X | XXX.XX | XXX.X | XXX.X | XXX.X | XXX | XXX.X | XXX.XX | XXX.X | XXX.X | XXX.X |
| Group 2 | XXX | XXX.X | XXX.XX | XXX.X | XXX.X | XXX.X | XXX | XXX.X | XXX.XX | XXX.X | XXX.X | XXX.X |
| ON TRT<br>WK XX | | | | | | | | | | | | |
| Group 1<br>Group 2 | XXX<br>XXX | XXX.X<br>XXX.X | XXX.XX<br>XXX.XX | XXX.X<br>XXX.X | XXX.X<br>XXX.X | XXX.X<br>XXX.X | XXX | XXX.X<br>XXX.X | XXX.XX<br>XXX.XX | XXX.X<br>XXX.X | XXX.X<br>XXX.X | XXX.X<br>XXX.X |
| <additional< td=""><td>L PERIODS A</td><td>AND VISITS</td><td>&gt;</td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td></additional<> | L PERIODS A | AND VISITS | > | | | | | | | | | |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_006 |
| Output File Name | rt-vl-sumchgs1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.5.6.1B |
| Title 1 | Summary Statistics for Values and Change from Baseline Over Time |
| Title 2 | HIV-1 RNA (log10 c/mL) |
| Title 3 | Overall and by Subgroup |
| Title 4 | Treated Subjects (Observed) - Stage 1 |
| Layout notes | The following weeks need to be included for the overall summary: baseline, Week 2, 4, 8, 12, 16, 24, 32, 40, 48, 60, 72, 84 and 96. The following weeks need to be included for the subgroup summaries: baseline, Week 24, 48 and 96. |

| | For the baseline Gag polymorphism: include also Week 4, 8 and 12. |
|---|---|
| Programming notes | Subgroups are: |
| | Baseline Gag Polymorphism |
| | Baseline Viral Load Category: HIV-1 RNA < 100,000 c/mL , >=100,000 c/mL |
| | • Baseline CD4 Category: < 100, 100 to < 200, 200 to < 350, 350 to < 500, >= 500 cells/uL |
| | Gender: Male, Female |
| | Race: White, Black/African American, American Indian/Alaska Native, Asian, Native Hawaiian/Other Pacific Islander, Other |
| | HIV-1 Clade: any clade available in the database |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_006 |
| Output File Name | rt-vl-sumchgs2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.5.6.2B |
| Title 1 | Summary Statistics for Values and Change from Baseline Over Time |
| Title 2 | HIV-1 RNA (log10 c/mL) |
| Title 3 | Overall and by Subgroup |
| Title 4 | Treated Subjects (Observed) - Stage 2 |
| Layout notes | The following weeks need to be included for the overall summary: baseline, Week 2, 4, 8, 12, 16, 24, 32, 40, 48, 60, 72, 84 and 96. The following weeks need to be included for the subgroup summaries: baseline, Week 24, 48 and 96. For the baseline Gag polymorphism: include also Week 4, 8 and 12. |
| Programming notes | <ul> <li>Subgroups are:</li> <li>Baseline Gag Polymorphism</li> <li>Baseline Viral Load Category: HIV-1 RNA &lt; 100,000 c/mL ,&gt;=100,000 c/mL</li> <li>Baseline CD4 Category: &lt; 100, 100 to &lt; 200, 200 to &lt; 350, 350 to &lt; 500, &gt;= 500 cells/uL</li> <li>Gender: Male, Female</li> <li>Race: White, Black/African American, American Indian/Alaska Native, Asian, Native Hawaiian/Other Pacific Islander, Other</li> <li>HIV-1 Clade: any clade available in the database</li> </ul> |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_006 |
| Output File Name | rt-lb-cd4s1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.5.7.1A |
| Title 1 | Summary Statistics for Values and Change from Baseline Over Time |
| Title 2 | CD4 Cell Count (cells/uL) |
| Title 3 | Overall and by Subgroup |
| Title 4 | Treated Subjects (Observed) - Stage 1 |
| Layout notes | The following weeks need to be included for the overall summary: baseline, Week 2, 4, 8, 12, 16, 24, 32, 40, 48, 60, 72, 84 and 96. The following weeks need to be included for the subgroup summaries: baseline, Week 24, 48 and 96. |
| Programming notes | Subgroups are: |
| | Baseline Viral Load Category: HIV-1 RNA < 100,000 c/mL , >=100,000 c/mL |
| | • Baseline CD4 Category: < 100, 100 to < 200, 200 to < 350, 350 to < 500, >= 500 cells/uL |
| | Gender: Male, Female |
| | Race: White, Black/African American, American Indian/Alaska Native, Asian, Native Hawaiian/Other Pacific Islander, Other |
| | HIV-1 Clade: any clade available in the database |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_006 |
| Output File Name | rt-lb-cd4s2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.5.7.2A |
| Title 1 | Summary Statistics for Values and Change from Baseline Over Time |
| Title 2 | CD4 Cell Count (cells/uL) |

| Title 3 | Overall and by Subgroup |
|---|---|
| Title 4 | Treated Subjects (Observed) - Stage 2 |
| Layout notes | The following weeks need to be included for the overall summary: baseline, Week 2, 4, 8, 12, 16, 24, 32, 40, 48, 60, 72, 84 and 96. |
| | The following weeks need to be included for the subgroup summaries: baseline, Week 24, 48 and 96. |
| Programming notes | Subgroups are: |
| | Baseline Viral Load Category: HIV-1 RNA < 100,000 c/mL , >=100,000 c/mL |
| | • Baseline CD4 Category: < 100, 100 to < 200, 200 to < 350, 350 to < 500, >= 500 cells/uL |
| | Gender: Male, Female |
| | Race: White, Black/African American, American Indian/Alaska Native, Asian, Native Hawaiian/Other Pacific Islander, Other |
| | HIV-1 Clade: any clade available in the database |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_006 |
| Output File Name | rt-lb-cd4pcts1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.5.8.1A |
| Title 1 | Summary Statistics for Values and Change from Baseline Over Time |
| Title 2 | CD4 Cell Percentage |
| Title 3 | Overall and by Subgroup |
| Title 4 | Treated Subjects (Observed) - Stage 1 |
| Layout notes | The following weeks need to be included for the overall summary: baseline, Week 2, 4, 8, 12, 16, 24, 32, 40, 48, 60, 72, 84 and 96. The following weeks need to be included for the subgroup summaries: baseline, Week 24, 48 and 96. |
| Programming notes | Subgroups are: |
| | Baseline Viral Load Category: HIV-1 RNA < 100,000 c/mL , >=100,000 c/mL |
| | • Baseline CD4 Category: < 100, 100 to < 200, 200 to < 350, 350 to < 500, >= 500 cells/uL |
| | Gender: Male, Female |
| | Race: White, Black/African American, American Indian/Alaska Native, Asian, Native Hawaiian/Other Pacific Islander, Other |

HIV-1 Clade: any clade available in the database

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_006 |
| Output File Name | rt-lb-cd4pcts2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.5.8.2A |
| Title 1 | Summary Statistics for Values and Change from Baseline Over Time |
| Title 2 | CD4 Cell Percentage |
| Title 3 | Overall and by Subgroup |
| Title 4 | Treated Subjects (Observed) - Stage 2 |
| Layout notes | The following weeks need to be included for the overall summary: baseline, Week 2, 4, 8, 12, 16, 24, 32, 40, 48, 60, 72, 84 and 96. The following weeks need to be included for the subgroup summaries: baseline, Week 24, 48 and 96. |
| Programming notes | Subgroups are: |
| | Baseline Viral Load Category: HIV-1 RNA < 100,000 c/mL , >=100,000 c/mL |
| | • Baseline CD4 Category: < 100, 100 to < 200, 200 to < 350, 350 to < 500, >= 500 cells/uL |
| | Gender: Male, Female |
| | Race: White, Black/African American, American Indian/Alaska Native, Asian, Native Hawaiian/Other Pacific Islander, Other |
| | HIV-1 Clade: any clade available in the database |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_006 |
| Output File Name | rt-lb-cd8s1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.5.9.1A |
| Title 1 | Summary Statistics for Values and Change from Baseline Over Time |

| Title 2 | CD8 Cell Count (cells/ul) |
|---|---|
| Title 3 | Overall and by Subgroup |
| Title 4 | Treated Subjects (Observed) - Stage 1 |
| Layout notes | The following weeks need to be included for the overall summary: baseline, Week 2, 4, 8, 12, 16, 24, 32, 40, 48, 60, 72, 84 and 96. The following weeks need to be included for the subgroup summaries: baseline, Week 24, 48 and 96. |
| Programming notes | <ul> <li>Subgroups are:</li> <li>Baseline Viral Load Category: HIV-1 RNA &lt; 100,000 c/mL , &gt;=100,000 c/mL</li> <li>Baseline CD4 Category: &lt; 100, 100 to &lt; 200, 200 to &lt; 350, 350 to &lt; 500, &gt;= 500 cells/uL</li> <li>Gender: Male, Female</li> <li>Race: White, Black/African American, American Indian/Alaska Native, Asian, Native Hawaiian/Other Pacific Islander, Other</li> <li>HIV-1 Clade: any clade available in the database</li> </ul> |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_006 |
| Output File Name | rt-lb-cd8s2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.5.9.2A |
| Title 1 | Summary Statistics for Values and Change from Baseline Over Time |
| Title 2 | CD8 Cell Count (cells/ul) |
| Title 3 | Overall and by Subgroup |
| Title 4 | Treated Subjects (Observed) - Stage 2 |
| Layout notes | The following weeks need to be included for the overall summary: baseline, Week 2, 4, 8, 12, 16, 24, 32, 40, 48, 60, 72, 84 and 96. The following weeks need to be included for the subgroup summaries: baseline, Week 24, 48 and 96. |
| Programming notes | Subgroups are: Baseline Viral Load Category: HIV-1 RNA < 100,000 c/mL , >=100,000 c/mL Baseline CD4 Category: < 100, 100 to < 200, 200 to < 350, 350 to < 500, >= 500 cells/uL Gender: Male, Female |

| • Race: White, Black/African American, American Indian/Alaska Native, Asian, Native Hawaiian/Other Pacific Islander, Other |
|---|
| HIV-1 Clade: any clade available in the database |

#### Template GS LB G 001: Box Plot



Duration computed as the difference between the last and first short-term dosing date plus on Program Path: /home/banckenf/sgtest/boxplot Program Name: box1.sas RUN DATE: 11SEP2008:15:29:12

| Parameter | Values |
|------------------|--------------------------------|
| Template ID | GS_LB_G_001 |
| Output File Name | rg-vl-box24s1 |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Figure S.5.6.1C |

| Title 1 | HIV-1 RNA (log10 c/mL) Change from Baseline to Week 24 |
|---|---|
| Title 2 | Treated Subjects - Stage 1 |
| Footnote 1 | N is the number of subjects with data at baseline and at Week 24. |
| Layout notes | Y-axis label: HIV-1 RNA Change from Baseline (log10 c/mL) |
| | X-axis label: Treatment Group |

| Parameter | Values |
|---|---|
| Template ID | GS_LB_G_001 |
| Output File Name | rg-vl-box24s2 |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Figure S.5.6.2C |
| Title 1 | HIV-1 RNA (log10 c/mL) Change from Baseline to Week 24 |
| Title 2 | Treated Subjects - Stage 2 |
| Footnote 1 | N is the number of subjects with data at baseline and at Week 24. |
| Layout notes | Y-axis label: HIV-1 RNA Change from Baseline (log10 c/mL) X-axis label: Treatment Group |

| Parameter | Values |
|---|---|
| Template ID | GS_LB_G_001 |
| Output File Name | rg-vl-box48s1 |
| Purpose | WK96S1, WK96S2 |
| Table No. | Figure S.5.6.1D |
| Title 1 | HIV-1 RNA (log10 c/mL) Change from Baseline to Week 48 |
| Title 2 | Treated Subjects - Stage 1 |
| Footnote 1 | N is the number of subjects with data at baseline and at Week 48. |

| Layout notes | Y-axis label: HIV-1 RNA Change from Baseline (log10 c/mL) |
|--------------|-----------------------------------------------------------|
| | X-axis label: Treatment Group |

| Parameter | Values |
|---|---|
| Template ID | GS_LB_G_001 |
| Output File Name | rg-vl-box48s2 |
| Purpose | WK48S2, WK96S2 |
| Table No. | Figure S.5.6.2D |
| Title 1 | HIV-1 RNA (log10 c/mL) Change from Baseline to Week 48 |
| Title 2 | Treated Subjects - Stage 2 |
| Footnote 1 | N is the number of subjects with data at baseline and at Week 48. |
| Layout notes | Y-axis label: HIV-1 RNA Change from Baseline (log10 c/mL) |
| | X-axis label: Treatment Group |

| Parameter | Values |
|---|---|
| Template ID | GS_LB_G_001 |
| Output File Name | rg-vl-box96s1 |
| Purpose | WK96S1, WK96S2 |
| Table No. | Figure S.5.6.1E |
| Title 1 | HIV-1 RNA (log10 c/mL) Change from Baseline to Week 96 |
| Title 2 | Treated Subjects - Stage 1 |
| Footnote 1 | N is the number of subjects with data at baseline and at Week 96. |
| Layout notes | Y-axis label: HIV-1 RNA Change from Baseline (log10 c/mL) X-axis label: Treatment Group |

| Parameter | Values |
|---|---|
| Template ID | GS_LB_G_001 |
| Output File Name | rg-vl-box96s2 |
| Purpose | WK96S2 |
| Table No. | Figure S.5.6.2E |
| Title 1 | HIV-1 RNA (log10 c/mL) Change from Baseline to Week 96 |
| Title 2 | Treated Subjects - Stage 2 |
| Footnote 1 | N is the number of subjects with data at baseline and at Week 96. |
| Layout notes | Y-axis label: HIV-1 RNA Change from Baseline (log10 c/mL) |
| | X-axis label: Treatment Group |

| Parameter | Values |
|---|---|
| Template ID | GS_LB_G_001 |
| Output File Name | rg-lb-cd4box24s1 |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Figure S.5.7.1B |
| Title 1 | CD4 Cell Count (cells/uL) Change from Baseline to Week 24 |
| Title 2 | Treated Subjects - Stage 1 |
| Footnote 1 | N is the number of subjects with data at baseline and at Week 24. |
| Layout notes | Y-axis label: CD4 Cell Count Change from Baseline (cells/uL) |
| | X-axis label: Treatment Group |

| Parameter | Values |
|------------------|------------------|
| Template ID | GS_LB_G_001 |
| Output File Name | rg-lb-cd4box24s2 |

| Purpose | WK24S2, WK48S2, WK96S2 |
|---|---|
| Table No. | Figure S.5.7.2B |
| Title 1 | CD4 Cell Count (cells/uL) Change from Baseline to Week 24 |
| Title 2 | Treated Subjects - Stage 2 |
| Footnote 1 | N is the number of subjects with data at baseline and at Week 24. |
| Layout notes | Y-axis label: CD4 Cell Count Change from Baseline (cells/uL) |
| | X-axis label: Treatment Group |

| Parameter | Values |
|---|---|
| Template ID | GS_LB_G_001 |
| Output File Name | rg-lb-cd4box48s1 |
| Purpose | WK96S1, WK96S2 |
| Table No. | Figure S.5.7.1C |
| Title 1 | CD4 Cell Count (cells/uL) Change from Baseline to Week 48 |
| Title 2 | Treated Subjects - Stage 1 |
| Footnote 1 | N is the number of subjects with data at baseline and at Week 48. |
| Layout notes | Y-axis label: CD4 Cell Count Change from Baseline (cells/uL) X-axis label: Treatment Group |

| Parameter | Values |
|------------------|-----------------------------------------------------------|
| Template ID | GS_LB_G_001 |
| Output File Name | rg-lb-cd4box48s2 |
| Purpose | WK48S2, WK96S2 |
| Table No. | Figure S.5.7.2C |
| Title 1 | CD4 Cell Count (cells/uL) Change from Baseline to Week 48 |

| Title 2 | Treated Subjects - Stage 2 |
|---|---|
| Footnote 1 | N is the number of subjects with data at baseline and at Week 48. |
| Layout notes | Y-axis label: CD4 Cell Count Change from Baseline (cells/uL) |
| | X-axis label: Treatment Group |

| Values |
|---|
| GS_LB_G_001 |
| rg-lb-cd4box96s1 |
| WK96S1, WK96S2 |
| Figure S.5.7.1D |
| CD4 Cell Count (cells/uL) Change from Baseline to Week 96 |
| Treated Subjects - Stage 1 |
| N is the number of subjects with data at baseline and at Week 96. |
| Y-axis label: CD4 Cell Count Change from Baseline (cells/uL) X-axis label: Treatment Group |

| Parameter | Values |
|---|---|
| Template ID | GS_LB_G_001 |
| Output File Name | rg-lb-cd4box96s2 |
| Purpose | WK96S2 |
| Table No. | Figure S.5.7.2D |
| Title 1 | CD4 Cell Count (cells/uL) Change from Baseline to Week 96 |
| Title 2 | Treated Subjects - Stage 2 |
| Footnote 1 | N is the number of subjects with data at baseline and at Week 96. |
| Layout notes | Y-axis label: CD4 Cell Count Change from Baseline (cells/uL) X-axis label: Treatment Group |

| Parameter | Values |
|---|---|
| Template ID | GS_LB_G_001 |
| Output File Name | rg-lb-cd8box24s1 |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Figure S.5.9.1B |
| Title 1 | CD8 Cell Count (cells/uL) Change from Baseline to Week 24 |
| Title 2 | Treated Subjects -Stage 1 |
| Footnote 1 | N is the number of subjects with data at baseline and at Week 24. |
| Layout notes | Y-axis label: CD8 Cell Count Change from Baseline (cells/uL) |
| | X-axis label: Treatment Group |

| Parameter | Values |
|---|---|
| Template ID | GS_LB_G_001 |
| Output File Name | rg-lb-cd8box24s2 |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Figure S.5.9.2B |
| Title 1 | CD8 Cell Count (cells/uL) Change from Baseline to Week 24 |
| Title 2 | Treated Subjects -Stage 2 |
| Footnote 1 | N is the number of subjects with data at baseline and at Week 24. |
| Layout notes | Y-axis label: CD8 Cell Count Change from Baseline (cells/uL) |
| | X-axis label: Treatment Group |

| Parameter | Values |
|-------------|-------------|
| Template ID | GS_LB_G_001 |

| Output File Name | rg-lb-cd8box48s1 |
|---|---|
| Purpose | WK96S1, WK96S2 |
| Table No. | Figure S.5.9.1C |
| Title 1 | CD8 Cell Count (cells/uL) Change from Baseline to Week 48 |
| Title 2 | Treated Subjects - Stage 1 |
| Footnote 1 | N is the number of subjects with data at baseline and at Week 48. |
| Layout notes | Y-axis label: CD8 Cell Count Change from Baseline (cells/uL) |
| | X-axis label: Treatment Group |

| Parameter | Values |
|---|---|
| Template ID | GS_LB_G_001 |
| Output File Name | rg-lb-cd8box48s2 |
| Purpose | WK48S2, WK96S2 |
| Table No. | Figure S.5.9.2C |
| Title 1 | CD8 Cell Count (cells/uL) Change from Baseline to Week 48 |
| Title 2 | Treated Subjects - Stage 2 |
| Footnote 1 | N is the number of subjects with data at baseline and at Week 48. |
| Layout notes | Y-axis label: CD8 Cell Count Change from Baseline (cells/uL) |
| | X-axis label: Treatment Group |

| Parameter | Values |
|------------------|------------------|
| Template ID | GS_LB_G_001 |
| Output File Name | rg-lb-cd8box96s1 |
| Purpose | WK96S1, WK96S2 |
| Table No. | Figure S.5.9.1D |

| Title 1 | CD8 Cell Count (cells/uL) Change from Baseline to Week 96 |
|---|---|
| Title 2 | Treated Subjects - Stage 1 |
| Footnote 1 | N is the number of subjects with data at baseline and at Week 96. |
| Layout notes | Y-axis label: CD8 Cell Count Change from Baseline (cells/uL) |
| | X-axis label: Treatment Group |

| Parameter | Values |
|---|---|
| Template ID | GS_LB_G_001 |
| Output File Name | rg-lb-cd8box96s2 |
| Purpose | WK96S2 |
| Table No. | Figure S.5.9.2D |
| Title 1 | CD8 Cell Count (cells/uL) Change from Baseline to Week 96 |
| Title 2 | Treated Subjects - Stage 2 |
| Footnote 1 | N is the number of subjects with data at baseline and at Week 96. |
| Layout notes | Y-axis label: CD8 Cell Count Change from Baseline (cells/uL) |
| | X-axis label: Treatment Group |

Template GS\_L\_G\_002: Longitudinal Line Plot Grouped by Treatment with Horizontal Shift and Reference Line



| Parameter | Values |
|---|---|
| Template ID | GS_LB_G_002 |
| Output File Name | rg-vl-times1 |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Figure S.5.6.1F |
| Title 1 | HIV-1 RNA (log10 c/mL) Mean Change from Baseline Over Time |
| Title 2 | Treated Subjects - Stage 1 |
| Layout notes | Y-axis label: HIV-1 RNA (log10 c/mL) Mean Change from Baseline (SE) |
| | X-axis label: Time (Weeks) |
| | Include horizontal reference line at Y=0. |

| Parameter | Values |
|-----------|--------|
|-----------|--------|

| Template ID | GS_LB_G_002 |
|---|---|
| Output File Name | rg-vl-times2 |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Figure S.5.6.2F |
| Title 1 | HIV-1 RNA (log10 c/mL) Mean Change from Baseline Over Time |
| Title 2 | Treated Subjects - Stage 2 |
| Layout notes | Y-axis label: HIV-1 RNA (log10 c/mL) Mean Change from Baseline (SE) |
| | X-axis label: Time (Weeks) |
| | Include horizontal reference line at Y=0. |

| Parameter | Values |
|------------------|----------------------------------------------------|
| Template ID | GS_LB_G_002 |
| Output File Name | rg-lb-cd4times1 |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Figure S.5.7.1E |
| Title 1 | CD4 (cells/uL) Mean Change from Baseline Over Time |
| Title 2 | Treated Subjects - Stage 1 |
| Layout notes | Y-axis label: CD4 Mean Change from Baseline (SE) |
| | X-axis label: Time (Weeks) |
| | Include horizontal reference line at Y=0. |

| Parameter | Values |
|------------------|------------------------|
| Template ID | GS_LB_G_002 |
| Output File Name | rg-lb-cd4times2 |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Figure S.5.7.2E |

| Title 1 | CD4 (cells/uL) Mean Change from Baseline Over Time |
|--------------|----------------------------------------------------|
| Title 2 | Treated Subjects - Stage 2 |
| Layout notes | Y-axis label: CD4 Mean Change from Baseline (SE) |
| | X-axis label: Time (Weeks) |
| | Include horizontal reference line at Y=0. |

| Parameter | Values |
|------------------|----------------------------------------------------|
| Template ID | GS_LB_G_002 |
| Output File Name | rg-lb-cd8times1 |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Figure S.5.9.1E |
| Title 1 | CD8 (cells/uL) Mean Change from Baseline Over Time |
| Title 2 | Treated Subjects - Stage 1 |
| Layout notes | Y-axis label: CD8 Mean Change from Baseline (SE) |
| | X-axis label: Time (Weeks) |
| | Include horizontal reference line at Y=0. |

| Parameter | Values |
|---|---|
| Template ID | GS_LB_G_002 |
| Output File Name | rg-lb-cd8times2 |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Figure S.5.9.2E |
| Title 1 | CD8 (cells/uL) Mean Change from Baseline Over Time |
| Title 2 | Treated Subjects - Stage 2 |
| Layout notes | Y-axis label: CD8 Mean Change from Baseline (SE) X-axis label: Time (Weeks) |

| Include horizontal reference line at Y=0. |
|-------------------------------------------|

## Template SS\_VL\_L\_004: Listing of Outcomes from Snapshot Analysis

\_\_\_\_\_

| Subject ID<br>(Age/Gender/Race | Randomized<br>) Treatment Group | Assessment Day<br>HIV-1 RNA (c/m | Response<br>L) | Specification | Disc.<br>Day | Disc.<br>Reason |
|---|---|---|---|---|---|---|
| <b>PPD</b> 25/M/C | BMS-986001 600 mg QD/<br>EFV/3TC | 01FEB2013/<br>8754 | NO VIROLOGIC DATA | DISC. STUDY/STUDY DRUG<br>DUE TO AE OR DEATH | 10FEB2013 | OTHER |
| PPD<br>24/F/B | BMS-986001 1200 mg QD/<br>EFV/3TC | / 20DEC2012<br><40 | RESPONDER | | | |
| PPD<br>26/M/C | BMS-986001 600 mg QD/<br>EFV/3TC | 01MAR2013<br>1350 | VIROLOGIC FAILURE | HIV-1 RNA >= 40 c/mL | | |

\_\_\_\_\_\_

| Parameter | Values |
|---|---|
| Template ID | SS_VL_L_004 |
| Output File Name | rl-vl-outcome24s1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Appendix 5.1.1A |
| Title 1 | Listing of Outcomes from HIV-1 RNA < 40 c/mL Snapshot Analysis |
| Title 2 | Data for Subjects in the Week 24 Snapshot |
| Title 3 | Treated Subjects - Stage 1 |
| Footnote 1 | HIV-1 RNA assessments used for the response evaluation are listed. |
| Programming notes | Listing should be sorted by Treatment group, response and specification. |

| Parameter | Values |
|------------------|------------------------|
| Template ID | SS_VL_L_004 |
| Output File Name | rl-vl-outcome24s2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |

| Table No. | Appendix 5.1.2A |
|---|---|
| Title 1 | Listing of Outcomes from HIV-1 RNA < 40 c/mL Snapshot Analysis |
| Title 2 | Data for Subjects in the Week 24 Snapshot |
| Title 3 | Treated Subjects - Stage 2 |
| Footnote 1 | HIV-1 RNA assessments used for the response evaluation are listed. |
| Programming notes | Listing should be sorted by Treatment group, response and specification. |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_L_004 |
| Output File Name | rl-vl-outcome48s1.lst |
| Purpose | WK96S1, WK96S2 |
| Table No. | Appendix 5.1.1B |
| Title 1 | Listing of Outcomes from HIV-1 RNA < 40 c/mL Snapshot Analysis |
| Title 2 | Data for Subjects in the Week 48 Snapshot |
| Title 3 | Treated Subjects - Stage 1 |
| Footnote 1 | HIV-1 RNA assessments used for the response evaluation are listed. |
| Programming notes | Listing should be sorted by Treatment group, response and specification. |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_L_004 |
| Output File Name | rl-vl-outcome48s2.lst |
| Purpose | WK48S2, WK96S2 |
| Table No. | Appendix 5.1.2B |
| Title 1 | Listing of Outcomes from HIV-1 RNA < 40 c/mL Snapshot Analysis |

| Title 2 | Data for Subjects in the Week 48 Snapshot |
|---|---|
| Title 3 | Treated Subjects - Stage 2 |
| Footnote 1 | HIV-1 RNA assessments used for the response evaluation are listed. |
| Programming notes | Listing should be sorted by Treatment group, response and specification. |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_L_004 |
| Output File Name | rl-vl-outcome96s1.lst |
| Purpose | WK96S1, WK96S2 |
| Table No. | Appendix 5.1.1C |
| Title 1 | Listing of Outcomes from HIV-1 RNA < 40 c/mL Snapshot Analysis |
| Title 2 | Data for Subjects in the Week 96 Snapshot |
| Title 3 | Treated Subjects - Stage 1 |
| Footnote 1 | HIV-1 RNA assessments used for the response evaluation are listed. |
| Programming notes | Listing should be sorted by Treatment group, response and specification. |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_L_004 |
| Output File Name | rl-vl-outcome96s2.lst |
| Purpose | WK96S2 |
| Table No. | Appendix 5.1.2C |
| Title 1 | Listing of Outcomes from HIV-1 RNA < 40 c/mL Snapshot Analysis |
| Title 2 | Data for Subjects in the Week 96 Snapshot |
| Title 3 | Treated Subjects - Stage 2 |
| Footnote 1 | HIV-1 RNA assessments used for the response evaluation are listed. |

| Programming notes | Listing should be sorted by Treatment group, response and specification. |
|---|---|

# $Template \ SS\_VL\_L\_005: Listing \ of \ Viral \ Load$

Treatment Group: DRUG A

| Subject ID<br>(Age/Gender/Race) | Current<br>Treatment | Period | Visit | Lab<br>Date | Treatment<br>Start<br>Study Day | HIV-1 RNA<br>(c/mL) | HIV-1 RNA<br>(log10 c/mL) | Assay |
|---|---|---|---|---|---|---|---|---|
| <br>PPD<br>(56/M/C) | DRUG A 250 MG DRUG A 300 MG DRUG A 200 MG DRUG A 200 MG | SCRN ON TRT ON TRT ON TRT ON TRT | A00<br>B01<br>B02<br>B03<br>B04 | PPD | -16<br>1<br>25<br>30<br>30 | 1500000<br>45000<br>23000<br>450<br>45 | 6.18<br>4.65<br>4.36<br>2.65<br>1.65 | U<br>S<br>U<br>S |
| PPD<br>(56/M/C) | DRUG A 250 MG DRUG A 300 MG DRUG A 200 MG DRUG A 300 MG DRUG A 200 MG DRUG A 200 MG DRUG A 200 MG DRUG A 300 MG DRUG A 200 MG DRUG A 200 MG DRUG A 200 MG DRUG A 200 MG DRUG A 200 MG | SCRN ON TRT | A00<br>B01<br>B02<br>B03<br>B02<br>B03<br>B04<br>B05<br>B06<br>B06 | | -16<br>1<br>2<br>5<br>6<br>7<br>36<br>62<br>90<br>118<br>146 | 1500000<br>45000<br>23000<br>450<br>23000<br>450<br>45<br>23000<br>450<br>45<br>45<br>45 | 6.18<br>4.65<br>4.36<br>2.65<br>4.36<br>2.65<br>1.65<br>4.36<br>2.65<br>1.65 | U<br>U<br>U<br>S<br>U<br>U<br>U<br>S<br>A<br>A |

ASSAY: S = ROCHE AMPLICOR STANDARD ASSAY U = ROCHE AMPLICOR ULTRA-SENSITIVE ASSAY A = ABBOTT REALTIME M2000 ASSAY

| Parameter | Values |
|------------------|--------------------------------|
| Template ID | SS_VL_L_005 |
| Output File Name | rl-vl-vllists1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Appendix 5.1.1D |
| Title 1 | Listing of HIV-1 RNA |
| Title 2 | Treated Subjects - Stage 1 |

| Parameter | Values |
|-----------|--------|
|-----------|--------|

| Template ID | SS_VL_L_005 |
|------------------|----------------------------|
| Output File Name | rl-vl-vllists2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Appendix 5.1.2D |
| Title 1 | Listing of HIV-1 RNA |
| Title 2 | Treated Subjects - Stage 2 |

## Template SS\_LB\_L\_002: Listing of CD4 and CD8

Treatment Group: DRUG A

| Subject<br>(Age/Gender/Race) | Period | Visit | Lab | Treatment<br>Start<br>Study Day | CD4+<br>(cells/ul) | CD4+<br>percentage | CD8+<br>(cells/ul) | CD8+<br>percentage |
|---|---|---|---|---|---|---|---|---|
| PPD (38/M/B) | PRE-TREATMENT STAGE 1 STAGE 2 STAGE 2 STAGE 2 | | PPD | -34 8 21 35 62 91 119 145 173 226 285 349 394 453 511 567 622 679 758 848 926 | 557 633 633 583 594 628 650 743 710 642 615 696 727 644 696 630 845 784 772 936 780 | 30.0<br>31.0<br>31.0<br>32.0<br>30.0<br>39.0<br>40.0<br>38.0<br>42.0<br>40.0<br>45.0<br>46.0<br>44.0<br>51.0<br>47.0<br>48.0<br>47.0 | 937 1025 998 842 844 660 613 761 571 567 503 506 515 443 465 399 474 479 491 555 479 | 51.0<br>51.0<br>49.0<br>46.0<br>43.0<br>40.0<br>38.0<br>39.0<br>34.0<br>35.0<br>34.0<br>33.0<br>31.0<br>28.0<br>29.0<br>29.0<br>29.0<br>29.0<br>29.0 |
| | STAGE 2 | WEEK 144 | | 1043 | 798 | 49.0 | 448 | 27.0 |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_L_005 |
| Output File Name | rl-lb-cd4cd8s1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Appendix 5.1.1E |
| Title 1 | Listing of CD4+ and CD8+ T-Cell Count and Percentages |
| Title 2 | Treated Subjects - Stage 1 |

| Parameter | Values |
|------------------|-------------------------------------------------------|
| Template ID | SS_VL_L_005 |
| Output File Name | rl-lb-cd4cd8s2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Appendix 5.1.2E |
| Title 1 | Listing of CD4+ and CD8+ T-Cell Count and Percentages |
| Title 2 | Treated Subjects - Stage 2 |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_001 |
| Output File Name | rt-gn-news1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.5.10.1A |
| Title 1 | Newly Emergent Genotypic Resistance Profile |
| Title 2 | Treated Subjects with On-Treatment Genotypic Resistance Testing - Stage 1 |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_001 |
| Output File Name | rt-gn-news2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.5.10.2A |
| Title 1 | Newly Emergent Genotypic Resistance Profile |
| Title 2 | Treated Subjects with On-Treatment Genotypic Resistance Testing - Stage 2 |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_001 |
| Output File Name | rt-gn-news12.lst |
| Purpose | WK96S2 |
| Table No. | Table S.5.10.3A |
| Title 1 | Newly Emergent Genotypic Resistance Profile |
| Title 2 | Treated Subjects with On-Treatment Genotypic Resistance Testing - Stage 1 and 2 |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_001 |
| Output File Name | rt-gn-newpdvfs1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.5.10.1B |
| Title 1 | Newly Emergent Genotypic Resistance Profile |
| Title 2 | Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 1 |
| Footnote 1 | Protocol Defined Virologic Failure is defined by a subject meeting one of the following criteria: |
| Footnote 2 | 1) Confirmed > 1 log <sub>10</sub> c/mL increase in HIV-1 RNA at anytime above nadir level where nadir is ≥ 40 c/mL |
| Footnote 3 | 2) Confirmed HIV-1 RNA ≥ 40 c/mL if prior suppression to < 40 c/mL |
| Footnote 4 | 3) Failure to have the last on-treatment HIV-1 RNA to < 400 c/mL within Week 24, 48, or 96 week snapshot window |
| Footnote 5 | 4) Failure to achieve > 1 log <sub>10</sub> c/mL decrease in HIV-1 RNA by Week 8 |

| Parameter | Values |
|------------------|------------------------|
| Template ID | SS_GN_T_001 |
| Output File Name | rt-gn-newpdvfs2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |

| Table No. | Table S.5.10.2B |
|---|---|
| Title 1 | Newly Emergent Genotypic Resistance Profile |
| Title 2 | Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 2 |
| Footnote 1 | Protocol Defined Virologic Failure is defined by a subject meeting one of the following criteria: |
| Footnote 2 | 1) Confirmed > 1 log <sub>10</sub> c/mL increase in HIV-1 RNA at anytime above nadir level where nadir is ≥ 40 c/mL |
| Footnote 3 | 2) Confirmed HIV-1 RNA ≥ 40 c/mL if prior suppression to < 40 c/mL |
| Footnote 4 | 3) Failure to have the last on-treatment HIV-1 RNA to < 400 c/mL within Week 24, 48, or 96 week snapshot window |
| Footnote 5 | 4) Failure to achieve > 1 log <sub>10</sub> c/mL decrease in HIV-1 RNA by Week 8 |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_001 |
| Output File Name | rt-gn-newpdvfs12.lst |
| Purpose | WK96S2 |
| Table No. | Table S.5.10.3B |
| Title 1 | Newly Emergent Genotypic Resistance Profile |
| Title 2 | Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 1 and 2 |
| Footnote 1 | Protocol Defined Virologic Failure is defined by a subject meeting one of the following criteria: |
| Footnote 2 | 1) Confirmed > 1 log <sub>10</sub> c/mL increase in HIV-1 RNA at anytime above nadir level where nadir is ≥ 40 c/mL |
| Footnote 3 | 2) Confirmed HIV-1 RNA ≥ 40 c/mL if prior suppression to < 40 c/mL |
| Footnote 4 | 3) Failure to have the last on-treatment HIV-1 RNA to < 400 c/mL within Week 24, 48, or 96 week snapshot window |
| Footnote 5 | 4) Failure to achieve > 1 log <sub>10</sub> c/mL decrease in HIV-1 RNA by Week 8 |

| Parameter | Values |
|------------------|-------------------|
| Template ID | SS_GN_L_001 |
| Output File Name | rl-gn-ontrts1.lst |

| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
|-----------|----------------------------------------------------------------|
| Table No. | Appendix 5.10.1A |
| Title 1 | Listing of Genotypic Substitutions |
| Title 2 | Treated Subjects with Baseline and On-Treatment Data - Stage 1 |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_L_001 |
| Output File Name | rl-gn-ontrts2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Appendix 5.10.2A |
| Title 1 | Listing of Genotypic Substitutions |
| Title 2 | Treated Subjects with Baseline and On-Treatment Data - Stage 2 |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_002 |
| Output File Name | rt-gn-newgags1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.5.10.1C |
| Title 1 | Emergent Gag Polymorphisms at Selected Positions |
| Title 2 | Treated Subjects with On-Treatment Gag Sequencing - Stage 1 |

| Parameter | Values |
|------------------|------------------------|
| Template ID | SS_GN_T_002 |
| Output File Name | rt-gn-newgags2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |

| Table No. | Table S.5.10.2C |
|-----------|-------------------------------------------------------------|
| Title 1 | Emergent Gag Polymorphisms at Selected Positions |
| Title 2 | Treated Subjects with On-Treatment Gag Sequencing - Stage 2 |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_002 |
| Output File Name | rt-gn-newgags12.lst |
| Purpose | WK96S2 |
| Table No. | Table S.5.10.3C |
| Title 1 | Emergent Gag Polymorphisms at Selected Positions |
| Title 2 | Treated Subjects with On-Treatment Gag Sequencing - Stage 1 and 2 |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_002 |
| Output File Name | rt-gn-newgagbysubtypes1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.5.10.1R |
| Title 1 | Emergent Gag Polymorphisms at Selected Positions |
| Title 2 | By HIV Subtype |
| Title 3 | Treated Subjects with On-Treatment Gag Sequencing - Stage 1 |

| Parameter | Values |
|------------------|-----------------------------|
| Template ID | SS_GN_T_002 |
| Output File Name | rt-gn-newgagbysubtypes2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |

| Table No. | Table S.5.10.2R |
|-----------|-------------------------------------------------------------|
| Title 1 | Emergent Gag Polymorphisms at Selected Positions |
| Title 2 | By HIV Subtype |
| Title 3 | Treated Subjects with On-Treatment Gag Sequencing - Stage 2 |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_002 |
| Output File Name | rt-gn-newgagbysubtypes12.lst |
| Purpose | WK96S2 |
| Table No. | Table S.5.10.3R |
| Title 1 | Emergent Gag Polymorphisms at Selected Positions |
| Title 2 | By HIV Subtype |
| Title 3 | Treated Subjects with On-Treatment Gag Sequencing - Stage 1 and 2 |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_002 |
| Output File Name | rt-gn-newgagpdvfs1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.5.10.1D |
| Title 1 | Emergent Gag Polymorphisms at Selected Positions |
| Title 2 | Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 1 |
| Footnote 1 | Protocol Defined Virologic Failure is defined by a subject meeting one of the following criteria: |
| Footnote 2 | 1) Confirmed > 1 log <sub>10</sub> c/mL increase in HIV-1 RNA at anytime above nadir level where nadir is ≥ 40 c/mL |
| Footnote 3 | 2) Confirmed HIV-1 RNA ≥ 40 c/mL if prior suppression to < 40 c/mL |
| Footnote 4 | 3) Failure to have the last on-treatment HIV-1 RNA to < 400 c/mL within Week 24, 48, or 96 week snapshot window |
| Footnote 5 | 4) Failure to achieve > 1 log <sub>10</sub> c/mL decrease in HIV-1 RNA by Week 8 |
|---|---|
|---|---|

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_002 |
| Output File Name | rt-gn-newgagpdvfs2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.5.10.2D |
| Title 1 | Emergent Gag Polymorphisms at Selected Positions |
| Title 2 | Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 2 |
| Footnote 1 | Protocol Defined Virologic Failure is defined by a subject meeting one of the following criteria: |
| Footnote 2 | 1) Confirmed > 1 log <sub>10</sub> c/mL increase in HIV-1 RNA at anytime above nadir level where nadir is ≥ 40 c/mL |
| Footnote 3 | 2) Confirmed HIV-1 RNA ≥ 40 c/mL if prior suppression to < 40 c/mL |
| Footnote 4 | 3) Failure to have the last on-treatment HIV-1 RNA to < 400 c/mL within Week 24, 48, or 96 week snapshot window |
| Footnote 5 | 4) Failure to achieve > 1 log <sub>10</sub> c/mL decrease in HIV-1 RNA by Week 8 |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_002 |
| Output File Name | rt-gn-newgagpdvfs12.lst |
| Purpose | WK96S2 |
| Table No. | Table S.5.10.3D |
| Title 1 | Emergent Gag Polymorphisms at Selected Positions |
| Title 2 | Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 1 and 2 |
| Footnote 1 | Protocol Defined Virologic Failure is defined by a subject meeting one of the following criteria: |
| Footnote 2 | 1) Confirmed > 1 log <sub>10</sub> c/mL increase in HIV-1 RNA at anytime above nadir level where nadir is ≥ 40 c/mL |
| Footnote 3 | 2) Confirmed HIV-1 RNA ≥ 40 c/mL if prior suppression to < 40 c/mL |

| Footnote 4 | 3) Failure to have the last on-treatment HIV-1 RNA to < 400 c/mL within Week 24, 48, or 96 week snapshot window |
|---|---|
| Footnote 5 | 4) Failure to achieve > 1 log <sub>10</sub> c/mL decrease in HIV-1 RNA by Week 8 |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_002 |
| Output File Name | rt-gn-newgagpdvfbysubtypes1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.5.10.1S |
| Title 1 | Emergent Gag Polymorphisms at Selected Positions |
| Title 2 | By HIV Subtype |
| Title 3 | Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 1 |
| Footnote 1 | Protocol Defined Virologic Failure is defined by a subject meeting one of the following criteria: |
| Footnote 2 | 1) Confirmed > 1 $\log_{10}$ c/mL increase in HIV-1 RNA at anytime above nadir level where nadir is $\geq 40$ c/mL |
| Footnote 3 | 2) Confirmed HIV-1 RNA ≥ 40 c/mL if prior suppression to < 40 c/mL |
| Footnote 4 | 3) Failure to have the last on-treatment HIV-1 RNA to < 400 c/mL within Week 24, 48, or 96 week snapshot window |
| Footnote 5 | 4) Failure to achieve > 1 log <sub>10</sub> c/mL decrease in HIV-1 RNA by Week 8 |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_002 |
| Output File Name | rt-gn-newgagpdvfbysubtypes2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.5.10.2S |
| Title 1 | Emergent Gag Polymorphisms at Selected Positions |
| Title 2 | By HIV Subtype |
| Title 3 | Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 2 |

| Footnote 1 | Protocol Defined Virologic Failure is defined by a subject meeting one of the following criteria: |
|---|---|
| Footnote 2 | 1) Confirmed > 1 log <sub>10</sub> c/mL increase in HIV-1 RNA at anytime above nadir level where nadir is ≥ 40 c/mL |
| Footnote 3 | 2) Confirmed HIV-1 RNA ≥ 40 c/mL if prior suppression to < 40 c/mL |
| Footnote 4 | 3) Failure to have the last on-treatment HIV-1 RNA to < 400 c/mL within Week 24, 48, or 96 week snapshot window |
| Footnote 5 | 4) Failure to achieve > 1 log <sub>10</sub> c/mL decrease in HIV-1 RNA by Week 8 |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_002 |
| Output File Name | rt-gn-newgagpdvfbysubtypes12.lst |
| Purpose | WK96S2 |
| Table No. | Table S.5.10.3S |
| Title 1 | Emergent Gag Polymorphisms at Selected Positions |
| Title 2 | By HIV Subtype |
| Title 3 | Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 1 and 2 |
| Footnote 1 | Protocol Defined Virologic Failure is defined by a subject meeting one of the following criteria: |
| Footnote 2 | 1) Confirmed > 1 log <sub>10</sub> c/mL increase in HIV-1 RNA at anytime above nadir level where nadir is ≥ 40 c/mL |
| Footnote 3 | 2) Confirmed HIV-1 RNA ≥ 40 c/mL if prior suppression to < 40 c/mL |
| Footnote 4 | 3) Failure to have the last on-treatment HIV-1 RNA to < 400 c/mL within Week 24, 48, or 96 week snapshot window |
| Footnote 5 | 4) Failure to achieve > 1 log <sub>10</sub> c/mL decrease in HIV-1 RNA by Week 8 |

| Parameter | Values |
|------------------|-------------------------------|
| Template ID | SS_GN_L_002 |
| Output File Name | rl-gn-gagontrts1.lst |
| Purpose | WK24S1, WK48S1 WK96S1, WK96S2 |
| Table No. | Appendix 5.10.1B |

| Title 1 | Listing of Gag Polymorphisms at Selected Positions |
|---------|----------------------------------------------------------------|
| Title 2 | Treated Subjects with Baseline and On-Treatment Data - Stage 1 |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_L_002 |
| Output File Name | rl-gn-gagontrts2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Appendix 5.10.2B |
| Title 1 | Listing of Gag Polymorphisms at Selected Positions |
| Title 2 | Treated Subjects with Baseline and On-Treatment Data - Stage 2 |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_003 |
| Output File Name | rt-gn-anygags1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.5.10.1E |
| Title 1 | Newly Emergent Gag Deviations |
| Title 2 | Treated Subjects with On-Treatment Gag Sequencing - Stage 1 |

| Parameter | Values |
|------------------|-------------------------------|
| Template ID | SS_GN_T_003 |
| Output File Name | rt-gn-anygags2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.5.10.2E |
| Title 1 | Newly Emergent Gag Deviations |

| Title 2 | Treated Subjects with On-Treatment Gag Sequencing - Stage 2 |
|---------|-------------------------------------------------------------|
|---------|-------------------------------------------------------------|

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_003 |
| Output File Name | rt-gn-anygags12.lst |
| Purpose | WK96S2 |
| Table No. | Table S.5.10.3E |
| Title 1 | Newly Emergent Gag Deviations |
| Title 2 | Treated Subjects with On-Treatment Gag Sequencing - Stage 1 and 2 |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_003 |
| Output File Name | rt-gn-anygagbysubtypes1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.5.10.1T |
| Title 1 | Newly Emergent Gag Deviations |
| Title 2 | By HIV Subtype |
| Title 3 | Treated Subjects with On-Treatment Gag Sequencing - Stage 1 |

| Parameter | Values |
|------------------|-------------------------------|
| Template ID | SS_GN_T_003 |
| Output File Name | rt-gn-anygagbysubtypes2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.5.10.2T |
| Title 1 | Newly Emergent Gag Deviations |

| Title 2 | By HIV Subtype |
|---------|-------------------------------------------------------------|
| Title 3 | Treated Subjects with On-Treatment Gag Sequencing - Stage 2 |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_003 |
| Output File Name | rt-gn-anygagbysubtypes12.lst |
| Purpose | WK96S2 |
| Table No. | Table S.5.10.3T |
| Title 1 | Newly Emergent Gag Deviations |
| Title 2 | By HIV Subtype |
| Title 3 | Treated Subjects with On-Treatment Gag Sequencing - Stage 1 and 2 |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_003 |
| Output File Name | rt-gn-anygagpdvfs1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.5.10.1F |
| Title 1 | Newly Emergent Gag Deviations |
| Title 2 | Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 1 |
| Footnote 1 | Protocol Defined Virologic Failure is defined by a subject meeting one of the following criteria: |
| Footnote 2 | 1) Confirmed > 1 log <sub>10</sub> c/mL increase in HIV-1 RNA at anytime above nadir level where nadir is ≥ 40 c/mL |
| Footnote 3 | 2) Confirmed HIV-1 RNA ≥ 40 c/mL if prior suppression to < 40 c/mL |
| Footnote 4 | 3) Failure to have the last on-treatment HIV-1 RNA to < 400 c/mL within Week 24, 48, or 96 week snapshot window |
| Footnote 5 | 4) Failure to achieve > 1 log <sub>10</sub> c/mL decrease in HIV-1 RNA by Week 8 |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_003 |
| Output File Name | rt-gn-anygagpdvfs2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.5.10.2F |
| Title 1 | Newly Emergent Gag Deviations |
| Title 2 | Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 2 |
| Footnote 1 | Protocol Defined Virologic Failure is defined by a subject meeting one of the following criteria: |
| Footnote 2 | 1) Confirmed > 1 log <sub>10</sub> c/mL increase in HIV-1 RNA at anytime above nadir level where nadir is ≥ 40 c/mL |
| Footnote 3 | 2) Confirmed HIV-1 RNA ≥ 40 c/mL if prior suppression to < 40 c/mL |
| Footnote 4 | 3) Failure to have the last on-treatment HIV-1 RNA to < 400 c/mL within Week 24, 48, or 96 week snapshot window |
| Footnote 5 | 4) Failure to achieve > 1 log <sub>10</sub> c/mL decrease in HIV-1 RNA by Week 8 |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_003 |
| Output File Name | rt-gn-anygagpdvfs12.lst |
| Purpose | WK96S2 |
| Table No. | Table S.5.10.3F |
| Title 1 | Newly Emergent Gag Deviations |
| Title 2 | Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 1 and 2 |
| Footnote 1 | Protocol Defined Virologic Failure is defined by a subject meeting one of the following criteria: |
| Footnote 2 | 1) Confirmed > 1 log <sub>10</sub> c/mL increase in HIV-1 RNA at anytime above nadir level where nadir is ≥ 40 c/mL |
| Footnote 3 | 2) Confirmed HIV-1 RNA ≥ 40 c/mL if prior suppression to < 40 c/mL |
| Footnote 4 | 3) Failure to have the last on-treatment HIV-1 RNA to < 400 c/mL within Week 24, 48, or 96 week snapshot window |
| Footnote 5 | 4) Failure to achieve > 1 log <sub>10</sub> c/mL decrease in HIV-1 RNA by Week 8 |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_003 |
| Output File Name | rt-gn-anygagpdvfbysubtypes1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.5.10.1U |
| Title 1 | Newly Emergent Gag Deviations |
| Title 2 | By HIV Subtype |
| Title 3 | Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 1 |
| Footnote 1 | Protocol Defined Virologic Failure is defined by a subject meeting one of the following criteria: |
| Footnote 2 | 1) Confirmed > 1 log <sub>10</sub> c/mL increase in HIV-1 RNA at anytime above nadir level where nadir is ≥ 40 c/mL |
| Footnote 3 | 2) Confirmed HIV-1 RNA ≥ 40 c/mL if prior suppression to < 40 c/mL |
| Footnote 4 | 3) Failure to have the last on-treatment HIV-1 RNA to < 400 c/mL within Week 24, 48, or 96 week snapshot window |
| Footnote 5 | 4) Failure to achieve > 1 log <sub>10</sub> c/mL decrease in HIV-1 RNA by Week 8 |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_003 |
| Output File Name | rt-gn-anygagpdvfbysubtypes2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.5.10.2U |
| Title 1 | Newly Emergent Gag Deviations |
| Title 2 | By HIV Subtype |
| Title 3 | Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 2 |
| Footnote 1 | Protocol Defined Virologic Failure is defined by a subject meeting one of the following criteria: |
| Footnote 2 | 1) Confirmed > 1 log <sub>10</sub> c/mL increase in HIV-1 RNA at anytime above nadir level where nadir is ≥ 40 c/mL |

| Footnote 3 | 2) Confirmed HIV-1 RNA ≥ 40 c/mL if prior suppression to < 40 c/mL |
|---|---|
| Footnote 4 | 3) Failure to have the last on-treatment HIV-1 RNA to < 400 c/mL within Week 24, 48, or 96 week snapshot window |
| Footnote 5 | 4) Failure to achieve > 1 log <sub>10</sub> c/mL decrease in HIV-1 RNA by Week 8 |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_003 |
| Output File Name | rt-gn-anygagpdvfbysubtypes12.lst |
| Purpose | WK96S2 |
| Table No. | Table S.5.10.3U |
| Title 1 | Newly Emergent Gag Deviations |
| Title 2 | By HIV Subtype |
| Title 3 | Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 1 and 2 |
| Footnote 1 | Protocol Defined Virologic Failure is defined by a subject meeting one of the following criteria: |
| Footnote 2 | 1) Confirmed > 1 log <sub>10</sub> c/mL increase in HIV-1 RNA at anytime above nadir level where nadir is ≥ 40 c/mL |
| Footnote 3 | 2) Confirmed HIV-1 RNA ≥ 40 c/mL if prior suppression to < 40 c/mL |
| Footnote 4 | 3) Failure to have the last on-treatment HIV-1 RNA to < 400 c/mL within Week 24, 48, or 96 week snapshot window |
| Footnote 5 | 4) Failure to achieve > 1 log <sub>10</sub> c/mL decrease in HIV-1 RNA by Week 8 |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_L_003 |
| Output File Name | rl-gn-gagontrts1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Appendix 5.10.1C |
| Title 1 | Listing of Newly Emergent Gag Deviations |
| Title 2 | Treated Subjects with Baseline and On-Treatment Data - Stage 1 |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_L_003 |
| Output File Name | rl-gn-gagontrts2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Appendix 5.10.2C |
| Title 1 | Listing of Newly Emergent Gag Deviations |
| Title 2 | Treated Subjects with Baseline and On-Treatment Data - Stage 2 |

| Parameter | Values |
|---|---|
| Template ID | SS_PN_T_001 |
| Output File Name | rt-pn-news1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.5.10.1G |
| Title 1 | Newly Emergent Phenotypic Resistance Profile |
| Title 2 | Treated Subjects with On-Treatment Phenotypic Resistance Profile - Stage 1 |
| Footnote 1 | Newly emergent phenotypic resistance to a drug is defined as a baseline fold change less than or equal to the cut-off for reduced susceptibility |
| Footnote 2 | and an on-treatment fold change greater than the cut-off for reduced susceptibility. |

| Parameter | Values |
|------------------|------------------------|
| Template ID | SS_PN_T_001 |
| Output File Name | rt-pn-news2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.5.10.2G |

| Title 1 | Newly Emergent Phenotypic Resistance Profile |
|---|---|
| Title 2 | Treated Subjects with On-Treatment Phenotypic Resistance Profile - Stage 2 |
| Footnote 1 | Newly emergent phenotypic resistance to a drug is defined as a baseline fold change less than or equal to the cut-off for reduced susceptibility |
| Footnote 2 | and an on-treatment fold change greater than the cut-off for reduced susceptibility. |

| Parameter | Values |
|---|---|
| Template ID | SS_PN_T_001 |
| Output File Name | rt-pn-news12.lst |
| Purpose | WK96S2 |
| Table No. | Table S.5.10.3G |
| Title 1 | Newly Emergent Phenotypic Resistance Profile |
| Title 2 | Treated Subjects with On-Treatment Phenotypic Resistance Profile - Stage 1 and 2 |
| Footnote 1 | Newly emergent phenotypic resistance to a drug is defined as a baseline fold change less than or equal to the cut-off for reduced susceptibility |
| Footnote 2 | and an on-treatment fold change greater than the cut-off for reduced susceptibility. |

| Parameter | Values |
|---|---|
| Template ID | SS_PN_T_001 |
| Output File Name | rt-pn-newpdvfs1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.5.10.1H |
| Title 1 | Newly Emergent Phenotypic Resistance Profile |
| Title 2 | Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 1 |
| Footnote 1 | Newly emergent phenotypic resistance to a drug is defined as a baseline fold change less than or equal to the cut-off for reduced susceptibility |

| Footnote 2 | and an on-treatment fold change greater than the cut-off for reduced susceptibility. |
|---|---|
| Footnote 3 | Protocol Defined Virologic Failure is defined by a subject meeting one of the following criteria: |
| Footnote 4 | 1) Confirmed > 1 log <sub>10</sub> c/mL increase in HIV-1 RNA at anytime above nadir level where nadir is ≥ 40 c/mL |
| Footnote 5 | 2) Confirmed HIV-1 RNA ≥ 40 c/mL if prior suppression to < 40 c/mL |
| Footnote 6 | 3) Failure to have the last on-treatment HIV-1 RNA to < 400 c/mL within Week 24, 48, or 96 week snapshot window |
| Footnote 7 | 4) Failure to achieve > 1 log <sub>10</sub> c/mL decrease in HIV-1 RNA by Week 8 |

| Parameter | Values |
|---|---|
| Template ID | SS_PN_T_001 |
| Output File Name | rt-pn-newpdvfs2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.5.10.2H |
| Title 1 | Newly Emergent Phenotypic Resistance Profile |
| Title 2 | Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 2 |
| Footnote 1 | Newly emergent phenotypic resistance to a drug is defined as a baseline fold change less than or equal to the cut-off for reduced susceptibility |
| Footnote 2 | and an on-treatment fold change greater than the cut-off for reduced susceptibility. |
| Footnote 3 | Protocol Defined Virologic Failure is defined by a subject meeting one of the following criteria: |
| Footnote 4 | 1) Confirmed > 1 log <sub>10</sub> c/mL increase in HIV-1 RNA at anytime above nadir level where nadir is ≥ 40 c/mL |
| Footnote 5 | 2) Confirmed HIV-1 RNA ≥ 40 c/mL if prior suppression to < 40 c/mL |
| Footnote 6 | 3) Failure to have the last on-treatment HIV-1 RNA to < 400 c/mL within Week 24, 48, or 96 week snapshot window |
| Footnote 7 | 4) Failure to achieve > 1 log <sub>10</sub> c/mL decrease in HIV-1 RNA by Week 8 |

| Parameter | Values |
|-------------|-------------|
| Template ID | SS_PN_T_001 |

| Output File Name | rt-pn-newpdvfs12.lst |
|---|---|
| Purpose | WK96S2 |
| Table No. | Table S.5.10.3H |
| Title 1 | Newly Emergent Phenotypic Resistance Profile |
| Title 2 | Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 1 and 2 |
| Footnote 1 | Newly emergent phenotypic resistance to a drug is defined as a baseline fold change less than or equal to the cut-off for reduced susceptibility |
| Footnote 2 | and an on-treatment fold change greater than the cut-off for reduced susceptibility. |
| Footnote 3 | Protocol Defined Virologic Failure is defined by a subject meeting one of the following criteria: |
| Footnote 4 | 1) Confirmed > 1 log <sub>10</sub> c/mL increase in HIV-1 RNA at anytime above nadir level where nadir is ≥ 40 c/mL |
| Footnote 5 | 2) Confirmed HIV-1 RNA ≥ 40 c/mL if prior suppression to < 40 c/mL |
| Footnote 6 | 3) Failure to have the last on-treatment HIV-1 RNA to < 400 c/mL within Week 24, 48, or 96 week snapshot window |
| Footnote 7 | 4) Failure to achieve > 1 log <sub>10</sub> c/mL decrease in HIV-1 RNA by Week 8 |

| Parameter | Values |
|---|---|
| Template ID | SS_PN_T_002 |
| Output File Name | rt-pn-newdrugs1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.5.10.1I |
| Title 1 | Newly Emergent Phenotypic Resistance by Class and Drug Name |
| Title 2 | Treated Subjects with On-Treatment Phenotypic Resistance Profile - Stage 1 |
| Footnote 1 | Newly emergent phenotypic resistance to a drug is defined as a baseline fold change less than or equal to the cut-off for reduced susceptibility |
| Footnote 2 | and an on-treatment fold change greater than the cut-off for reduced susceptibility. |

| Parameter | Values |
|-----------|--------|
|-----------|--------|

| Template ID | SS_PN_T_002 |
|---|---|
| Output File Name | rt-pn-newdrugs2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.5.10.2I |
| Title 1 | Newly Emergent Phenotypic Resistance by Class and Drug Name |
| Title 2 | Treated Subjects with On-Treatment Phenotypic Resistance Profile - Stage 2 |
| Footnote 1 | Newly emergent phenotypic resistance to a drug is defined as a baseline fold change less than or equal to the cut-off for reduced susceptibility |
| Footnote 2 | and an on-treatment fold change greater than the cut-off for reduced susceptibility. |

| Parameter | Values |
|---|---|
| Template ID | SS_PN_T_002 |
| Output File Name | rt-pn-newdrugs12.lst |
| Purpose | WK96S2 |
| Table No. | Table S.5.10.3I |
| Title 1 | Newly Emergent Phenotypic Resistance by Class and Drug Name |
| Title 2 | Treated Subjects with On-Treatment Phenotypic Resistance Profile - Stage 1 and 2 |
| Footnote 1 | Newly emergent phenotypic resistance to a drug is defined as a baseline fold change less than or equal to the cut-off for reduced susceptibility |
| Footnote 2 | and an on-treatment fold change greater than the cut-off for reduced susceptibility. |

| Parameter | Values |
|------------------|--------------------------------|
| Template ID | SS_PN_T_002 |
| Output File Name | rt-pn-newdrugpdvfs1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.5.10.1J |

| Title 1 | Newly Emergent Phenotypic Resistance by Class and Drug Name |
|---|---|
| Title 2 | Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 1 |
| Footnote 1 | Newly emergent phenotypic resistance to a drug is defined as a baseline fold change less than or equal to the cut-off for reduced susceptibility |
| Footnote 2 | and an on-treatment fold change greater than the cut-off for reduced susceptibility. |
| Footnote 3 | Protocol Defined Virologic Failure is defined by a subject meeting one of the following criteria: |
| Footnote 4 | 1) Confirmed > 1 log <sub>10</sub> c/mL increase in HIV-1 RNA at anytime above nadir level where nadir is ≥ 40 c/mL |
| Footnote 5 | 2) Confirmed HIV-1 RNA ≥ 40 c/mL if prior suppression to < 40 c/mL |
| Footnote 6 | 3) Failure to have the last on-treatment HIV-1 RNA to < 400 c/mL within Week 24, 48, or 96 week snapshot window |
| Footnote 7 | 4) Failure to achieve > 1 log <sub>10</sub> c/mL decrease in HIV-1 RNA by Week 8 |

| Parameter | Values |
|---|---|
| Template ID | SS_PN_T_002 |
| Output File Name | rt-pn-newdrugpdvfs2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.5.10.2J |
| Title 1 | Newly Emergent Phenotypic Resistance by Class and Drug Name |
| Title 2 | Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 2 |
| Footnote 1 | Newly emergent phenotypic resistance to a drug is defined as a baseline fold change less than or equal to the cut-off for reduced susceptibility |
| Footnote 2 | and an on-treatment fold change greater than the cut-off for reduced susceptibility. |
| Footnote 3 | Protocol Defined Virologic Failure is defined by a subject meeting one of the following criteria: |
| Footnote 4 | 1) Confirmed > 1 log <sub>10</sub> c/mL increase in HIV-1 RNA at anytime above nadir level where nadir is ≥ 40 c/mL |
| Footnote 5 | 2) Confirmed HIV-1 RNA ≥ 40 c/mL if prior suppression to < 40 c/mL |
| Footnote 6 | 3) Failure to have the last on-treatment HIV-1 RNA to < 400 c/mL within Week 24, 48, or 96 week snapshot window |
| Footnote 7 | 4) Failure to achieve > 1 log <sub>10</sub> c/mL decrease in HIV-1 RNA by Week 8 |

| Parameter | Values |
|---|---|
| Template ID | SS_PN_T_002 |
| Output File Name | rt-pn-newdrugpdvfs12.lst |
| Purpose | WK96S2 |
| Table No. | Table S.5.10.3J |
| Title 1 | Newly Emergent Phenotypic Resistance by Class and Drug Name |
| Title 2 | Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 1 and 2 |
| Footnote 1 | Newly emergent phenotypic resistance to a drug is defined as a baseline fold change less than or equal to the cut-off for reduced susceptibility |
| Footnote 2 | and an on-treatment fold change greater than the cut-off for reduced susceptibility. |
| Footnote 3 | Protocol Defined Virologic Failure is defined by a subject meeting one of the following criteria: |
| Footnote 4 | 1) Confirmed > 1 log <sub>10</sub> c/mL increase in HIV-1 RNA at anytime above nadir level where nadir is ≥ 40 c/mL |
| Footnote 5 | 2) Confirmed HIV-1 RNA ≥ 40 c/mL if prior suppression to < 40 c/mL |
| Footnote 6 | 3) Failure to have the last on-treatment HIV-1 RNA to < 400 c/mL within Week 24, 48, or 96 week snapshot window |
| Footnote 7 | 4) Failure to achieve > 1 log <sub>10</sub> c/mL decrease in HIV-1 RNA by Week 8 |

| Parameter | Values |
|---|---|
| Template ID | SS_PN_L_001 |
| Output File Name | rl-pn-ontrts1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Appendix 5.10.1D |
| Title 1 | Listing of Phenotypic Resistance |
| Title 2 | Treated Subjects with Baseline and On-Treatment Data - Stage 1 |
| Footnote 1 | Susc = Susceptibility |

| Footnote 2 | P = Partial, R = Resistance, S = Susceptible |
|------------|----------------------------------------------|
|------------|----------------------------------------------|

| Parameter | Values |
|---|---|
| Template ID | SS_PN_L_001 |
| Output File Name | rl-pn-ontrts2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Appendix 5.10.2D |
| Title 1 | Listing of Phenotypic Resistance |
| Title 2 | Treated Subjects with Baseline and On-Treatment Data - Stage 2 |
| Footnote 1 | Susc = Susceptibility |
| Footnote 2 | P = Partial, R = Resistance, S = Susceptible |

# Template SS\_PN\_T\_003: Maximum Change in IC50 Summary

| ASSESSMENT | TRT A N = 10 | TRT B<br>N = 15 | TRT C<br>N = 14 | TRT D<br>N = 15 |
|---|---|---|---|---|
| BASELINE<br>N<br>MEAN (SD)<br>GEOMETRIC MEAN<br>(COEFFICIENT OF VARIATION) | 3<br>0.042480 (0.0276698)<br>0.033159 (65.1) | 11<br>0.012479 (0.0220447)<br>0.001733 (176.7) | | 5<br>0.009394 (0.0149333)<br>0.001608 (159.0) |
| MAXIMUM ON TREATMENT<br>N<br>MEAN (SD)<br>GEOMETRIC MEAN<br>(COEFFICIENT OF VARIATION) | 2<br>0.096295 (0.1327734)<br>0.021409 (137.9) | 9<br>0.718214 (1.6357205)<br>0.019219 (227.7) | 6<br>0.121485 (0.2291942)<br>0.006114 (188.7) | 5<br>1.038524 (2.2150816)<br>0.022420 (213.3) |
| MAXIMUM CHANGE FROM BASELINE<br>MEAN (SD)<br>MEDIAN<br>MIN , MAX | 0.063335 (0.1013496)<br>0.063335<br>-0.00833 , 0.13500 | 0.703029 (1.6328842)<br>0.007120<br>-0.00007 , 4.98500 | 0.118785 (0.2306211)<br>0.003155<br>-0.00005 , 0.57797 | 1.029130 (2.2200751)<br>0.041980<br>-0.00011 , 4.99979 |

| Parameter | Values |
|---|---|
| Template ID | SS_PN_T_003 |
| Output File Name | rt-pn-maxic50s1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.5.10.1K |
| Title 1 | Maximum Change from Baseline Summary for BMS-955176 IC50 |
| Title 2 | Treated Subjects with On-Treatment Phenotypic Resistance Profile - Stage 1 |
| Layout notes | Assessment = BMS-955176 IC50 |

| Parameter | Values |
|-------------|-------------|
| Template ID | SS_PN_T_003 |

| Output File Name | rt-pn-maxic50s2.lst |
|---|---|
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.5.10.2K |
| Title 1 | Maximum Change from Baseline Summary for BMS-955176 IC50 |
| Title 2 | Treated Subjects with On-Treatment Phenotypic Resistance Profile - Stage 2 |
| Layout notes | Assessment = BMS-955176 IC50 |

| Parameter | Values |
|---|---|
| Template ID | SS_PN_T_003 |
| Output File Name | rt-pn-maxic50pdvfs1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.5.10.1L |
| Title 1 | Maximum Change from Baseline Summary for BMS-955176 IC50 |
| Title 2 | Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 1 |
| Footnote 1 | Protocol Defined Virologic Failure is defined by a subject meeting one of the following criteria: |
| Footnote 2 | 1) Confirmed > 1 log <sub>10</sub> c/mL increase in HIV-1 RNA at anytime above nadir level where nadir is ≥ 40 c/mL |
| Footnote 3 | 2) Confirmed HIV-1 RNA ≥ 40 c/mL if prior suppression to < 40 c/mL |
| Footnote 4 | 3) Failure to have the last on-treatment HIV-1 RNA to < 400 c/mL within Week 24, 48, or 96 week snapshot window |
| Footnote 5 | 4) Failure to achieve > 1 log <sub>10</sub> c/mL decrease in HIV-1 RNA by Week 8 |
| Layout notes | Assessment = BMS-955176 IC50 |

| Parameter | Values |
|------------------|-------------------------|
| Template ID | SS_PN_T_003 |
| Output File Name | rt-pn-maxic50pdvfs2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |

| Table No. | Table S.5.10.2L |
|---|---|
| Title 1 | Maximum Change from Baseline Summary for BMS-955176 IC50 |
| Title 2 | Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 2 |
| Footnote 1 | Protocol Defined Virologic Failure is defined by a subject meeting one of the following criteria: |
| Footnote 2 | 1) Confirmed > 1 log <sub>10</sub> c/mL increase in HIV-1 RNA at anytime above nadir level where nadir is ≥ 40 c/mL |
| Footnote 3 | 2) Confirmed HIV-1 RNA ≥ 40 c/mL if prior suppression to < 40 c/mL |
| Footnote 4 | 3) Failure to have the last on-treatment HIV-1 RNA to < 400 c/mL within Week 24, 48, or 96 week snapshot window |
| Footnote 5 | 4) Failure to achieve > 1 log <sub>10</sub> c/mL decrease in HIV-1 RNA by Week 8 |
| Layout notes | Assessment = BMS-955176 IC50 |

| Parameter | Values |
|---|---|
| Template ID | SS_PN_T_003 |
| Output File Name | rt-pn-maxic50fcs1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.5.10.1M |
| Title 1 | Summary for Maximum BMS-955176 IC50 Fold Change |
| Title 2 | Treated Subjects with On-Treatment Phenotypic Resistance Profile - Stage 1 |
| Layout notes | Assessment = BMS-955176 IC50 Fold Change |
| | Only include the 'MAXIMUM ON TREATMENT' part |

| Parameter | Values |
|------------------|------------------------|
| Template ID | SS_PN_T_003 |
| Output File Name | rt-pn-maxic50fcs2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.5.10.2M |

| Title 1 | Summary for Maximum BMS-955176 IC50 Fold Change |
|---|---|
| Title 2 | Treated Subjects with On-Treatment Phenotypic Resistance Profile - Stage 2 |
| Layout notes | Assessment = BMS-955176 IC50 Fold Change |
| | Only include the 'MAXIMUM ON TREATMENT' part |

| Parameter | Values |
|---|---|
| Template ID | SS_PN_T_003 |
| Output File Name | rt-pn-maxic50fcpdvfs1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.5.10.1N |
| Title 1 | Summary for Maximum BMS-955176 IC50 Fold Change |
| Title 2 | Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 1 |
| Footnote 1 | Protocol Defined Virologic Failure is defined by a subject meeting one of the following criteria: |
| Footnote 2 | 1) Confirmed > 1 log <sub>10</sub> c/mL increase in HIV-1 RNA at anytime above nadir level where nadir is ≥ 40 c/mL |
| Footnote 3 | 2) Confirmed HIV-1 RNA ≥ 40 c/mL if prior suppression to < 40 c/mL |
| Footnote 4 | 3) Failure to have the last on-treatment HIV-1 RNA to < 400 c/mL within Week 24, 48, or 96 week snapshot window |
| Footnote 5 | 4) Failure to achieve > 1 log <sub>10</sub> c/mL decrease in HIV-1 RNA by Week 8 |
| Layout notes | Assessment = BMS-955176 IC50 Fold Change Only include the 'MAXIMUM ON TREATMENT' part |

| Parameter | Values |
|------------------|---------------------------|
| Template ID | SS_PN_T_003 |
| Output File Name | rt-pn-maxic50fcpdvfs2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.5.10.2N |

| Title 1 | Summary for Maximum BMS-955176 IC50 Fold Change |
|---|---|
| Title 2 | Treated Subjects Identified as Protocol Defined Virologic Failures - Stage 2 |
| Footnote 1 | Protocol Defined Virologic Failure is defined by a subject meeting one of the following criteria: |
| Footnote 2 | 1) Confirmed > 1 log <sub>10</sub> c/mL increase in HIV-1 RNA at anytime above nadir level where nadir is ≥ 40 c/mL |
| Footnote 3 | 2) Confirmed HIV-1 RNA ≥ 40 c/mL if prior suppression to < 40 c/mL |
| Footnote 4 | 3) Failure to have the last on-treatment HIV-1 RNA to < 400 c/mL within Week 24, 48, or 96 week snapshot window |
| Footnote 5 | 4) Failure to achieve > 1 log <sub>10</sub> c/mL decrease in HIV-1 RNA by Week 8 |
| Layout notes | Assessment = BMS-955176 IC50 Fold Change |
| | Only include the 'MAXIMUM ON TREATMENT' part |

### Template SS\_PN\_T\_004: Proportion of Subjects with > 3 Fold Increase in IC50 Fold Change

| Parameter | Values |
|---|---|
| Template ID | SS_PN_T_004 |
| Output File Name | rt-pn-props1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.5.10.1O |
| Title 1 | Proportion of Subjects with Greater than 3 Fold Increase in BMS-955176 IC50 Fold Change |
| Title 2 | Treated Subjects with Baseline and On-Treatment Phenotypic Resistance Profile - Stage 1 |
| Footnote 1 | A > 3 fold increase from baseline in BMS-955176 FC-IC50 is defined as BMS-955176 FC-IC50 on-treatment divided by BMS-955176 FC-IC50 at baseline >3. |

| Parameter | Values |
|---|---|
| Template ID | SS_PN_T_004 |
| Output File Name | rt-pn-props2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.5.10.2O |
| Title 1 | Proportion of Subjects with Greater than 3 Fold Increase in BMS-955176 IC50 Fold Change |
| Title 2 | Treated Subjects with Baseline and On-Treatment Phenotypic Resistance Profile - Stage 2 |
| Footnote 1 | A > 3 fold increase from baseline in BMS-955176 FC-IC50 is defined as BMS-955176 FC-IC50 on-treatment divided by BMS-955176 FC-IC50 at baseline >3. |

| Parameter | Values |
|---|---|
| Template ID | SS_PN_T_004 |
| Output File Name | rt-pn-props12.lst |
| Purpose | WK96S2 |
| Table No. | Table S.5.10.3O |
| Title 1 | Proportion of Subjects with Greater than 3 Fold Increase in BMS-955176 IC50 Fold Change |
| Title 2 | Treated Subjects with Baseline and On-Treatment Phenotypic Resistance Profile - Stage 1 and 2 |
| Footnote 1 | A > 3 fold increase from baseline in BMS-955176 FC-IC50 is defined as BMS-955176 FC-IC50 on-treatment divided by BMS-955176 FC-IC50 at baseline >3. |

| Parameter | Values |
|---|---|
| Template ID | SS_PN_T_004 |
| Output File Name | rt-pn-proppdvfs1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.5.10.1P |
| Title 1 | Proportion of Subjects with Greater than 3 Fold Increase in BMS-955176 IC50 Fold Change |
| Title 2 | Treated Subjects Identified as Protocol Defined Virologic Failures |
| Title 3 | with Baseline and On-Treatment Phenotypic Resistance Profile - Stage 1 |
| Footnote 1 | A > 3 fold increase from baseline in BMS-955176 FC-IC50 is defined as BMS-955176 FC-IC50 on-treatment divided by BMS-955176 FC-IC50 at baseline >3. |
| Footnote 2 | Protocol Defined Virologic Failure is defined by a subject meeting one of the following criteria: |
| Footnote 3 | 1) Confirmed > 1 log <sub>10</sub> c/mL increase in HIV-1 RNA at anytime above nadir level where nadir is ≥ 40 c/mL |
| Footnote 4 | 2) Confirmed HIV-1 RNA ≥ 40 c/mL if prior suppression to < 40 c/mL |
| Footnote 5 | 3) Failure to have the last on-treatment HIV-1 RNA to < 400 c/mL within Week 24, 48, or 96 week snapshot window |
| Footnote 6 | 4) Failure to achieve > 1 log <sub>10</sub> c/mL decrease in HIV-1 RNA by Week 8 |

| Parameter | Values |
|---|---|
| Template ID | SS_PN_T_004 |
| Output File Name | rt-pn-proppdvfs2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.5.10.2P |
| Title 1 | Proportion of Subjects with Greater than 3 Fold Increase in BMS-955176 IC50 Fold Change |
| Title 2 | Treated Subjects Identified as Protocol Defined Virologic Failures |
| Title 3 | with Baseline and On-Treatment Phenotypic Resistance Profile - Stage 2 |
| Footnote 1 | A > 3 fold increase from baseline in BMS-955176 FC-IC50 is defined as BMS-955176 FC-IC50 on-treatment divided by BMS-955176 FC-IC50 at baseline >3. |
| Footnote 2 | Protocol Defined Virologic Failure is defined by a subject meeting one of the following criteria: |
| Footnote 3 | 1) Confirmed > 1 log <sub>10</sub> c/mL increase in HIV-1 RNA at anytime above nadir level where nadir is ≥ 40 c/mL |
| Footnote 4 | 2) Confirmed HIV-1 RNA ≥ 40 c/mL if prior suppression to < 40 c/mL |
| Footnote 5 | 3) Failure to have the last on-treatment HIV-1 RNA to < 400 c/mL within Week 24, 48, or 96 week snapshot window |
| Footnote 6 | 4) Failure to achieve > 1 log <sub>10</sub> c/mL decrease in HIV-1 RNA by Week 8 |

| Parameter | Values |
|---|---|
| Template ID | SS_PN_T_004 |
| Output File Name | rt-pn-proppdvfs12.lst |
| Purpose | WK96S2 |
| Table No. | Table S.5.10.3P |
| Title 1 | Proportion of Subjects with Greater than 3 Fold Increase in BMS-955176 IC50 Fold Change |
| Title 2 | Treated Subjects Identified as Protocol Defined Virologic Failures |
| Title 3 | with Baseline and On-Treatment Phenotypic Resistance Profile - Stage 1 and 2 |
| Footnote 1 | A > 3 fold increase from baseline in BMS-955176 FC-IC50 is defined as BMS-955176 FC-IC50 on-treatment divided by BMS-955176 FC-IC50 at baseline >3. |

| Footnote 2 | Protocol Defined Virologic Failure is defined by a subject meeting one of the following criteria: |
|---|---|
| Footnote 3 | 1) Confirmed > 1 log <sub>10</sub> c/mL increase in HIV-1 RNA at anytime above nadir level where nadir is ≥ 40 c/mL |
| Footnote 4 | 2) Confirmed HIV-1 RNA ≥ 40 c/mL if prior suppression to < 40 c/mL |
| Footnote 5 | 3) Failure to have the last on-treatment HIV-1 RNA to < 400 c/mL within Week 24, 48, or 96 week snapshot window |
| Footnote 6 | 4) Failure to achieve > 1 log <sub>10</sub> c/mL decrease in HIV-1 RNA by Week 8 |

| Parameter | Values |
|---|---|
| Template ID | SS_PN_T_004 |
| Output File Name | rt-pn-propnews1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.5.10.1V |
| Title 1 | Proportion of Subjects with Newly Emergent Phenotypic Resistance to BMS-955176 |
| Title 2 | Treated Subjects with Baseline and On-Treatment Phenotypic Resistance Profile - Stage 1 |
| Footnote 1 | Newly emergent phenotypic resistance to BMS-955176 is defined as a baseline fold change <= 3 |
| Footnote 2 | and an on-treatment fold change >3 |

| Parameter | Values |
|---|---|
| Template ID | SS_PN_T_004 |
| Output File Name | rt-pn-propnews2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.5.10.2V |
| Title 1 | Proportion of Subjects with Newly Emergent Phenotypic Resistance to BMS-955176 |
| Title 2 | Treated Subjects with Baseline and On-Treatment Phenotypic Resistance Profile - Stage 2 |
| Footnote 1 | Newly emergent phenotypic resistance to BMS-955176 is defined as a baseline fold change <= 3 |
| Footnote 2 | and an on-treatment fold change >3 |

| Parameter | Values |
|---|---|
| Template ID | SS_PN_T_004 |
| Output File Name | rt-pn-propnews12.lst |
| Purpose | WK96S2 |
| Table No. | Table S.5.10.3V |
| Title 1 | Proportion of Subjects with Newly Emergent Phenotypic Resistance to BMS-955176 |
| Title 2 | Treated Subjects with Baseline and On-Treatment Phenotypic Resistance Profile - Stage 1 and 2 |
| Footnote 1 | Newly emergent phenotypic resistance to BMS-955176 is defined as a baseline fold change <= 3 |
| Footnote 2 | and an on-treatment fold change >3 |

| Parameter | Values |
|---|---|
| Template ID | SS_PN_T_004 |
| Output File Name | rt-pn-propnewpdvfs1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.5.10.1W |
| Title 1 | Proportion of Subjects with Newly Emergent Phenotypic Resistance to BMS-955176 |
| Title 2 | Treated Subjects Identified as Protocol Defined Virologic Failures |
| Title 3 | with Baseline and On-Treatment Phenotypic Resistance Profile - Stage 1 |
| Footnote 1 | Protocol Defined Virologic Failure is defined by a subject meeting one of the following criteria: |
| Footnote 2 | 1) Confirmed > 1 log <sub>10</sub> c/mL increase in HIV-1 RNA at anytime above nadir level where nadir is ≥ 40 c/mL |
| Footnote 3 | 2) Confirmed HIV-1 RNA ≥ 40 c/mL if prior suppression to < 40 c/mL |
| Footnote 4 | 3) Failure to have the last on-treatment HIV-1 RNA to < 400 c/mL within Week 24, 48, or 96 week snapshot window |
| Footnote 5 | 4) Failure to achieve > 1 log <sub>10</sub> c/mL decrease in HIV-1 RNA by Week 8 |
| Footnote 6 | Newly emergent phenotypic resistance to BMS-955176 is defined as a baseline fold change <= 3 |

| Footnote 7 | and an on-treatment fold change >3 |
|------------|------------------------------------|
|------------|------------------------------------|

| Parameter | Values |
|---|---|
| Template ID | SS_PN_T_004 |
| Output File Name | rt-pn-propnewpdvfs2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.5.10.2W |
| Title 1 | Proportion of Subjects with Newly Emergent Phenotypic Resistance to BMS-955176 |
| Title 2 | Treated Subjects Identified as Protocol Defined Virologic Failures |
| Title 3 | with Baseline and On-Treatment Phenotypic Resistance Profile - Stage 2 |
| Footnote 1 | Protocol Defined Virologic Failure is defined by a subject meeting one of the following criteria: |
| Footnote 2 | 1) Confirmed > 1 log <sub>10</sub> c/mL increase in HIV-1 RNA at anytime above nadir level where nadir is ≥ 40 c/mL |
| Footnote 3 | 2) Confirmed HIV-1 RNA ≥ 40 c/mL if prior suppression to < 40 c/mL |
| Footnote 4 | 3) Failure to have the last on-treatment HIV-1 RNA to < 400 c/mL within Week 24, 48, or 96 week snapshot window |
| Footnote 5 | 4) Failure to achieve > 1 log <sub>10</sub> c/mL decrease in HIV-1 RNA by Week 8 |
| Footnote 6 | Newly emergent phenotypic resistance to BMS-955176 is defined as a baseline fold change <= 3 |
| Footnote 7 | and an on-treatment fold change >3 |

| Parameter | Values |
|---|---|
| Template ID | SS_PN_T_004 |
| Output File Name | rt-pn-propnewpdvfs12.lst |
| Purpose | WK96S2 |
| Table No. | Table S.5.10.3W |
| Title 1 | Proportion of Subjects with Newly Emergent Phenotypic Resistance to BMS-955176 |
| Title 2 | Treated Subjects Identified as Protocol Defined Virologic Failures |

| Title 3 | with Baseline and On-Treatment Phenotypic Resistance Profile - Stage 1 and 2 |
|---|---|
| Footnote 1 | Protocol Defined Virologic Failure is defined by a subject meeting one of the following criteria: |
| Footnote 2 | 1) Confirmed > 1 log <sub>10</sub> c/mL increase in HIV-1 RNA at anytime above nadir level where nadir is ≥ 40 c/mL |
| Footnote 3 | 2) Confirmed HIV-1 RNA ≥ 40 c/mL if prior suppression to < 40 c/mL |
| Footnote 4 | 3) Failure to have the last on-treatment HIV-1 RNA to < 400 c/mL within Week 24, 48, or 96 week snapshot window |
| Footnote 5 | 4) Failure to achieve > 1 log <sub>10</sub> c/mL decrease in HIV-1 RNA by Week 8 |
| Footnote 6 | Newly emergent phenotypic resistance to BMS-955176 is defined as a baseline fold change <= 3 |
| Footnote 7 | and an on-treatment fold change >3 |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_002 |
| Output File Name | rt-gn-newgagincs1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.5.10.1Q |
| Title 1 | Emergent Gag Polymorphisms |
| Title 2 | Treated Subjects with Greater than 3 Fold Increase in BMS-955176 IC50 Fold Change- Stage 1 |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_002 |
| Output File Name | rt-gn-newgagincs2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.5.10.2Q |
| Title 1 | Emergent Gag Polymorphisms |
| Title 2 | Treated Subjects with Greater than 3 Fold Increase in BMS-955176 IC50 Fold Change- Stage 2 |

| Parameter | Values |
|---|---|
| Template ID | SS_GN_T_002 |
| Output File Name | rt-gn-newgagincs12.lst |
| Purpose | WK96S2 |
| Table No. | Table S.5.10.3Q |
| Title 1 | Emergent Gag Polymorphisms |
| Title 2 | Treated Subjects with Greater than 3 Fold Increase in BMS-955176 IC50 Fold Change- Stage 1 and 2 |

#### Template SS\_VL\_T\_007: Proportion of Responders (mITT) - Futility Analysis

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_007 |
| Output File Name | rt-vl-futw24s1.lst |
| Purpose | WK24S1 |
| Table No. | Table S.5.11.1 |
| Title 1 | Test for Virologic Futility Based on HIV-1 RNA < 40 c/mL |
| Title 2 | Proportion of Responders at Week 24 (mITT) |
| Title 3 | Treated Subjects - Stage 1 |
| Footnote 1 | (a) Response is assessed using the last plasma HIV-1 RNA value in the predefined visit window to classify a subject's response status. |
| Footnote 2 | (b) Based on one-sided Fisher's exact test. |

| Parameter | Values |
|------------------|--------------------|
| Template ID | SS_VL_T_007 |
| Output File Name | rt-vl-futw24s2.lst |
| Purpose | WK24S2 |
| Table No. | Table S.5.11.2 |

| Title 1 | Test for Virologic Futility Based on HIV-1 RNA < 40 c/mL |
|---|---|
| Title 2 | Proportion of Responders at Week 24 (mITT) |
| Title 3 | Treated Subjects - Stage 2 |
| Footnote 1 | (a) Response is assessed using the last plasma HIV-1 RNA value in the predefined visit window to classify a subject's response status. |
| Footnote 2 | (b) Based on one-sided Fisher's exact test. |

# 4.6 Safety Results

## 4.6.1 All Adverse Events

## Template SS\_AE\_T\_001: Overall Adverse Events Summary

| | TRT A | TRT B | TRT C | All Subjects |
|---|---|---|---|---|
| | N = XXX | N = XXX | N = XXX | N = XXXX |
| SUBJECTS WITH ONE OR MORE ADVERSE EVENTS SUBJECTS WHO DIED SUBJECTS WITH SERIOUS ADVERSE EVENTS SUBJECTS WITH RELATED ADVERSE EVENTS SUBJECTS WITH ADVERSE EVENT LEADING TO DISCONTINUATION | XXX ( XX.X) | XXX ( XX.X) | XX ( XX.X) | XXXX ( XX.X) |
| | XXX ( XX.X) | XXX ( XX.X) | XX ( XX.X) | XXXX ( XX.X) |

| Parameter | Values |
|------------------|--------------------------------|
| Template ID | SS_AE_T_001 |
| Output File Name | rt-ae-overallsums1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.6.7.1 |
| Title 1 | Adverse Events |
| Title 2 | Overall Adverse Events Summary |
| Title 3 | Treated Subjects - Stage 1 |

| Parameter | Values |
|------------------|--------------------------------|
| Template ID | SS_AE_T_001 |
| Output File Name | rt-ae-overallsums2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.6.7.2 |
| Title 1 | Adverse Events |
| Title 2 | Overall Adverse Events Summary |
| Title 3 | Treated Subjects - Stage 2 |

| Parameter | Values |
|------------------|----------------------------------|
| Template ID | SS_AE_T_001 |
| Output File Name | rt-ae-overallsums12.lst |
| Purpose | WK96S2 |
| Table No. | Table S.6.7.3 |
| Title 1 | Adverse Events |
| Title 2 | Overall Adverse Events Summary |
| Title 3 | Treated Subjects - Stage 1 and 2 |

## 4.6.2 Deaths

### Template SS\_AE\_L\_001: Listing of Death

\_\_\_\_\_\_

Subject ID (Age/Gender/Race) Treatment Group

Current Trt Period

Death Date

Death Day

Cause of Death

| Parameter | Values |
|------------------|--------------------------------|
| Template ID | SS_AE_L_001 |
| Output File Name | rl-ae-deaths1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.6.1.1 |
| Title 1 | Death Listing |
| Title 2 | Enrolled Subjects - Stage 1 |

| Parameter | Values |
|------------------|-----------------------------|
| Template ID | SS_AE_L_001 |
| Output File Name | rl-ae-deaths2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.6.1.2 |
| Title 1 | Death Listing |
| Title 2 | Enrolled Subjects - Stage 2 |

#### 4.6.3 Serious Adverse Events

| Parameter | Values |
|-----------|--------|
|-----------|--------|

| Template ID | GS_AE_T_X_001 |
|------------------|--------------------------------|
| Output File Name | rt-ae-saes1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.6.2.1A |
| Title 1 | Adverse Event Summary |
| Title 2 | Serious Adverse Events |
| Title 3 | Treated Subjects - Stage 1 |

| Parameter | Values |
|------------------|----------------------------|
| Template ID | GS_AE_T_X_001 |
| Output File Name | rt-ae-saes2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.6.2.2A |
| Title 1 | Adverse Event Summary |
| Title 2 | Serious Adverse Events |
| Title 3 | Treated Subjects - Stage 2 |

| Parameter | Values |
|------------------|-----------------------|
| Template ID | GS_AE_T_X_001 |
| Output File Name | rt-ae-saes12.lst |
| Purpose | WK96S2 |
| Table No. | Table S.6.2.3A |
| Title 1 | Adverse Event Summary |
| Title 2 | Serious Adverse Events |
|------------|----------------------------------|
| Title 3 | Treated Subjects - Stage 1 and 2 |

| Parameter | Values |
|---|---|
| Template ID | GS_AE_T_X_001 |
| Output File Name | rt-ae-saeconts1.lst |
| Purpose | WK96S1, WK96S2 |
| Table No. | Table S.6.2.1B |
| Title 1 | Adverse Event Summary |
| Title 2 | Serious Adverse Events After Switch to Continuation Dose |
| Title 3 | Treated Subjects - Stage 1 |

| Parameter | Values |
|------------------|----------------------------------------------------------|
| Template ID | GS_AE_T_X_001 |
| Output File Name | rt-ae-saeconts2.lst |
| Purpose | WK96S2 |
| Table No. | Table S.6.2.2B |
| Title 1 | Adverse Event Summary |
| Title 2 | Serious Adverse Events After Switch to Continuation Dose |
| Title 3 | Treated Subjects - Stage 2 |

| Template ID | GS_AE_T_X_001 |
|------------------|------------------------------------------------|
| Output File Name | rt-ae-saeldeaths1eu.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.6.2.1C |
| Title 1 | Adverse Event Summary |
| Title 2 | Serious Adverse Event With Death As An Outcome |
| Title 3 | Treated Subjects - Stage 1 |

| Parameter | Values |
|------------------|------------------------------------------------|
| Template ID | GS_AE_T_X_001 |
| Output File Name | rt-ae-saeldeaths2eu.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.6.2.2C |
| Title 1 | Adverse Event Summary |
| Title 2 | Serious Adverse Event With Death As An Outcome |
| Title 3 | Treated Subjects - Stage 2 |

| Parameter | Values |
|------------------|--------------------------------|
| Template ID | GS_AE_T_X_001 |
| Output File Name | rt-ae-relsaeldeaths1eu.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.6.2.1D |
| Title 1 | Adverse Event Summary |

| Title 2 | Drug Related Serious Adverse Event With Death As An Outcome |
|------------|-------------------------------------------------------------|
| Title 3 | Treated Subjects - Stage 1 |

| Parameter | Values |
|---|---|
| Template ID | GS_AE_T_X_001 |
| Output File Name | rt-ae-relsaeldeaths2eu.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.6.2.2D |
| Title 1 | Adverse Event Summary |
| Title 2 | Drug Related Serious Adverse Event With Death As An Outcome |
| Title 3 | Treated Subjects - Stage 2 |

#### Template GS AE L S 001: Adverse Event Listing (by Subject)

Protocol: IM101031 

Adverse Event All Treated Subjects

| Subject ID<br>(Age/Gender/Race)<br>Treatment Group | Current Trt<br>Period<br>Visit | Onset<br>Resolutio<br>Study I | | Dur<br>TRD<br>Type | System Organ Class<br>Preferred Term<br>Reported Term | REL<br>INT | TRT<br>ACT |
|---|---|---|---|---|---|---|---|
| PPD<br>(55/F/C)<br>ABATACEPT | ABA 10<br>ON TRT<br>Day 1 | PPD | 1 | 1D<br>7H<br>SAE | GASTROINTESTINAL DISORDERS<br>NAUSEA<br>NAUSEA | 5<br>2 | 0 |
| | ABA 10<br>ON TRT<br>Day 1 | PPD | 1 | 1D<br>5H<br>AE | SKIN AND SUBCUTANEOUS TISSUE DISORDERS<br>NIGHT SWEATS<br>NIGHT SWEAT | 5<br>2 | 0 1 |
| | ABA 15<br>ON TRT<br>Day 58 | PPD | 58 | 54D<br>14H<br>AE | GASTROINTESTINAL DISORDERS STOMATITIS MOUTH SORES | 5<br>1 | 1 1 |
| | ABA 20<br>ON TRT<br>Day 167 | PPD<br>1 | L67 | 6D<br>6H<br>AE | GASTROINTESTINAL DISORDERS STOMATITIS MOUTH SORES | 5<br>2 | 1 1 |
| | ABA 30<br>ON TRT<br>Day 218 | PPD 2 | 218 | 4D<br>45M<br>AE | GASTROINTESTINAL DISORDERS<br>STOMATITIS<br>MOUTH SORES | 5<br>1 | 0 1 |
| PPD<br>(60/M/C)<br>PLACEBO | PLACEBO<br>ON TRT<br>Day 15 | PPD | 15 | 1D<br>10H<br>AE | MUSCULOSKELETAL AND CONNECTIVE TISSUE<br>DISORDERS<br>BACK PAIN<br>PAIN IN BACK | 5<br>3 | 1<br>5 |

REL (RELATIONSHIP): 5 = NOT RELATED 6 = RELATED

2 = MODERATEINT (INTENSITY): 1 = MILD3 = SEVERE4 = VERY SEVERE

TRT (TREATMENT REQUIRED): 0 = NO 1 = YES

2 = DOSE REDUCED 3 = DOSE INCREASED 4 = DRUG INTERRUPTED 5 = DRUG DISCONTINUED ACT (ACTION): 1 = NONEDUR (DURATION OF EVENT): D = DAYS H = HOURSM = MINUTESS = SECONDS

TRD (TIME RELATIVE TO MOST RECENT DOSE): D = DAYS H = HOURSM = MINUTESS = SECONDS

MedDRA Version: 7.1

Program Source: /wwbdm/ndp/prime/msr/devtest/test/sample21.sas

14JAN2005:16:49:00

| Parameter | Values |
|---|---|
| Template ID | GS_AE_L_S_001 |
| Output File Name | rl-ae-saes1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.6.2.1E |
| Title 1 | Adverse Event |
| Title 2 | Serious Adverse Events |
| Title 3 | Enrolled Subjects - Stage 1 |
| Footnote 1 | REL (RELATIONSHIP): 5 = NOT RELATED 6 = RELATED |
| Footnote 2 | INT (INTENSITY): 1 = MILD 2 = MODERATE 3 = SEVERE 4 = VERY SEVERE |
| Footnote 3 | TRT (TREATMENT REQUIRED): 0 = NO 1 = YES |
| Footnote 4 | ACT (ACTION): 1 = NONE 2 = DOSE REDUCED 3 = DOSE INCREASED 4 = DRUG INTERRUPTED 5 = DRUG DISCONTINUED |
| Footnote 5 | DUR (DURATION OF EVENT): D = DAYS H = HOURS M = MINUTES S = SECONDS |
| Footnote 6 | TRD (TIME RELATIVE TO MOST RECENT DOSE): D = DAYS H = HOURS M = MINUTES S = SECONDS |
| Footnote 7 | MedDRA Version XX.X |

| Parameter | Values |
|------------------|------------------------|
| Template ID | GS_AE_L_S_001 |
| Output File Name | rl-ae-saes2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.6.2.2E |
| Title 1 | Adverse Event |
| Title 2 | Serious Adverse Events |

| Title 3 | Enrolled Subjects - Stage 2 |
|---|---|
| Footnote 1 | REL (RELATIONSHIP): 5 = NOT RELATED 6 = RELATED |
| Footnote 2 | INT (INTENSITY): $1 = MILD$ $2 = MODERATE$ $3 = SEVERE$ $4 = VERY SEVERE$ |
| Footnote 3 | TRT (TREATMENT REQUIRED): 0 = NO 1 = YES |
| Footnote 4 | ACT (ACTION): 1 = NONE 2 = DOSE REDUCED 3 = DOSE INCREASED 4 = DRUG INTERRUPTED 5 = DRUG DISCONTINUED |
| Footnote 5 | DUR (DURATION OF EVENT): D = DAYS H = HOURS M = MINUTES S = SECONDS |
| Footnote 6 | TRD (TIME RELATIVE TO MOST RECENT DOSE): D = DAYS H = HOURS M = MINUTES S = SECONDS |

## 4.6.4 Adverse Events Leading to Discontinuation of Study Therapy

| Parameter | Values |
|---|---|
| Template ID | GS_AE_T_X_001 |
| Output File Name | rt-ae-aediscs1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.6.3.1A |
| Title 1 | Adverse Event Summary |
| Title 2 | Adverse Events Leading to Discontinuation of Study Medication |
| Title 3 | Treated Subjects - Stage 1 |

| Parameter | Values |
|------------------|------------------------|
| Template ID | GS_AE_T_X_001 |
| Output File Name | rt-ae-aediscs2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |

| Table No. | Table S.6.3.2A |
|------------|---------------------------------------------------------------|
| Title 1 | Adverse Event Summary |
| Title 2 | Adverse Events Leading to Discontinuation of Study Medication |
| Title 3 | Treated Subjects - Stage 2 |

| Parameter | Values |
|---|---|
| Template ID | GS_AE_T_X_001 |
| Output File Name | rt-ae-aediscs12.lst |
| Purpose | WK96S2 |
| Table No. | Table S.6.3.3A |
| Title 1 | Adverse Event Summary |
| Title 2 | Adverse Events Leading to Discontinuation of Study Medication |
| Title 3 | Treated Subjects - Stage 1 and 2 |

| Parameter | Values |
|---|---|
| Template ID | GS_AE_T_X_001 |
| Output File Name | rt-ae-aediscconts1.lst |
| Purpose | WK96S1, WK96S2 |
| Table No. | Table S.6.3.1B |
| Title 1 | Adverse Event Summary |
| Title 2 | Adverse Events Leading to Discontinuation of Study Medication After Switch to Continuation Dose |
| Title 3 | Treated Subjects - Stage 1 |

| Parameter | Values |
|---|---|
| Template ID | GS_AE_T_X_001 |
| Output File Name | rt-ae-aediscconts2.lst |
| Purpose | WK96S2 |
| Table No. | Table S.6.3.2B |
| Title 1 | Adverse Event Summary |
| Title 2 | Adverse Events Leading to Discontinuation of Study Medication After Switch to Continuation Dose |
| Title 3 | Treated Subjects - Stage 2 |

#### Template GS\_AE\_L\_X\_001: Adverse Event Listing (by Treatment Group)

Protocol: IM101031 
Adverse Event

All Treated Subjects

Treatment Group: ABATACEPT

| Subject ID<br>(Age/Gender/Race) | Current Trt<br>Period<br>Visit | Onset<br>Resolution<br>Study Day | Dur<br>TRD<br>Type | System Organ Class<br>Preferred Term<br>Reported Term | REL TRT<br>INT ACT |
|---|---|---|---|---|---|
| PPD<br>(55/F/C) | ABA 10<br>ON TRT<br>Day 1 | PPD 1 | 1D<br>7H<br>SAE | GASTROINTESTINAL DISORDERS<br>NAUSEA<br>NAUSEA | 5 0 2 1 |
| | ABA 10<br>ON TRT<br>Day 1 | 1 | 1D<br>5H<br>AE | SKIN AND SUBCUTANEOUS TISSUE DISORDERS<br>NIGHT SWEATS<br>NIGHT SWEAT | 5 0 2 1 |
| | ABA 15<br>ON TRT<br>Day 58 | 58 | 54D<br>14H<br>AE | GASTROINTESTINAL DISORDERS<br>STOMATITIS<br>MOUTH SORES | 5 1<br>1 1 |
| | ABA 20<br>ON TRT<br>Day 167 | <b>PPD</b> 167 | 6D<br>6H<br>AE | GASTROINTESTINAL DISORDERS<br>STOMATITIS<br>MOUTH SORES | 5 1<br>2 1 |
| | ABA 30<br>ON TRT<br>Day 218 | <b>PPD</b> 218 | 4D<br>45M<br>AE | GASTROINTESTINAL DISORDERS<br>STOMATITIS<br>MOUTH SORES | 5 0<br>1 1 |
| | ABA 30<br>ON TRT<br>Day 297 | <b>PPD</b> 297 | 15D<br>1H<br>AE | SKIN AND SUBCUTANEOUS TISSUE DISORDERS<br>INGROWN HAIR<br>INGROWN HAIR FOLLICLE | 5 1<br>2 1 |
| PPD<br>(60/M/C) | ABA 10<br>ON TRT<br>Day 15 | <b>PPD</b> 15 | 1D<br>10H<br>AE | MUSCULOSKELETAL AND CONNECTIVE TISSUE<br>DISORDERS<br>BACK PAIN<br>PAIN IN BACK | 5 1<br>3 5 |

REL (RELATIONSHIP): 5 = NOT RELATED 6 = RELATED

TRT (TREATMENT REQUIRED): 0 = NO 1 = YES

ACT (ACTION): 1 = NONE 2 = DOSE REDUCED 3 = DOSE INCREASED 4 = DRUG INTERRUPTED 5 = DRUG DISCONTINUED DUR (DURATION OF EVENT): D = DAYS H = HOURS M = MINUTES S = SECONDS

TRD (TIME RELATIVE TO MOST RECENT DOSE): D = DAYS H = HOURS M = MINUTES S = SECONDS

MedDRA Version: 7.1

Program Source: /wwbdm/ndp/prime/msr/devtest/test/sample21.sas

14JAN2005:16:49:00

| Parameter | Values |
|---|---|
| Template ID | GS_AE_L_X_001 |
| Output File Name | rl-ae-discs1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.6.3.1C |
| Title 1 | Adverse Event |
| Title 2 | Adverse Events Leading to Discontinuation of Study Medication |
| Title 3 | Treated Subjects - Stage 1 |
| Footnote 1 | REL (RELATIONSHIP): 5 = NOT RELATED 6 = RELATED |
| Footnote 2 | INT (INTENSITY): 1 = MILD 2 = MODERATE 3 = SEVERE 4 = VERY SEVERE |
| Footnote 3 | TRT (TREATMENT REQUIRED): 0 = NO 1 = YES |
| Footnote 4 | ACT (ACTION): 1 = NONE 2 = DOSE REDUCED 3 = DOSE INCREASED 4 = DRUG INTERRUPTED 5 = DRUG DISCONTINUED |
| Footnote 5 | DUR (DURATION OF EVENT): D = DAYS H = HOURS M = MINUTES S = SECONDS |
| Footnote 6 | TRD (TIME RELATIVE TO MOST RECENT DOSE): D = DAYS H = HOURS M = MINUTES S = SECONDS |

| Parameter | Values |
|---|---|
| Template ID | GS_AE_L_X_001 |
| Output File Name | rl-ae-discs2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.6.3.2C |
| Title 1 | Adverse Event |
| Title 2 | Adverse Events Leading to Discontinuation of Study Medication |

| Title 3 | Treated Subjects - Stage 2 |
|---|---|
| Footnote 1 | REL (RELATIONSHIP): 5 = NOT RELATED 6 = RELATED |
| Footnote 2 | INT (INTENSITY): 1 = MILD 2 = MODERATE 3 = SEVERE 4 = VERY SEVERE |
| Footnote 3 | TRT (TREATMENT REQUIRED): 0 = NO 1 = YES |
| Footnote 4 | ACT (ACTION): 1 = NONE 2 = DOSE REDUCED 3 = DOSE INCREASED 4 = DRUG INTERRUPTED 5 = DRUG DISCONTINUED |
| Footnote 5 | DUR (DURATION OF EVENT): D = DAYS H = HOURS M = MINUTES S = SECONDS |
| Footnote 6 | TRD (TIME RELATIVE TO MOST RECENT DOSE): D = DAYS H = HOURS M = MINUTES S = SECONDS |

## 4.6.5 Other Significant Adverse Events

| Parameter | Values |
|---|---|
| Template ID | GS_AE_T_X_001 |
| Output File Name | rt-ae-nsae5pcts1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.6.5.1A |
| Title 1 | Adverse Event Summary |
| Title 2 | Non-Serious Adverse Events Occurring in at Least 5 Percent of Treated Subjects |
| Title 3 | Treated Subjects - Stage 1 |
| Programming notes | Apply the 5% cut to preferred terms only, not "TOTAL SUBJECTS WITH AN EVENT" and SOCs. |

| Parameter | Values |
|------------------|----------------------|
| Template ID | GS_AE_T_X_001 |
| Output File Name | rt-ae-nsae5pcts2.lst |

| Purpose | WK24S2, WK48S2, WK96S2 |
|---|---|
| Table No. | Table S.6.5.2A |
| Title 1 | Adverse Event Summary |
| Title 2 | Non-Serious Adverse Events Occurring in at Least 5 Percent of Treated Subjects |
| Title 3 | Treated Subjects - Stage 2 |
| Programming notes | Apply the 5% cut to preferred terms only, not "TOTAL SUBJECTS WITH AN EVENT" and SOCs. |

| Parameter | Values |
|------------------|--------------------------------|
| Template ID | GS_AE_T_X_001 |
| Output File Name | rt-ae-grade1to4s1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.6.5.1B |
| Title 1 | Adverse Event Summary |
| Title 2 | Grade 1 to 4 Adverse Events |
| Title 3 | Treated Subjects - Stage 1 |

| Parameter | Values |
|------------------|-----------------------------|
| Template ID | GS_AE_T_X_001 |
| Output File Name | rt-ae-grade1to4s2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.6.5.2B |
| Title 1 | Adverse Event Summary |
| Title 2 | Grade 1 to 4 Adverse Events |

| Title 3 | Treated Subjects - Stage 2 |
|------------|----------------------------|

| Parameter | Values |
|------------------|--------------------------------|
| Template ID | GS_AE_T_X_001 |
| Output File Name | rt-ae-grade2to4s1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.6.5.1C |
| Title 1 | Adverse Event Summary |
| Title 2 | Grade 2 to 4 Adverse Events |
| Title 3 | Treated Subjects - Stage 1 |

| Parameter | Values |
|------------------|-----------------------------|
| Template ID | GS_AE_T_X_001 |
| Output File Name | rt-ae-grade2to4s2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.6.5.2C |
| Title 1 | Adverse Event Summary |
| Title 2 | Grade 2 to 4 Adverse Events |
| Title 3 | Treated Subjects - Stage 2 |

| Parameter | Values |
|-------------|---------------|
| Template ID | GS_AE_T_X_001 |

| Output File Name | rt-ae-grade3to4s1.lst |
|------------------|--------------------------------|
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.6.5.1D |
| Title 1 | Adverse Event Summary |
| Title 2 | Grade 3 to 4 Adverse Events |
| Title 3 | Treated Subjects - Stage 1 |

| Parameter | Values |
|------------------|-----------------------------|
| Template ID | GS_AE_T_X_001 |
| Output File Name | rt-ae-grade3to4s2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.6.5.2D |
| Title 1 | Adverse Event Summary |
| Title 2 | Grade 3 to 4 Adverse Events |
| Title 3 | Treated Subjects - Stage 2 |

| Parameter | Values |
|------------------|-----------------------------|
| Template ID | GS_AE_T_X_001 |
| Output File Name | rt-ae-grade3to4s12.lst |
| Purpose | WK96S2 |
| Table No. | Table S.6.5.3D |
| Title 1 | Adverse Event Summary |
| Title 2 | Grade 3 to 4 Adverse Events |

| Title 3 | Treated Subjects - Stage 1 and 2 |
|------------|----------------------------------|

| Parameter | Values |
|------------------|-------------------------------------|
| Template ID | GS_AE_T_X_001 |
| Output File Name | rt-ae-relateds1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.6.5.1E |
| Title 1 | Adverse Event Summary |
| Title 2 | Grade 1 to 4 Related Adverse Events |
| Title 3 | Treated Subjects - Stage 1 |

| Parameter | Values |
|------------------|-------------------------------------|
| Template ID | GS_AE_T_X_001 |
| Output File Name | rt-ae-relateds2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.6.5.2E |
| Title 1 | Adverse Event Summary |
| Title 2 | Grade 1 to 4 Related Adverse Events |
| Title 3 | Treated Subjects - Stage 2 |

| Parameter | Values |
|-------------|---------------|
| Template ID | GS_AE_T_X_001 |

| Output File Name | rt-ae-relgrade2to4s1.lst |
|------------------|-------------------------------------|
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.6.5.1F |
| Title 1 | Adverse Event Summary |
| Title 2 | Grade 2 to 4 Related Adverse Events |
| Title 3 | Treated Subjects - Stage 1 |

| Parameter | Values |
|------------------|-------------------------------------|
| Template ID | GS_AE_T_X_001 |
| Output File Name | rt-ae-relgrade2to4s2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.6.5.2F |
| Title 1 | Adverse Event Summary |
| Title 2 | Grade 2 to 4 Related Adverse Events |
| Title 3 | Treated Subjects - Stage 2 |

| Parameter | Values |
|------------------|-------------------------------------|
| Template ID | GS_AE_T_X_001 |
| Output File Name | rt-ae-relgrade2to4s12.lst |
| Purpose | WK96S2 |
| Table No. | Table S.6.5.3F |
| Title 1 | Adverse Event Summary |
| Title 2 | Grade 2 to 4 Related Adverse Events |

| Title 3 | Treated Subjects - Stage 1 and 2 |
|------------|----------------------------------|

| Parameter | Values |
|------------------|-------------------------------------|
| Template ID | GS_AE_T_X_001 |
| Output File Name | rt-ae-relgrade3to4s1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.6.5.1G |
| Title 1 | Adverse Event Summary |
| Title 2 | Grade 3 to 4 Related Adverse Events |
| Title 3 | Treated Subjects - Stage 1 |

| Parameter | Values |
|------------------|-------------------------------------|
| Template ID | GS_AE_T_X_001 |
| Output File Name | rt-ae-relgrade3to4s2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.6.5.2G |
| Title 1 | Adverse Event Summary |
| Title 2 | Grade 3 to 4 Related Adverse Events |
| Title 3 | Treated Subjects - Stage 2 |

| Parameter | Values |
|-------------|--------------|
| Template ID | GS_AEL_X_001 |

| Output File Name | rl-ae-lists1.lst |
|---|---|
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Appendix 6.5.1 |
| Title 1 | Adverse Event |
| Title 2 | Treated Subjects - Stage 1 |
| Footnote 1 | REL (RELATIONSHIP): 5 = NOT RELATED 6 = RELATED |
| Footnote 2 | INT (INTENSITY): 1 = MILD 2 = MODERATE 3 = SEVERE 4 = VERY SEVERE |
| Footnote 3 | TRT (TREATMENT REQUIRED): 0 = NO 1 = YES |
| Footnote 4 | ACT (ACTION): 1 = NONE 2 = DOSE REDUCED 3 = DOSE INCREASED 4 = DRUG INTERRUPTED 5 = DRUG DISCONTINUED |
| Footnote 5 | DUR (DURATION OF EVENT): D = DAYS H = HOURS M = MINUTES S = SECONDS |
| Footnote 6 | TRD (TIME RELATIVE TO MOST RECENT DOSE): D = DAYS H = HOURS M = MINUTES S = SECONDS |

| Parameter | Values |
|---|---|
| Template ID | GS_AEL_X_001 |
| Output File Name | rl-ae-lists2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Appendix 6.5.2 |
| Title 1 | Adverse Event |
| Title 2 | Treated Subjects - Stage 2 |
| Footnote 1 | REL (RELATIONSHIP): 5 = NOT RELATED 6 = RELATED |
| Footnote 2 | INT (INTENSITY): 1 = MILD 2 = MODERATE 3 = SEVERE 4 = VERY SEVERE |
| Footnote 3 | TRT (TREATMENT REQUIRED): 0 = NO 1 = YES |
| Footnote 4 | ACT (ACTION): 1 = NONE 2 = DOSE REDUCED 3 = DOSE INCREASED 4 = DRUG INTERRUPTED 5 = |

| | DRUG DISCONTINUED |
|---|---|
| Footnote 5 | DUR (DURATION OF EVENT): D = DAYS H = HOURS M = MINUTES S = SECONDS |
| Footnote 6 | TRD (TIME RELATIVE TO MOST RECENT DOSE): D = DAYS H = HOURS M = MINUTES S = SECONDS |

| Parameter | Values |
|------------------|--------------------------------|
| Template ID | GS_AE_T_X_001 |
| Output File Name | rt-ae-cdcaes1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.6.4.1A |
| Title 1 | Adverse Event Summary |
| Title 2 | CDC Class C AIDS Events |
| Title 3 | Treated Subjects - Stage 1 |

| Parameter | Values |
|------------------|----------------------------|
| Template ID | GS_AE_T_X_001 |
| Output File Name | rt-ae-cdcaes2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.6.4.2A |
| Title 1 | Adverse Event Summary |
| Title 2 | CDC Class C AIDS Events |
| Title 3 | Treated Subjects - Stage 2 |

| Parameter | Values |
|------------------|----------------------------------|
| Template ID | GS_AE_T_X_001 |
| Output File Name | rt-ae-cdcaes12.lst |
| Purpose | WK96S2 |
| Table No. | Table S.6.4.3A |
| Title 1 | Adverse Event Summary |
| Title 2 | CDC Class C AIDS Events |
| Title 3 | Treated Subjects - Stage 1 and 2 |

| Parameter | Values |
|---|---|
| Template ID | GS_AEL_X_001 |
| Output File Name | rl-ae-cdcaes1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.6.4.1B |
| Title 1 | Adverse Event |
| Title 2 | CDC Class C AIDS Events |
| Title 3 | Treated Subjects - Stage 1 |
| Footnote 1 | REL (RELATIONSHIP): 5 = NOT RELATED 6 = RELATED |
| Footnote 2 | INT (INTENSITY): 1 = MILD 2 = MODERATE 3 = SEVERE 4 = VERY SEVERE |
| Footnote 3 | TRT (TREATMENT REQUIRED): 0 = NO 1 = YES |
| Footnote 4 | ACT (ACTION): 1 = NONE 2 = DOSE REDUCED 3 = DOSE INCREASED 4 = DRUG INTERRUPTED 5 = DRUG DISCONTINUED |
| Footnote 5 | DUR (DURATION OF EVENT): D = DAYS H = HOURS M = MINUTES S = SECONDS |
| Footnote 6 | TRD (TIME RELATIVE TO MOST RECENT DOSE): D = DAYS H = HOURS M = MINUTES S = SECONDS |

| Footnote 7 |
|------------|
|------------|

| Parameter | Values |
|---|---|
| Template ID | GS_AEL_X_001 |
| Output File Name | rl-ae-cdcaes2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.6.4.2B |
| Title 1 | Adverse Event |
| Title 2 | CDC Class C AIDS Events |
| Title 3 | Treated Subjects - Stage 2 |
| Footnote 1 | REL (RELATIONSHIP): 5 = NOT RELATED 6 = RELATED |
| Footnote 2 | INT (INTENSITY): 1 = MILD 2 = MODERATE 3 = SEVERE 4 = VERY SEVERE |
| Footnote 3 | TRT (TREATMENT REQUIRED): 0 = NO 1 = YES |
| Footnote 4 | ACT (ACTION): 1 = NONE 2 = DOSE REDUCED 3 = DOSE INCREASED 4 = DRUG INTERRUPTED 5 = DRUG DISCONTINUED |
| Footnote 5 | DUR (DURATION OF EVENT): D = DAYS H = HOURS M = MINUTES S = SECONDS |
| Footnote 6 | TRD (TIME RELATIVE TO MOST RECENT DOSE): D = DAYS H = HOURS M = MINUTES S = SECONDS |

| Parameter | Values |
|------------------|--------------------------------|
| Template ID | GS_AE_T_X_001 |
| Output File Name | rt-ae-giaes1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.6.4.1C |
| Title 1 | Adverse Event Summary |

| Title 2 | Gastrointestinal Events of Special Interest |
|------------|---------------------------------------------|
| Title 3 | Treated Subjects - Stage 1 |

| Parameter | Values |
|------------------|---------------------------------------------|
| Template ID | GS_AE_T_X_001 |
| Output File Name | rt-ae-giaes2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.6.4.2C |
| Title 1 | Adverse Event Summary |
| Title 2 | Gastrointestinal Events of Special Interest |
| Title 3 | Treated Subjects - Stage 2 |

| Parameter | Values |
|------------------|---------------------------------------------|
| Template ID | GS_AE_T_X_001 |
| Output File Name | rt-ae-giaes12.lst |
| Purpose | WK96S2 |
| Table No. | Table S.6.4.3C |
| Title 1 | Adverse Event Summary |
| Title 2 | Gastrointestinal Events of Special Interest |
| Title 3 | Treated Subjects - Stage 1 and 2 |

| Template ID | GS_AE_L_X_001 |
|---|---|
| Output File Name | rl-ae-giaes1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.6.4.1D |
| Title 1 | Adverse Event |
| Title 2 | Gastrointestinal Events of Special Interest |
| Title 3 | Treated Subjects - Stage 1 |
| Footnote 1 | REL (RELATIONSHIP): 5 = NOT RELATED 6 = RELATED |
| Footnote 2 | INT (INTENSITY): 1 = MILD 2 = MODERATE 3 = SEVERE 4 = VERY SEVERE |
| Footnote 3 | TRT (TREATMENT REQUIRED): 0 = NO 1 = YES |
| Footnote 4 | ACT (ACTION): 1 = NONE 2 = DOSE REDUCED 3 = DOSE INCREASED 4 = DRUG INTERRUPTED 5 = DRUG DISCONTINUED |
| Footnote 5 | DUR (DURATION OF EVENT): D = DAYS H = HOURS M = MINUTES S = SECONDS |
| Footnote 6 | TRD (TIME RELATIVE TO MOST RECENT DOSE): D = DAYS H = HOURS M = MINUTES S = SECONDS |

| Parameter | Values |
|------------------|-------------------------------------------------|
| Template ID | GS_AE_L_X_001 |
| Output File Name | rl-ae-giaes2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.6.4.2D |
| Title 1 | Adverse Event |
| Title 2 | Gastrointestinal Events of Special Interest |
| Title 3 | Treated Subjects - Stage 2 |
| Footnote 1 | REL (RELATIONSHIP): 5 = NOT RELATED 6 = RELATED |

| Footnote 2 | INT (INTENSITY): 1 = MILD 2 = MODERATE 3 = SEVERE 4 = VERY SEVERE |
|---|---|
| Footnote 3 | TRT (TREATMENT REQUIRED): 0 = NO 1 = YES |
| Footnote 4 | ACT (ACTION): 1 = NONE 2 = DOSE REDUCED 3 = DOSE INCREASED 4 = DRUG INTERRUPTED 5 = DRUG DISCONTINUED |
| Footnote 5 | DUR (DURATION OF EVENT): $D = DAYS$ $H = HOURS$ $M = MINUTES$ $S = SECONDS$ |
| Footnote 6 | TRD (TIME RELATIVE TO MOST RECENT DOSE): D = DAYS H = HOURS M = MINUTES S = SECONDS |

# 4.6.6 Multiple Adverse Events

#### Template GS\_AE\_T\_M\_001: Exposure Adjusted Adverse Events Summary by SOC and Preferred Term

Protocol: TA123456 Page 1 of 20

Exposure Adjusted Adverse Event Summary Including Multiple Occurrences of Unique Events All Treated Subjects

TRT A TRT B TOTAL (N=477)(N=472)(N=949)(P-Y = 218.9)(P-Y = 218.3)(P-Y = 437.2)System Organ Class Rate: Event Rate: Event Event Rate: Preferred Term Count (IR/100 P-Y)Count (IR/100 P-Y) Count (IR/100 P-Y)TOTAL EVENTS 6138 2804.0 6128 2807.3 12266 5611.6 259.3 INFECTIONS AND INFESTATIONS 616 281.4 566 1182 271.7 URINARY TRACT INFECTION 179 81.8 179 82.0 358 81.8 39 17.8 40 18.3 79 18.1 CYTOMEGALOVIRUS INFECTION UPPER RESPIRATORY TRACT 27 12.3 26 11.9 53 11.2 INFECTION 8.3 NASOPHARYNGITIS 26 11.9 18 44 10.2 ORAL CANDIDIASIS 10.5 14 6.4 37 8.9 23 36 25 21 10.5 13 6.0 8.5 BRONCHITIS GASTROENTERITIS 14 6.4 11 5.0 5.4 HERPES ZOSTER 14 6.4 7 3.2 4.6 12 5.5 1.8 16 3.9 SINUSITIS 4 **INFLUENZA** 11 5.0 13 2.0 24 3.5 7 9 3.2 16 3.3 HERPES SIMPLEX 4.1 5 2 UROSEPSIS

P-Y = person-years of exposure

Incidence rate per 100 person-years of exposure (IR/100 P-Y) = event count \* 100 /person-years of exposure

MedDRA Version: 13.0

Program Source: /qbs/prod/clin/programs/im/103/maa-renal/emea150/scs/rpt/rt-adae-ae-inc2-m36-v01.sas

02MAR2011:11:04:59

| Parameter | Values |
|------------------|--------------------------------|
| Template ID | GS_AE_T_M_001 |
| Output File Name | rt-ae-expadjusts1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |

| Table No. | Table S.6.6.1A |
|---|---|
| Title 1 | Exposure Adjusted Adverse Events Summary |
| Title 2 | Treated Subjects - Stage 1 |
| Footnote 1 | P-Y = person-years of exposure |
| Footnote 2 | Incidence rate per 100 person-years of exposure (IR/100 P-Y) = event count * 100 /person-years of exposure |
| Footnote 3 | MedDRA Version: x.x |

| Parameter | Values |
|---|---|
| Template ID | GS_AE_T_M_001 |
| Output File Name | rt-ae-expadjusts2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.6.6.2A |
| Title 1 | Exposure Adjusted Adverse Events Summary |
| Title 2 | Treated Subjects - Stage 2 |
| Footnote 1 | P-Y = person-years of exposure |
| Footnote 2 | Incidence rate per 100 person-years of exposure (IR/100 P-Y) = event count * 100 /person-years of exposure |

| Parameter | Values |
|------------------|---------------------------------------------------------|
| Template ID | GS_AE_T_M_001 |
| Output File Name | rt-ae-expadjsaes1eu.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.6.6.1B |
| Title 1 | Exposure Adjusted Adverse Events Summary |
| Title 2 | Including Multiple Occurrences of Unique Adverse Events |

| Title 3 | Treated Subjects - Stage 1 |
|---|---|
| Title 4 | Serious Adverse Events |
| Footnote 1 | P-Y = person-years of exposure |
| Footnote 2 | Incidence rate per 100 person-years of exposure (IR/100 P-Y) = event count * 100 /person-years of exposure |
| Programming notes | Subset SAEs then collapse using multiple events macro. |

| Parameter | Values |
|---|---|
| Template ID | GS_AE_T_M_001 |
| Output File Name | rt-ae-expadjsaes2eu.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.6.6.2B |
| Title 1 | Exposure Adjusted Adverse Events Summary |
| Title 2 | Including Multiple Occurrences of Unique Adverse Events |
| Title 3 | Treated Subjects - Stage 2 |
| Title 4 | Serious Adverse Events |
| Footnote 1 | P-Y = person-years of exposure |
| Footnote 2 | Incidence rate per 100 person-years of exposure (IR/100 P-Y) = event count * 100 /person-years of exposure |
| Programming notes | Subset SAEs then collapse using multiple events macro. |

| Parameter | Values |
|------------------|--------------------------------|
| Template ID | GS_AE_T_M_001 |
| Output File Name | rt-ae-expadjrelsaes1eu.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |

| Table No. | Table S.6.6.1C |
|---|---|
| Title 1 | Exposure Adjusted Adverse Events Summary |
| Title 2 | Including Multiple Occurrences of Unique Adverse Events |
| Title 3 | Treated Subjects - Stage 1 |
| Title 4 | Drug Related Serious Adverse Events |
| Footnote 1 | P-Y = person-years of exposure |
| Footnote 2 | Incidence rate per 100 person-years of exposure (IR/100 P-Y) = event count * 100 /person-years of exposure |
| Programming notes | Subset SAEs then collapse using multiple events macro. |

| Parameter | Values |
|---|---|
| Template ID | GS_AE_T_M_001 |
| Output File Name | rt-ae-expadjrelsaes2eu.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.6.6.2C |
| Title 1 | Exposure Adjusted Adverse Events Summary |
| Title 2 | Including Multiple Occurrences of Unique Adverse Events |
| Title 3 | Treated Subjects - Stage 2 |
| Title 4 | Drug Related Serious Adverse Events |
| Footnote 1 | P-Y = person-years of exposure |
| Footnote 2 | Incidence rate per 100 person-years of exposure (IR/100 P-Y) = event count * 100 /person-years of exposure |
| Programming notes | Subset SAEs then collapse using multiple events macro. |

| Parameter | Values |
|-----------|--------|
|-----------|--------|

| Template ID | GS_AE_T_M_001 |
|---|---|
| Output File Name | rt-ae-expadjnsae5pcts1eu.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.6.6.1D |
| Title 1 | Exposure Adjusted Adverse Event Summary |
| Title 2 | Including Multiple Occurrences of Unique Adverse Events |
| Title 3 | Treated Subjects - Stage 1 |
| Title 4 | Non-Serious Adverse Events Using a Global Cutoff of 5 Percent |
| Footnote 1 | P-Y = person-years of exposure. Only events occurring in at least 5% of treated subjects in any group are displayed. |
| Footnote 2 | Incidence rate per 100 person-years of exposure (IR/100 P-Y) = event count * 100 /person-years of exposure |
| Programming notes | Display perferred terms with frequency ≥ 5% of treated subjects per rt-ae-nsae5pct.lst. Do not apply the 5% cut to "TOTAL EVENTS" and SOCs |
| | Subset NSAEs then collapse using multiple events macro. |

| Parameter | Values |
|---|---|
| Template ID | GS_AE_T_M_001 |
| Output File Name | rt-ae-expadjnsae5pcts2eu.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.6.6.2D |
| Title 1 | Exposure Adjusted Adverse Event Summary |
| Title 2 | Including Multiple Occurrences of Unique Adverse Events |
| Title 3 | Treated Subjects - Stage 2 |
| Title 4 | Non-Serious Adverse Events Using a Global Cutoff of 5 Percent |
| Footnote 1 | P-Y = person-years of exposure. Only events occurring in at least 5% of treated subjects in any group are displayed. |
| Footnote 2 | Incidence rate per 100 person-years of exposure (IR/100 P-Y) = event count * 100 /person-years of exposure |

|---|---|
| Programming notes | Display perferred terms with frequency ≥ 5% of treated subjects per rt-ae-nsae5pct.lst. Do not apply the 5% cut to "TOTAL EVENTS" and SOCs |
| | Subset NSAEs then collapse using multiple events macro. |

#### Template GS\_AE\_L\_U\_002: Unique Adverse Event Listing

Protocol: IM101031 

Adverse Event Unique Events All Treated Subjects

Treatment Group: ABATACEPT

| Subject ID<br>(Age/Gender/Race) | Current Trt<br>Period<br>Visit | Onset<br>Resolution<br>Study Day | Dur<br>TRD<br>Type | System Organ Class<br>Preferred Term | REL TRT<br>INT ACT |
|---|---|---|---|---|---|
| PPD<br>(55/F/C) | ABA 10<br>ON TRT<br>Day 1 | PPD 1 | 1D<br>7H<br>SAE | GASTROINTESTINAL DISORDERS<br>NAUSEA | 5 0<br>2 1 |
| | ABA 10<br>ON TRT<br>Day 1 | 1 | 1D<br>5H<br>AE | SKIN AND SUBCUTANEOUS TISSUE DISORDERS NIGHT SWEATS | 5 0<br>2 1 |
| | ABA 15<br>ON TRT<br>Day 58 | 58 | 54D<br>14H<br>AE | GASTROINTESTINAL DISORDERS<br>STOMATITIS | 5 1<br>1 1 |
| | ABA 20<br>ON TRT<br>Day 167 | <b>PPD</b> 167 | 6D<br>6H<br>AE | GASTROINTESTINAL DISORDERS<br>STOMATITIS | 5 1<br>2 1 |
| | ABA 30<br>ON TRT<br>Day 218 | <b>PPD</b> 218 | 4D<br>45M<br>AE | GASTROINTESTINAL DISORDERS<br>STOMATITIS | 5 0<br>1 1 |
| PPD<br>(60/M/C) | PLACEBO<br>ON TRT<br>Day 15 | <b>PPD</b> 15 | 1D<br>10H<br>AE | MUSCULOSKELETAL AND CONNECTIVE TISSUE<br>DISORDERS<br>BACK PAIN | 5 1<br>3 5 |
| REL (RELATIONSHIP): INT (INTENSITY): TRT (TREATMENT REQUI ACT (ACTION): DUR (DURATION OF EVE TRD (TIME RELATIVE T | 1 = MILD RED): $0 = NO$ $1 = NONE$ NT): $D = DAYS$ | 2 = DOSE REDUCE<br>H = HOURS | M = MINUTES | 4 = VERY SEVERE CREASED 4 = DRUG INTERRUPTED 5 = DRUG DISCO S = SECONDS M = MINUTES S = SECONDS | ONTINUED |

MedDRA Version: 7.1 Program Source: /wwbdm/ndp/prime/msr/devtest/test/sample21.sas

14JAN2005:16:49:00

| Parameter | Values |
|-----------|--------|
|-----------|--------|

| Template ID | GS_AE_L_U_002 |
|---|---|
| Output File Name | rl-ae-uniques1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Appendix 6.6.1 |
| Title 1 | Adverse Event |
| Title 2 | Unique Events |
| Title 3 | Treated Subjects - Stage 1 |
| Footnote 1 | REL (RELATIONSHIP): 5 = NOT RELATED 6 = RELATED |
| Footnote 2 | INT (INTENSITY): 1 = MILD 2 = MODERATE 3 = SEVERE 4 = VERY SEVERE |
| Footnote 3 | TRT (TREATMENT REQUIRED): 0 = NO 1 = YES |
| Footnote 4 | ACT (ACTION): 1 = NONE 2 = DOSE REDUCED 3 = DOSE INCREASED 4 = DRUG INTERRUPTED 5 = DRUG DISCONTINUED |
| Footnote 5 | DUR (DURATION OF EVENT): D = DAYS H = HOURS M = MINUTES S = SECONDS |
| Footnote 6 | TRD (TIME RELATIVE TO MOST RECENT DOSE): D = DAYS H = HOURS M = MINUTES S = SECONDS |

| Parameter | Values |
|------------------|-------------------------------------------------|
| Template ID | GS_AE_L_U_002 |
| Output File Name | rl-ae-uniques2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Appendix 6.6.2 |
| Title 1 | Adverse Event |
| Title 2 | Unique Events |
| Title 3 | Treated Subjects - Stage 2 |
| Footnote 1 | REL (RELATIONSHIP): 5 = NOT RELATED 6 = RELATED |

| Footnote 2 | INT (INTENSITY): 1 = MILD 2 = MODERATE 3 = SEVERE 4 = VERY SEVERE |
|---|---|
| Footnote 3 | TRT (TREATMENT REQUIRED): 0 = NO 1 = YES |
| Footnote 4 | ACT (ACTION): 1 = NONE 2 = DOSE REDUCED 3 = DOSE INCREASED 4 = DRUG INTERRUPTED 5 = DRUG DISCONTINUED |
| Footnote 5 | DUR (DURATION OF EVENT): $D = DAYS$ $H = HOURS$ $M = MINUTES$ $S = SECONDS$ |
| Footnote 6 | TRD (TIME RELATIVE TO MOST RECENT DOSE): D = DAYS H = HOURS M = MINUTES S = SECONDS |

# 4.6.7 Clinical Laboratory Evaluations

### Template SS\_LB\_T\_001: Laboratory Test Worst Abnormalities Table by Baseline


Laboratory Test Summary of <Toxicity Grade Description> Abnormalities <Title 2>

| | | Number With Abnormality/Number With Measurement (%) | |
|---|---|---|---|
| <lab type=""></lab> | Baseline | Group 1<br>N = XXX | Group 2<br>N = XXX |
| <test 1=""></test> | | XXX/XXX (XXX.X) | XXX/XXX (XXX.X) |
| <additional tests=""></additional> | | | |
| <test x=""></test> | | XXX/XXX (XXX.X) | XXX/XXX (XXX.X) |

... < ADDITIONAL LAB TYPES AND TESTS ON SEPARATE PAGES>

Toxicity Scale: DAIDS Version 1.0 <Footnote 2>

<Footnote 3>

Program Source: <TBD> DDMMYYYYY:HR:MM:SS

| Parameter | Values |
|------------------|-----------------|
| Template ID | SS_LB_T_001 |
| Output File Name | rt-lb-toxs1.lst |

| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
|---|---|
| Table No. | Table S.7.1.1A |
| Title 1 | Laboratory Test Results Summary of Worst Toxicity Grade |
| Title 2 | Treated Subjects - Stage 1 |
| Footnote 1 | Toxicity Scale: DAIDS |
| Programming notes | The laboratory tests to be included in this output are specified in the SAP. |

| Parameter | Values |
|---|---|
| Template ID | SS_LB_T_001 |
| Output File Name | rt-lb-toxs2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.7.1.2A |
| Title 1 | Laboratory Test Results Summary of Worst Toxicity Grade |
| Title 2 | Treated Subjects - Stage 2 |
| Footnote 1 | Toxicity Scale: DAIDS |
| Programming notes | The laboratory tests to be included in this output are specified in the SAP. |

| Parameter | Values |
|------------------|--------------------------------|
| Template ID | SS_LB_T_001 |
| Output File Name | rt-lb-g34toxs1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.7.1.1B |
| Title 1 | Laboratory Test Results |
| Title 2 | Summary of Grade 3-4 Toxicity |
| Title 3 | Treated Subjects - Stage 1 |

| Footnote 1 | Toxicity Scale: DAIDS |
|---|---|
| Programming notes | The laboratory tests to be included in this output are specified in the SAP. |

| Parameter | Values |
|---|---|
| Template ID | SS_LB_T_001 |
| Output File Name | rt-lb-g34toxs2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.7.1.2B |
| Title 1 | Laboratory Test Results |
| Title 2 | Summary of Grade 3-4 Toxicity |
| Title 3 | Treated Subjects - Stage 2 |
| Footnote 1 | Toxicity Scale: DAIDS |
| Programming notes | The laboratory tests to be included in this output are specified in the SAP. |

| Parameter | Values |
|---|---|
| Template ID | SS_LB_T_001 |
| Output File Name | rt-lb-g34toxs12.lst |
| Purpose | WK96S2 |
| Table No. | Table S.7.1.3B |
| Title 1 | Laboratory Test Results |
| Title 2 | Summary of Grade 3-4 Toxicity |
| Title 3 | Treated Subjects - Stage 1 and 2 |
| Footnote 1 | Toxicity Scale: DAIDS |
| Programming notes | The laboratory tests to be included in this output are specified in the SAP. |
#### Template SS\_LB\_T\_002: Laboratory Test Treatment Emergent Abnormalities Table

Protocol: AI438XXX Laboratory Test Summary of Treatment Emergent Abnormalities <Title 2>

Page 1 of X

| | | Number With Abnormality/Number With Measurement (%) | | | | (응) | |
|---|---|---|---|---|---|---|---|
| | Group 1<br>N = XXX | | | | | | |
| <lab type=""></lab> | Baseline | n | Increased to<br>Grade 1 | Increased to<br>Grade 2 | Increased to<br>Grade 3 | Increased to<br>Grade 4 | Increased to<br>Any Grade |
| <test 1=""></test> | TOTAL<br>NORMAL<br>GRADE 1 TO 4<br>NOT REPORTED | XXX<br>XXX<br>XXX<br>XXX | XXX (XXX.X)<br>XXX (XXX.X)<br>XXX (XXX.X)<br>XXX (XXX.X) | XXX (XXX.X)<br>XXX (XXX.X)<br>XXX (XXX.X)<br>XXX (XXX.X) | XXX (XXX.X)<br>XXX (XXX.X)<br>XXX (XXX.X)<br>XXX (XXX.X) | XXX (XXX.X)<br>XXX (XXX.X)<br>XXX (XXX.X)<br>XXX (XXX.X) | XXX (XXX.X)<br>XXX (XXX.X)<br>XXX (XXX.X)<br>XXX (XXX.X) |
| <additio< td=""><td>NAL TESTS&gt;</td><td></td><td></td><td></td><td></td><td></td><td></td></additio<> | NAL TESTS> | | | | | | |
| <test x=""></test> | TOTAL<br>NORMAL<br>GRADE 1 TO 4<br>NOT REPORTED | XXX<br>XXX<br>XXX<br>XXX | XXX (XXX.X)<br>XXX (XXX.X)<br>XXX (XXX.X)<br>XXX (XXX.X) | XXX (XXX.X)<br>XXX (XXX.X)<br>XXX (XXX.X)<br>XXX (XXX.X) | XXX (XXX.X)<br>XXX (XXX.X)<br>XXX (XXX.X)<br>XXX (XXX.X) | XXX (XXX.X)<br>XXX (XXX.X)<br>XXX (XXX.X)<br>XXX (XXX.X) | XXX (XXX.X)<br>XXX (XXX.X)<br>XXX (XXX.X)<br>XXX (XXX.X) |

<... ADDITIONAL TREATMENT GROUPS AND LAB TYPES ON SEPARATE PAGES>

Toxicity Scale: DAIDS Version 1.0

<Footnote 2>
<Footnote 3>
Program Source: <TBD>

Program Source: <TBD>
DDMMYYYY:HR:MM:SS

| Parameter | Values |
|------------------|--------------------------------|
| Template ID | SS_LB_T_001 |
| Output File Name | rt-lb-etoxs1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.7.1.1C |

| Title 1 | Laboratory Test Results Summary of Treatment-Emergent Abnormalities |
|---|---|
| Title 2 | Treated Subjects - Stage 1 |
| Footnote 1 | Toxicity Scale: DAIDS |
| Programming notes | The laboratory tests to be included in this output are specified in the SAP. |

| Parameter | Values |
|---|---|
| Template ID | SS_LB_T_001 |
| Output File Name | rt-lb-etoxs2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.7.1.2C |
| Title 1 | Laboratory Test Results Summary of Treatment-Emergent Abnormalities |
| Title 2 | Treated Subjects - Stage 2 |
| Footnote 1 | Toxicity Scale: DAIDS |
| Programming notes | The laboratory tests to be included in this output are specified in the SAP. |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_006 |
| Output File Name | rt-lb-renals1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.7.2.1A |
| Title 1 | Laboratory Test Results |
| Title 2 | Summary Statistics for Renal Function Values and Change from Baseline - SI Units |
| Title 3 | Treated Subjects - Stage 1 |
| Programming notes | Include creatinine and creatinine clearance as renal tests. |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_006 |
| Output File Name | rt-lb-renals2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.7.2.2A |
| Title 1 | Laboratory Test Results |
| Title 2 | Summary Statistics for Renal Function Values and Change from Baseline - SI Units |
| Title 3 | Treated Subjects - Stage 2 |
| Programming notes | Include creatinine and creatinine clearance as renal tests. |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_006 |
| Output File Name | rt-zl-renals1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.7.2.1B |
| Title 1 | Laboratory Test Results |
| Title 2 | Summary Statistics for Renal Function Values and Change from Baseline - US Units |
| Title 3 | Treated Subjects - Stage 1 |
| Programming notes | Include creatinine and creatinine clearance as renal tests. |

| Parameter | Values |
|------------------|------------------------|
| Template ID | SS_VL_T_006 |
| Output File Name | rt-zl-renals2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.7.2.2B |

| Title 1 | Laboratory Test Results |
|---|---|
| Title 2 | Summary Statistics for Renal Function Values and Change from Baseline - US Units |
| Title 3 | Treated Subjects - Stage 2 |
| Programming notes | Include creatinine and creatinine clearance as renal tests. |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_006 |
| Output File Name | rt-lb-lipidss1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.7.2.1C |
| Title 1 | Laboratory Test Results |
| Title 2 | Summary Statistics for Fasting Lipid Values and Change from Baseline - SI Units |
| Title 3 | Treated Subjects - Stage 1 |
| Footnote 1 | Values obtained after the start of serum lipid-reducing agents are excluded from the summary. |
| Programming notes | Include fasting Total cholesterol, HDL-cholesterol, LDL-cholesterol, triglycerides and total:HDL cholesterol ratio |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_006 |
| Output File Name | rt-lb-lipidss2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.7.2.2C |
| Title 1 | Laboratory Test Results |
| Title 2 | Summary Statistics for Fasting Lipid Values and Change from Baseline - SI Units |
| Title 3 | Treated Subjects - Stage 2 |
| Footnote 1 | Values obtained after the start of serum lipid-reducing agents are excluded from the summary. |

| Programming notes | Include fasting Total cholesterol, HDL-cholesterol, LDL-cholesterol, triglycerides and total:HDL cholesterol ratio |
|---|---|
|---|---|

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_006 |
| Output File Name | rt-zl-lipidss1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.7.2.1D |
| Title 1 | Laboratory Test Results |
| Title 2 | Summary Statistics for Fasting Lipid Values and Change from Baseline - US Units |
| Title 3 | Treated Subjects - Stage 1 |
| Footnote 1 | Values obtained after the start of serum lipid-reducing agents are excluded from the summary. |
| Programming notes | Include fasting Total cholesterol, HDL-cholesterol, LDL-cholesterol, triglycerides and total:HDL cholesterol ratio |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_006 |
| Output File Name | rt-zl-lipidss2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.7.2.2D |
| Title 1 | Laboratory Test Results |
| Title 2 | Summary Statistics for Fasting Lipid Values and Change from Baseline - US Units |
| Title 3 | Treated Subjects - Stage 2 |
| Footnote 1 | Values obtained after the start of serum lipid-reducing agents are excluded from the summary. |
| Programming notes | Include fasting Total cholesterol, HDL-cholesterol, LDL-cholesterol, triglycerides and total:HDL cholesterol ratio |

| Parameter | Values |
|-----------|--------|
|-----------|--------|

| Template ID | SS_VL_T_006 |
|---|---|
| Output File Name | rt-lb-pchglipidss1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.7.2.1E |
| Title 1 | Laboratory Test Results |
| Title 2 | Summary Statistics for Fasting Lipid Values and Percent Change from Baseline - SI Units |
| Title 3 | Treated Subjects - Stage 1 |
| Footnote 1 | Values obtained after the start of serum lipid-reducing agents are excluded from the summary. |
| Layout notes | Change spanning header to "Percent Change From Baseline". |
| Programming notes | Include fasting Total cholesterol, HDL-cholesterol, LDL-cholesterol, triglycerides and total:HDL cholesterol ratio |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_006 |
| Output File Name | rt-lb-pchglipidss2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.7.2.2E |
| Title 1 | Laboratory Test Results |
| Title 2 | Summary Statistics for Fasting Lipid Values and Percent Change from Baseline - SI Units |
| Title 3 | Treated Subjects - Stage 2 |
| Footnote 1 | Values obtained after the start of serum lipid-reducing agents are excluded from the summary. |
| Layout notes | Change spanning header to "Percent Change From Baseline". |
| Programming notes | Include fasting Total cholesterol, HDL-cholesterol, LDL-cholesterol, triglycerides and total:HDL cholesterol ratio |

| Parameter | Values |
|-------------|-------------|
| Template ID | SS_VL_T_006 |

| Output File Name | rt-zl-pchglipidss1.lst |
|---|---|
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Table S.7.2.1F |
| Title 1 | Laboratory Test Results |
| Title 2 | Summary Statistics for Fasting Lipid Values and Percent Change from Baseline - US Units |
| Title 3 | Treated Subjects - Stage 1 |
| Footnote 1 | Values obtained after the start of serum lipid-reducing agents are excluded from the summary. |
| Layout notes | Change spanning header to "Percent Change From Baseline". |
| Programming notes | Include fasting Total cholesterol, HDL-cholesterol, LDL-cholesterol, triglycerides and total:HDL cholesterol ratio |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_006 |
| Output File Name | rt-zl-pchglipidss2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Table S.7.2.2F |
| Title 1 | Laboratory Test Results |
| Title 2 | Summary Statistics for Fasting Lipid Values and Percent Change from Baseline - US Units |
| Title 3 | Treated Subjects - Stage 2 |
| Footnote 1 | Values obtained after the start of serum lipid-reducing agents are excluded from the summary. |
| Layout notes | Change spanning header to "Percent Change From Baseline". |
| Programming notes | Include fasting Total cholesterol, HDL-cholesterol, LDL-cholesterol, triglycerides and total:HDL cholesterol ratio |

| Parameter | Values |
|------------------|---------------|
| Template ID | GS_LB_G_002 |
| Output File Name | rg-lb-tchols1 |

| WK24S1, WK96S1, WK96S2 |
|---|
| Figure S.7.2.1A |
| Fasting Total Cholesterol (mg/dL) Mean Percent Change from Baseline Over Time |
| Treated Subjects - Stage 1 |
| Y-axis label: Fasting Total Cholesterol Mean Percent Change from Baseline (SE) |
| X-axis label: Time (Weeks) Include horizontal reference line at Y=0. |

| Parameter | Values |
|---|---|
| Template ID | GS_LB_G_002 |
| Output File Name | rg-lb-tchols2 |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Figure S.7.2.2A |
| Title 1 | Fasting Total Cholesterol (mg/dL) Mean Percent Change from Baseline Over Time |
| Title 2 | Treated Subjects - Stage 2 |
| Layout notes | Y-axis label: Fasting Total Cholesterol Mean Percent Change from Baseline (SE) |
| | X-axis label: Time (Weeks) |
| | Include horizontal reference line at Y=0. |

| Parameter | Values |
|---|---|
| Template ID | GS_LB_G_002 |
| Output File Name | rg-lb-ldlcs1 |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Figure S.7.2.1B |
| Title 1 | Fasting LDL-Cholesterol (mg/dL) Mean Percent Change from Baseline Over Time |
| Title 2 | Treated Subjects - Stage 1 |

| Layout notes | Y-axis label: Fasting LDL-Cholesterol Mean Percent Change from Baseline (SE) |
|---|---|
| | X-axis label: Time (Weeks) |
| | Include horizontal reference line at Y=0. |

| Parameter | Values |
|---|---|
| Template ID | GS_LB_G_002 |
| Output File Name | rg-lb-ldlcs2 |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Figure S.7.2.2B |
| Title 1 | Fasting LDL-Cholesterol (mg/dL) Mean Percent Change from Baseline Over Time |
| Title 2 | Treated Subjects - Stage 2 |
| Layout notes | Y-axis label: Fasting LDL-Cholesterol Mean Percent Change from Baseline (SE) |
| | X-axis label: Time (Weeks) |
| | Include horizontal reference line at Y=0. |

| Parameter | Values |
|---|---|
| Template ID | GS_LB_G_002 |
| Output File Name | rg-lb-hdlcs1 |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Figure S.7.2.1C |
| Title 1 | Fasting HDL-Cholesterol (mg/dL) Mean Percent Change from Baseline Over Time |
| Title 2 | Treated Subjects - Stage 1 |
| Layout notes | Y-axis label: Fasting HDL-Cholesterol Mean Percent Change from Baseline (SE) X-axis label: Time (Weeks) Include horizontal reference line at Y=0. |

| Parameter | Values |
|---|---|
| Template ID | GS_LB_G_002 |
| Output File Name | rg-lb-hdlcs2 |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Figure S.7.2.2C |
| Title 1 | Fasting HDL-Cholesterol (mg/dL) Mean Percent Change from Baseline Over Time |
| Title 2 | Treated Subjects - Stage 2 |
| Layout notes | Y-axis label: Fasting HDL-Cholesterol Mean Percent Change from Baseline (SE) |
| | X-axis label: Time (Weeks) |
| | Include horizontal reference line at Y=0. |

| Parameter | Values |
|---|---|
| Template ID | GS_LB_G_002 |
| Output File Name | rg-lb-trigs1 |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Figure S.7.2.1D |
| Title 1 | Fasting Total Triglycerides (mg/dL) Mean Percent Change from Baseline Over Time |
| Title 2 | Treated Subjects - Stage 1 |
| Layout notes | Y-axis label: Fasting Triglycerides Mean Percent Change from Baseline (SE) |
| | X-axis label: Time (Weeks) |
| | Include horizontal reference line at Y=0. |

| Parameter | Values |
|------------------|------------------------|
| Template ID | GS_LB_G_002 |
| Output File Name | rg-lb-trigs2 |
| Purpose | WK24S2, WK48S2, WK96S2 |

| Table No. | Figure S.7.2.2D |
|---|---|
| Title 1 | Fasting Total Triglycerides (mg/dL) Mean Percent Change from Baseline Over Time |
| Title 2 | Treated Subjects - Stage 2 |
| Layout notes | Y-axis label: Fasting Triglycerides Mean Percent Change from Baseline (SE) |
| | X-axis label: Time (Weeks) |
| | Include horizontal reference line at Y=0. |

### Template SS\_LB\_L\_001: Laboratory Test Results Listing With Toxicity Grades


Treatment Group: XXXXXXXX

| Subject ID<br>(Age/Gender/Race) | Current Trt<br>Period<br>Visit | Lab Date<br>Study<br>Day | <test 1=""><br/>(<units)></units)></test> | <br><test x=""><br/>(<units>)</units></test> |
|---|---|---|---|---|
| PPD<br>(AAA/G/R) | XXXXXXX<br>XXXXXXX<br>XXXXXXX | DDMMYYYY<br>XXX | XX.X L | XXX.X (X) |
| | <additio< td=""><td>NAL PERIODS</td><td>AND VISITS&gt;</td><td></td></additio<> | NAL PERIODS | AND VISITS> | |
| | XXXXXXX<br>XXXXXXX<br>XXXXXXX | DDMMYYYY<br>XXX | XX.X H | XXX.X (XE) |

... <ADDITIONAL SUBJECTS>

Normal range flag: L = low, H = high Toxicity Scale: DAIDS Version 1.0(Toxicity Grade; E = Emergent on treatment) Program Source: <TBD>

DDMMMYYYY:HR:MM:SS

| Parameter | Values |
|---|---|
| Template ID | SS_LB_L_001 |
| Output File Name | rl-lb-hems1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Appendix 7.1.1A |
| Title 1 | Hematology - SI Units |
| Title 2 | Treated Subjects - Stage 1 |
| Footnote 1 | Normal range flag: L = low, H = high |
| Footnote 2 | Toxicity Scale: DAIDS Version 1.0 (Toxicity Grade; E = Emergent on treatment) |
| Layout notes | Hematology: White Blood Cells (WBC); Neutrophils + Bands, absolute; Red Blood Cells (RBC); Hematocrit; Hemoglobin; Platelets |

| Parameter | Values |
|---|---|
| Template ID | SS_LB_L_001 |
| Output File Name | rl-lb-hems2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Appendix 7.1.2A |
| Title 1 | Hematology - SI Units |
| Title 2 | Treated Subjects - Stage 2 |
| Footnote 1 | Normal range flag: L = low, H = high |
| Layout notes | Hematology: White Blood Cells (WBC); Neutrophils + Bands, absolute; Red Blood Cells (RBC); Hematocrit; Hemoglobin; Platelets |

| Parameter | Values |
|-------------|-------------|
| Template ID | SS_LB_L_001 |

| Output File Name | rl-lb-lfts1.lst |
|---|---|
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Appendix 7.1.1B |
| Title 1 | Liver Function Tests - SI Units |
| Title 2 | Treated Subjects - Stage 1 |
| Footnote 1 | Normal range flag: L = low, H = high |
| Layout notes | <u>Liver Function Tests:</u> Alanine Aminotransferase (ALT); Aspartate Aminotransferase (AST); Total Protein; Albumin; Alkaline Phosphatase; Total Bilirubin; Direct Bilirubin; Indirect Bilirubin |

| Parameter | Values |
|---|---|
| Template ID | SS_LB_L_001 |
| Output File Name | rl-lb-lfts2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Appendix 7.1.2B |
| Title 1 | Liver Function Tests - SI Units |
| Title 2 | Treated Subjects - Stage 2 |
| Footnote 1 | Normal range flag: L = low, H = high |
| Layout notes | <u>Liver Function Tests:</u> Alanine Aminotransferase (ALT); Aspartate Aminotransferase (AST); Total Protein; Albumin; Alkaline Phosphatase; Total Bilirubin; Direct Bilirubin; Indirect Bilirubin |

| Parameter | Values |
|------------------|--------------------------------|
| Template ID | SS_LB_L_001 |
| Output File Name | rl-lb-enzs1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |

| Table No. | Appendix 7.1.1C |
|---|---|
| Title 1 | Enzymes - SI Units |
| Title 2 | Treated Subjects - Stage 1 |
| Footnote 1 | Normal range flag: L = low, H = high |
| Layout notes | Enzymes: Amylase; Creatinine Kinase (CK); Lipase |

| Parameter | Values |
|---|---|
| Template ID | SS_LB_L_001 |
| Output File Name | rl-lb-enzs2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Appendix 7.1.2C |
| Title 1 | Enzymes - SI Units |
| Title 2 | Treated Subjects - Stage 2 |
| Footnote 1 | Normal range flag: L = low, H = high |
| Layout notes | Enzymes: Amylase; Creatinine Kinase (CK); Lipase |

| Parameter | Values |
|------------------|---------------------------------|
| Template ID | SS_LB_L_001 |
| Output File Name | rl-lb-rfts1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Appendix 7.1.1D |
| Title 1 | Renal Function Tests - SI Units |
| Title 2 | Treated Subjects - Stage 1 |

| Footnote 1 | Normal range flag: L = low, H = high |
|---|---|
| Layout notes | Renal Function Tests: Blood Urea Nitrogen (BUN); Creatinine; Creatinine Clearance; Uric Acid; Estimated Glomerular Filtration Rate (eGFR) using Cockcroft-Gault |

| Parameter | Values |
|---|---|
| Template ID | SS_LB_L_001 |
| Output File Name | rl-lb-rfts2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Appendix 7.1.2D |
| Title 1 | Renal Function Tests - SI Units |
| Title 2 | Treated Subjects - Stage 2 |
| Footnote 1 | Normal range flag: L = low, H = high |
| Layout notes | Renal Function Tests: Blood Urea Nitrogen (BUN); Creatinine; Creatinine Clearance; Uric Acid; Estimated Glomerular Filtration Rate (eGFR) using Cockcroft-Gault |

| Parameter | Values |
|---|---|
| Template ID | SS_LB_L_001 |
| Output File Name | rl-lb-elcs1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Appendix 7.1.1E |
| Title 1 | Electrolytes - SI Units |
| Title 2 | Treated Subjects - Stage 1 |
| Footnote 1 | Normal range flag: L = low, H = high |

| Layout notes <u>Electrolytes:</u> I | Bicarbonate, serum; Calcium, serum; Chloride, serum; Potassium, serum; Sodium, serum |
|---|---|
|---|---|

| Parameter | Values |
|---|---|
| Template ID | SS_LB_L_001 |
| Output File Name | rl-lb-elcs2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Appendix 7.1.2E |
| Title 1 | Electrolytes - SI Units |
| Title 2 | Treated Subjects - Stage 2 |
| Footnote 1 | Normal range flag: L = low, H = high |
| Layout notes | Electrolytes: Bicarbonate, serum; Calcium, serum; Chloride, serum; Potassium, serum; Sodium, serum |

| Parameter | Values |
|---|---|
| Template ID | SS_LB_L_001 |
| Output File Name | rl-lb-flgs1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Appendix 7.1.1F |
| Title 1 | Fasting Lipids and Glucose - SI Units |
| Title 2 | Treated Subjects - Stage 1 |
| Footnote 1 | Normal range flag: L = low, H = high |
| Layout notes | <u>Fasting Lipids:</u> Total Cholesterol; LDL Cholesterol; HDL Cholesterol; Triglycerides; Total:HDL Cholesterol <u>Fasting Glucose:</u> Glucose, serum |

| Parameter | Values |
|---|---|
| Template ID | SS_LB_L_001 |
| Output File Name | rl-lb-flgs2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Appendix 7.1.2F |
| Title 1 | Fasting Lipids and Glucose - SI Units |
| Title 2 | Treated Subjects - Stage 2 |
| Footnote 1 | Normal range flag: L = low, H = high |
| Layout notes | <u>Fasting Lipids:</u> Total Cholesterol; LDL Cholesterol; HDL Cholesterol; Triglycerides; Total:HDL Cholesterol <u>Fasting Glucose:</u> Glucose, serum |

| Parameter | Values |
|---|---|
| Template ID | SS_LB_L_001 |
| Output File Name | rl-zl-hems1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Appendix 7.1.1G |
| Title 1 | Hematology - US Units |
| Title 2 | Treated Subjects - Stage 1 |
| Footnote 1 | Normal range flag: L = low, H = high |
| Layout notes | Hematology: White Blood Cells (WBC); Neutrophils + Bands, absolute; Red Blood Cells (RBC); Hematocrit; Hemoglobin; Platelets |

| Parameter | Values |
|-------------|-------------|
| Template ID | SS_LB_L_001 |

| Output File Name | rl-zl-hems2.lst |
|---|---|
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Appendix 7.1.2G |
| Title 1 | Hematology - US Units |
| Title 2 | Treated Subjects - Stage 2 |
| Footnote 1 | Normal range flag: L = low, H = high |
| Layout notes | Hematology: White Blood Cells (WBC); Neutrophils + Bands, absolute; Red Blood Cells (RBC); Hematocrit; Hemoglobin; Platelets |

| Parameter | Values |
|---|---|
| Template ID | SS_LB_L_001 |
| Output File Name | rl-zl-lfts1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Appendix 7.1.1H |
| Title 1 | Liver Function Tests - US Units |
| Title 2 | Treated Subjects - Stage 1 |
| Footnote 1 | Normal range flag: L = low, H = high |
| Layout notes | <u>Liver Function Tests:</u> Alanine Aminotransferase (ALT); Aspartate Aminotransferase (AST); Total Protein; Albumin; Alkaline Phosphatase; Total Bilirubin; Direct Bilirubin; Indirect Bilirubin |

| Parameter | Values |
|------------------|------------------------|
| Template ID | SS_LB_L_001 |
| Output File Name | rl-zl-lfts2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |

| Table No. | Appendix 7.1.2H |
|---|---|
| Title 1 | Liver Function Tests - US Units |
| Title 2 | Treated Subjects - Stage 2 |
| Footnote 1 | Normal range flag: L = low, H = high |
| Layout notes | <u>Liver Function Tests:</u> Alanine Aminotransferase (ALT); Aspartate Aminotransferase (AST); Total Protein; Albumin; Alkaline Phosphatase; Total Bilirubin; Direct Bilirubin; Indirect Bilirubin |

| Parameter | Values |
|---|---|
| Template ID | SS_LB_L_001 |
| Output File Name | rl-zl-enzs1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Appendix 7.1.1I |
| Title 1 | Enzymes - US Units |
| Title 2 | Treated Subjects - Stage 1 |
| Footnote 1 | Normal range flag: $L = low$ , $H = high$ |
| Layout notes | Enzymes: Amylase; Creatinine Kinase (CK); Lipase |

| Parameter | Values |
|------------------|------------------------|
| Template ID | SS_LB_L_001 |
| Output File Name | rl-zl-enzs2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Appendix 7.1.2I |
| Title 1 | Enzymes - US Units |

| Title 2 | Treated Subjects - Stage 2 |
|---|---|
| Footnote 1 | Normal range flag: L = low, H = high |
| Layout notes | Enzymes: Amylase; Creatinine Kinase (CK); Lipase |

| Parameter | Values |
|---|---|
| Template ID | SS_LB_L_001 |
| Output File Name | rl-zl-rfts1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Appendix 7.1.1J |
| Title 1 | Renal Function Tests - US Units |
| Title 2 | Treated Subjects - Stage 1 |
| Footnote 1 | Normal range flag: L = low, H = high |
| Layout notes | Renal Function Tests: Blood Urea Nitrogen (BUN); Creatinine; Creatinine Clearance; Uric Acid; Estimated Glomerular Filtration Rate (eGFR) using Cockcroft-Gault |

| Parameter | Values |
|------------------|--------------------------------------|
| Template ID | SS_LB_L_001 |
| Output File Name | rl-zl-rfts2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Appendix 7.1.2J |
| Title 1 | Renal Function Tests - US Units |
| Title 2 | Treated Subjects - Stage 2 |
| Footnote 1 | Normal range flag: L = low, H = high |

|---|---|
| Layout notes | Renal Function Tests: Blood Urea Nitrogen (BUN); Creatinine; Creatinine Clearance; Uric Acid; Estimated Glomerular Filtration Rate (eGFR) using Cockcroft-Gault |

| Parameter | Values |
|---|---|
| Template ID | SS_LB_L_001 |
| Output File Name | rl-zl-elcs1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Appendix 7.1.1K |
| Title 1 | Electrolytes - US Units |
| Title 2 | Treated Subjects - Stage 1 |
| Footnote 1 | Normal range flag: L = low, H = high |
| Layout notes | Electrolytes: Bicarbonate, serum; Calcium, serum; Chloride, serum; Potassium, serum; Sodium, serum |

| Parameter | Values |
|---|---|
| Template ID | SS_LB_L_001 |
| Output File Name | rl-zl-elcs2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Appendix 7.1.2K |
| Title 1 | Electrolytes - US Units |
| Title 2 | Treated Subjects - Stage 2 |
| Footnote 1 | Normal range flag: L = low, H = high |
| Layout notes | Electrolytes: Bicarbonate, serum; Calcium, serum; Chloride, serum; Potassium, serum; Sodium, serum |

| Parameter | Values |
|---|---|
| Template ID | SS_LB_L_001 |
| Output File Name | rl-zl-flgs1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Appendix 7.1.1L |
| Title 1 | Fasting Lipids and Glucose - US Units |
| Title 2 | Treated Subjects - Stage 1 |
| Footnote 1 | Normal range flag: L = low, H = high |
| Layout notes | Fasting Lipids: Total Cholesterol; LDL Cholesterol; HDL Cholesterol; Total:HDL Cholesterol Ratio; Triglycerides |
| | Fasting Glucose: Glucose, serum |

| Parameter | Values |
|---|---|
| Template ID | SS_LB_L_001 |
| Output File Name | rl-zl-flgs2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Appendix 7.1.2L |
| Title 1 | Fasting Lipids and Glucose - US Units |
| Title 2 | Treated Subjects - Stage 2 |
| Footnote 1 | Normal range flag: L = low, H = high |
| Layout notes | Fasting Lipids: Total Cholesterol; LDL Cholesterol; HDL Cholesterol; Total: HDL Cholesterol Ratio; Triglycerides Fasting Glucose: Glucose, serum |

#### Template GS LB L S 008: Differences in Categorization of SI and US units

Protocol: AI463022 

Draft
Differences in Categorization of SI and US Laboratory Test Results
Treated Subjects

Lab Test: Glucose (SI units: mmol/L, US Std Units: mg/dL)

| | | | SI Unit | | | | | US Standard Unit | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Subject ID | Period | Lab Date | Standard<br>Lab<br>Result | Normal Range | | | | Standard<br>Lab | Normal Range | | | |
| (Age/Gender/Race)<br>Treatment Group | | Study Day | | Low | High | Flag | Toxicity | Result | Low | High | Flag | Toxicity |
| PPD (59/F/O) | BASELINE<br>A00 | <b>PPD</b> -28 | 2.1 | 4.0 | 5.0 | L | GRADE 0 | 37.8 | 52.0 | 65.0 | L | GRADE 1 |
| ENTECAVIR | ON TREATMENT<br>B01 | PPD 1 | 3.1 | 4.0 | 5.0 | L | GRADE 1 | 45.8 | 52.0 | 65.0 | L | GRADE 2 |
| PPD (43/F/C) | ON TREATMENT<br>B02 | PPD 14 | 4.1 | 4.0 | 5.0 | | GRADE 1 | 53.1 | 52.0 | 65.0 | | GRADE 2 |
| PLACEBO | ON TREATMENT<br>B03 | <b>PPD</b> 27 | 5.6 | 4.0 | 5.0 | | GRADE 2 | 66.6 | 39.0 | 65.0 | Н | GRADE 3 |

NORMAL RANGE FLAG: L = LOW H = HIGH+ = NO NORMAL RANGES

Toxicity Scale : Descriptive text of toxicity scale

| Parameter | Values |
|---|---|
| Template ID | GS_LB_L_S_008 |
| Output File Name | rl-lb-diffunits1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Appendix 7.1.1M |
| Title 1 | Differences in Categorization of SI and US Laboratory Test Results |
| Title 2 | Treated Subjects - Stage 1 |
| Footnote 1 | NORMAL RANGE FLAG: L = LOW H = HIGH + = NO NORMAL RANGES |
| Footnote 2 | Toxicity Scale : DAIDS |

| Parameter | Values |
|---|---|
| Template ID | GS_LB_L_S_008 |
| Output File Name | rl-lb-diffunits2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Appendix 7.1.2M |
| Title 1 | Differences in Categorization of SI and US Laboratory Test Results |
| Title 2 | Treated Subjects - Stage 2 |
| Footnote 1 | NORMAL RANGE FLAG: L = LOW H = HIGH + = NO NORMAL RANGES |
| Footnote 2 | Toxicity Scale : DAIDS |

## Template GS\_LB\_L\_X\_006: Pregnancy Listing by Treatment Group

Protocol: TA123456 

Pregnancy Test
All Treated Female Subjects

Treatment Group: TRT B

| Subject ID<br>(Age/Gender, | /Race) Period | Test Date | Study<br>Day | Method | Result | Reason Not done |
|---|---|---|---|---|---|---|
| PPD<br>(59/F/O) | X<br>Y | PPD | -1<br>28 | URINE HCG<br>SERUM HCG | NEGATIVE<br>0 | |
| PPD<br>(34/F/B) | X<br>Y | | -1<br>24<br>46 | URINE HCG<br>URINE HCG<br>SERUM HCG | NEGATIVE<br>NEGATIVE<br>O | |
| PPD<br>(44/F/C) | X<br>Y | | -1<br>7 | | | SURGICALLY STERILE<br>SURGICALLY STERILE |

Program Source: /wwbdm/ndp/prime/gssr/devtest/prg/test/prg lst.sas

07SEP2004:14:35:00

| Parameter | Values |
|------------------|-----------------------------------|
| Template ID | GS_LB_L_X_006 |
| Output File Name | rl-lb-pregs1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Appendix 7.1.1N |
| Title 1 | Pregnancy Test |
| Title 2 | Treated Female Subjects - Stage 1 |

| Parameter | Values |
|------------------|------------------------|
| Template ID | GS_LB_L_X_006 |
| Output File Name | rl-lb-pregs2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |

| Table No. | Appendix 7.1.2N |
|-----------|-----------------------------------|
| Title 1 | Pregnancy Test |
| Title 2 | Treated Female Subjects - Stage 2 |

## 4.6.8 Electrocardiograms

## Template SS\_EG\_T\_003: ECG Summary Table with 95% CI


| Period<br>Visit | Percentiles | | | | | | Change From Baseline | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Group | N | Mean | SD | Q1 | Median | Q3 | N | Mean | SD | 95% CI for Mean | Q1 | Median | Q3 |
| PRE-TRT<br>B/L<br>Group 1<br>Group 2 | XXX<br>XXX | XXX.X<br>XXX.X | XXX.XX<br>XXX.XX | XXX.X<br>XXX.X | XXX.X<br>XXX.X | XXX.X<br>XXX.X | XXX<br>XXX | XXX.X<br>XXX.X | XXX.XX<br>XXX.XX | (XXX.XX, XXX.XX)<br>(XXX.XX, XXX.XX) | XXX.X<br>XXX.X | XXX.X<br>XXX.X | XXX.X<br>XXX.X |
| ON TRT<br>WK XX<br>Group 1<br>Group 2 | XXX<br>XXX | XXX.X<br>XXX.X | XXX.XX<br>XXX.XX | XXX.X<br>XXX.X | XXX.X<br>XXX.X | XXX.X<br>XXX.X | XXX<br>XXX | XXX.X<br>XXX.X | XXX.XX<br>XXX.XX | (XXX.XX, XXX.XX)<br>(XXX.XX, XXX.XX) | XXX.X<br>XXX.X | XXX.X<br>XXX.X | XXX.X<br>XXX.X |

... <ADDITIONAL PERIODS AND VISITS>

| Parameter | Values |
|---|---|
| Template ID | SS_EG_T_003 |
| Output File Name | rt-eg-sumchgs1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Appendix 7.3.1A |
| Title 1 | Electrocardiogram Summary of Values and Changes from Baseline over Time |
| Title 2 | Treated Subjects - Stage 1 |
| Layout notes | Parameters are specified in SAP, Section 7.6.14. |

| Parameter | Values |
|-------------|-------------|
| Template ID | SS_EG_T_003 |

| Output File Name | rt-eg-sumchgs2.lst |
|---|---|
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Appendix 7.3.2A |
| Title 1 | Electrocardiogram Summary of Values and Changes from Baseline over Time |
| Title 2 | Treated Subjects - Stage 2 |
| Layout notes | Parameters are specified in SAP, Section 7.6.14. |

Template SS\_EG\_T\_001: ECG Change from Baseline Category Summary

| ECG Parameter (unit)<br>Category (%) | BMS-663068<br>400 mg BID/<br>RAL/TDF<br>N = 50 | BMS-663068<br>800 mg BID/<br>RAL/TDF<br>N = 49 | BMS-663068<br>600 mg QD/<br>RAL/TDF<br>N = 51 | BMS-663068<br>1200 mg QD/<br>RAL/TDF<br>N = 50 | ATV/r/<br>RAL/TDF<br>N = 51 |
|---|---|---|---|---|---|
| PR INTERVAL (MSEC) <0 0 to <20 20 to <40 40 to <60 60 to <80 >=80 NOT REPORTED | 4 ( 8.0)<br>33 ( 66.0)<br>11 ( 22.0)<br>0<br>0<br>0<br>2 ( 4.0) | 8 (16.3)<br>30 (61.2)<br>11 (22.4)<br>0<br>0 | 4 ( 7.8)<br>35 ( 68.6)<br>11 ( 21.6)<br>1 ( 2.0)<br>0 | 7 (14.0)<br>33 (66.0)<br>7 (14.0)<br>1 (2.0)<br>0<br>0<br>2 (4.0) | 8 ( 15.7)<br>28 ( 54.9)<br>13 ( 25.5)<br>1 ( 2.0)<br>0<br>0<br>1 ( 2.0) |
| QRS (MSEC) <0 0 to <10 10 to <20 20 to <30 30 to <40 >=40 NOT REPORTED | 4 ( 8.0)<br>33 ( 66.0)<br>9 ( 18.0)<br>2 ( 4.0)<br>0<br>0<br>2 ( 4.0) | 6 ( 12.2)<br>32 ( 65.3)<br>9 ( 18.4)<br>2 ( 4.1)<br>0 | 3 ( 5.9)<br>37 ( 72.5)<br>10 ( 19.6)<br>1 ( 2.0)<br>0 | 2 ( 4.0)<br>38 ( 76.0)<br>6 ( 12.0)<br>2 ( 4.0)<br>0<br>2 ( 4.0) | 6 ( 11.8)<br>29 ( 56.9)<br>15 ( 29.4)<br>0<br>0<br>0<br>1 ( 2.0) |
| QTC [FRIDERICIA] (MSEC) <0 0 to <10 10 to <20 20 to <30 30 to <40 >=40 NOT REPORTED | 6 ( 12.0)<br>7 ( 14.0)<br>17 ( 34.0)<br>11 ( 22.0)<br>6 ( 12.0)<br>1 ( 2.0)<br>2 ( 4.0) | 6 (12.2)<br>8 (16.3)<br>21 (42.9)<br>9 (18.4)<br>2 (4.1)<br>3 (6.1) | 4 ( 7.8)<br>13 ( 25.5)<br>18 ( 35.3)<br>7 ( 13.7)<br>4 ( 7.8)<br>5 ( 9.8) | 3 ( 6.0)<br>11 ( 22.0)<br>20 ( 40.0)<br>10 ( 20.0)<br>1 ( 2.0)<br>3 ( 6.0)<br>2 ( 4.0) | 9 ( 17.6)<br>13 ( 25.5)<br>15 ( 29.4)<br>7 ( 13.7)<br>5 ( 9.8)<br>1 ( 2.0)<br>1 ( 2.0) |

ParameterValuesTemplate IDSS\_EG\_T\_001Output File Namert-eg-changecats1.lstPurposeWK24S1, WK48S1, WK96S1, WK96S2Table No.Appendix 7.3.1BTitle 1Electrocardiogram Change from Baseline Category Summary

| Title 2 | Treated Subjects - Stage 1 |
|---|---|
| Footnote 1 | Each subject is counted only once using the longest change observed. |

| Parameter | Values |
|---|---|
| Template ID | SS_EG_T_001 |
| Output File Name | rt-eg-changecats2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Appendix 7.3.2B |
| Title 1 | Electrocardiogram Change from Baseline Category Summary |
| Title 2 | Treated Subjects - Stage 2 |
| Footnote 1 | Each subject is counted only once using the longest change observed. |

Template SS\_EG\_T\_002: ECG Category Summary

| ECG Parameter (unit)<br>Category (%) | BMS-663068<br>400 mg BID/<br>RAL/TDF<br>N = 50 | BMS-663068<br>800 mg BID/<br>RAL/TDF<br>N = 49 | BMS-663068<br>600 mg QD/<br>RAL/TDF<br>N = 51 | BMS-663068<br>1200 mg QD/<br>RAL/TDF<br>N = 50 | ATV/r/<br>RAL/TDF<br>N = 51 |
|---|---|---|---|---|---|
| PR INTERVAL (MSEC) <200 200 to <220 220 to <240 240 to <260 260 to <280 280 to <300 >=300 NOT REPORTED | 44 ( 88.0)<br>4 ( 8.0)<br>0<br>0<br>0<br>0<br>0<br>2 ( 4.0) | 46 ( 93.9)<br>1 ( 2.0)<br>2 ( 4.1)<br>0<br>0<br>0 | 46 ( 90.2)<br>5 ( 9.8)<br>0<br>0<br>0<br>0 | 43 ( 86.0) 5 ( 10.0) 0 0 0 0 0 2 ( 4.0) | 49 ( 96.1)<br>1 ( 2.0)<br>0<br>0<br>0<br>0<br>0<br>1 ( 2.0) |
| QRS (MSEC) <100 100 to <110 110 to <120 120 to <130 130 to <140 >=140 NOT REPORTED | 39 ( 78.0)<br>8 ( 16.0)<br>1 ( 2.0)<br>0<br>0<br>0<br>2 ( 4.0) | 40 ( 81.6)<br>8 ( 16.3)<br>1 ( 2.0)<br>0<br>0 | 38 ( 74.5)<br>12 ( 23.5)<br>1 ( 2.0)<br>0<br>0 | 38 ( 76.0)<br>5 ( 10.0)<br>5 ( 10.0)<br>0<br>0<br>0<br>2 ( 4.0) | 33 ( 64.7)<br>12 ( 23.5)<br>5 ( 9.8)<br>0<br>0<br>1 ( 2.0) |
| QTC [FRIDERICIA] (MSEC) <400 400 to <425 425 to <450 450 to <460 460 to <470 470 to <480 480 to <490 >=490 NOT REPORTED | 1 ( 2.0)<br>17 ( 34.0)<br>27 ( 54.0)<br>3 ( 6.0)<br>0<br>0<br>0<br>0<br>2 ( 4.0) | 4 ( 8.2)<br>14 ( 28.6)<br>25 ( 51.0)<br>1 ( 2.0)<br>5 ( 10.2)<br>0<br>0 | 2 ( 3.9)<br>25 ( 49.0)<br>17 ( 33.3)<br>5 ( 9.8)<br>0<br>0<br>1 ( 2.0)<br>1 ( 2.0) | 2 ( 4.0)<br>29 (58.0)<br>13 (26.0)<br>2 ( 4.0)<br>1 ( 2.0)<br>0<br>0<br>1 ( 2.0)<br>2 ( 4.0) | 8 ( 15.7)<br>21 ( 41.2)<br>16 ( 31.4)<br>3 ( 5.9)<br>2 ( 3.9)<br>0<br>0<br>0 |

-----

| Parameter | Values |
|------------------|-----------------|
| Template ID | SS_EG_T_002 |
| Output File Name | rt-eg-cats1.lst |

| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
|---|---|
| Table No. | Appendix 7.3.1C |
| Title 1 | Electrocardiogram Category Summary |
| Title 2 | Treated Subjects - Stage 1 |
| Footnote 1 | Each subject is counted only once using the longest interval observed. |

| Parameter | Values |
|---|---|
| Template ID | SS_EG_T_002 |
| Output File Name | rt-eg-cats2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Appendix 7.3.2C |
| Title 1 | Electrocardiogram Category Summary |
| Title 2 | Treated Subjects - Stage 2 |
| Footnote 1 | Each subject is counted only once using the longest interval observed. |

Template GS\_EG\_L\_X\_001: ECG Listing

Protocol: CN138112  Draft

Electrocardiogram
All Treated Subjects

Treatment Group: TRT A

| Subject ID | | | | Study | | | HR | I | nterv | al (mse | ec) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| (Age/Gender/Race) | Period | Visit | Date | Day | Time | TRD# | (bpm) | PR | QRS | QΤ | QTC | Interpretation |
| PPD (54/M/C) | SCREENING | Day -1 | PPD | -1 | 09:50 | -30D | 66 | 169 | 91 | 402 | 421 | NORMAL |
| PPD (44/F/C) | SCREENING | Day -1 | | -1 | 16 <b>:</b> 47 | -1H | 103 | 180 | 78 | 346 | 405 | ABNORMAL |
| PPD<br>(42/M/C) | SCREENING | Day -1 | | -1 | 17:11 | -32D | 87 | 200 | 70 | 334 | | |
| PPD<br>(55/M/C) | SCREENING<br>SCREENING | Day -30<br>Day -1 | | -44<br>-1 | 09:50<br>13:53 | -29D<br>-2H | 65<br>77 | 165<br>173 | 92<br>93 | 383<br>383 | 399<br>434 | NORMAL<br>ABNORMAL |

# Time relative to most recent dose
Program Source: /wwbdm/ndp/prime/gssr/devtest/ecg/test/eg\_st.sas

07OCT2004:17:58:00

| Parameter | Values |
|------------------|-------------------------------------|
| Template ID | GS_EG_L_X_001 |
| Output File Name | rl-eg-ecgs1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Appendix 7.3.1D |
| Title 1 | Electrocardiogram |
| Title 2 | Treated Subjects - Stage 1 |
| Footnote 1 | # Time relative to most recent dose |

| Parameter | Values |
|-----------|--------|
|-----------|--------|

| Template ID | GS_EG_L_X_001 |
|------------------|-------------------------------------|
| Output File Name | rl-eg-ecgs2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Appendix 7.3.2D |
| Title 1 | Electrocardiogram |
| Title 2 | Treated Subjects - Stage 2 |
| Footnote 1 | # Time relative to most recent dose |

# 4.6.9 Vital Signs and Physical Findings

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_006 |
| Output File Name | rt-vs-sums1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Appendix 7.4.1A |
| Title 1 | Vital Sign Summary of Values and Changes from Baseline over Time |
| Title 2 | Treated Subjects - Stage 1 |
| Layout notes | Parameters are: Sitting Systolic Blood Pressure, Sitting Diastolic Blood Pressure, Sitting Heart Rate (beats/min), Respiration Rate (/min) and Temperature (C). |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_006 |
| Output File Name | rt-vs-sums2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Appendix 7.4.2A |
| Title 1 | Vital Sign Summary of Values and Changes from Baseline over Time |

| Title 2 | Treated Subjects - Stage 2 |
|---|---|
| Layout notes | Parameters are: Sitting Systolic Blood Pressure, Sitting Diastolic Blood Pressure, Sitting Heart Rate (beats/min), Respiration Rate (/min) and Temperature (C). |
## Template GS\_VS\_L\_X\_006: Vital Signs Listing by Treatment Group

Draft Vital Signs All Treated Subjects Protocol: IM101031 

Treatment Group: DRUG A

| Subject ID<br>(Age/Gender/Race) | Period | Visit | Date | Study<br>Day | Position | Blood<br>Pressure<br>(mmHg) | Heart<br>Rate<br>(bpm) | Temp<br>(C) | Resp<br>Rate<br>(/Min) |
|---|---|---|---|---|---|---|---|---|---|
| PPD (46/M/C) | SCREENING<br>PHASE I | DAY -26<br>DAY 1 | PPD | -26<br>1 | SITTING<br>SITTING<br>SITTING | 138 / 90<br>120 / 65<br>126 / 70 | 64<br>68<br>72 | 36.2<br>36.2<br>36.5 | 32<br>34<br>33<br>31 |
| | PHASE II | DAY 13<br>DAY 31 | | 13<br>31 | SITTING<br>SITTING<br>SITTING | 116 / 82<br>120 / 84<br>110 / 70 | 72<br>68<br>72 | 36.7<br>36.6<br>36.6 | 31<br>30<br>33<br>32 |
| | PHASE III | DAY 59 | | 59 | SITTING<br>SITTING<br>SITTING | 122 / 75<br>118 / 76<br>122 / 68 | 80<br>68<br>68 | 36.7<br>36.7<br>36.7 | 32<br>31<br>32 |
| | | DAY 87 | | 87 | STANDING<br>SITTING | 134 / 78<br>134 / 84 | 70<br>72<br>70 | 36.9 | 32 |
| | | DAY 122 | | 122 | SITTING<br>SITTING<br>SITTING | 130 / 80<br>128 / 86<br>124 / 82 | 70<br>70<br>70 | 36.6<br>36.9<br>37.3 | 33<br>32<br>31 |
| | | DAY 142 | | 142 | SITTING<br>SITTING<br>SITTING | 124 / 82<br>126 / 86<br>130 / 80 | 70<br>70<br>78 | 36.7<br>36.7 | 32<br>32 |
| | | DAY 167 | | 167 | SITTING<br>SITTING<br>SITTING | 130 / 80<br>128 / 84<br>132 / 80 | 68<br>70 | 37.2<br>36.9 | 32<br>33<br>33<br>32<br>32 |
| | | DAY 199 | | 199 | SITTING<br>SITTING<br>SITTING | 132 / 84<br>130 / 86 | 80<br>78 | 36.5<br>36.6 | 32<br>30 |
| | POST ST | DAY 223 | | 223 | SITTING | 128 / 84 | 76 | 36.9 | 32 |
| <b>PPD</b> (56/F/C) | SCREENING | DAY -1 | | <b>-</b> 26<br>1 | SITTING<br>SITTING<br>SITTING | 138 / 90<br>/ 80<br>126 / 70 | 64<br>68<br>72 | 36.2<br>36.2<br>36.5 | 32<br>34<br>33 |
| | PHASE I | DAY 7 | | 13 | SITTING<br>SITTING | 116 / 82<br>122 / 75 | 72<br>80 | 36.7<br>36.6 | 31<br>32 |
| | PHASE II<br>PHASE III | DAY 14<br>DAY 21 | | 31<br>87 | SITTING<br>SITTING<br>SITTING | 110 / 70<br>134 / 84<br>130 / 80 | 72<br>72<br>70 | 36.6<br>37.2<br>36.9 | 32<br>32<br>33 |

Program Source: /wwbdm/ndp/prime/gssr/devtest/dem/test/vs\_st.sas

07SEP2004:14:35:00

| Parameter | Values |
|-------------|---------------|
| Template ID | GS_VS_L_X_006 |

| Output File Name | rl-vs-lists1.lst |
|------------------|--------------------------------|
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Appendix 7.4.1B |
| Title 1 | Vital Signs |
| Title 2 | Treated Subjects - Stage 1 |

| Parameter | Values |
|------------------|----------------------------|
| Template ID | GS_VS_L_X_006 |
| Output File Name | rl-vs-lists2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Appendix 7.4.2B |
| Title 1 | Vital Signs |
| Title 2 | Treated Subjects - Stage 2 |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_006 |
| Output File Name | rt-pm-sums1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Appendix 7.4.1C |
| Title 1 | Physical Measurements Summary of Values and Changes from Baseline over Time |
| Title 2 | Treated Subjects - Stage 1 |
| Layout notes | Parameters are: Weight (kg) and BMI (kg/m2). |

| Parameter | Values |
|-------------|-------------|
| Template ID | SS_VL_T_006 |

| Output File Name | rt-pm-sums2.lst |
|---|---|
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Appendix 7.4.2C |
| Title 1 | Physical Measurements Summary of Values and Changes from Baseline over Time |
| Title 2 | Treated Subjects - Stage 2 |
| Layout notes | Parameters are: Weight (kg) and BMI (kg/m2). |

# 4.6.10 Other Observations Related to Safety

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_006 |
| Output File Name | rt-lb-bmrenals1.lst |
| Purpose | WK96S1, WK96S2 |
| Table No. | Table S.7.5.1A |
| Title 1 | Laboratory Test Results |
| Title 2 | Summary Statistics for Renal Biomarker Values and Change from Baseline - US Units |
| Title 3 | Treated Subjects - Stage 1 |
| Programming notes | Include urinary beta-2-microglobilin/creatinine and fractional excretion of phosphorous. |

| Parameter | Values |
|------------------|-------------------------|
| Template ID | SS_VL_T_006 |
| Output File Name | rt-lb-bmrenals2.lst |
| Purpose | WK96S2 |
| Table No. | Table S.7.5.2A |
| Title 1 | Laboratory Test Results |

| Title 2 | Summary Statistics for Renal Biomarker Values and Change from Baseline - US Units |
|---|---|
| Title 3 | Treated Subjects - Stage 2 |
| Programming notes | Include urinary beta-2-microglobilin/creatinine and fractional excretion of phosphorous. |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_006 |
| Output File Name | rt-zl-bmrenals1.lst |
| Purpose | WK96S1, WK96S2 |
| Table No. | Table S.7.5.1B |
| Title 1 | Laboratory Test Results |
| Title 2 | Summary Statistics for Renal Biomarker Values and Change from Baseline - SI Units |
| Title 3 | Treated Subjects - Stage 1 |
| Programming notes | Include urinary beta-2-microglobilin/creatinine and fractional excretion of phosphorous. |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_006 |
| Output File Name | rt-zl-bmrenals2.lst |
| Purpose | WK96S2 |
| Table No. | Table S.7.5.2B |
| Title 1 | Laboratory Test Results |
| Title 2 | Summary Statistics for Renal Biomarker Values and Change from Baseline - SI Units |
| Title 3 | Treated Subjects - Stage 2 |
| Programming notes | Include urinary beta-2-microglobilin/creatinine and fractional excretion of phosphorous. |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_006 |
| Output File Name | rt-lb-pchbmrenals1.lst |
| Purpose | WK96S1, WK96S2 |
| Table No. | Table S.7.5.1C |
| Title 1 | Laboratory Test Results |
| Title 2 | Summary Statistics for Renal Biomarker Values and Percent Change from Baseline - US Units |
| Title 3 | Treated Subjects - Stage 1 |
| Layout notes | Change spanning header to "Percent Change From Baseline". |
| Programming notes | Include urinary beta-2-microglobilin/creatinine and fractional excretion of phosphorous. |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_006 |
| Output File Name | rt-lb-pchbmrenals2.lst |
| Purpose | WK96S2 |
| Table No. | Table S.7.5.2C |
| Title 1 | Laboratory Test Results |
| Title 2 | Summary Statistics for Renal Biomarker Values and Percent Change from Baseline - US Units |
| Title 3 | Treated Subjects - Stage 2 |
| Layout notes | Change spanning header to "Percent Change From Baseline". |
| Programming notes | Include urinary beta-2-microglobilin/creatinine and fractional excretion of phosphorous. |

| Parameter | Values |
|------------------|------------------------|
| Template ID | SS_VL_T_006 |
| Output File Name | rt-zl-pchbmrenals1.lst |

| Purpose | WK96S1, WK96S2 |
|---|---|
| Table No. | Table S.7.5.1D |
| Title 1 | Laboratory Test Results |
| Title 2 | Summary Statistics for Renal Biomarker Values and Percent Change from Baseline - SI Units |
| Title 3 | Treated Subjects - Stage 1 |
| Layout notes | Change spanning header to "Percent Change From Baseline". |
| Programming notes | Include urinary beta-2-microglobilin/creatinine and fractional excretion of phosphorous. |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_006 |
| Output File Name | rt-zl-pchbmrenals2.lst |
| Purpose | WK96S2 |
| Table No. | Table S.7.5.2D |
| Title 1 | Laboratory Test Results |
| Title 2 | Summary Statistics for Renal Biomarker Values and Percent Change from Baseline - SI Units |
| Title 3 | Treated Subjects - Stage 2 |
| Layout notes | Change spanning header to "Percent Change From Baseline". |
| Programming notes | Include urinary beta-2-microglobilin/creatinine and fractional excretion of phosphorous. |

| Parameter | Values |
|------------------|-------------------------|
| Template ID | SS_VL_T_006 |
| Output File Name | rt-lb-bmbones1.lst |
| Purpose | WK24S1 |
| Table No. | Table S.7.5.1E |
| Title 1 | Laboratory Test Results |

| Title 2 | Summary Statistics for Bone Biomarker Values and Change from Baseline - US Units |
|---|---|
| Title 3 | Treated Subjects - Stage 1 |
| Programming notes | Include N-terminal Propeptide of Type 1 procollagen (P1NP) and Cross-linked C-telopeptide of Type 1 collagen (CTx). |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_006 |
| Output File Name | rt-lb-bmbones2.lst |
| Purpose | WK24S2 |
| Table No. | Table S.7.5.2E |
| Title 1 | Laboratory Test Results |
| Title 2 | Summary Statistics for Bone Biomarker Values and Change from Baseline - US Units |
| Title 3 | Treated Subjects - Stage 2 |
| Programming notes | Include N-terminal Propeptide of Type 1 procollagen (P1NP) and Cross-linked C-telopeptide of Type 1 collagen (CTx). |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_006 |
| Output File Name | rt-zl-bmbones1.lst |
| Purpose | WK24S1 |
| Table No. | Table S.7.5.1F |
| Title 1 | Laboratory Test Results |
| Title 2 | Summary Statistics for Bone Biomarker Values and Change from Baseline - SI Units |
| Title 3 | Treated Subjects - Stage 1 |
| Programming notes | Include N-terminal Propeptide of Type 1 procollagen (P1NP) and Cross-linked C-telopeptide of Type 1 collagen (CTx). |

| Parameter | Values |
|-----------|--------|
|-----------|--------|

| Template ID | SS_VL_T_006 |
|---|---|
| Output File Name | rt-zl-bmbones2.lst |
| Purpose | WK24S2 |
| Table No. | Table S.7.5.2F |
| Title 1 | Laboratory Test Results |
| Title 2 | Summary Statistics for Bone Biomarker Values and Change from Baseline - SI Units |
| Title 3 | Treated Subjects - Stage 2 |
| Programming notes | Include N-terminal Propeptide of Type 1 procollagen (P1NP) and Cross-linked C-telopeptide of Type 1 collagen (CTx). |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_006 |
| Output File Name | rt-lb-pchbmbones1.lst |
| Purpose | WK24S1 |
| Table No. | Table S.7.5.1G |
| Title 1 | Laboratory Test Results |
| Title 2 | Summary Statistics for Bone Biomarker Values and Percent Change from Baseline - US Units |
| Title 3 | Treated Subjects - Stage 1 |
| Layout notes | Change spanning header to "Percent Change From Baseline". |
| Programming notes | Include N-terminal Propeptide of Type 1 procollagen (P1NP) and Cross-linked C-telopeptide of Type 1 collagen (CTx). |

| Parameter | Values |
|------------------|-----------------------|
| Template ID | SS_VL_T_006 |
| Output File Name | rt-lb-pchbmbones2.lst |
| Purpose | WK24S2 |
| Table No. | Table S.7.5.2G |

| Title 1 | Laboratory Test Results |
|---|---|
| Title 2 | Summary Statistics for Bone Biomarker Values and Percent Change from Baseline - US Units |
| Title 3 | Treated Subjects - Stage 2 |
| Layout notes | Change spanning header to "Percent Change From Baseline". |
| Programming notes | Include N-terminal Propeptide of Type 1 procollagen (P1NP) and Cross-linked C-telopeptide of Type 1 collagen (CTx). |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_006 |
| Output File Name | rt-zl-pchbmbones1.lst |
| Purpose | WK24S1 |
| Table No. | Table S.7.5.1H |
| Title 1 | Laboratory Test Results |
| Title 2 | Summary Statistics for Bone Biomarker Values and Percent Change from Baseline - SI Units |
| Title 3 | Treated Subjects - Stage 1 |
| Layout notes | Change spanning header to "Percent Change From Baseline". |
| Programming notes | Include N-terminal Propeptide of Type 1 procollagen (P1NP) and Cross-linked C-telopeptide of Type 1 collagen (CTx). |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_006 |
| Output File Name | rt-zl-pchbmbones2.lst |
| Purpose | WK24S2 |
| Table No. | Table S.7.5.2H |
| Title 1 | Laboratory Test Results |
| Title 2 | Summary Statistics for Bone Biomarker Values and Percent Change from Baseline - SI Units |
| Title 3 | Treated Subjects - Stage 2 |

| Layout notes | Change spanning header to "Percent Change From Baseline". |
|---|---|
| Programming notes | Include N-terminal Propeptide of Type 1 procollagen (P1NP) and Cross-linked C-telopeptide of Type 1 collagen (CTx). |

| Parameter | Values |
|---|---|
| Template ID | GS_LB_G_002 |
| Output File Name | rg-lb-ub2s1 |
| Purpose | WK24S1 |
| Table No. | Figure S.7.5.1A |
| Title 1 | Urinary Beta-2-Microglobulin/Creatinine Median Percent Change from Baseline Over Time |
| Title 2 | Treated Subjects - Stage 1 |
| Layout notes | Y-axis label: Urinary Beta-2-Microglobulin/Creatinine Median Percent Change from Baseline (IQR) X-axis label: Time (Weeks) Include horizontal reference line at Y=0. |

| Parameter | Values |
|---|---|
| Template ID | GS_LB_G_002 |
| Output File Name | rg-lb-ub2s2 |
| Purpose | WK24S2 |
| Table No. | Figure S.7.5.2A |
| Title 1 | Urinary Beta-2-Microglobulin/Creatinine Median Percent Change from Baseline Over Time |
| Title 2 | Treated Subjects - Stage 2 |
| Layout notes | Y-axis label: Urinary Beta-2-Microglobulin/Creatinine Median Percent Change from Baseline (IQR) |
| | X-axis label: Time (Weeks) |
| | Include horizontal reference line at Y=0. |

| Parameter | Values |
|---|---|
| Template ID | GS_LB_G_002 |
| Output File Name | rg-lb-feps1 |
| Purpose | WK24S1 |
| Table No. | Figure S.7.5.1B |
| Title 1 | Fractional Excretion of Phosphorous Median Change from Baseline Over Time |
| Title 2 | Treated Subjects - Stage 1 |
| Layout notes | Y-axis label: Fractional Excretion of Phosphorous Median Change from Baseline (IQR) |
| | X-axis label: Time (Weeks) |
| | Include horizontal reference line at Y=0. |

| Parameter | Values |
|---|---|
| Template ID | GS_LB_G_002 |
| Output File Name | rg-lb-feps2 |
| Purpose | WK24S2 |
| Table No. | Figure S.7.5.2B |
| Title 1 | Fractional Excretion of Phosphorous Median Change from Baseline Over Time |
| Title 2 | Treated Subjects - Stage 2 |
| Layout notes | Y-axis label: Fractional Excretion of Phosphorous Median Change from Baseline (IQR) |
| | X-axis label: Time (Weeks) |
| | Include horizontal reference line at Y=0. |

| Parameter | Values |
|------------------|-----------------|
| Template ID | GS_LB_G_002 |
| Output File Name | rg-lb-pchp1nps1 |
| Purpose | WK96S1, WK96S2 |

| Table No. | Figure S.7.5.1C |
|---|---|
| Title 1 | N-Terminal Propeptide of Type 1 Procollagen Median Percent Change from Baseline Over Time |
| Title 2 | Treated Subjects - Stage 1 |
| Layout notes | Y-axis label: P1NP Median Percent Change from Baseline (IQR) |
| | X-axis label: Time (Weeks) |
| | Include horizontal reference line at Y=0. |

| Parameter | Values |
|---|---|
| Template ID | GS_LB_G_002 |
| Output File Name | rg-lb-pchp1nps2 |
| Purpose | WK96S2 |
| Table No. | Figure S.7.5.2C |
| Title 1 | N-Terminal Propeptide of Type 1 Procollagen Median Percent Change from Baseline Over Time |
| Title 2 | Treated Subjects - Stage 2 |
| Layout notes | Y-axis label: P1NP Median Percent Change from Baseline (IQR) |
| | X-axis label: Time (Weeks) |
| | Include horizontal reference line at Y=0. |

| Parameter | Values |
|---|---|
| Template ID | GS_LB_G_002 |
| Output File Name | rg-lb-pchctxs1 |
| Purpose | WK96S1, WK96S2 |
| Table No. | Figure S.7.5.1D |
| Title 1 | Cross-Linked C-Telopeptide of Type 1 Collagen Median Percent Change from Baseline Over Time |
| Title 2 | Treated Subjects - Stage 1 |
| Layout notes | Y-axis label: CTx Median Percent Change from Baseline (IQR) |

| X-axis label: Time (Weeks) |
|-------------------------------------------|
| Include horizontal reference line at Y=0. |

| Parameter | Values |
|---|---|
| Template ID | GS_LB_G_002 |
| Output File Name | rg-lb-pchctxs2 |
| Purpose | WK96S2 |
| Table No. | Figure S.7.5.2D |
| Title 1 | Cross-Linked C-Telopeptide of Type 1 Collagen Median Percent Change from Baseline Over Time |
| Title 2 | Treated Subjects - Stage 2 |
| Layout notes | Y-axis label: CTx Median Percent Change from Baseline (IQR) |
| | X-axis label: Time (Weeks) |
| | Include horizontal reference line at Y=0. |

## 4.7 Pharmacokinetic Results

Template MS\_PK\_T\_004: Summary Statistics for PK Parameters

| | | | | TREATI | ÆNT |
|---------------|---------------|-----------|---------|---------|---------|
| <br>PARAMETER | UNIT | STATISTIC | A | В | ( |
| Cmax | ng/mL | N | XX | XX | XX |
| | 9, | MEAN | XXXX.XX | XXXX.XX | XXXX.XX |
| | | S.D. | XXXX.XX | XXXX.XX | XXXX.X |
| | | GEO.MEAN | XXXX.XX | XXXX.XX | XXXX.X |
| | | %CV | XX | XX | X |
| | | MEDIAN | XXXX.XX | XXXX.XX | XXXX.X |
| | | MIN | XXXX.XX | XXXX.XX | XXXX.X |
| | | MAX | XXXX.XX | XXXX.XX | XXXX.X |
| Tmax | h | N | XX | XX | X |
| | | MEAN | XXXX.XX | XXXX.XX | XXXX.X |
| | | S.D. | XXXX.XX | XXXX.XX | XXXX.XX |
| | | GEO.MEAN | XXXX.XX | XXXX.XX | XXXX.X |
| | | %CV | XX | XX | X |
| | | MEDIAN | XXXX.XX | XXXX.XX | XXXX.X |
| | | MIN | XXXX.XX | XXXX.XX | XXXX.X |
| | | MAX | XXXX.XX | XXXX.XX | XXXX.X |
| AUC | ng.h/mL | N | XX | XX | XX |
| 1100 | 119 •11/ 1100 | MEAN | XXXX.XX | XXXX.XX | XXXX.X |
| | | S.D. | XXXX.XX | XXXX.XX | XXXX.XX |
| | | GEO.MEAN | XXXX.XX | XXXX.XX | XXXX.X |
| | | %CV | XX | XX | X |
| | | MEDIAN | XXXX.XX | XXXX.XX | XXXX.X |
| | | MIN | XXXX.XX | XXXX.XX | XXXX.X |
| | | MAX | XXXX.XX | XXXX.XX | XXXX.X |

------

| Parameter | Values |
|-------------|-------------|
| Template ID | MS_PK_T_004 |

| Output File Name | rt-pk-sumbmss1.lst |
|---|---|
| Purpose | WK24S1 |
| Table No. | Table S.8.1.1A |
| Title 1 | Summary Statistics of BMS-955176 Pharmacokinetic Parameters |
| Title 2 | Evaluable PK Population - Stage 1 |
| Footnote 1 | A = BMS 955176 120 mg QD + ATV/r + DTG |
| Layout notes | PK parameters: Cmax, Tmax, Ctau, C0, AUC(TAU) |

| Parameter | Values |
|---|---|
| Template ID | MS_PK_T_004 |
| Output File Name | rt-pk-sumbmss2.lst |
| Purpose | WK24S2 |
| Table No. | Table S.8.1.2A |
| Title 1 | Summary Statistics of BMS-955176 Pharmacokinetic Parameters |
| Title 2 | Evaluable PK Population - Stage 2 |
| Footnote 1 | C = BMS 955176 120 mg QD + ATV + DTG |
| | D = BMS 955176 180 mg QD + ATV + DTG |
| Layout notes | PK parameters: Cmax, Tmax, Ctau, C0, AUC(TAU) |

| Parameter | Values |
|------------------|--------------------|
| Template ID | MS_PK_T_004 |
| Output File Name | rt-pk-sumatvs1.lst |
| Purpose | WK24S1 |
| Table No. | Table S.8.1.1B |

| Title 1 | Summary Statistics of ATV Pharmacokinetic Parameters |
|---|---|
| Title 2 | Evaluable PK Population - Stage 1 |
| Footnote 1 | A = BMS 955176 120 mg QD + ATV/r + DTG<br>B = TDF + ATV/r + DTG |
| Layout notes | PK parameters: Cmax, Tmax, Ctau, C0, AUC(TAU) |

| Parameter | Values |
|---|---|
| Template ID | MS_PK_T_004 |
| Output File Name | rt-pk-sumatvs2.lst |
| Purpose | WK24S2 |
| Table No. | Table S.8.1.2B |
| Title 1 | Summary Statistics of ATV Pharmacokinetic Parameters |
| Title 2 | Evaluable PK Population - Stage 2 |
| Footnote 1 | C = BMS 955176 120 mg QD + ATV + DTG<br>D = BMS 955176 180 mg QD + ATV + DTG<br>E = TDF + ATV/r + DTG |
| Layout notes | PK parameters: Cmax, Tmax, Ctau, C0, AUC(TAU) |

| Parameter | Values |
|------------------|------------------------------------------------------|
| Template ID | MS_PK_T_004 |
| Output File Name | rt-pk-sumdtgs1.lst |
| Purpose | WK24S1 |
| Table No. | Table S.8.1.1C |
| Title 1 | Summary Statistics of DTG Pharmacokinetic Parameters |

| Title 2 | Evaluable PK Population - Stage 1 |
|---|---|
| Footnote 1 | A = BMS 955176 120 mg QD + ATV/r + DTG $B = TDF + ATV/r + DTG$ |
| Layout notes | PK parameters: Cmax, Tmax, Ctau, C0, AUC(TAU) |

| Parameter | Values |
|---|---|
| Template ID | MS_PK_T_004 |
| Output File Name | rt-pk-sumdtgs2.lst |
| Purpose | WK24S2 |
| Table No. | Table S.8.1.2C |
| Title 1 | Summary Statistics of DTG Pharmacokinetic Parameters |
| Title 2 | Evaluable PK Population - Stage 2 |
| Footnote 1 | C = BMS 955176 120 mg QD + ATV + DTG<br>D = BMS 955176 180 mg QD + ATV + DTG<br>E = TDF + ATV/r + DTG |
| Layout notes | PK parameters: Cmax, Tmax, Ctau, C0, AUC(TAU) |

# Template MS\_PK\_T\_005: In-text Table for Summary Statistics for PK Parameters

| DA DAMERIUD | | TREATMENT | |
|---|---|---|---|
| PARAMETER<br>STATISTIC | A | В | С |
| Cmax (ng/mL)<br>Geo.Mean [N]<br>(%CV) | 199 [12]<br>(25) | 640 [12]<br>(21) | 493 [12]<br>(27) |
| AUC(0-T)(ng.h/mL)<br>Geo.Mean[N]<br>(%CV) | 721 [12]<br>(15) | 534 [12]<br>(27) | 503 [12]<br>(23) |
| AUC(INF)(ng.h/mL)<br>Geo.Mean[N]<br>(%CV) | 696 [12]<br>(22) | 612 [12]<br>(23) | 523 [12]<br>(21) |
| Tmax (h)<br>Median [N]<br>(Min - Max) | | 1.75 [16]<br>(1.00 - 5.00) | |
| T-HALF (h)<br>Mean [N]<br>(SD) | 9.70 [15]<br>(2.862) | 8.71 [16]<br>(3.912) | 8.90 [16]<br>(3.762) |

| Parameter | Values |
|---|---|
| Template ID | MS_PK_T_005 |
| Output File Name | rt-pk-itsumbmss1.lst |
| Purpose | WK24S1 |
| Table No. | Table 9.2.1A |
| Title 1 | Summary Statistics of BMS-955176 Pharmacokinetic Parameters |
| Title 2 | Evaluable PK Population - Stage 1 |
| Footnote 1 | A = BMS 955176 120 mg QD + ATV/r + DTG |
| Programming notes | This is an in-text table |

| Parameter | Values |
|---|---|
| Template ID | MS_PK_T_005 |
| Output File Name | rt-pk-itsumbmss2.lst |
| Purpose | WK24S2 |
| Table No. | Table 9.2.2A |
| Title 1 | Summary Statistics of BMS-955176 Pharmacokinetic Parameters |
| Title 2 | Evaluable PK Population - Stage 2 |
| Footnote 1 | C = BMS 955176 120 mg QD + ATV + DTG |
| | D = BMS 955176 180 mg QD + ATV + DTG |
| Programming notes | This is an in-text table |

| Parameter | Values |
|---|---|
| Template ID | MS_PK_T_005 |
| Output File Name | rt-pk-itsumdtgs1.lst |
| Purpose | WK24S1 |
| Table No. | Table 9.3.1A |
| Title 1 | Summary Statistics of DTG Pharmacokinetic Parameters |
| Title 2 | Evaluable PK Population - Stage 1 |
| Footnote 1 | A = BMS 955176 120 mg QD + ATV/r + DTG $B = TDF + ATV/r + DTG$ |
| Programming notes | This is an in-text table |

| Parameter | Values |
|------------------|----------------------|
| Template ID | MS_PK_T_005 |
| Output File Name | rt-pk-itsumdtgs2.lst |

| Purpose | WK24S2 |
|---|---|
| Table No. | Table 9.3.2A |
| Title 1 | Summary Statistics of DTG Pharmacokinetic Parameters |
| Title 2 | Evaluable PK Population - Stage 2 |
| Footnote 1 | C = BMS 955176 120 mg QD + ATV + DTG<br>D = BMS 955176 180 mg QD + ATV + DTG<br>E = TDF + ATV/r + DTG |
| Programming notes | This is an in-text table |

| Parameter | Values |
|-------------------|------------------------------------------------------|
| Template ID | MS_PK_T_005 |
| Output File Name | rt-pk-itsumatvs1.lst |
| Purpose | WK24S1 |
| Table No. | Table 9.4.1A |
| Title 1 | Summary Statistics of ATV Pharmacokinetic Parameters |
| Title 2 | Evaluable PK Population - Stage 1 |
| Footnote 1 | A = BMS 955176 120 mg QD + ATV/r + DTG |
| | B = TDF + ATV/r + DTG |
| Programming notes | This is an in-text table |

| Parameter | Values |
|------------------|------------------------------------------------------|
| Template ID | MS_PK_T_005 |
| Output File Name | rt-pk-itsumatvs2.lst |
| Purpose | WK24S2 |
| Table No. | Table 9.4.2A |
| Title 1 | Summary Statistics of ATV Pharmacokinetic Parameters |

| Title 2 | Evaluable PK Population - Stage 2 |
|-------------------|--------------------------------------|
| Footnote 1 | C = BMS 955176 120 mg QD + ATV + DTG |
| | D = BMS 955176 180 mg QD + ATV + DTG |
| | E = TDF + ATV/r + DTG |
| Programming notes | This is an in-text table |

### Template MS PK T 006: Statistical Analysis for PK Parameters

#### PK Parameter

| | | | | On Natural | Logarithmic S | | | on Original Scale |
|---|---|---|---|---|---|---|---|---|
| TREATMENT AND COMPARISON | ADJUSTED S<br>MEAN | STANDARD<br>ERROR | DF | Т | Pr > T | 90% CI | ADJUSTED<br>GEO MEAN | 90% CI |
| A<br>B<br>B vs A | X.XXX<br>X.XXX<br>X.XXX | X.XXX<br>X.XXX<br>X.XXX | X.X<br>X.X<br>X.X | XX.XX<br>XX.XX<br>X.XX | 0.XXXX<br>0.XXXX<br>0.XXXX | (X.XXX,X.XXX)<br>(X.XXX,X.XXX)<br>(X.XXX,X.XXX) | XXXX.XXX<br>XXXX.XXX<br>X.XXX | (XXXX.XXX,XXXX.XXX)<br>(XXXX.XXX,XXXX.XXX)<br>(X.XXX,X.XXX) |

#### MODEL INFORMATION

Covariance Structure - Unstructured Subject Effect - USUBJID Estimation Method - REML Residual Variance Method - None

Fixed Effects SE Method - Prasad-Rao-Jeske-Kackar-Harville

Degrees of Freedom Method - Kenward-Roger Fixed Effects - TRI SEQ PERIOD USUBJID

Covariance Matrix Block

| Row | Col 1 | Col 2 | COL 3 |
|-----|-------|-------|-------|
| 1 | X.XXX | X.XXX | X.XXX |
| 2 | X.XXX | X.XXX | X.XXX |
| 3 | X.XXX | X.XXX | X.XXX |

| Parameter | Values |
|---|---|
| Template ID | MS_PK_T_006 |
| Output File Name | rt-pk-mixedbmsdtgs1.lst |
| Purpose | WK24S1 |
| Table No. | Table S.8.2.5.1A |
| Title 1 | Effect of BMS-955176 on Exposure of DTG |
| Title 2 | PK Parameters DTG Cmax, Ctau and AUC(TAU) |
| Title 3 | BMS-955176 120 mg QD+ ATV/r + DTG versus TDF + ATV/r + DTG |
| Title 4 | Evaluable PK Population - Stage 1 |

| Footnote 1 | A = BMS 955176 120 mg QD + ATV/r + DTG |
|------------|-----------------------------------------|
| | B = TDF + ATV/r + DTG |

| Parameter | Values |
|---|---|
| Template ID | MS_PK_T_006 |
| Output File Name | rt-pk-mixedbms120dtgs2.lst |
| Purpose | WK24S2 |
| Table No. | Table S.8.2.5.2A |
| Title 1 | Effect of BMS-955176 on Exposure of DTG |
| Title 2 | PK Parameters DTG Cmax, Ctau and AUC(TAU) |
| Title 3 | BMS-955176 120 mg QD+ ATV + DTG versus Historical Data |
| Title 4 | Evaluable PK Population - Stage 2 |
| Footnote 1 | C = BMS 955176 120 mg QD + ATV + DTG<br>F = Historical Data |

| Parameter | Values |
|---|---|
| Template ID | MS_PK_T_006 |
| Output File Name | rt-pk-mixedbms180dtgs2.lst |
| Purpose | WK24S2 |
| Table No. | Table S.8.2.5.2B |
| Title 1 | Effect of BMS-955176 on Exposure of DTG |
| Title 2 | PK Parameters DTG Cmax, Ctau and AUC(TAU) |
| Title 3 | BMS-955176 180 mg QD+ ATV + DTG versus Historical Data |
| Title 4 | Evaluable PK Population - Stage 2 |
| Footnote 1 | D = BMS 955176 180 mg QD + ATV + DTG |
| | F = Historical Data |

## Template MS\_PK\_T\_007: In-text Table for Statistical Analysis for PK Parameters

| PK<br>PARAMETER | TREATMENT AND COMPARISON | ADJUSTED<br>GEOMETRIC MEAN | 90% CI |
|---|---|---|---|
| CMAX (ng/mL) | A | XX.XX | (XX.XX, XX.XX) |
| | B | XX.XX | (XX.XX, XX.XX) |
| | B vs A | X.XXX | (X.XXX, X.XXX) |
| CTAU (ng/mL) | A | XX.XX | (XX.XX, XX.XX) |
| | B | XX.XX | (XX.XX, XX.XX) |
| | B vs A | X.XXX | (X.XXX, X.XXX) |
| AUC(TAU)(ng.h/mL) | A | XX.XX | (XX.XX, XX.XX) |
| | B | XX.XX | (XX.XX, XX.XX) |
| | B vs A | X.XXX | (X.XXX, X.XXX) |

-----

| Parameter | Values |
|---|---|
| Template ID | MS_PK_T_007 |
| Output File Name | rt-pk-itmixedbmss1.lst |
| Purpose | WK24S1 |
| Table No. | Table 9.3.1.1A |
| Title 1 | In-text Table of Effect of BMS-955176 on Exposure of DTG |
| Title 2 | PK Parameters DTG Cmax, Ctau and AUC(TAU) |
| Title 3 | BMS-955176 120 mg QD+ ATV/r + DTG versus TDF + ATV/r + DTG |
| Title 4 | Evaluable PK Population - Stage 1 |
| Footnote 1 | A = BMS 955176 120 mg QD + ATV/r + DTG |
| | B = TDF + ATV/r + DTG |
| Footnote 2 | Source: Table S.8.2.5.1A |
| Programming notes | This is an in-text table |

| Parameter | Values |
|-------------------|----------------------------------------------------------|
| Template ID | MS_PK_T_007 |
| Output File Name | rt-pk-itmixedbms120s2.lst |
| Purpose | WK24S2 |
| Table No. | Table 9.3.1.2A |
| Title 1 | In-text Table of Effect of BMS-955176 on Exposure of DTG |
| Title 2 | PK Parameters DTG Cmax, Ctau and AUC(TAU) |
| Title 3 | BMS-955176 120 mg QD+ ATV + DTG versus TDF + ATV/r + DTG |
| Title 4 | Evaluable PK Population - Stage 2 |
| Footnote 1 | C = BMS 955176 120 mg QD + ATV + DTG |
| | F = Historical Data |
| Footnote 2 | Source: Table S.8.2.5.2A |
| Programming notes | This is an in-text table |

| Parameter | Values |
|------------------|----------------------------------------------------------|
| Template ID | MS_PK_T_007 |
| Output File Name | rt-pk-itmixedbms180s2.lst |
| Purpose | WK24S2 |
| Table No. | Table 9.3.1.2B |
| Title 1 | In-text Table of Effect of BMS-955176 on Exposure of DTG |
| Title 2 | PK Parameters DTG Cmax, Ctau and AUC(TAU) |
| Title 3 | BMS-955176 180 mg QD+ ATV + DTG versus TDF + ATV/r + DTG |
| Title 4 | Evaluable PK Population - Stage 2 |
| Footnote 1 | D = BMS 955176 180 mg QD + ATV + DTG |
| | F = Historical Data |
| Footnote 2 | Source: Table S.8.2.5.2B |

| Programming notes | This is an in-text table |
|-------------------|--------------------------|

# Template MS\_PK\_L\_005: Listing for PK Parameters

| Subject | Treatment | Study<br>Day | Cmax<br>(ng/mL) | Tmax<br>(h) | Ctau<br>(ng*h/mL) | CO<br>(ng*h/mL) | AUC (TAU) | Exclusion<br>Flag |
|---|---|---|---|---|---|---|---|---|
| XXXXXXXX-X-X | А | 1<br>14 | XX.XX<br>XX.XX | XX.XX<br>XX.XX | XX.XX<br>XX.XX | XX.XX<br>XX.XX | XX.XX<br>XX.XX | 3 |
| XXXXXXX-X-X | В | 1<br>14 | XX.XX<br>XX.XX | XX.XX<br>XX.XX | XX.XX<br>XX.XX | XX.XX<br>XX.XX | XX.XX<br>XX.XX | |

| Parameter | Values |
|---|---|
| Template ID | MS_PK_L_005 |
| Output File Name | rl-pk-listbms01s1.lst |
| Purpose | WK24S1 |
| Table No. | Appendix 8.2.5A |
| Title 1 | Listing of BMS-955176 Pharmacokinetic Parameters |
| Title 2 | PK Population - Stage 1 |
| Footnote 1 | A = BMS 955176 120 mg QD + ATV/r + DTG $B = TDF + ATV/r + DTG$ |
| Footnote 2 | Note:# Values are excluded from PK Summary Statistics |
| Footnote 3 | Exclusion Flag Definitions: 1= All Parameters, 2= CMAX, 3= Tmax, 4= Ctau, 5= C0, 6= AUC(TAU) |

| Parameter | Values |
|------------------|-----------------------|
| Template ID | MS_PK_L_005 |
| Output File Name | rl-pk-listbms01s2.lst |
| Purpose | WK24S2 |
| Table No. | Appendix 8.2.5A |

| Title 1 | Listing of BMS-955176 Pharmacokinetic Parameters |
|---|---|
| Title 2 | X Population - Stage 2 |
| Footnote 1 | C = BMS 955176 120 mg QD + ATV + DTG |
| | D = BMS 955176 180 mg QD + ATV + DTG |
| | E = TDF + ATV/r + DTG |
| Footnote 2 | Note:# Values are excluded from PK Summary Statistics |
| Footnote 3 | Exclusion Flag Definitions: 1= All Parameters, 2= CMAX, 3= Tmax, 4= Ctau, 5= C0, 6= AUC(TAU) |

| Parameter | Values |
|---|---|
| Template ID | MS_PK_L_005 |
| Output File Name | rl-pk-listatv01s1.lst |
| Purpose | WK24S1 |
| Table No. | Appendix 8.2.5B |
| Title 1 | Listing of ATV Pharmacokinetic Parameters |
| Title 2 | PK Population - Stage 1 |
| Footnote 1 | A = BMS 955176 120 mg QD + ATV/r + DTG |
| | B = TDF + ATV/r + DTG |
| Footnote 2 | note 2 Note:# Values are excluded from PK Summary Statistics |
| Footnote 3 | Exclusion Flag Definitions: 1= All Parameters, 2= CMAX, 3= Tmax, 4= Ctau, 5= C0, 6= AUC(TAU) |

| Parameter | Values |
|-------------------------|-----------------------|
| Template ID MS_PK_L_005 | |
| Output File Name | rl-pk-listatv01s2.lst |
| Purpose | WK24S2 |
| Table No. | |
| Title 1 | |

| Title 2 | PK Population - Stage 2 |
|---|---|
| Footnote 1 | C = BMS 955176 120 mg QD + ATV + DTG<br>D = BMS 955176 180 mg QD + ATV + DTG<br>E = TDF + ATV/r + DTG |
| Footnote 2 | Note:# Values are excluded from PK Summary Statistics |
| Footnote 3 | Exclusion Flag Definitions: 1= All Parameters, 2= CMAX, 3= Tmax, 4= Ctau, 5= C0, 6= AUC(TAU) |

| Parameter | Values |
|---|---|
| Template ID | MS_PK_L_005 |
| Output File Name | rl-pk-listdtg01s1.lst |
| Purpose | WK24S1 |
| Table No. | Appendix 8.2.5C |
| Title 1 | Listing of DTG Pharmacokinetic Parameters |
| Title 2 | PK Population - Stage 1 |
| Footnote 1 | A = BMS 955176 120 mg QD + ATV/r + DTG |
| | B = TDF + ATV/r + DTG |
| Footnote 2 | Note:# Values are excluded from PK Summary Statistics |
| Footnote 3 | Exclusion Flag Definitions: 1= All Parameters, 2= CMAX, 3= Tmax, 4= Ctau, 5= C0, 6= AUC(TAU) |

| Parameter | Values |
|------------------|-----------------------|
| Template ID | MS_PK_L_005 |
| Output File Name | rl-pk-listdtg01s2.lst |
| Purpose | WK24S2 |
| Table No. | Appendix 8.2.5C |
| Title 1 | |
| Title 2 | |

| Footnote 1 | C = BMS 955176 120 mg QD + ATV + DTG<br>D = BMS 955176 180 mg QD + ATV + DTG |
|---|---|
| | E = TDF + ATV/r + DTG |
| Footnote 2 | Note:# Values are excluded from PK Summary Statistics |
| Footnote 3 | Exclusion Flag Definitions: 1= All Parameters, 2= CMAX, 3= Tmax, 4= Ctau, 5= C0, 6= AUC(TAU) |

# $Template\ MS\_PK\_L\_001:\ Listing\ of\ Plasma\ Concentration-Time\ Data$

| SUBJECT | TREATMENT | STUDY<br>DAY | NOMINAL<br>TIME (h) | ACTUAL<br>TIME (h) | CONCENTRATION<br>(ng/mL) | EXCLUSION<br>FLAG |
|---|---|---|---|---|---|---|
| PPD | A | 14 | 0.00<br>1.00<br>1.50<br>2.00<br>3.00<br>4.00<br>8.00<br>12.00<br>18.00<br>24.00<br>48.00<br>72.00<br>96.00<br>120.00<br>144.00 | 0.00<br>1.00<br>1.50<br>2.00<br>3.00<br>4.00<br>8.00<br>12.00<br>18.00<br>24.00<br>48.00<br>72.00<br>96.00<br>120.02 | <pre><llq 1.12="" 100.02="" 108.94="" 11.73="" 15.75="" 22.94="" 3.30="" 36.39="" 46.23="" 79.14="" 99.00="" <="" pre=""> <pre><llq< pre=""> <pre><llq< pre=""> <pre><llq< pre=""></llq<></pre></llq<></pre></llq<></pre></llq></pre> | |

\_\_\_\_\_\_

| Parameter | Values |
|---|---|
| Template ID | MS_PK_L_001 |
| Output File Name | rl-pk-cpar1bmss1.lst |
| Purpose | WK24S1 |
| Table No. | Appendix 8.2.1A |
| Title 1 | Listing of BMS-955176 Plasma Concentration – Time Data |
| Title 2 | PK Population - Stage 1 |
| Footnote 1 | A = BMS 955176 120 mg QD + ATV/r + DTG $B = TDF + ATV/r + DTG$ |
| Footnote 2 | Note: <llq (xx="" =="" below="" limit="" lower="" ml)<="" ng="" of="" quantification="" td=""></llq> |

| Parameter | Values |
|---|---|
| Template ID | MS_PK_L_001 |
| Output File Name | rl-pk-cpar1bmss2.lst |
| Purpose | WK24S2 |
| Table No. | Appendix 8.2.1A |
| Title 1 | Listing of BMS-955176 Plasma Concentration – Time Data |
| Title 2 | PK Population - Stage 2 |
| Footnote 1 | C = BMS 955176 120 mg QD + ATV + DTG<br>D = BMS 955176 180 mg QD + ATV + DTG<br>E = TDF + ATV/r + DTG |
| Footnote 2 Note: <llq (xx="" =="" below="" limit="" lower="" ml)<="" ng="" of="" quantification="" td=""></llq> | |

| Parameter | Values |
|---|---|
| Template ID | MS_PK_L_001 |
| Output File Name | -pk-cparlatvs1.lst |
| Purpose | WK24S1 |
| Table No. | Appendix 8.2.1B |
| Title 1 | Listing of ATV Plasma Concentration – Time Data |
| Title 2 | PK Population - Stage 1 |
| Footnote 1 | A = BMS 955176 120 mg QD + ATV/r + DTG $B = TDF + ATV/r + DTG$ |
| Footnote 2 Note: <llq (xx="" =="" below="" limit="" lower="" ml)<="" ng="" of="" quantification="" td=""></llq> | |

| Parameter | Values |
|-------------|-------------|
| Template ID | MS_PK_L_001 |

| Output File Name | rl-pk-cpar1atvs2.lst |
|---|---|
| Purpose | WK24S2 |
| Table No. | Appendix 8.2.1B |
| Title 1 | Listing of ATV Plasma Concentration – Time Data |
| Title 2 | PK Population - Stage 2 |
| Footnote 1 | C = BMS 955176 120 mg QD + ATV + DTG<br>D = BMS 955176 180 mg QD + ATV + DTG<br>E = TDF + ATV/r + DTG |
| Footnote 2 | Note: <llq (xx="" =="" below="" limit="" lower="" ml)<="" ng="" of="" quantification="" td=""></llq> |

| Parameter | Values |
|---|---|
| Template ID | MS_PK_L_001 |
| Output File Name | rl-pk-cpar1dtgs1.lst |
| Purpose | WK24S1 |
| Table No. | Appendix 8.2.1C |
| Title 1 | Listing of DTG Plasma Concentration – Time Data |
| Title 2 | PK Population - Stage 1 |
| Footnote 1 | A = BMS 955176 120 mg QD + ATV/r + DTG $B = TDF + ATV/r + DTG$ |
| Footnote 2 | Note: <llq (xx="" =="" below="" limit="" lower="" ml)<="" ng="" of="" quantification="" td=""></llq> |

| Parameter | Values |
|------------------|----------------------|
| Template ID | MS_PK_L_001 |
| Output File Name | rl-pk-cpar1dtgs2.lst |
| Purpose | WK24S2 |

| Table No. | Appendix 8.2.1C |
|---|---|
| Title 1 | Listing of DTG Plasma Concentration – Time Data |
| Title 2 | PK Population - Stage 2 |
| Footnote 1 | C = BMS 955176 120 mg QD + ATV + DTG |
| | D = BMS 955176 180 mg QD + ATV + DTG |
| | E = TDF + ATV/r + DTG |
| Footnote 2 | Note: <llq (xx="" =="" below="" limit="" lower="" ml)<="" ng="" of="" quantification="" td=""></llq> |

# Template MS\_PK\_G\_002: Individual Plot of Plasma Concentrations vs. Time



| Parameter | Values |
|---|---|
| Template ID | MS_PK_G_002 |
| Output File Name | rg-pk-cpar3bmss1.lst |
| Purpose | WK24S1 |
| Table No. | Figure S.8.2.3A |
| Title 1 | Plots of Individual BMS-955176 Plasma Concentration Profiles vs. Time |
| Title 2 | Evaluable PK Population - Stage 1 |
| Footnote 1 | A = BMS 955176 120 mg QD + ATV/r + DTG |
| | B = TDF + ATV/r + DTG |
| Footnote 2 | Notes: LLOQ – xx ng/mL; <lloq "missing"="" as="" calculation="" for="" mean="" of="" td="" treated="" values="" values<="" were=""></lloq> |
| Layout notes | x-axis label: time |
| | y-axis label: BMS-955176 concentration (ng/mL) |
| Programming notes | 1. There should be two plots (on same page): |
| | a. Cartesian Plot over 24 h or tau (to show Cmax differences) |
| | b. Semi-Log Plot over entire time range (to show terminal phase differences |
| | 2. Treatment and/or Study Day overlay, as appropriate |
| | 3. Add in dotted line for LLOQ value |
| | 4. Cartesian and semi-log plots for each individual subject on the same page |

| Parameter | Values |
|---|---|
| Template ID | MS_PK_G_002 |
| Output File Name | rg-pk-cpar3bmss2.lst |
| Purpose | WK24S2 |
| Table No. | Figure S.8.2.3A |
| Title 1 | Plots of Individual BMS-955176 Plasma Concentration Profiles vs. Time |
| Title 2 | Evaluable PK Population - Stage 2 |
| Footnote 1 | C = BMS 955176 120 mg QD + ATV + DTG |
| | D = BMS 955176 180 mg QD + ATV + DTG |
|---|---|
| | E = TDF + ATV/r + DTG |
| Footnote 2 | Notes: LLOQ – xx ng/mL; <lloq "missing"="" as="" calculation="" for="" mean="" of="" td="" treated="" values="" values<="" were=""></lloq> |
| Layout notes | x-axis label: time |
| | y-axis label: BMS-955176 concentration (ng/mL) |
| Programming notes | 1. There should be two plots (on same page): |
| | a. Cartesian Plot over 24 h or tau (to show Cmax differences) |
| | b. Semi-Log Plot over entire time range (to show terminal phase differences |
| | 2. Treatment and/or Study Day overlay, as appropriate |
| | 3. Add in dotted line for LLOQ value |
| | 4. Cartesian and semi-log plots for each individual subject on the same page |

| Parameter | Values |
|---|---|
| Template ID | MS_PK_G_002 |
| Output File Name | rg-pk-cpar3atvs1.lst |
| Purpose | WK24S1 |
| Table No. | Figure S.8.2.3B |
| Title 1 | Plots of Individual ATV Plasma Concentration Profiles vs. Time |
| Title 2 | Evaluable PK Population- Stage 1 |
| Footnote 1 | A = BMS 955176 120 mg QD + ATV/r + DTG |
| | B = TDF + ATV/r + DTG |
| Footnote 2 | Notes: LLOQ – xx ng/mL; <lloq "missing"="" as="" calculation="" for="" mean="" of="" td="" treated="" values="" values<="" were=""></lloq> |
| Layout notes | x-axis label: time |
| | y-axis label: ATV concentration (ng/mL) |
| Programming notes | 1. There should be two plots (on same page): |
| | a. Cartesian Plot over 24 h or tau (to show Cmax differences) |

| b. Semi-Log Plot over entire time range (to show terminal phase differences |
|------------------------------------------------------------------------------|
| 2. Treatment and/or Study Day overlay, as appropriate |
| 3. Add in dotted line for LLOQ value |
| 4. Cartesian and semi-log plots for each individual subject on the same page |

| Parameter | Values |
|---|---|
| Template ID | MS_PK_G_002 |
| Output File Name | rg-pk-cpar3atvs2.lst |
| Purpose | WK24S2 |
| Table No. | Figure S.8.2.3B |
| Title 1 | Plots of Individual ATV Plasma Concentration Profiles vs. Time |
| Title 2 | Evaluable PK Population- Stage 2 |
| Footnote 1 | C = BMS 955176 120 mg QD + ATV + DTG<br>D = BMS 955176 180 mg QD + ATV + DTG<br>E = TDF + ATV/r + DTG |
| Footnote 2 | Notes: LLOQ – xx ng/mL; <lloq "missing"="" as="" calculation="" for="" mean="" of="" td="" treated="" values="" values<="" were=""></lloq> |
| Layout notes | x-axis label: time y-axis label: ATV concentration (ng/mL) |
| Programming notes | 1. There should be two plots (on same page): a. Cartesian Plot over 24 h or tau (to show Cmax differences) b. Semi-Log Plot over entire time range (to show terminal phase differences 2. Treatment and/or Study Day overlay, as appropriate 3. Add in dotted line for LLOQ value 4. Cartesian and semi-log plots for each individual subject on the same page |

| Parameter | Values |
|-----------|--------|
|-----------|--------|

| Template ID | MS_PK_G_002 |
|---|---|
| Output File Name | rg-pk-cpar3dtgs1.lst |
| Purpose | WK24S1 |
| Table No. | Figure S.8.2.3C |
| Title 1 | Plots of Individual DTG Plasma Concentration Profiles vs. Time |
| Title 2 | Evaluable PK Population - Stage 1 |
| Footnote 1 | A = BMS 955176 120 mg QD + ATV/r + DTG |
| | B = TDF + ATV/r + DTG |
| Footnote 2 | Notes: LLOQ – xx ng/mL; <lloq "missing"="" as="" calculation="" for="" mean="" of="" td="" treated="" values="" values<="" were=""></lloq> |
| Layout notes | x-axis label: time |
| | y-axis label: DTG concentration (ng/mL) |
| Programming notes | 1. There should be two plots (on same page): |
| | a. Cartesian Plot over 24 h or tau (to show Cmax differences) |
| | b. Semi-Log Plot over entire time range (to show terminal phase differences |
| | 2. Treatment and/or Study Day overlay, as appropriate |
| | 3. Add in dotted line for LLOQ value |
| | 4. Cartesian and semi-log plots for each individual subject on the same page |

| Parameter | Values |
|---|---|
| Template ID | MS_PK_G_002 |
| Output File Name | rg-pk-cpar3dtgs2.lst |
| Purpose | WK24S2 |
| Table No. | Figure S.8.2.3C |
| Title 1 | Plots of Individual DTG Plasma Concentration Profiles vs. Time |
| Title 2 | Evaluable PK Population - Stage 2 |
| Footnote 1 | C = BMS 955176 120 mg QD + ATV + DTG<br>D = BMS 955176 180 mg QD + ATV + DTG |

| | E = TDF + ATV/r + DTG |
|---|---|
| Footnote 2 | Notes: LLOQ – xx ng/mL; <lloq "missing"="" as="" calculation="" for="" mean="" of="" td="" treated="" values="" values<="" were=""></lloq> |
| Layout notes | x-axis label: time |
| | y-axis label: DTG concentration (ng/mL) |
| Programming notes | 1. There should be two plots (on same page): |
| | a. Cartesian Plot over 24 h or tau (to show Cmax differences) |
| | b. Semi-Log Plot over entire time range (to show terminal phase differences |
| | 2. Treatment and/or Study Day overlay, as appropriate |
| | 3. Add in dotted line for LLOQ value |
| | 4. Cartesian and semi-log plots for each individual subject on the same page |

## Template MS\_PK\_G\_001: Overlay of Individual Matrix Concentration vs. Time

Gamma-Secretase Inhibitor CN156008 BMS-708163 Final Clinical Study Report

Appendix 8.1.3

Spaghetti Plot Overlay by Treatment followed by Individual Plots with Treatment Overlay for Donepesil

Treatment = TRT A Analyte = donepezil StudyDay = 14



TREATMENT CODES:

PROGRAM SOURCE: eToolBox/DataXchange\BMS-708163\CN156008\GENERIC\_PK\_1\_2.0009 RUN DATE:29JUN2010 15:14

| Parameter | Values |
|---|---|
| Template ID | MS_PK_G_001 |
| Output File Name | rg-pk-cpar1bmss1.lst |
| Purpose | WK24S1 |
| Table No. | Figure S.8.2.1A |
| Title 1 | Overlay of Individual BMS-955176 Plasma Concentration Profile vs. Time by Treatment |
| Title 2 | Evaluable PK Population - Stage 1 |
| Footnote 1 | A = BMS 955176 120 mg QD + ATV/r + DTG |

| | B = TDF + ATV/r + DTG |
|---|---|
| Layout notes | x-axis label: time |
| | y-axis label: BMS955176 concentration (ng/mL) |
| Programming notes | 1. Treatment and/or Study Day overlay, as appropriate. |
| | 2. There should be two plots (on same page): |
| | a. Cartesian Plot over 24 h or tau (to show Cmax differences) |
| | b. Semi-Log Plot over entire time range (to show terminal phase differences |
| | 3. Cartesian and semi-log plots on the same page (sometimes referred to as a spaghetti plot as there are no symbols in the profiles) |

| Parameter | Values |
|---|---|
| Template ID | MS_PK_G_001 |
| Output File Name | rg-pk-cpar1bmss2.lst |
| Purpose | WK24S2 |
| Table No. | Figure S.8.2.1A |
| Title 1 | Overlay of Individual BMS-955176 Plasma Concentration Profile vs. Time by Treatment |
| Title 2 | Evaluable PK Population - Stage 2 |
| Footnote 1 | C = BMS 955176 120 mg QD + ATV + DTG |
| | D = BMS 955176 180 mg QD + ATV + DTG |
| | E = TDF + ATV/r + DTG |
| Layout notes | x-axis label: time |
| | y-axis label: BMS955176 concentration (ng/mL) |
| Programming notes | 1. Treatment and/or Study Day overlay, as appropriate. |
| | 2. There should be two plots (on same page): |
| | a. Cartesian Plot over 24 h or tau (to show Cmax differences) |
| | b. Semi-Log Plot over entire time range (to show terminal phase differences |
| | 3. Cartesian and semi-log plots on the same page (sometimes referred to as a spaghetti plot as there are no symbols in the profiles) |

| Parameter | Values |
|---|---|
| Template ID | MS_PK_G_001 |
| Output File Name | rg-pk-cparlatvs1.lst |
| Purpose | WK24S1 |
| Table No. | Figure S.8.2.1B |
| Title 1 | Overlay of Individual ATV Plasma Concentration Profile vs. Time by Treatment |
| Title 2 | Evaluable PK Population - Stage 1 |
| Footnote 1 | A = BMS 955176 60 mg QD + TDF/FTC B = BMS 955176 120 mg QD + TDF/FTC C = BMS 955176 180 mg QD + TDF/FTC D = EFV 600 mg QD + TDF/FTC |
| Layout notes | x-axis label: time y-axis label: ATV concentration (ng/mL) |
| Programming notes | <ol> <li>Treatment and/or Study Day overlay, as appropriate.</li> <li>There should be two plots (on same page): <ul> <li>Cartesian Plot over 24 h or tau (to show Cmax differences)</li> <li>Semi-Log Plot over entire time range (to show terminal phase differences)</li> </ul> </li> <li>Cartesian and semi-log plots on the same page (sometimes referred to as a spaghetti plot as there are no symbols in the profiles)</li> </ol> |

| Parameter | Values |
|---|---|
| Template ID | MS_PK_G_001 |
| Output File Name | rg-pk-cparlatvs2.lst |
| Purpose | WK24S2 |
| Table No. | Figure S.8.2.1B |
| Title 1 | Overlay of Individual ATV Plasma Concentration Profile vs. Time by Treatment |
| Title 2 | Evaluable PK Population - Stage 2 |
| Footnote 1 | C = BMS 955176 120 mg QD + ATV + DTG |

| | D = BMS 955176 180 mg QD + ATV + DTG |
|---|---|
| | E = TDF + ATV/r + DTG |
| Layout notes | x-axis label: time |
| | y-axis label: ATV concentration (ng/mL) |
| Programming notes | 1. Treatment and/or Study Day overlay, as appropriate. |
| | 2. There should be two plots (on same page): |
| | a. Cartesian Plot over 24 h or tau (to show Cmax differences) |
| | b. Semi-Log Plot over entire time range (to show terminal phase differences |
| | 3. Cartesian and semi-log plots on the same page (sometimes referred to as a spaghetti plot as there are no symbols in the profiles) |

| Parameter | Values |
|---|---|
| Template ID | MS_PK_G_001 |
| Output File Name | rg-pk-cpar1dtgs1.lst |
| Purpose | WK24S1 |
| Table No. | Figure S.8.2.1A |
| Title 1 | Overlay of Individual DTG Plasma Concentration Profile vs. Time by Treatment |
| Title 2 | Evaluable PK Population - Stage 1 |
| Footnote 1 | A = BMS 955176 120 mg QD + ATV/r + DTG |
| | B = TDF + ATV/r + DTG |
| Layout notes | x-axis label: time |
| | y-axis label: DTG concentration (ng/mL) |
| Programming notes | 1. Treatment and/or Study Day overlay, as appropriate. |
| | 2. There should be two plots (on same page): |
| | a. Cartesian Plot over 24 h or tau (to show Cmax differences) |
| | b. Semi-Log Plot over entire time range (to show terminal phase differences |
| | 3. Cartesian and semi-log plots on the same page (sometimes referred to as a spaghetti plot as there are no symbols in the profiles) |

| Parameter | Values |
|-----------|--------|
|-----------|--------|

| Template ID | MS_PK_G_001 |
|---|---|
| Output File Name | rg-pk-cpar1dtgs2.lst |
| Purpose | WK24S2 |
| Table No. | Figure S.8.2.1A |
| Title 1 | Overlay of Individual DTG Plasma Concentration Profile vs. Time by Treatment |
| Title 2 | Evaluable PK Population - Stage 2 |
| Footnote 1 | C = BMS 955176 120 mg QD + ATV + DTG<br>D = BMS 955176 180 mg QD + ATV + DTG<br>E = TDF + ATV/r + DTG |
| Layout notes | x-axis label: time y-axis label: DTG concentration (ng/mL) |
| Programming notes | <ol> <li>Treatment and/or Study Day overlay, as appropriate.</li> <li>There should be two plots (on same page): <ul> <li>Cartesian Plot over 24 h or tau (to show Cmax differences)</li> <li>Semi-Log Plot over entire time range (to show terminal phase differences)</li> </ul> </li> <li>Cartesian and semi-log plots on the same page (sometimes referred to as a spaghetti plot as there are no symbols in the profiles)</li> </ol> |

## Template MS\_PK\_G\_006: Mean Plot of Matrix Concentration vs. Time





| Parameter | Values |
|---|---|
| Template ID | MS_PK_G_006 |
| Output File Name | rg-pk-cpar6bmss1.lst |
| Purpose | WK24S1 |
| Table No. | Figure S.8.2.6A |
| Title 1 | Mean (+SD) BMS-955176 Plasma Concentration Profile vs. Time |
| Title 2 | Evaluable PK Population - Stage 1 |
| Footnote 1 | A = BMS 955176 120 mg QD + ATV/r + DTG |
| | B = TDF + ATV/r + DTG |
| Layout notes | x-axis label: time |
| | y-axis label: BMS-955176 concentration (ng/mL) |
| Programming notes | 1. Including SD bar |
| | 2. Treatment and/or Study Day overlay, as appropriate |
| | 3. There should be two plots (both on same page): |
| | a. Linear plot over 24 h or tau (to show Cmax differences) |
| | b. Semi-log plot over entire time range if longer than tau (to show terminal phase differences) |
| | 4. Add in dotted line for LLOQ |
| | 5. in-text figure required (Figure 9.1) |

| Parameter | Values |
|---|---|
| Template ID | MS_PK_G_006 |
| Output File Name | rg-pk-cpar6bmss2.lst |
| Purpose | WK24S2 |
| Table No. | Figure S.8.2.6A |
| Title 1 | Mean (+SD) BMS-955176 Plasma Concentration Profile vs. Time |
| Title 2 | Evaluable PK Population - Stage 2 |
| Footnote 1 | C = BMS 955176 120 mg QD + ATV + DTG |

| | D = BMS 955176 180 mg QD + ATV + DTG |
|---|---|
| | E = TDF + ATV/r + DTG |
| Layout notes | x-axis label: time |
| | y-axis label: BMS-955176 concentration (ng/mL) |
| Programming notes | 1. Including SD bar |
| | 2. Treatment and/or Study Day overlay, as appropriate |
| | 3. There should be two plots (both on same page): |
| | a. Linear plot over 24 h or tau (to show Cmax differences) |
| | b. Semi-log plot over entire time range if longer than tau (to show terminal phase differences) |
| | 4. Add in dotted line for LLOQ |
| | 5. in-text figure required (Figure 9.1) |

| Parameter | Values |
|---|---|
| Template ID | MS_PK_G_006 |
| Output File Name | rg-pk-cpar6atvs1.lst |
| Purpose | WK24S1 |
| Table No. | Figure S.8.2.6B |
| Title 1 | Mean (+SD) ATV Plasma Concentration Profile vs. Time |
| Title 2 | Evaluable PK Population - Stage 1 |
| Footnote 1 | A = BMS 955176 120 mg QD + ATV/r + DTG |
| | B = TDF + ATV/r + DTG |
| Layout notes | x-axis label: time |
| | y-axis label: ATV concentration (ng/mL) |
| Programming notes | 1. Including SD bar |
| | 2. Treatment and/or Study Day overlay, as appropriate |
| | 3. There should be two plots (both on same page): |
| | a. Linear plot over 24 h or tau (to show Cmax differences) |
| | b. Semi-log plot over entire time range if longer than tau (to show terminal phase differences) |

| 4. Add in dotted line for LLOQ |
|-----------------------------------------|
| 5. in-text figure required (Figure 9.1) |

| Parameter | Values |
|---|---|
| Template ID | MS_PK_G_006 |
| Output File Name | rg-pk-cpar6atvs2.lst |
| Purpose | WK24S2 |
| Table No. | Figure S.8.2.6B |
| Title 1 | Mean (+SD) ATV Plasma Concentration Profile vs. Time |
| Title 2 | Evaluable PK Population - Stage 2 |
| Footnote 1 | C = BMS 955176 120 mg QD + ATV + DTG<br>D = BMS 955176 180 mg QD + ATV + DTG<br>E = TDF + ATV/r + DTG |
| Layout notes | x-axis label: time y-axis label: ATV concentration (ng/mL) |
| Programming notes | <ol> <li>Including SD bar</li> <li>Treatment and/or Study Day overlay, as appropriate</li> <li>There should be two plots (both on same page): <ul> <li>a. Linear plot over 24 h or tau (to show Cmax differences)</li> <li>b. Semi-log plot over entire time range if longer than tau (to show terminal phase differences)</li> </ul> </li> <li>Add in dotted line for LLOQ</li> <li>in-text figure required (Figure 9.1)</li> </ol> |

| Parameter | Values |
|------------------|----------------------|
| Template ID | MS_PK_G_006 |
| Output File Name | rg-pk-cpar6dtgs1.lst |
| Purpose | WK24S1 |

| Table No. | Figure S.8.2.6C |
|---|---|
| Title 1 | Mean (+SD) DTG Plasma Concentration Profile vs. Time |
| Title 2 | Evaluable PK Population - Stage 1 |
| Footnote 1 | A = BMS 955176 120 mg QD + ATV/r + DTG $B = TDF + ATV/r + DTG$ |
| Layout notes | x-axis label: time y-axis label: DTG concentration (ng/mL) |
| Programming notes | <ol> <li>Including SD bar</li> <li>Treatment and/or Study Day overlay, as appropriate</li> <li>There should be two plots (both on same page): <ul> <li>Linear plot over 24 h or tau (to show Cmax differences)</li> <li>Semi-log plot over entire time range if longer than tau (to show terminal phase differences)</li> </ul> </li> <li>Add in dotted line for LLOQ</li> <li>in-text figure required (Figure 9.1)</li> </ol> |

| Parameter | Values |
|---|---|
| Template ID | MS_PK_G_006 |
| Output File Name | rg-pk-cpar6dtgs2.lst |
| Purpose | WK24S2 |
| Table No. | Figure S.8.2.6C |
| Title 1 | Mean (+SD) DTG Plasma Concentration Profile vs. Time |
| Title 2 | Evaluable PK Population - Stage 2 |
| Footnote 1 | C = BMS 955176 120 mg QD + ATV + DTG<br>D = BMS 955176 180 mg QD + ATV + DTG<br>E = TDF + ATV/r + DTG |
| Layout notes | x-axis label: time y-axis label: DTG concentration (ng/mL) |

| Programming notes | 1. Including SD bar |
|---|---|
| | 2. Treatment and/or Study Day overlay, as appropriate |
| | 3. There should be two plots (both on same page): |
| | a. Linear plot over 24 h or tau (to show Cmax differences) |
| | b. Semi-log plot over entire time range if longer than tau (to show terminal phase differences) |
| | 4. Add in dotted line for LLOQ |
| | 5. in-text figure required (Figure 9.1) |

## 4.8 Pharmacodynamic Results

Not applicable

## 4.9 Other Study Results

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_006 |
| Output File Name | rt-qs-eq5ds1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Appendix 10.1.1 |
| Title 1 | EQ-5D-3L Summary of US and UK Centric Scores and Changes From Baseline Over Time on Treatment |
| Title 2 | Treated Subjects - Stage 1 |
| Layout notes | Parameters: US Centric Score, UK Centric Score No units. |

| Parameter | Values |
|------------------|------------------------|
| Template ID | SS_VL_T_006 |
| Output File Name | rt-qs-eq5ds2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |

| Table No. | Appendix 10.1.2 |
|---|---|
| Title 1 | EQ-5D-3L Summary of US and UK Centric Scores and Changes From Baseline Over Time on Treatment |
| Title 2 | Treated Subjects - Stage 2 |
| Layout notes | Parameters: US Centric Score, UK Centric Score |
| | No units. |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_006 |
| Output File Name | rt-qs-fahis1.lst |
| Purpose | WK24S1, WK48S1, WK96S1, WK96S2 |
| Table No. | Appendix 10.2.1 |
| Title 1 | FAHI Summary of Total Scores Over Time on Treatment |
| Title 2 | Treated Subjects - Stage 1 |
| Layout notes | Do not show title row "Parameter (Units)". Do not show changes from baseline. No units. |

| Parameter | Values |
|---|---|
| Template ID | SS_VL_T_006 |
| Output File Name | rt-qs-fahis2.lst |
| Purpose | WK24S2, WK48S2, WK96S2 |
| Table No. | Appendix 10.2.2 |
| Title 1 | FAHI Summary of Total Scores Over Time on Treatment |
| Title 2 | Treated Subjects - Stage 2 |
| Layout notes | Do not show title row "Parameter (Units)". Do not show changes from baseline. No units. |